

Activated: 12/08/14 Version Date: 12/19/2019 Closed: 09/30/19 Amendment #10A

### CHILDREN'S ONCOLOGY GROUP

### **AALL1331**

Risk-Stratified Randomized Phase III Testing of Blinatumomab (NSC# 765986) in First Relapse of Childhood B-Lymphoblastic Leukemia (B-ALL)

IND Sponsor for Blinatumomab: DCTD, NCI

### A Groupwide Phase III Study

Participating Countries: Australia, Canada, New Zealand and United States

THIS PROTOCOL IS FOR RESEARCH PURPOSES ONLY, AND SHOULD NOT BE COPIED, REDISTRIBUTED OR USED FOR ANY OTHER PURPOSE. MEDICAL AND SCIENTIFIC INFORMATION CONTAINED WITHIN THIS PROTOCOL IS NOT INCLUDED TO AUTHORIZE OR FACILITATE THE PRACTICE OF MEDICINE BY ANY PERSON OR ENTITY. RESEARCH MEANS A SYSTEMATIC INVESTIGATION, INCLUDING RESEARCH DEVELOPMENT, TESTING AND EVALUATION, DESIGNED TO DEVELOP OR CONTRIBUTE TO GENERALIZABLE KNOWLEDGE. THIS PROTOCOL IS THE RESEARCH PLAN DEVELOPED BY THE CHILDREN'S ONCOLOGY GROUP TO INVESTIGATE A PARTICULAR STUDY QUESTION OR SET OF STUDY QUESTIONS AND SHOULD NOT BE USED TO DIRECT THE PRACTICE OF MEDICINE BY ANY PERSON OR TO PROVIDE INDIVIDUALIZED MEDICAL CARE, TREATMENT, OR ADVICE TO ANY PATIENT OR STUDY SUBJECT. THE PROCEDURES IN THIS PROTOCOL ARE INTENDED ONLY FOR USE BY CLINICAL ONCOLOGISTS IN CAREFULLY STRUCTURED SETTINGS, AND MAY NOT PROVE TO BE MORE EFFECTIVE THAN STANDARD TREATMENT. ANY PERSON WHO REQUIRES MEDICAL CARE IS URGED TO CONSULT WITH HIS OR HER PERSONAL PHYSICIAN OR TREATING PHYSICIAN OR VISIT THE NEAREST LOCAL HOSPITAL OR HEALTHCARE INSTITUTION.

## **STUDY CHAIR**

Patrick Brown, MD 1650 Orleans Street, CRB1 RM 2M49 Baltimore, MD. 21231

Fax: (410) 955-8897 E-mail: pbrown2@jhmi.edu

Phone: (410) 614-4915

2



# **ABBREVIATIONS**

| Abbreviation | Term |
|--------------|------------------------------------|
| aGVHD | Acute graft versus host disease |
| B-ALL | B-Lymphoblastic Leukemia |
| CR | Complete remission |
| DFS | Disease free survival |
| GVHD | Graft vs. host disease |
| HR | High risk |
| HSCT | Hematopoietic stem cell transplant |
| IEM | Isolated extramedullary |
| IR | Intermediate risk |
| IS | Immune suppression |
| LR | Low risk |
| MRD | Minimal residual disease |
| PFS | Progression free survival |
| $Ph^+$ | Philadelphia chromosome positive |
| TF | Treatment failure |
| TKI | Tyrosine kinase inhibitor |
| URD | Unrelated Donor |



# TABLE OF CONTENTS

| <u>SECT</u> | <u> ION</u> | | <u>P.</u> | <u>AGE</u> |
|---|---|---|---|---|
| STUI | OY CON | MMITTI | <b>EE</b> | 12 |
| ABST | <b>TRACT</b> | | | 15 |
| EXPI | ERIME | NTAL D | ESIGN SCHEMA | 16 |
| 1.0 | GOALS AND OBJECTIVES (SCIENTIFIC AIMS) | | | |
| | 1.1 | 1.1 Primary Aims | | |
| | | 1.1.1 | To compare disease free survival (DFS) of HR and IR relapse B-ALL patien who are randomized following Induction Block 1 chemotherapy to receive etwo intensive chemotherapy blocks or two 5-week blocks of blinatumomab (HR/IR Randomization). (Closed effective September 18, 2019) To compare DFS of LR relapse B-ALL patients who are randomized following the survival of | ither<br>17 |
| | | | Block 1 chemotherapy to receive either chemotherapy alone or chemotherapy plus blinatumomab (LR Randomization). | |
| | 1.2 | Secon | dary Aims | 17 |
| | | 1.2.1 | To compare overall survival (OS) of HR and IR relapse B-ALL patients who randomized following Induction Block 1 chemotherapy to receive either two intensive chemotherapy blocks or two 5 week blocks of blinatumomab (HR/Randomization). (Closed effective September 18, 2019) | ) |
| | | 1.2.2 | To compare OS of LR relapse B-ALL patients who are randomized followin Block 1 chemotherapy to receive either chemotherapy alone or chemotherapy plus blinatumomab (LR Randomization). | _ |
| | 1.3 | Explo | ratory Aims | |
| | | 1.3.1 | To compare the rates of MRD $\geq$ 0.01% at the end of Block 2 and Block 3 for and IR relapse B-ALL patients in HR/IR randomization. (Closed effective September 18, 2019) | r HR<br>17 |
| | | 1.3.2 | To estimate, for treatment failure (TF) patients not previously receiving blinatumomab, the hematologic complete remission rate (CR), rate of MRD < 0.01%, and proportion able to proceed to hematopoietic stem cell transplar (HSCT) in CR after treatment with blinatumomab. | nt<br>17 |
| | | 1.3.3 | To assess the feasibility and safety of rapid taper of immune suppression for subset of HSCT patients with MRD $\geq$ 0.01% pre- and/or post-HSCT with no acute graft versus host disease (aGVHD). | |
| | | 1.3.4 | To evaluate blinatumomab pharmacokinetics (PK) and explore exposure-response relationships for measures of safety and effectiveness. | 17 |
| 2.0 | BACKGROUND | | | |
| | 2.1 | Overv | view | 18 |
| | 2.2 | Ration | nale for Selected Approach and Trial Design | 18 |
| | | 2.2.1 | Rationale for Consolidated First Relapse B-ALL Trial | 18 |
| | | 2.2.2 | Rationale for Studying Blinatumomab in First Relapse of B-ALL | 19 |
| | | 2.2.3 | Rationale for Risk Stratification | 21 |
| | | 2.2.4 | Rationale for Backbone Chemotherapy Treatment (Blocks 1, 2 and 3) | 22 |
| | | 2.2.5 | Rationale for Backbone Chemotherapy Treatment (post-Block 3) | 24 |
| | | 2.2.6 | Therapy for CNS3 Patients | 24 |
| | | 2.2.7 | Treatment of Testicular Relapse | 25 |



| | | 2.2.8 | Treatment Failure (TF) | 26 |
|---|---|---|---|---|
| | | 2.2.9 | Additional non-randomized Pilot Intervention for Very High Risk Subset of HSCT Recipients based on MRD and aGVHD | 26 |
| | | 2.2.10 | Rationale for closure of the HR/IR Randomization (Amendment #10) | 27 |
| 3.0 | STUI | DY ENR | OLLMENT PROCEDURES AND PATIENT ELIGIBILITY | 28 |
| | 3.1 | Study | Enrollment | 28 |
| | | 3.1.1 | Patient Registration | 28 |
| | | 3.1.2 | IRB Approval | 28 |
| | | 3.1.3 | Study Enrollment | 29 |
| | | 3.1.4 | Timing | 30 |
| | | 3.1.5 | Staged Consent | 30 |
| | | 3.1.6 | Risk Assignment, Randomization, and Treatment Assignment | 31 |
| | | 3.1.7 | Callbacks | 32 |
| | | 3.1.8 | Drug Preparation and Administration | 33 |
| | | 3.1.9 | Inclusion of Women and Minorities | 33 |
| | 3.2 | Patien | nt Eligibility Criteria | 33 |
| | | 3.2.1 | Age | 33 |
| | | 3.2.2 | Diagnosis | 33 |
| | | 3.2.3 | Prior Therapy | 34 |
| | | 3.2.4 | Performance Status | 34 |
| | | 3.2.5 | Organ Function Requirements | 34 |
| | | 3.2.6 | Exclusion Criteria | 35 |
| | | 3.2.7 | Regulatory Requirements | 36 |
| | 3.3 | Defini | itions | 36 |
| 4.0 | TRE | ATMEN | T PLAN | 40 |
| | 4.1 | Overv | view of Treatment Plan | 40 |
| | | 4.1.1 | TREATMENT ASSIGNMENTS | 41 |
| | | 4.1.2 | Concomitant Therapy Restrictions | 42 |
| | | 4.1.3 | Supportive Care for Patients 15 Years and Older | 43 |
| | 4.2 | Block | 1 (All patients) - 4 Weeks Duration | 44 |
| | | 4.2.1 | Disease Evaluation Pre-Treatment | 44 |
| | | 4.2.2 | General Chemotherapy Guidelines | 44 |
| | | 4.2.3 | Block 1 Chemotherapy | 44 |
| | | 4.2.4 | Disease Evaluation End Block 1 | 46 |
| | | 4.2.5 | Research Studies Block 1 | 46 |
| | | 4.2.6 | HLA Tissue Typing for Hematopoietic Stem Cell Transplant | 46 |
| | | 4.2.7 | Evaluation 1 (Risk Assessment following Block 1) | 46 |
| | 4.3 | Block | 2 (LR Patients: Post-randomization) – 4 weeks duration | 48 |
| | | 4.3.1 | Criteria to Begin Block 2 Therapy | 48 |
| | | 4.3.2 | Testicular Radiation Therapy (TRT) | 48 |
| | | 4.3.3 | General Chemotherapy Guidelines | 48 |
| | | 4.3.4 | Block 2 Chemotherapy | 49 |
| | | 4.3.5 | Evaluation 2 (Disease Evaluation End Block 2) | 51 |



| | 4.3.6 | Following Completion of Block 2: | 51 |
|---|---|---|---|
| 4.4 | Block | 3 (LR Patients on Arm C) - 4 weeks | 52 |
| | 4.4.1 | Criteria to Begin Block 3 Therapy | 52 |
| | 4.4.2 | General Chemotherapy Guidelines | 52 |
| | 4.4.3 | Block 3 Chemotherapy | 52 |
| | 4.4.4 | Disease Evaluation End Block 3 (HR/IR Patients ONLY): | 54 |
| | 4.4.5 | Following completion of Block 3: | 54 |
| 4.5 | Blinati | umomab Block: Cycle 1 (HR/IR Patients in Arm B) - 5 weeks | 55 |
| | 4.5.1 | Criteria to Begin Blinatumomab Block: Cycle 1 | 55 |
| | 4.5.2 | Testicular Radiation Therapy (TRT) | 56 |
| | 4.5.3 | General Chemotherapy Guidelines | 56 |
| | 4.5.4 | Blinatumomab Block: Cycle 1 Chemotherapy | 56 |
| | 4.5.5 | Disease Evaluation End-Blinatumomab Block: Cycle 1 | 57 |
| | 4.5.6 | Following completion of Blinatumomab Block: Cycle 1 (Arm B) | 57 |
| 4.6 | Blinati | umomab Block: Cycle 2 (HR/IR Patients in Arm B) - 5 weeks | 58 |
| | 4.6.1 | Criteria to Begin Blinatumomab Block: Cycle 2 | 58 |
| | 4.6.2 | General Chemotherapy Guidelines | 58 |
| | 4.6.3 | Blinatumomab Block: Cycle 2 Administration Guidelines | 59 |
| | 4.6.4 | Disease Evaluation End-Blinatumomab Block: Cycle 2 | 59 |
| | 4.6.5 | Following completion of Blinatumomab Block: Cycle 2 (Arm B): | 60 |
| 4.7 | Blinati | umomab-S: Cycle 1 (Salvage Therapy) - 5 weeks | 61 |
| | 4.7.1 | Criteria to Begin Blinatumomab-S: Cycle 1 | 61 |
| | 4.7.2 | Testicular Radiation Therapy (TRT) | 61 |
| | 4.7.3 | General Chemotherapy Guidelines | 62 |
| | 4.7.4 | Blinatumomab-S: Cycle 1 Chemotherapy Guidelines | 62 |
| | 4.7.5 | Disease Evaluation End Blinatumomab-S Cycle 1: | 63 |
| | 4.7.6 | Following completion of Blinatumomab-S: Cycle 1: | 63 |
| 4.8 | Blinati | umomab-S: Cycle 2 (Salvage Therapy) - 5 weeks | 64 |
| | 4.8.1 | Criteria to Begin Blinatumomab-S: Cycle 2 | 64 |
| | 4.8.2 | General Chemotherapy Guidelines | 64 |
| | 4.8.3 | Blinatumomab-S: Cycle 2 Chemotherapy | 65 |
| | 4.8.4 | Disease Evaluation End-Blinatumomab-S: Cycle 2 | 65 |
| | 4.8.5 | Following completion of Blinatumomab-S: Cycle 2: | 65 |
| 4.9 | Hemat | topoietic Stem Cell Transplant | 67 |
| | 4.9.1 | Overview | 67 |
| | 4.9.2 | Preparative Regimen Administration | 71 |
| | 4.9.3 | Preparative Regimen Administration Tables | 71 |
| | 4.9.4 | Sanctuary Site Therapy (see Section 14.0) | 73 |
| | 4.9.5 | Growth Factor Administration | 73 |
| | 4.9.6 | GVHD Prophylaxis | 74 |
| | 4.9.7 | Standard Taper of Immune Suppression | 76 |
| | 4.9.8 | Accelerated Taper of Immune Suppression | 76 |
| 4.10 | _ | ng Maintenance Therapy (All HR/IR Patients, as required) – up to 6 weeks | 77 |
| | 4.10.1 | Criteria to Begin Bridging Maintenance Therapy | 77 |



| | 4.10.2 | General Chemotherapy Guidelines | 77 |
|---|---|---|---|
| | 4.10.3 | Bridging Maintenance Chemotherapy Guidelines | 77 |
| 4.11 | Contin | nuation 1/Continuation 2 (All LR Patients) - 8 weeks | 78 |
| | 4.11.1 | Criteria to Begin and During Continuation Therapy | 78 |
| | 4.11.2 | General Chemotherapy Guidelines | 79 |
| | 4.11.3 | Continuation 1/Continuation 2 Chemotherapy Guidelines | 79 |
| | 4.11.4 | Following Continuation 1: | 82 |
| | 4.11.5 | Following Continuation 2: | 82 |
| 4.12 | Mainto | enance Cycle 1 (All LR patients) – 12 weeks | 83 |
| | 4.12.1 | Criteria to Begin Maintenance Therapy | 83 |
| | 4.12.2 | Duration of Cycles in Maintenance Therapy | 83 |
| | 4.12.3 | General Chemotherapy Guidelines | 83 |
| | 4.12.4 | Maintenance Chemotherapy Cycle 1 | 84 |
| | | Following Maintenance Cycle 1: | 85 |
| 4.13 | | enance Chemoradiation - 3 weeks | 86 |
| | | Criteria to Begin Maintenance Chemoradiation | 86 |
| | | Cranial Radiation Therapy | 86 |
| | | General Chemotherapy Guidelines | 86 |
| | | Chemotherapy Guidelines for Maintenance Chemoradiation | 86 |
| | | Following Maintenance Chemoradiation: | 87 |
| 4.14 | | enance-Post Cycle 1 (All LR patients) | 88 |
| | | Criteria to Continue Maintenance Therapy | 88 |
| | | Duration of Cycles in Maintenance Chemotherapy | 88 |
| | | General Chemotherapy Guidelines | 88 |
| | | Chemotherapy Guidelines for Maintenance-Post Cycle 1 | 88 |
| 4.15 | | umomab Block: Cycle 1 (Patients in Arm D) - 5 weeks | 90 |
| | | Criteria to Begin Blinatumomab | 90 |
| | | General Chemotherapy Guidelines | 90 |
| | | Blinatumomab Block: Cycle 1 (Patients in Arm D) Chemotherapy | 91 |
| | | Following Blinatumomab Block: Cycle 1 (Arm D) | 91 |
| 4.16 | | umomab Block: Cycle 2/3 (LR Patients in Arm D) - 5 weeks | 92 |
| | | Criteria to Begin Blinatumomab Block: Cycle 2/3 | 92 |
| | | General Chemotherapy Guidelines | 92 |
| | | Blinatumomab Block: Cycle 2/3: Chemotherapy Guidelines | 92 |
| | | Following Blinatumomab Block Cycle 2: | 93 |
| | 4.16.5 | Following Blinatumomab Block Cycle 3: | 93 |
| DOSE | E MODII | FICATIONS FOR TOXICITIES | 94 |
| 5.1 | Aspara | aginase [Pegaspargase (PEG-Asparaginase) or Erwinia] | 94 |
| 5.2 | Blinatumomab | | |
| 5.3 | Cyclophosphamide | | |
| 5.4 | Cytarabine (ARAC) | | |
| 5.5 | | acycline-Mitoxantrone | 100 |
| 5.6 | Etopos | | 101 |
| 5.7 | Intratl | necal Methotrexate/Triple Intrathecal Therapy | 101 |

5.0



| | 5.8 | Intermediate-Dose Methotrexate (ID MTX) and Leucovorin Rescue | 103 |
|---|---|---|---|
| | | 5.8.1 ID MTX Infusion Guidelines and dose modifications for toxicity | 103 |
| | 5.9 | PO Methotrexate (MTX) and 6-Mercaptopurine (MP) | 106 |
| | 5.10 | Steroids (Dexamethasone) | 109 |
| | 5.11 | PO 6-Thioguanine (TG) | 110 |
| | 5.12 | Vincristine | 110 |
| | 5.13 | Stem Cell Transplant Regimen Agents | 111 |
| | | 5.13.1 Tacrolimus | 111 |
| | | 5.13.2 Cyclosporine | 112 |
| | | 5.13.3 Methotrexate | 112 |
| | | 5.13.4 Guidelines for Leucovorin Rescue | 113 |
| | | 5.13.5 Mycophenolate Mofetil (MMF) | 113 |
| | | 5.13.6 Adjustment of TBI/chemotherapy During the Preparative Regimen. | 113 |
| | | 5.13.7 Dose Adjustment of Chemotherapy for Patients Whose Weight Exceeds > | 125% |
| | | Ideal Body Weight (IBW) | 113 |
| 6.0 | DRU | G INFORMATION | 115 |
| | 6.1 | BLINATUMOMAB (11/18/2019) | 115 |
| | 6.2 | ASPARAGINASE Erwinia chrysanthemi (05/07/19) | 128 |
| | 6.3 | CYCLOPHOSPHAMIDE INJECTION (03/13/13) | 130 |
| | 6.4 | CYCLOSPORINE A (11/16/17) | 132 |
| | 6.5 | CYTARABINE - ALL ROUTES (07/13/15) | 134 |
| | 6.6 | DEXAMETHASONE (05/07/19) | 136 |
| | 6.7 | ETOPOSIDE – INJECTION (11/15/2016) | 138 |
| | 6.8 | FILGRASTIM, TBO-FILGRATIM, FILGRATIM-SNDZ (05/13/2019) | 141 |
| | 6.9 | FLUDARABINE (01/10/18) | 142 |
| | 6.10 | INTRATHECAL TRIPLES (05/08/12) | 146 |
| | 6.11 | LEUCOVORIN CALCIUM (05/07/19) | 147 |
| | 6.12 | MERCAPTOPURINE (11/27/17) | 149 |
| | 6.13 | METHOTREXATE-ALL ROUTES (05/07/19) | 150 |
| | 6.14 | MITOXANTRONE (11/27/17) | 154 |
| | 6.15 | MYCOPHENOLATE MOFETIL (12/06/18) | 156 |
| | 6.16 | PEGASPARGASE (06/05/17) | 160 |
| | 6.17 | TACROLIMUS (11/27/17) | 162 |
| | 6.18 | THIOGUANINE (12/05/2016) | 165 |
| | 6.19 | THIOTEPA (01/23/18) | 166 |
| | 6.20 | VINCRISTINE SULFATE (08/16/12) | 168 |
| 7.0 | | LUATIONS/MATERIAL AND DATA TO BE ACCESSIONED | 171 |
| 7.0 | 7.1 | | 171 |
| | 7.1<br>7.2 | Required and Optional Clinical, Laboratory and Disease Evaluations Research Studies | 171 |
| | 7.2 | At Relapse | 174 |
| | 7.3<br>7.4 | Follow-up | 175 |
| | | · | 1/5 |
| 8.0 | | TERIA FOR REMOVAL FROM PROTOCOL THERAPY AND OFF STUDY | 175 |
| | 1 14 1 | II.IX I A | |



| | 8.1 | Criter | ia for Removal from Protocol Therapy | 175 |
|---|---|---|---|---|
| | 8.2 | Off St | udy Criteria | 176 |
| 9.0 | STAT | TISTICA | L CONSIDERATIONS | 176 |
| | 9.1 | Statist | tical Design | 176 |
| | | 9.1.1 | Primary Endpoint | 176 |
| | | 9.1.2 | Secondary Endpoints | 176 |
| | | 9.1.3 | Exploratory Endpoints | 177 |
| | 9.2 | Patien | t Accrual and Expected Duration of Trial | 177 |
| | | 9.2.1 | Stratification to be used in the randomization | 177 |
| | | 9.2.2 | Sample size with power calculation (Activation Protocol) | 178 |
| | | 9.2.3 | Extension of accrual duration for both the LR cohort and the HR/IR cohort (Amendment #8) | 179 |
| | 9.3 | Statist | tical Analysis Methods | 183 |
| | | 9.3.1 | HR/IR Randomization for HR and IR relapse patients | 183 |
| | | 9.3.2 | LR Randomization for LR relapse patients | 189 |
| | | 9.3.3 | Pilot intervention for very high risk subset of HSCT recipients based on MF and aGVHD | RD<br>193 |
| | | 9.3.4 | Treatment Failure (TF) patients who are non-randomly assigned to blinatumomab | 195 |
| | | 9.3.5 | Blinatumomab related reportable adverse event (RAE) | 196 |
| | | 9.3.6 | Monitoring for infection rate of 96-hour bag changes in Blinatumomab administration (Amendment #2) | 196 |
| | | 9.3.7 | Monitoring for infection rate of 7-day bag changes in Blinatumomab administration (Amendment #8) | 196 |
| | 9.4 | Gende | er and Minority Accrual Estimates | 197 |
| 10.0 | EVAI | LUATIO | ON CRITERIA | 198 |
| | 10.1 | | non Terminology Criteria for Adverse Events (CTCAE) | 198 |
| | 10.2 | | nse Criteria | 198 |
| 11.0 | ADVI | ERSE EV | VENT REPORTING REQUIREMENTS | 199 |
| | 11.1 | Purpo | - | 199 |
| | 11.2 | | mination of reporting requirements | 199 |
| | 11.3 | | lited Reporting Requirements – Serious Adverse Events (SAEs) | 199 |
| | 11.4 | _ | al Situations for Expedited Reporting | 200 |
| | | - | SAEs Occurring More than 30 Days After Last Dose of Study Drug | 200 |
| | | | Persistent or Significant Disabilities/Incapacities | 200 |
| | | | Death | 200 |
| | | 11.4.4 | Secondary Malignancy | 201 |
| | | | Second Malignancy | 201 |
| | | | Pregnancy, Pregnancy Loss, and Death Neonatal | 201 |
| | | | Baseline AEs | 202 |
| | | | Persistent AEs | 202 |
| | | 11.5.3 | Recurrent AEs | 203 |
| | 11.6 | | tions to Expedited Reporting | 203 |
| | | _ | Specific Protocol Exceptions to Expedited Reporting (SPEER) | 203 |



| | | 11.6.2 | Special Situations as Exceptions to Expedited Reporting | 203 |
|---|---|---|---|---|
| | 11.7 | Report | ing Requirements - Investigator Responsibility | 203 |
| | 11.8 | Genera | al Instructions for Expedited Reporting via CTEP-AERS | 203 |
| | 11.9 | Report | ring Table for Late Phase 2 and Phase 3 Studies – Table A | 205 |
| | 11.10 | Protoc | ol Specific Additional Instructions and Reporting Exceptions | 206 |
| | 11.11 | Report | ting of Adverse Events for commercial agents – CTEP-AERS abbreviated | i |
| | | pathwa | ay | 206 |
| | 11.12 | Routin | e Adverse Event Reporting | 207 |
| 12.0 | RECO | RDS AN | ND REPORTING | 209 |
| | 12.1 | <b>CDUS</b> | | 209 |
| | 12.2 | CTA/C | CRADA | 209 |
| 13.0 | SPEC | IAL STU | UDIES AND SPECIMEN REQUIREMENTS | 211 |
| | 13.1 | Bankir | ng for Future Research (optional) | 211 |
| | 13.2 | Local l | Bone Marrow: Central review of cytogenetics/FISH | 212 |
| | 13.3 | Bone N | Marrow for Central Flow-Immunophenotyping and MRD (required) | 213 |
| | 13.4 | Bone N | Marrow for CRLF2 expression (optional) | 214 |
| | 13.5 | Blinatu | ımomab Pharmacodynamics (PD) (optional) | 215 |
| | 13.6 | Proteir | n Cell Stress Pathways (optional) | 216 |
| | 13.8 | Blinatı | ımomab PK (required) | 218 |
| 14.0 | RADI | ATION ' | THERAPY GUIDELINES FOR ALL PATIENTS | 219 |
| | 14.1 | Genera | al Guidelines | 219 |
| | | 14.1.1 | Required Benchmark and Questionnaires | 220 |
| | 14.2 | Indicat | tions for Radiation Therapy | 220 |
| | | 14.2.1 | Total Body Irradiation | 220 |
| | | 14.2.2 | Cranial Irradiation | 220 |
| | | 14.2.3 | Testicular Irradiation | 221 |
| | 14.3 | Timing | Ţ | 221 |
| | | 14.3.1 | All patients who might require irradiation should be seen in consultation by a radiation oncologist in advance of treatment. The purpose of the consultation to participate in planning the sequence of treatment and to determine the need extra medullary (cranial, testicular and other) and supplemental irradiation in conjunction with HSCT. | n is<br>d for |
| | | 14.3.2 | The timing of TBI and supplemental irradiation will be determined in part by TBI fractionation regimen. Supplemental irradiation should precede TBI and performed during weekdays. | |
| | 14.4 | Emerg | ency Irradiation | 221 |
| | 14.5 | Equipr | nent and Methods of Delivery | 221 |
| | 14.6 | Treatn | nent Volumes | 221 |
| | | 14.6.1 | Total Body Irradiation | 221 |
| | | 14.6.2 | Cranial Irradiation | 222 |
| | | 14.6.3 | Testicular Irradiation | 222 |
| | 14.7 | Target | Dose | 222 |
| | | 14.7.1 | Dose Definition | 222 |
| | | 1472 | Prescribed Dose Fractionation and Dose Rate for TRI | 222 |

| | | • | • | 4 | _ | _ | 4 |
|---|---|---|---|---|----|---|---|
| Α | А | L | Л | Л | -3 | 3 | 1 |

| | 14.7.3 Prescribed Dose and Fractionation for Cranial Irradiation | 222 |
|---|---|---|
| 14.8 | Treatment Technique | 223 |
| | 14.8.1 TBI | 223 |
| | 14.8.2 TBI - Lung Shielding | 223 |
| | 14.8.3 Cranial Irradiation | 224 |
| | 14.8.4 Testicular Irradiation | 224 |
| 14.9 | Organs at Risk | 224 |
| | 14.9.1 Normal tissue sparing for TBI | 224 |
| | 14.9.2 Normal tissue sparing for cranial irradiation | 224 |
| | 14.9.3 Normal tissue sparing for testicular irradiation | 224 |
| 14.10 | Dose Calculation and Reporting | 224 |
| | 14.10.1 Dose calculations for TBI | 224 |
| | 14.10.2 Dose Uniformity and Treatment Site Coverage | 226 |
| | 14.10.3 Tissue heterogeneity | 227 |
| | 14.10.4 Interruption of therapy | 227 |
| 14.11 | <b>Quality Assurance Documentation and Review</b> | 227 |
| 14.12 | <b>Definitions of Deviation in Protocol Performance</b> | 227 |
| | 14.12.1 TBI | 227 |
| | 14.12.2 Deviations for Cranial Irradiation Dose | 228 |
| | 14.12.3 Deviations for Testicular Irradiation Dose | 228 |
| APPENDIX I: | SUPPORTIVE CARE | 229 |
| APPENDIX II | : THERAPY DELIVERY MAPS | 233 |
| APPENDIX II | II: MERCAPTOPURINE DOSING GUIDELINES | 257 |
| APPENDIX I | V: THIOGUANINE DOSING GUIDELINES | 259 |
| APPENDIX V | YOUTH INFORMATION SHEETS | 260 |
| APPENDIX V | I: ADDITIONAL INFORMATION FOR BANKING FOR FUTURE | |
| RESE | ARCH CORRELATIVE BIOLOGY STUDY | 262 |
| | II-A: CLINICAL SITE MANAGEMENT OF OUT-PATIENT<br>TMENT USING CTEP-SUPPLIED BLINATUMOMAB | 264 |
| | TI-B: SHIPMENT OF BLINATUMOMAB IV BAG FROM PHARMACY TO PATIENT'S HOME | 268 |
| | III: ADDITIONAL INFORMATION FOR MRD CORRELATIVE OGY STUDY | 269 |
| | X: ADDITIONAL INFORMATION FOR CRLF2 CORRELATIVE OGY STUDY | 270 |
| | : ADDITIONAL INFORMATION FOR BLINATUMOMAB MACODYNAMICS CORRELATIVE BIOLOGY STUDY | 273 |
| APPENDIX X | I: ADDITIONAL INFORMATION FOR PROTEIN CELL STRESS WAYS CORRELATIVE BIOLOGY STUDY | 279 |
| ESTA1 | II: COG STEM CELL COMMITTEE CONSENSUS GUIDELINES FOR BLISHING ORGAN STAGE AND OVERALL GRADE OF ACUTE GRAFT | |
| VERS | US HOST DISEASE (GVHD) | 285 |





#### STUDY COMMITTEE

STUDY CHAIR

Patrick Brown, MD

Hematology/Oncology

Johns Hopkins Univ./Sidney Kimmel Cancer Center

1650 Orleans St. CRB 2M49

Baltimore, MD. 21231

Phone: (410) 614-4915 Fax: (410) 955-8897

Fax: (410) 955-8897 E-mail: pbrown2@jhmi.edu

STUDY VICE CHAIR

James A. Whitlock, MD

Hematology/Oncology

Hospital for Sick Children

555 University Ave, Room 9409 Black

Toronto, ON M5G 1X8

Phone: (416) 813-8885

Fax: (416) 813-5327

E-mail: jim.whitlock@sickkids.ca

STUDY STATISTICIAN

Lingyun Ji, PhD

Children's Oncology Group

Statistics and Data Center

222 E. Huntington Drive, #100

Monrovia, CA 91016

Phone: (626) 241-1519

Fax: (626) 445-4334

E-mail: lji@childrensoncologygroup.org

STUDY COMMITTEE MEMBERS

Michael Borowitz, MD PhD

Pathology

Johns Hopkins Univ./Sidney Kimmel Cancer Center

401 N. Broadway, Weinberg 2237

Baltimore, MD. 21231

Phone: (410) 614-2889

Fax: (410) 502-1493

E-mail: mborowit@jhmi.edu

Stephen Hunger, MD

Hematology/Oncology

Children's Hospital of Philadelphia

Colket Translational Research Building

3501 Civic Center Blvd

Room 3060

Philadelphia, PA 19104

Phone: (267) 425-0197

E-mail: hungers@email.chop.edu

STUDY COMMITTEE MEMBERS

Andrew Carroll, PhD.

Cytogenetics

Children's Hospital of Alabama

Department of Genetics

1530 3<sup>rd</sup> Ave. South Kaul Bldg. Rm 314B

Birmingham, AL 35294

Phone: (205) 934-0665

Fax: (205) 934-1078

E-mail: acarroll@uab.edu

M. Brooke Bernhardt, PharmD

Pharmacy

Baylor College of Medicine

1102 Bates St. Suite 1025.17

Houston, TX 77030

Phone: (832) 824-7702

E-mail: mbbernha@txch.org

Kala Kamdar, MD

Hematology/Oncology

Baylor College of Medicine

6621 Fannin St. CC1410.00

Houston, TX 77030

Phone: (832) 824-4163

E-mail: kykamdar@txch.org

Mignon Lee-Cheun Loh, MD

Hematology/Oncology

UCSF Medical Center-Mission Bay

Loh Laboratory

Helen Diller Family Comprehensive Cancer Center

1450 3rd Street, Room 284

San Francisco CA 94158

Phone: (415) 476-3831

Fax: (415) 353-2657

E-mail: mignon.loh@ucsf.edu

Lia Gore MD

Hematology/Oncology

Children's Hospital Colorado

Center for Cancer & Blood Disorders

Pediatrics, Mail Stop 8302

PO Box 6511

Aurora, CO 80045

Phone: (720) 777-4159

Fax: (720) 777-7279

E-mail: lia.gore@ucdenver.edu

13



STUDY COMMITTEE MEMBERS

Jennifer McNeer, MD Hematology/Oncology

University of Chicago Comprehensive Cancer Center

Pediatrics

5841 S. Maryland Ave

MC 4060

Chicago, IL. 60637 Phone: (773) 702-5782 Fax: (773) 702-9881

E-mail: jmcneer@peds.bsd.uchicago.edu

Maureen Megan O'Brien, MD

Hematology/Oncology

Cincinnati Children's Hospital Medical Center

3333 Burnet Avenue

MLC 7015

Cincinnati, OH. 45229 Phone: (513) 803-1678 Fax: (513) 636-3549

E-mail: maureen.obrien@cchmc.org

Michael Pulsipher, MD

Cellular Therapy

Children's Hospital of Los Angeles Blood and Marrow Transplantation

4650 Sunset Blvd, MS#54 Los Angeles, CA 90027 Phone: (323) 361-2546 Fax: (323) 361-8068

E-mail: mpulsipher@chla.usc.edu

Susan Rheingold, MD

Hematology/Oncology

Children's Hospital of Philadelphia

Division of Oncology 34 & Civic Center Blvd. Philadelphia, PA. 19104 Phone: (215) 590-3079 Fax: (215) 590-4183

E-mail: Rheingold@email.chop.edu

Richard Tower, MD MS

Hematology/Oncology

Children's Hospital of Wisconsin Pediatric/Hematology/Oncology/BMT

MACC Fund Research Center 8701 Watertown Plank Road. Milwaukee, WI. 53226

Phone: (414) 955-5653 Fax: (414) 955-6543 E-mail: rtower@mcw.edu Fady Mikhail, MD PhD

Cytogenetics

Children's Hospital of Alabama

Genetics

720 20th Street South, Kaul Bldg. Rm. 314A

Birmingham, AL 35294 Phone: (205) 934-9588 Fax: (205) 934-1078 E-mail: fmikhail@uab.edu

Julie M. Gastier-Foster, PhD.

Laboratory Science

Nationwide Children's Hospital

Laboratory Medicine

700 Children's Drive, CO988A

Columbus, OH. 43205 Phone: (614) 722-2866 Fax: (614) 722-2887

E-mail: Julie.Gastier-Foster@nationwidechildrens.org

Terzah Horton, MD PhD Hematology/Oncology Baylor College of Medicine

Pediatrics

1102 Bates Avenue, Suite 750

Houston, TX. 77030 Phone: (832) 824-4269 Fax: (832) 824-1206 E-mail: tmhorton@txch.org

Stephanie Terezakis, MD.

Radiation Oncology

Johns Hopkins Univ./Sidney Kimmel Cancer Center

Department of Radiation 401 N. Broadway, Ste 1440 Baltimore, MD. 21231 Phone: (443) 287-7889 Fax: (410) 502-1419 E-mail: stereza1@jhmi.edu

Christopher Henchen, BS, CCRP Clinical Research Associates Children's Hospital of Wisconsin 8701 Watertown Plank Road Milwaukee, WI, 53226 Phone: (414) 266-8913 E-mail: chenchen@mcw.edu

e, W1. 53226 114) 955-5653



Meenakshi Devidas, PhD

Statistics

St. Jude Children's Research Hospital Department of Global Pediatric Medicine 262 Danny Thomas Place Mail Stop 721

Memphis, TN 38105 Phone: (904) 595-1764

E-mail: mini.devidas@stjude.org

Sarah Tasian, MD Hematology/Oncology

Children's Hospital of Philadelphia

Division of Oncology 3501 Civic Center Blvd CTRB, 3<sup>rd</sup> Floor Room 3010 Philadelphia, PA 19104 Phone: (267) 425-0118 Fax: (215) 590-3770

Email: tasians@email.chop.edu

Teena Bhatla, MD Hematology/Oncology

Newark Beth Israel Medical Center

201 Lyons Avenue Newark, NJ 07112 Phone: (973) 926-7161 Fax: (973) 282-0395

E-mail: teena.bhatla@rwjbh.org

Debra Marie Schissel, RN CCRP CPON

Nursing

Children's Hospital Colorado Center for Cancer & Blood Disorders 13123 East 16<sup>th</sup> Avenue B115

Aurora, CO 80218 Phone: (720) 777-2879 Fax: (720) 777-7289

Email: Debra.schissel@childrenscolorado.org

Laura Hogan, MD Hematology/Oncology

Stony Brook University Medical Center

**Pediatrics** 

HSC T11-029, Stony Brook, NY 11794

Phone: (631) 444-7720 Fax: (631) 444-2785

E-mail: laura.hogan@stonybrookmedicine.edu

Susan Zupanec, MN NP

Nursing

Hospital for Sick Children 555 University Avenue Toronto, ON M5G1X8 Phone: (416) 813-3488 Fax: (416) 813-5574

E-mail: sue.zupanec@sickkids.ca

## COG RESEARCH COORDINATOR

| AGENT | NSC# | IND# |
|---|---|---|
| Blinatumomab | 765986 | |
| (IND Sponsor: <u>CTEP</u> ) | | |
| Asparaginase E. chrysanthemi | 106977 | Exempt |
| Cyclophosphamide | 26271 | Exempt |
| Cyclosporine | 290193 | Exempt |
| Cytarabine | 63878 | Exempt |
| Dexamethasone | 34521 | Exempt |
| Etoposide | 141540 | Exempt |
| Filgrastim | 614629 | Exempt |
| Fludarabine | 312887 | Exempt |
| Hydrocortisone | 10483 | Exempt |
| Leucovorin | 003590 | Exempt |
| Mercaptopurine | 000755 | Exempt |
| Methotrexate | 000740 | Exempt |
| Mitoxantrone | 301739 | Exempt |
| Mycophenolate Mofetil | 724229 | Exempt |
| Pegaspargase | 624239 | Exempt |
| Tacrolimus | 717865 | Exempt |
| Thioguanine | 00752 | Exempt |
| Thiotepa | 6396 | Exempt |
| Vincristine | 67574 | Exempt |
| | Blinatumomab (IND Sponsor: CTEP) Asparaginase E. chrysanthemi Cyclophosphamide Cyclosporine Cytarabine Dexamethasone Etoposide Filgrastim Fludarabine Hydrocortisone Leucovorin Mercaptopurine Methotrexate Mitoxantrone Mycophenolate Mofetil Pegaspargase Tacrolimus Thioguanine Thiotepa | Blinatumomab 765986 (IND Sponsor: CTEP) 765986 Asparaginase E. chrysanthemi 106977 Cyclophosphamide 26271 Cyclosporine 290193 Cytarabine 63878 Dexamethasone 34521 Etoposide 141540 Filgrastim 614629 Fludarabine 312887 Hydrocortisone 10483 Leucovorin 003590 Mercaptopurine 000755 Methotrexate 000740 Mitoxantrone 301739 Mycophenolate Mofetil 724229 Pegaspargase 624239 Tacrolimus 717865 Thiotepa 6396 |

SEE **SECTION 13.0** FOR SPECIMEN SHIPPING ADDRESSES.



The Children's Oncology Group has received a Certificate of Confidentiality from the federal government, which will help us protect the privacy of our research subjects. The Certificate protects against the involuntary release of information about your subjects collected during the course of our covered studies. The researchers involved in the studies cannot be forced to disclose the identity or any information collected in the study in any legal proceedings at the federal, state, or local level, regardless of whether they are criminal, administrative, or legislative proceedings. However, the subject or the researcher may choose to voluntarily disclose the protected information under certain circumstances. For example, if the subject or his/her guardian requests the release of information in writing, the Certificate does not protect against that voluntary disclosure. Furthermore, federal agencies may review our records under limited circumstances, such as a DHHS request for information for an audit or program evaluation or an FDA request under the Food, Drug and Cosmetics Act. The Certificate of Confidentiality will not protect against mandatory disclosure by the researchers of information on suspected child abuse, reportable communicable diseases, and/or possible threat of harm to self or others.

### **ABSTRACT**

AALL1331 is a group wide risk-stratified, randomized Phase III study to test whether incorporation of blinatumomab into the treatment of patients with childhood B-Lymphoblastic Leukemia (B-ALL) at first relapse will improve disease free survival. Blinatumomab is being tested in this population based on its demonstrated safety profile and single agent activity (induction of MRD-negative remissions in children with multiple relapsed refractory B-ALL).

AALL1331 risk stratification is determined based on site of relapse [marrow versus isolated extramedullary (IEM)], time to relapse and minimal residual disease (MRD) status following a uniform first block of chemotherapy. High risk (HR) and intermediate risk (IR) patients will be eligible for randomization to either a control arm with two additional blocks of chemotherapy, or an experimental arm with two blocks of blinatumomab. Both arms will proceed to protocol-specified hematopoietic stem cell transplant (HSCT) that includes a rapid taper of immune suppression for patients with residual disease and no graft vs. host disease (GVHD). Low risk (LR) patients will be eligible for randomization to either a control arm with two blocks of chemotherapy followed by continuation and maintenance chemotherapy, or an experimental arm with one block of chemotherapy, 2 blocks of blinatumomab, each followed by continuation and a third additional block of blinatumomab followed by maintenance.

AALL1331 includes correlative laboratory studies to refine risk stratification, identify new targets for therapy, identify biomarkers to predict response to chemotherapy and blinatumomab, and to link host polymorphisms with various disease characteristics and toxicities.

Amendment #10 incorporates the High Risk/Intermediate Risk randomization closure as a result of COG DSMC's recommendation based on data that determined the experimental arm with blinatumomab (Arm B) has a significantly more favorable tolerability profile and similar or superior EFS/OS. Effective September 18, 2019, accrual and randomization on the HR/IR arms closed. At completion of Block 1, if patient is found to be HR/IR the patient comes off protocol therapy. HR/IR patients already assigned to Arm A (standard chemotherapy) who are at an appropriate point in their treatment program (prior to receiving Day 22 treatment on Block 3) will be offered the opportunity to cross over to Arm B to receive blinatumomab.







## 1.0 GOALS AND OBJECTIVES (SCIENTIFIC AIMS)

# 1.1 **Primary Aims**

- 1.1.1 To compare disease free survival (DFS) of HR and IR relapse B-ALL patients who are randomized following Induction Block 1 chemotherapy to receive either two intensive chemotherapy blocks or two 5-week blocks of blinatumomab (HR/IR Randomization). (Closed effective September 18, 2019)
- 1.1.2 To compare DFS of LR relapse B-ALL patients who are randomized following Block 1 chemotherapy to receive either chemotherapy alone or chemotherapy plus blinatumomab (LR Randomization).

## 1.2 Secondary Aims

- 1.2.1 To compare overall survival (OS) of HR and IR relapse B-ALL patients who are randomized following Induction Block 1 chemotherapy to receive either two intensive chemotherapy blocks or two 5 week blocks of blinatumomab (HR/IR Randomization). (Closed effective September 18, 2019)
- 1.2.2 To compare OS of LR relapse B-ALL patients who are randomized following Block 1 chemotherapy to receive either chemotherapy alone or chemotherapy plus blinatumomab (LR Randomization).

## 1.3 Exploratory Aims

- 1.3.1 To compare the rates of MRD  $\geq$  0.01% at the end of Block 2 and Block 3 for HR and IR relapse B-ALL patients in HR/IR randomization. (Closed effective September 18, 2019)
- 1.3.2 To estimate, for treatment failure (TF) patients not previously receiving blinatumomab, the hematologic complete remission rate (CR), rate of MRD < 0.01%, and proportion able to proceed to hematopoietic stem cell transplant (HSCT) in CR after treatment with blinatumomab.
- 1.3.3 To assess the feasibility and safety of rapid taper of immune suppression for the subset of HSCT patients with MRD  $\geq$  0.01% pre- and/or post-HSCT with no acute graft versus host disease (aGVHD).
- 1.3.4 To evaluate blinatumomab pharmacokinetics (PK) and explore exposure-response relationships for measures of safety and effectiveness.



### 2.0 BACKGROUND

## 2.1 **Overview**

First relapse of childhood B-ALL is a vexing clinical problem with high rates of subsequent relapse and death with current treatment approaches. This trial will determine if blinatumomab can reduce rates of second relapse, and improve survival. If successful, these interventions could become standard of care for this disease. Additionally, success in relapsed B-ALL will identify interventions that can subsequently be studied in patients with newly diagnosed B-ALL in order to reduce rates of first relapse.

This study also is a paradigm shift away from the non-randomized historical control outcome comparisons pursued in recent COG trials for patients with early relapse of B-ALL (ADVL04P2 and AALL07P1). Those trials were designed to screen promising new agents for possible activity in order to identify which agents should be tested further in more definitive trials. Because of the remarkable efficacy of blinatumomab in adult trials<sup>2</sup> and in the Phase I portion of COG AALL1121,<sup>6</sup> this study will directly test the efficacy of blinatumomab in two risk groups of relapsed B-ALL in a randomized fashion.

This trial also seeks to enhance accrual to relapse childhood ALL trials within COG. Prior to this trial, COG has used a fragmented approach that has required institutions to open a different protocol for each of the many subsets of first relapse ALL. This trial will address this issue by studying first relapse B-ALL in a single, comprehensive protocol.

Importantly, this study will establish an infrastructure for systematic studies of the classification and biology of relapsed childhood B-ALL. Due to the fragmented nature of previous trials and poor accrual, these types of studies have not been possible in the COG until now.

## 2.2 Rationale for Selected Approach and Trial Design

## 2.2.1 Rationale for Consolidated First Relapse B-ALL Trial

This study alters the approach to clinical investigation of relapsed B-ALL in COG. Previous treatment protocols for the 3 major risk groups of first relapse ALL based on duration of 1st complete remission (CR1) and site of relapse (see Table 1) have been separate.

Table 1: Risk groups by duration of CR1, and site of relapse.

| g g y y y | | |
|---|---|---|
| Risk group | CR1 duration and site | Studies |
| Low | ≥ 18 mo isolated extramedullary (Late IEM) | AALL02P2<br>(closed) |
| Intermediate | ≥ 36 mo marrow (Late marrow),<br>< 18 mo isolated extramedullary (Early IEM) | AALL0433<br>(closed) |
| High | < 36 mo marrow (Early marrow),<br>all T-ALL/T-LL relapses | ADVL04P2<br>(completed)<br>AALL07P1 |

The approach for HR patients has been a series of single arm, limited accrual/duration Phase II re-Induction studies of novel agents (epratuzumab for ADVL04P2, bortezomib for AALL07P1) added to the 3-block backbone of chemotherapy established by AALL01P2 (see <u>Table 2</u>) with the primary endpoint being CR2 at end Block 1 as compared to historical control data using the

19



backbone alone. Use of historical control data is problematic for a number of reasons. COG trials for IR and LR patients have each utilized a unique multiagent chemotherapy regimen with or without randomized interventions with a 3-year event free survival (EFS) endpoint.

Table 2: Backbone Chemotherapy for relapse B-ALL

| Block 1 | Block 2 | Block 3 |
|---|---|---|
| PRED 40 mg/m <sup>2</sup> /day, Days 1-29<br>VCR 1.5 mg/m <sup>2</sup> , Days 1, 7, 15, 21<br>PEG 2500 IU/m <sup>2</sup> , Days 2, 9, 16, 23<br>DOXO 60 mg/m <sup>2</sup> , on Day 1<br>IT ARAC Day 1<br>IT MTX Days 15, 29 (or ITT if CNS positive) | ETOP Days 1-5<br>CPM Days 1-5<br>HDMTX Day 22<br>with leucovorin<br>rescue | HD ARAC Days 1, 2, 8, 9<br>L-ASP Days 2, 9<br>IT MTX or ITT Days 1, 22 |

This fragmented approach has been associated with problems in meeting accrual goals and/or completion of studies in a timely and efficient manner. A major obstacle to accrual is the reluctance of COG sites to open all of the relapse studies. Since relapsed ALL is significantly less common than newly diagnosed ALL, the annual accrual to each individual study is expected to be low enough at most COG sites that it may not justify the regulatory burden involved in opening several studies. This is exacerbated for the HR group by the limited accrual/duration of each study, since individual COG sites may be unlikely to enroll any patients during the conduct of such a study. For example, major frontline COG ALL trials are typically open at 190 - 200 sites. In contrast the HR relapse trials have been open in only about 100 sites, and the IR and LR trials at 125 to 150 sites.

We therefore are addressing these issues with a consolidated approach to the classification and initial treatment of first relapse B-ALL, in which all patients are eligible to enroll in a single trial. This approach has been successful in other cooperative groups, including the International Berlin Frankfurt Munster (I-BFM)<sup>8</sup> and United Kingdom Children's Cancer and Leukemia Group (UK CCLG)/Australia/New Zealand<sup>9</sup> consortia.

# 2.2.2 Rationale for Studying Blinatumomab in First Relapse of B-ALL

Survival for first relapse of B-ALL is suboptimal. Blinatumomab is a promising novel agent for the treatment of B-lineage lymphoid malignancies. Blinatumomab is a bispecific single-chain antibody that targets the CD19 antigen and redirects CD3+ T cells for selective lysis of tumor cells. In a Phase II trial of adult B-ALL, patients with MRD persistence or relapse after Induction and Consolidation therapy received blinatumomab as a 4 week continuous intravenous infusion at a dose of 15  $\mu$ g/m²/24 hours. Of 21 treated patients, 16 patients became MRD negative as assessed by quantitative polymerase chain reaction for either rearrangements of immunoglobulin or T-cell receptor genes, or specific genetic aberrations. Among the 16 responders, 12 patients had been molecularly refractory to previous chemotherapy. Probability for relapse-free survival was 78% at a median follow-up of 405 days. Blinatumomab was similarly effective and well tolerated in an anecdotal report of a small series of pediatric cases.  $^2$ 



Blinatumomab is presently being evaluated in children with relapsed/refractory ALL in an Amgen-sponsored Phase I/II study being conducted by COG (MT103-205/AALL1121) and the I-BFM European childhood leukemia cooperative group with extremely promising early results. As of September 2013, 34 patients have been treated in the Phase I portion. Across all dose levels, 11 (32%) patients had CR, 1 (3%) had hypocellular blast-free bone marrow, and 2 (6%) had partial remission within the first two treatment cycles. All patients with CR also experienced molecular remission (MRD level < 10<sup>-4</sup>) after one 4 week block of blinatumomab. 10 The recommended Phase 2 dose for patients with untreated relapse has been determined to be a 4 week continuous IV infusion of 5 µg/m<sup>2</sup>/day for the first week of Cycle 1 and 15 µg/m<sup>2</sup>/day thereafter (i.e. Weeks 2 - 4 of Cycle 1 and Weeks 1 - 4 of all subsequent cycles), with a 2 week break between each cycle. The Phase 2 portion of the study is being conducted at 20 COG and 20 European institutions and began accrual in September 2013. A 2 week rest period between 4 week cycles was selected arbitrarily in early studies of blinatumomab. To preserve the symmetry of timing between arms as much as possible, in AALL1331, a "block" of blinatumomab will be 5 weeks in duration, and will consist of a 4 week continuous infusion followed by a 1 week break. AALL1331 will also use a flat dose of 15 µg/m<sup>2</sup>/day for all blinatumomab cycles except for the first cycle for TF patients (who, like the Phase I/II study patients, will have bulk disease at the time of initiating treatment), where the Phase 2 escalating dosing strategy will be used.

The level of single agent activity seen with blinatumomab has not been seen in recent Phase I ALL studies outside the use of tyrosine kinase inhibitors (TKI) in patients with Philadelphia chromosome positive (Ph<sup>+</sup>) ALL, thus supporting a Phase III randomized clinical trial with DFS endpoints. AALL1331 uses a risk-stratified approach to test whether incorporating blinatumomab into treatment of first relapse B-ALL will reduce rates of second relapse and improve DFS. If successful, inclusion of blinatumomab could become standard of care for this disease. Additionally, success in relapsed B-ALL will provide additional rationale to test blinatumomab in newly diagnosed B-ALL patients in order to reduce rates of first relapse.

As experience with blinatumomab remains relatively limited, this study will include close early monitoring for uncommon but significant adverse events in patients receiving blinatumomab. In addition, the potential for adverse effects from long term depletion of CD19+ normal lymphocytes following blinatumomab treatment is unknown and so monitoring for lymphocyte recovery and for potential adverse effects related to delayed recovery are included.

Neurological adverse events have been described with blinatumomab and will be closely monitored on this study. One potential concern regards the safety of combining blinatumomab with IT chemotherapy. In the current Phase I/II pediatric study cited above, IT methotrexate or IT triples are included prior to Cycle 1, at Day 15 of Cycle 1 and at Day 29 of each cycle. No unusual or increased CNS side effects have been seen in this setting. <sup>10</sup>

Cytokine release syndrome (CRS) has also been described. This is more prevalent in patients with higher leukemia burden, however can occur in any patient treated



with blinatumomab. Pre-medication with dexamethasone is mandated in the protocol, and at the suggestion of the development of CRS, even after the premedication doses, additional dexamethasone administration is suggested. There is a published case report suggesting that for cases of life-threatening cytokine release syndrome for which dexamethasone and supportive care measures are not adequate, consideration may be given to the administration of tocilizumab, the anti-IL-6 monoclonal antibody. 11

## 2.2.3 Rationale for Risk Stratification

Long term survival rates for B-ALL early marrow (15% - 30%) and B-ALL early IEM (30% - 50%) relapses are very poor, and HSCT is generally considered to provide the best chance for cure. This group of patients will be classified as HR and will be eligible to participate in HR/IR randomization upon recovery from Block 1 unless they meet TF criteria (see <u>Table 6</u>).

Late B-ALL marrow relapse patients have excellent end-reinduction CR2 rates (>95%), but long term EFS is suboptimal at about 50 - 60%. For these late B-ALL marrow relapse patients, end-Block 1 MRD has been identified in multiple studies to be a strong prognostic factor. 7,12-14 In AALL01P2, for example, the 5 year EFS for late marrow/MRD-negative patients (< 0.01% by flow at end-Block 1, occurring in about 50% of patients) was 57% vs. 24% for those with MRD  $\geq 0.01\%$ . Thus, AALL1331 will use MRD response to stratify late pre-B marrow relapse patients into those for whom HSCT is or is not indicated. We will use an MRD threshold of 0.1% at end-Block 1 for this HSCT allocation (see Table 3 below). This is based on data from AALL01P2 and the ongoing AALL0433 trial, in which MRD data (end Blocks 1, 2 and 3) have been collected for a large cohort (~150) of late B-ALL marrow relapse patients. The AALL0433 cohort is especially informative since the post-Block 3 therapy given in the context of AALL0433 is uniform (this is not true for AALL01P2). Recent analyses of MRD and outcome from patients enrolled on COG AALL0433 with BM or combined relapse and available end Induction MRD data (n = 175) showed 3 year EFS  $80.2 \pm 5.2\%$  vs.  $40.9 \pm 8.4\%$ , and 3year OS of  $87.1 \pm 4.3\%$  vs.  $56.2 \pm 9.0\%$ for those below (n = 112) or above (n = 63) an MRD cutoff of 0.1%. Thus far, about 62% of late BM relapse patients enrolled in AALL0433 attain MRD < 0.1% by end Block 1. Summarily, for late B-ALL marrow relapse patients, post-Block 1 treatment will be risk-stratified, based on end-Block 1 MRD. MRD analysis will be performed centrally in Dr. Borowitz's laboratory at Johns Hopkins using flow cytometry and a cutoff for MRD positivity of  $\geq 0.1\%$  will be used. Patients with end-Block 1 MRD levels of  $\geq 0.1\%$  will be classified as IR and will be eligible to participate in HR/IR randomization. Those with end-Block 1 MRD levels of < 0.1% will be classified as LR and will be eligible to participate in LR Randomization (see Table 3 below).

For B-ALL IEM relapses, expected outcomes with chemotherapy and radiation for those relapsing at least 18 months from diagnosis are similar to those for late marrow LR patients. It is generally agreed that HSCT is not indicated for B-ALL late IEM relapses. An exception to this will be patients found to have detectable minimal marrow disease at study entry that does not clear to < 0.1% by the end of Block 1, based on published literature that minimal marrow disease in the setting of extramedullary relapse is associated with increased risk of



subsequent marrow relapse.  $^{18,19}$  Thus, B-ALL late IEM relapses that have MRD < 0.1% (or uninterpretable MRD results) at end Block 1 will be classified as LR and will be eligible to participate in LR Randomization. B-ALL late IEM/end Block 1 MRD  $\geq$  0.1% relapses will be classified as IR and will be eligible to participate in HR/IR randomization. Effective September 18, 2019, accrual and randomization on the HR/IR arms closed. With Amendment #10, at completion of Block 1, if patient is found to be HR/IR the patient comes off protocol therapy. HR/IR patients already assigned to Arm A (standard chemotherapy) who are at an appropriate point in their treatment program (prior to receiving Day 22 treatment on Block 3) will be offered the opportunity to cross over to Arm B to receive blinatumomab.

**Table 3: Risk Classification on AALL1331** 

| Risk Group | Definition | Randomization<br>Eligibility | HSCT Treatment |
|---|---|---|---|
| Low | <ul> <li>Late (≥ 36 months) marrow, end-Block 1 MRD &lt; 0.1%</li> <li>Late (≥ 18 months) Isolated extramedullary (IEM), end-Block 1 MRD &lt; 0.1%</li> </ul> | LR<br>Randomization | No HSCT<br>(Treatment includes<br>Continuation and<br>Maintenance) |
| Intermediate | <ul> <li>Late (≥ 36 months) marrow, end-Block 1 MRD ≥ 0.1%</li> <li>Late (≥ 18 months) IEM, end-Block 1 MRD ≥ 0.1%</li> </ul> | HR/IR<br>Randomization | HSCT |
| High | <ul><li>Early (&lt; 36 months)<br/>marrow</li><li>Early (&lt; 18 months) IEM</li></ul> | HR/IR<br>Randomization | HSCT |
| Treatment<br>Failure | Failure to achieve the following at end Block 1: • M2 or better • CNS remission (clearance of CSF blasts, i.e. CNS1) | None (Possible<br>treatment<br>assignment to<br>Salvage<br>Therapy) | HSCT |

# 2.2.4 Rationale for Backbone Chemotherapy Treatment (Blocks 1, 2 and 3)

AALL1331 adopts the chemotherapy used in the recently published international collaborative United Kingdom Medical Research Council ALLR3 study (mitoxantrone arm). These results are the most promising for relapsed childhood ALL published to date, and need to be confirmed using data from the standard arms of this trial. In addition, adopting ALLR3 will pave the way for the international collaboration that we know will be necessary as we begin to test agents targeted to small molecularly-defined subsets of patients (i.e., JAK2 mutant). The first 3 blocks of therapy will serve as the control arm for all patients on this study. These 3 blocks are quite similar to the AALL01P2 Blocks (Table 4).

Table 4: Comparison of AALL01P2 and AALLR3

| COG AALL01P2 | ALLR3 (mitoxantrone arm) |
|---|---|
| VCR 1.5 mg/m <sup>2</sup> , Days 1, 8, 15, 22 | DEX 20 mg/m²/day Days 1-5, 15-19<br>VCR1.5 mg/m² Days 3, 10, 17, 24<br>PEG 1000 IU/m² Day 3 of weeks 1 & 3<br>Mitoxantrone 10 mg/m² Days 1, 2 |



| | IT MTX Days 15, 29 (or ITT if CNS positive) | IT MTX Days 1, 8 (or weekly if CNS positive until 2 clear samples are obtained) |
|---|---|---|
| Block 2 | ETOP 100 mg/m <sup>2</sup> Days 1-5<br>CPM 440 mg/m <sup>2</sup> Days 1-5<br>MTX 5 g/m <sup>2</sup> Day 22<br>IT MTX Days 1, 8 | DEX 6 mg/m²/day Days 1-5<br>VCR 1.5 mg/m² Day 3<br>MTX 1 g/m² Day 8<br>PEG 1000 IU/m² Day 9<br>CPM 440 mg/m² Days 15-19<br>ETOP 100 mg/m² Days 15-19<br>IT MTX Day 8 |
| Block 3 | ARAC 3000 mg/m <sup>2</sup> q12h<br>Days 1, 2, 8, 9<br>L-ASP 6000 IU/m <sup>2</sup> Days 2, 9 | DEX 6 mg/m²/day Days 1-5<br>VCR 1.5 mg/m² Day 3<br>ARAC 3000 mg/m² q12 Days 1, 2, 8, 9<br>Erwinia asparaginase 20,000 IU/m²<br>Days 2, 4, 9, 11, 23<br>MTX 1 g/m² Day 22<br>IT MTX Days 1, 22 |
| CR2 end<br>Block 1 | 96% for IR, 67% for HR (31% for CR1 < 18 mo), 29% for T-ALL | 92% for IR, 58% for HR |
| MRD+<br>end<br>Block 1 | 51% for IR, 75% for HR | 59% for IR, 100% for HR (small numbers) |
| Survival | 12 month EFS: 80% for IR, 35% for HR 3-year EFS: 55% for IR, 15% for HR | 3-year PFS: 65% for mitoxantrone arm (includes HR and IR patients) |

The ALLR3 trial randomized patients to mitoxantrone versus idarubicin in Block 1, and found that the mitoxantrone arm with a 3 year progression free survival (PFS) of 65% was superior to the idarubicin arm in both 3 year PFS (65% vs. 36%, p = 0.0004) and 3 year overall survival (69% vs. 45%, p = 0.004). The major differences between Block 1 in ALLR3 and in the COG AALL01P2 backbone are the replacement of doxorubicin with mitoxantrone and 28 days of prednisone with two 5-day pulses of high-dose dexamethasone. Dexamethasone was used in ALLR3 based on evidence in prior studies of superior CNS activity and survival when compared with prednisone. 20-22 For Block 2, the major differences are the inclusion of a "prophase" week of dexamethasone and vincristine, a lower dose of methotrexate (MTX; 1 g/m<sup>2</sup> vs. 5 g/m<sup>2</sup>), and the inclusion of a dose of PEG asparaginase in combination with MTX. For Block 3, the major differences are the addition of dexamethasone and vincristine to the first week of high dose cytarabine, the addition of intravenous (IV) MTX (1 g/m<sup>2</sup>) and 2 doses of intrathecal (IT) MTX, the use of Erwinia asparaginase instead of E.coli asparaginase and the inclusion of 3 additional doses of Erwinia asparaginase. AALL1331 differs from ALLR3 in several ways:

- AALL1331 administers vincristine beginning on Day 1 of Block 1, rather than beginning on Day 3.
- The pegaspargase preparation utilized in the ALLR3 trial, which is supplied by Medac, differs from that utilized in North America, which is supplied by Sigma Tau. Thus, it is possible that the pharmacokinetics (PK) and/or activity profiles of the pegaspargase preparation utilized in Europe differ from that



used in North America. As the Medac pegaspargase product is not available for use in North America, AALL1331 will use the COG standard dose (2,500 IU/m²) of intravenous Oncospar pegaspargase given on the same schedule utilized in ALLR3. Recent and ongoing COG relapse ALL trials utilize 4 doses of pegaspargase (2,500 IU/m²) given weekly in Block 1, and the most recent and current UKALL 2003/2011 trials and current frontline AIEOP-BFM 2009 ALL trial use 2 doses of pegaspargase during a 4-drug Induction, so this change is expected to be safe.

# 2.2.5 Rationale for Backbone Chemotherapy Treatment (post-Block 3)

One attractive aspect of the post-Block 3 chemotherapy given in the ALLR3 protocol is that it is significantly less intensive than that given to similar patients on the current COG study, AALL0433 (Table 5), affording us an opportunity to decrease short and long term toxicity for relapsed patients with a relatively good prognosis.

**Table 5\* Comparative Cumulative Dosing** 

| Drug | AALL0433 | ALLR3 |
|---|---|---|
| Intravenous methotrexate (IV MTX) | 40 | |
| Cytarabine (ARAC) | 48 | 0.6 |
| Etoposide (ETOP) | 2.4 | 0.6 |
| Cyclophosphamide (CPM) | 10 | 1.2 |
| Vincristine (VCR) | 0.0525 | 0.030 |
| Mercaptopurine (MP) | 18 | 44 |
| Dexamethasone (DEX) | 0.39 | 0.24 |
| Doxorubicin (DOXO) | 0.075 | |
| Pegaspargase (PEG) | 6 doses (2500 IU/m <sup>2</sup> ) | |
| Intrathecal methotrexate (IT MTX) - CNS | 15 doses | 10 doses |
| negative | | |
| Oral Methotrexate (PO MTX) | 1.2 | 1.7 |

<sup>\*</sup>Units are cumulative grams/m<sup>2</sup> of indicated drug unless otherwise indicated.

### 2.2.6 Therapy for CNS3 Patients

The majority of patients with isolated CNS relapse on the ALLR3 trial proceeded to HSCT, so data regarding the efficacy of ALLR3 chemotherapy and radiation alone are lacking. However, Pediatric Oncology Group (POG) studies demonstrated excellent outcomes for late isolated CNS relapse with the incorporation of drugs with both systemic and CNS efficacy (intermediate-dose MTX 1 g/m<sup>2</sup> and high-dose ARAC 3 g/m<sup>2</sup>) and delayed CNS-directed radiation. 16.17 On these trials, coordinated systemic and intrathecal therapy (IT) were given early in therapy to target both the CNS relapse and the high risk for subsequent marrow relapse. On POG 9061, radiation therapy (cranial 24 Gy, spinal 15 Gy) was given after 6 months of intensive chemotherapy and then followed by maintenance chemotherapy, resulting in 84% EFS for late EM relapse patients. The chemotherapy used on POG 9061 was similar to the proposed backbone for this study but included additional CNS-directed therapy. The successor trial, POG 9412, successfully reduced radiation to 18 Gy cranial and eliminated spinal radiation for late CNS relapse patients but included maximal intensity chemotherapy for 12 months prior to radiation. 16



On AALL1331, the backbone described above will be modified to include increased CNS-directed therapy. Throughout therapy, intrathecal triples (ITT) will replace IT MTX. During Block 1, two additional ITT doses will be given. During Block 2, one additional ITT dose will be given. Late B-ALL isolated CNS or late B-ALL CNS3 combined relapse patients with MRD < 0.1% after Block 1 will be LR and eligible for randomization to receive either standard Block 3, Continuation Maintenance Blinatumomab, Continuation/Blinatumomab or Maintenance. We will further intensify CNS-directed therapy for these patients by replacing lower dose oral MTX (25 mg/m<sup>2</sup> every 6 hours x 4 doses) with intermediate-dose IV MTX (1,000 mg/m<sup>2</sup> over 36 hours) during the each of the 2 continuation phases. All of these patients will then receive 1800 cGy cranial radiation and concurrent chemotherapy (including high-dose dexamethasone) between and the first and second 12 week blocks of Maintenance. Radiation will be administered later on the current study (approximately Week 40 for the control arm and Week 54 for the experimental arm) as compared to the ALLR3 trial (Week 14) to maximize delivery of early intensive chemotherapy; this is similar to the timing of radiation in POG 9412 (Week 51).

All other CNS3 relapse patients that meet IR or HR criteria will proceed to total body irradiation (TBI) based HSCT as described in <u>Section 14.5</u>. In addition to the TBI, these patients will also receive a protocol-specified cranial radiation boost as part of their HSCT preparative regimen.

## 2.2.7 <u>Treatment of Testicular Relapse</u>

Although historically testicular irradiation has been used for patients with testicular leukemia at relapse, there are no studies that prove the necessity of this approach. Studies conducted by St. Jude and the European Organization for Research and Treatment of Cancer (EORTC) show that the prognostic significance of overt testicular disease at first diagnosis of ALL has declined on modern treatment protocols. 23,24 The EORTC no longer irradiates any of these patients. 24 The Dutch Childhood Oncology Group has shown that it is possible to effectively treat patients with isolated testicular relapse without radiation. 25,26 The COG has been steadily decreasing the percentage of newly diagnosed and relapsed patients with testicular leukemia that receive testicular irradiation due to the intensified chemotherapeutic regimens and the associated long-term morbidity of testicular irradiation. The findings described above, along with those that show testicular relapses have decreased as chemotherapy regimens for newly diagnosed ALL have intensified, patients with testicular relapse often have detectable disease in the bone marrow, and patients with initial testicular disease usually relapse in the bone marrow, suggest that cure of patients with testicular leukemia is a systemic control problem, not a local control problem. Much of the decrease in testicular relapse has been attributed to intermediate and high-dose MTX. 27-29 Patients will receive intermediate-dose MTX in Blocks 2 and 3 of AALL1331. Since the ALLR3 protocol has shown superior outcomes to previous relapsed leukemia therapies, we believe the improved chemotherapy backbone on this protocol will allow the elimination of testicular irradiation (beyond that which may be used in the HSCT preparative regimen) for those patients that have a complete response of testicular leukemia by end Block 1.



### 2.2.8 <u>Treatment Failure (TF)</u>

Recent COG early marrow relapse ALL studies have defined TF as not achieving M1 marrow by Day 15 of Block 2. In both ALLR3 and in this study, the order of Block 2 chemotherapy differs from that of prior COG studies and non-cross-resistant therapy is not given until Day 15; thus in this study, TF is assessed at the Blocks 1 and 2.

Patients failing to achieve pre-defined response criteria at end-Block 1, end-Block 2/Blinatumomab Cycle 1 (Table 6) will be categorized as having TF (an event). Such patients will be eligible to receive up to 2 blocks of blinatumomab if they had not previously received it on study and do not have residual CNS disease, and will be eligible to continue on study to HSCT if they achieve a CR. Otherwise they will be removed from protocol therapy. Patients who achieve remission at end of Block 1 or Block 2 but are no longer in remission on a subsequent evaluation will be removed from protocol therapy for relapse and will not be eligible to receive blinatumomab. TF is assessed at the end of Blocks 1 and 2.

Table 6: Response criteria required to continue on study

| | Marrow | CNS | Testicular |
|---|---|---|---|
| End-Block 1<br>(All patients) | M2 or<br>better | Remission<br>(clearance of CSF<br>blasts) | None; patients with persistent testicular disease will receive testicular radiation in Block 2 (LR and HR/IR randomized to the control arm) or during Blinatumomab Block: Cycle 1 (HR/IR randomized to the experimental arm) |
| End-Block 2 or End<br>Blinatumomab Block:<br>Cycle 1(HR/IR only) | M1 | Continued remission | Remission (clearance of testicular disease) |

# 2.2.9 Additional non-randomized Pilot Intervention for Very High Risk Subset of HSCT Recipients based on MRD and aGVHD

Relapse rates for patients with relapsed B-ALL who are MRD+ immediately prior to HSCT or are MRD+ in the first 100 days post HSCT are exceedingly high, particularly if there is no aGVHD. Table 7 below shows the relative risk of relapse in the recently closed COG ASCT0431 trial according to MRD (using 0.01% as a threshold) and aGVHD status by Day +55. 33

Table 7 Relapse risk on ASCT0431 per MRD and aGVHD status

| Factor | RR (95% CI) |
|----------------------|------------------|
| Pre-MRD+ vs Pre-MRD- | 1.9 (0.9-4.1) |
| aGVHD Yes vs No | 0.29 (0.12-0.72) |
| Any post-MRD+ | 2.8 (1.2-6.5) |



Patients who were MRD+ pre-HSCT who did not develop acute GVHD and patients with any MRD+ detected after HSCT had a relapse rate of 83%. Given this unacceptably high relapse rate, including a post-HSCT immunological intervention for such patients could potentially address this high relapse rate, and should help standardize post-HSCT interventions and decrease dropout of MRD+ patients prior to HSCT. While the optimal immunological intervention is not known, AALL1331 will include a relatively simple intervention (accelerated taper of immune suppression as detailed in Section 4.9) that is designed to gather additional data to set the stage for more definitive interventions in future trials (e.g. post-HSCT blinatumomab, moxetumomab or other immunotherapy). Trials both in Europe and the US have shown that patients defined as high risk for relapse based upon increasing recipient chimerism (i.e., increased percentage of recipient DNA markers) can successfully undergo withdrawal of immune suppression (IS) without excessive toxicity, and their survival is improved. Out of 46 patients with increasing recipient chimerism (a group at very high risk for relapse), Bader et al intervened in 31 patients with immune suppression (IS) withdrawal, donor lymphocyte infusions (DLI), or both. Three-year EFS was 37% vs. 0% in the intervention vs. non-intervention groups (p < 0.001). $^{34}$  Of the 31 patients, 11 received IS withdrawal alone; 2 relapsed and 1 died of TRM with 8/11 surviving. Three, 2, and 2 patients developed Grades 1, 2, and 3 aGHVD respectively, with no Grade IV or chronic GVHD. A smaller portion of patients responded to DLI (4/17) or a combination of both (1/3). Follow up publications by the Bader group and American groups have shown that patients defined at high risk for relapse by chimerism can safely undergo immune withdrawal with a survival benefit to the patient. 35,36 It is reasonable, therefore, to hypothesize that IS withdrawal may provide benefit, and it is necessary to do this in a standardized manner in the context of this trial. In addition, understanding the proportion of high risk patients who can successfully discontinue IS vital to future trial planning, as many interventions to prevent relapse under consideration require patients to be on no or minimal IS.

# 2.2.10 Rationale for closure of the HR/IR Randomization (Amendment #10)

The DSMC decision was made in the interest of current and future patients despite the monitoring rule for DFS in the AALL1331 protocol not being crossed. The DSMC decision was made based on following four key points:

- The profound difference in toxicity between Arm A chemotherapy and blinatumomab as given on Arm B.
- The DFS and OS results favoring Arm B (blinatumomab) that make it highly likely that Arm B (blinatumomab) has an impact on DFS and OS that is as good as or better than that achieved with the chemotherapy of Arm A.
- The highly significant difference in MRD levels favoring Arm B (blinatumomab) over the chemotherapy of Arm A that support high level anti-leukemia activity for blinatumomab as given on Arm B.
- The comparison of DFS and OS for Arm A and B of the original AALL1331 protocol can still be made with longer follow-up. The original comparison was based on 170 patients. As a result of an amendment to the protocol in 2018, accrual was extended to a target enrollment of 220 patients. The number of patients randomized as of the June 30, 2019 report was 208.



### 3.0 STUDY ENROLLMENT PROCEDURES AND PATIENT ELIGIBILITY

## 3.1 **Study Enrollment**

Note: This study is not on the CTSU Menu (i.e. it is not posted to the CTSU web site) but is supported by the CTSU Regulatory Office, OPEN and Rave.

## 3.1.1 Patient Registration

Prior to enrollment on this study, patients must be assigned a COG patient ID number. This number is obtained via the Patient Registry module in OPEN once authorization for the release of protected health information (PHI) has been obtained. The COG patient ID number is used to identify the patient in all future interactions with COG. If you have problems with the registration, please refer to the online help. For additional help or information, please contact the CTSU Help Desk at 1-888-823-5923 or ctsucontact@westat.com.

In order for an institution to maintain COG membership requirements, every patient with a known or suspected neoplasm needs to be offered participation in APEC14B1, *Project:EveryChild A Registry, Eligibility Screening, Biology and Outcome Study.* 

A Biopathology Center (BPC) number will be assigned as part of the registration process. Each patient will be assigned only one BPC number per COG Patient ID. For additional information about the labeling of specimens please refer to the Pathology and/or Biology Guidelines in this protocol.

Please see <u>Appendix XIII</u> for detailed CTEP Registration Procedures for Investigators and Associates, and Cancer Trials Support Unit (CTSU) Registration Procedures including: how to download site registration documents; requirements for site registration, submission of regulatory documents and how to check your site's registration status.

## 3.1.2 IRB Approval

Each investigator or group of investigators at a clinical site must obtain IRB approval for this protocol and submit IRB approval and supporting documentation to the CTSU Regulatory Office before they can be approved to enroll patients. Assignment of site registration status in the CTSU Regulatory Support System (RSS) uses extensive data to make a determination of whether a site has fulfilled all regulatory criteria including but not limited to the following:

- An active Federal Wide Assurance (FWA) number
- An active roster affiliation with the Lead Network or a participating organization
- A valid IRB approval
- Compliance with all protocol specific requirements.

In addition, the site-protocol Principal Investigator (PI) must meet the following criteria:

- Active registration status
- The IRB number of the site IRB of record listed on their Form FDA 1572
- An active status on a participating roster at the registering site.



For information about the submission of IRB/REB approval documents and other regulatory documents as well as checking the status of study center registration packets, please see <u>Appendix I</u>.

Institutions with patients waiting that are unable to use the Portal should alert the CTSU Regulatory Office immediately at 1-866-651-2878 in order to receive further instruction and support. For general (non-regulatory) questions call the CTSU General Helpdesk at: 1-888-823-5923.

Note: Sites participating on the NCI CIRB initiative and accepting CIRB approval for the study are not required to submit separate IRB approval documentation to the CTSU Regulatory Office for initial, continuing or amendment review. For sites using the CIRB, IRB approval information is received from the CIRB and applied to the RSS in an automated process. Signatory Institutions must submit a Study Specific Worksheet for Local Context (SSW) to the CIRB via IRBManager to indicate their intent to open the study locally. The CIRB's approval of the SSW is then communicated to the CTSU Regulatory Office. In order for the SSW approval to be processed, the Signatory Institution must inform the CTSU which CIRB-approved institutions aligned with the Signatory Institution are participating in the study. Other site registration requirements (i.e., laboratory certifications, protocol-specific training certifications, or modality credentialing) must be submitted to the CTSU Regulatory Office or compliance communicated per protocol instructions.

## 3.1.3 Study Enrollment

Patient enrollment will be facilitated using the Oncology Patient Enrollment Network (OPEN). OPEN is a web-based registration system available on a 24/7 basis. To access OPEN, the site user must have an active CTEP-IAM account (check at <a href="https://ctepcore.nci.nih.gov/iam">https://ctepcore.nci.nih.gov/iam</a>) and a 'Registrar' role on either the lead protocol organization (LPO) or participating organization roster. Registrars must hold a minimum of an AP registration type. If a DTL is required for the study, the registrar(s) must also be assigned the OPEN Registrar task on the DTL.

All site staff will use OPEN to enroll patients to this study. It is integrated with the CTSU Enterprise System for regulatory and roster data and, upon enrollment, initializes the patient position in the Rave database. OPEN can be accessed at <a href="https://open.ctsu.org">https://open.ctsu.org</a> or from the OPEN tab on the CTSU members' side of the website at <a href="https://www.ctsu.org">https://www.ctsu.org</a>. To assign an IVR or NPIVR as the treating, crediting, consenting, drug shipment (IVR only), or investigator receiving a transfer in OPEN, the IVR or NPIVR must list on their Form FDA 1572 in RCR the IRB number used on the site's IRB approval. If a DTL is required for the study, the IVR or NPIVR must also be assigned the appropriate OPEN-related tasks on the DTL.

Prior to accessing OPEN, site staff should verify the following:

- All eligibility criteria have been met within the protocol stated timeframes.
- All patients have signed an appropriate consent form and HIPAA authorization form (if applicable).



Note: The OPEN system will provide the site with a printable confirmation of registration and treatment information. Please print this confirmation for your records.

Further instructional information is provided on the CTSU members' web site OPEN tab or within the OPEN URL (<a href="https://open.ctsu.org">https://open.ctsu.org</a>). For any additional questions contact the CTSU Help Desk at 1-888-823-5923 or <a href="https://open.ctsu.org">ctsucontact@westat.com</a>.

See <u>Section 3.1.6</u> below for details regarding randomization and treatment assignment for patients.

## 3.1.4 <u>Timing</u>

<u>Informed consent</u>: Except for administration of intrathecal chemotherapy (methotrexate strongly preferred) administered at the time of the required diagnostic lumbar puncture to establish baseline CNS status, *informed consent/parental permission* MUST be signed before protocol therapy begins. See <u>Section 3.1.5</u> for summary of time points to obtain informed consent.

Study enrollment: Study enrollment must take place no later than *five* (5) calendar days after beginning protocol therapy. If study enrollment takes place *before* starting protocol therapy, the date that protocol therapy is projected to start must be no later than *five* (5) calendar days after enrollment.

<u>Eligibility studies</u>: Patients must meet all eligibility criteria prior to the start of protocol therapy or enrollment, whichever occurs first. All clinical and laboratory studies to determine eligibility must be performed within 7 days prior to enrollment.

### 3.1.5 Staged Consent

Informed consent will be obtained at critical stages of treatment for the different groups of patients on this study (see summary table below). Informed consent that describes Block 1 therapy (common to all patients on study) will be obtained before starting treatment, with the exception of intrathecal chemotherapy (methotrexate strongly preferred) administered at the time of the required diagnostic lumbar puncture to establish baseline CNS status. At the end of Block 1 therapy, after risk groups have been assigned, subsequent informed consent that describes further therapy will be obtained at the various time points detailed in Table 8 below. Also see Experimental Design Schema

Effective September 18, 2019 the HR/IR randomization closed. Patients who meet criteria for HR/IR randomization should not be approached for post-Induction therapy on AALL1331 and will be removed from protocol therapy at the completion of Block 1.



Table 8: Summary of required consents for AALL1331

| Table 6. Summary of required consents for AALL1331 | | |
|---|---|---|
| Consent Form | Time point to Obtain Consent | Population for<br>Consent |
| Consent 5 – Consent for collection | Before study entry (prior to | All potential |
| of additional marrow | collection of bone marrow) | subjects |
| Consent 1 – Re-induction (block 1) | Study Entry (Prior to shipment | All subjects |
| therapy for all subjects | of bone marrow sample, enrollment, and initiation of | |
| | therapy) | |
| Consent 2: All High-Risk and | Evaluation 1 (prior to HR/IR | HR/IR subjects |
| Intermediate-Risk patients eligible | randomization) | |
| to take part in HR/IR | | |
| randomization | | |
| Closed effective 09/18/2019 | | |
| Consent 3: All lovy right nationts | Evaluation 1 (prior to start of I D | I D subjects |
| • | • | LIX subjects |
| randomization | Tandonnization) | |
| Consent 4: Patients who did not | Prior to start of Salvage | Treatment Failures |
| respond to therapy after Block 1 (all | Therapy (Blinatumomab-S): | (TF) |
| patients) or Block 2 (HR/IR Patients | ●End Block 1 | |
| on Treatment Arm A) | ●End Block 2 | |
| randomization Closed effective 09/18/2019 Consent 3: All low-risk patients eligible to take part in LR randomization Consent 4: Patients who did not respond to therapy after Block 1 (all patients) or Block 2 (HR/IR Patients | Therapy (Blinatumomab-S): ●End Block 1 | |

# 3.1.6 Risk Assignment, Randomization, and Treatment Assignment

• Evaluation 1 (detailed in <u>Section 4.2.7).</u>



\*Exception: 14 days for HR/IR patients with M1 marrow assigned to Arm B



Evaluation 1 must occur <u>no earlier than Day 29 ( $\pm$  1 day)</u>; the evaluation may be delayed until <u>no later than Day 36 ( $\pm$  1 day)</u> if ANC < 500 and/or platelets < 50,000 on Day 29.

Completion of <u>risk group/stratum assignment</u> must occur within <u>5 calendar days</u> of Evaluation 1.

- Step 1: site enters results of local morphologic assessment (marrow/CSF/testes) using Block 1 RP form (form may be saved while incomplete)
- o Step 2: central lab enters marrow flow MRD result using Block 1 MRD form
- Step 3: Study chair confirms risk group/stratum assignment using SC
   Risk Assignment form (using criteria outlined in Section 3.3)

Submission of <u>end-Block 1 callback</u> form must occur within <u>5 calendar days of risk group/stratum assignment.</u>

Components of callback

- 1) Risk group/stratum
- 2) Confirmation that patient does not have severe residual toxicities
- 3) Confirmation that consent has been signed

Upon submission, site receives <u>treatment assignment</u>: Consenting LR patients will be randomized according to LR Randomization; HR/IR patients are not eligible for post-Induction treatment on AALL1331 and are removed from protocol therapy following completion of Block 1; patients deemed Treatment Failure at Evaluation 1 who are eligible for and consent to Salvage Therapy will be assigned to Salvage Therapy.

NOTE: Patients with residual non-heme toxicities that are likely to prevent beginning post-Block 1 treatment within required time frames should NOT submit the End-Block 1 callback.

## 3.1.7 Callbacks

Callback is performed using the Oncology Patient Enrollment Network (OPEN).

| Callback | Timing | Population for<br>Callback | Purpose |
|---|---|---|---|
| End Block 1 | Evaluation 1* | Consenting LR | Randomize LR patients to |
| Callback | | patients not off | either of 2 treatment |
| (ALL | | protocol therapy | arms: |
| patients | | after completion of | <b>Arm C</b> (Control Arm) or |
| continuing to | | Block 1 therapy. | <b>Arm D</b> (Experimental |
| post-Block 1 | | | Arm). |
| therapy) | | | |
| | | Treatment Failure | Assign patients to |
| | | patients who are | Salvage Therapy |
| | | eligible for and | (Blinatumomab-S) |
| | | consent to Salvage | |
| | | Therapy | |

<sup>\*</sup>See Section 3.1.6 for timing details

33



## 3.1.8 Drug Preparation and Administration

Blinatumomab must be prepared in an ISO Class 5 containment device, ideally in an ISO Class 7 room as described in USP <797>, but ISO Class 7 is not required. US sites must attest that their drug preparation and administration guidelines comply with the USP 797. Documentation of participating site training with regard to the preparation and administration of blinatumomab must be submitted via RSS as protocol specific requirement at the time of site activation for participation on the trial.

### 3.1.9 Inclusion of Women and Minorities

Both men and women of all races and ethnic groups are eligible for this study. To allow non-English speaking patients to participate in the study, bilingual health care services will be provided in the appropriate language.

## 3.2 Patient Eligibility Criteria

<u>Important note</u>: The eligibility criteria listed below are interpreted literally and cannot be waived (per COG policy posted 5/11/01). All clinical and laboratory data required for determining eligibility of a patient enrolled on this trial must be available in the patient's medical/research record which will serve as the source document for verification at the time of audit.

All clinical and laboratory studies to determine eligibility must be performed within 7 days prior to enrollment unless otherwise indicated. Laboratory values used to assess eligibility must be no older than seven (7) days at the start of therapy. Laboratory tests need not be repeated if therapy starts within seven (7) days of obtaining labs to assess eligibility. If a post-enrollment lab value is outside the limits of eligibility, or laboratory values are > 7 days old, then the following laboratory evaluations must be re-checked within 48 hours prior to initiating therapy: CBC with differential, bilirubin, ALT (SGPT) and serum creatinine. If the recheck is outside the limits of eligibility, the patient may not receive protocol therapy and will be considered off protocol therapy. Imaging studies, if applicable, must be obtained within 2 weeks prior to start of protocol therapy (repeat the tumor imaging if necessary).

See <u>Section 7.1</u> for required studies to be obtained prior to starting protocol therapy.

# **INCLUSION CRITERIA**

# 3.2.1 Age

Patients  $\ge 1$  year and < 31 years of age at the time of relapse will be eligible.

### 3.2.2 Diagnosis

First relapse of B-ALL, allowable sites of disease include isolated bone marrow, combined bone marrow and CNS and/or testicular, and isolated CNS and/or testicular.



Extramedullary sites are limited to the CNS and testicles. Please refer to Section 3.3 for definitions of relapse and criteria for risk classification.

### 3.2.3 Prior Therapy

Please see <u>Section 4.1.2</u> for the concomitant therapy restrictions for patients during treatment.

- 3.2.3.1 No waiting period for patients who relapse while receiving standard Maintenance therapy
- 3.2.3.2 Patients who relapse on frontline therapy in phases other than Maintenance must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study.
- 3.2.3.3 Cytotoxic therapy: At least 14 days since the completion of cytotoxic therapy with the exception of hydroxyurea, which is permitted up to 24 hours prior to the start of protocol therapy, or Maintenance chemotherapy (see Section 3.2.3.1), or intrathecal chemotherapy (methotrexate strongly preferred) administered at the time of the required diagnostic lumbar puncture to establish baseline CNS status.
- 3.2.3.4 Biologic (anti-neoplastic) agent: At least 7 days since the completion of therapy with a biologic agent. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur.
- 3.2.3.5 Stem cell transplant or rescue: Patient has not had a prior stem cell transplant or rescue.
- 3.2.3.6 Patient has not had prior treatment with blinatumomab.
- 3.2.3.7 With the exception of intrathecal chemotherapy (methotrexate strongly preferred; cytarabine is permissible) administered at the time of the required diagnostic lumbar puncture to establish baseline CNS status, patient has not received prior relapse-directed therapy (i.e., this protocol is intended as the INITIAL treatment of first relapse).

### 3.2.4 Performance Status

Patients must have a performance status corresponding to ECOG scores of 0, 1, or 2. Use Karnofsky for patients > 16 years of age and Lansky for patients ≤ 16 years of age. Please refer to performance status scale at: <a href="https://members.childrensoncologygroup.org/files/protocol/Standard/PerformanceStatusScalesScoring.pdf">https://members.childrensoncologygroup.org/files/protocol/Standard/PerformanceStatusScalesScoring.pdf</a>

# 3.2.5 Organ Function Requirements

3.2.5.1 Adequate Renal Function Defined As:

35



- Creatinine clearance or radioisotope GFR  $\geq 70 \text{ mL/min/1.73 m}^2 \text{ or}$
- A serum creatinine based on age/gender as follows:

| Age | | Maximum Serum<br>Creatinine (mg/dL) |
|------------------|------|-------------------------------------|
| | Male | Female |
| 1 to < 2 years | 0.6 | 0.6 |
| 2 to < 6 years | 0.8 | 0.8 |
| 6 to < 10 years | 1 | 1 |
| 10 to < 13 years | 1.2 | 1.2 |
| 13 to < 16 years | 1.5 | 1.4 |
| ≥ 16 years | 1.7 | 1.4 |

The threshold creatinine values in this Table were derived from the Schwartz formula for estimating GFR utilizing child length and stature data published by the CDC. $^{37}$ 

- 3.2.5.2 Adequate liver function defined as a direct bilirubin < 3.0 mg/dL.
- 3.2.5.3 Adequate Cardiac Function Defined As:
  - Shortening fraction of  $\geq 27\%$  by echocardiogram, or
  - Ejection fraction of  $\geq 50\%$  by radionuclide angiogram.

# 3.2.6 Exclusion Criteria

- 3.2.6.1 Patients with Philadelphia chromosome positive/BCR-ABL1+ ALL are not eligible
- 3.2.6.2 Patients with Burkitt Leukemia/Lymphoma or mature B-cell leukemia are not eligible
- 3.2.6.3 Patients with T-Lymphoblastic Leukemia (T-ALL)/Lymphoblastic Lymphoma (T-LL) are not eligible
- 3.2.6.4 Patients with B-Lymphoblastic Lymphoma (B-LL) are not eligible
- 3.2.6.5 Patients with known optic nerve and/or retinal involvement are not eligible. Patients who are presenting with visual disturbances should have an ophthalmologic exam and, if indicated, an MRI to determine optic nerve or retinal involvement.
- 3.2.6.6 Patients known to have one of the following concomitant genetic syndromes: Down syndrome, Bloom syndrome, ataxia-telangiectasia, Fanconi anemia, Kostmann syndrome, Shwachman syndrome or any other known bone marrow failure syndrome.
- 3.2.6.7 Patients with known HIV infection.
- 3.2.6.8 Patients with known allergy to mitoxantrone, cytarabine, or both etoposide and etoposide phosphate (Etopophos).


- 3.2.6.9 Lactating females who plan to breastfeed.
- 3.2.6.10 Patients who are pregnant since fetal toxicities and teratogenic effects have been noted for several of the study drugs. A pregnancy test is required for female patients of childbearing potential.
- 3.2.6.11 Sexually active patients of reproductive potential who have not agreed to use an effective contraceptive method for the duration of their study participation.

# 3.2.6.12

- a) Patients with pre-existing significant central nervous system pathology that would preclude treatment with blinatumomab, including: history of severe brain injury, dementia, cerebellar disease, organic brain syndrome, psychosis, coordination /movement disorder, or autoimmune disease with CNS involvement are not eligible. Patients with a history of cerebrovascular ischemia/hemorrhage with residual deficits are not eligible. (Patients with a history of cerebrovascular ischemia/hemorrhage remain eligible provided all neurologic deficits have resolved)
- b) Patients with uncontrolled seizure disorder are not eligible. (Patients with seizure disorders that do not require antiepileptic drugs, or are well controlled with stable doses of antiepileptic drugs remain eligible.)

# 3.2.7 Regulatory Requirements

- 3.2.7.1 All patients and/or their parent or legal guardian must sign a written informed consent.
- 3.2.7.2 All institutional, FDA, and NCI requirements for human studies must be met.

#### 3.3 **Definitions**

# Acute Lymphoblastic Leukemia (ALL)

Bone marrow with > 25% L1 or L2 lymphoblasts (M3 marrow). Patients with > 25% L3 marrow lymphoblasts and/or evidence of c-myc translocation are considered to have Burkitt or mature B-cell leukemia and are ineligible for this study.

# **Definitions of Relapse**

- <u>RELAPSE</u>: Any recurrence of disease whether in marrow or extramedullary. For the purposes of eligibility for this trial, extramedullary sites are limited to the CNS and testicles. Relapse should be confirmed by pathology examination of appropriate tissue.
- <u>ISOLATED BONE MARROW RELAPSE</u>: Patients with an M3 marrow at any point after achieving remission without involvement of the CNS and/or testicles. Every effort



should be made to confirm morphologic relapse using flow cytometry, FISH and/or cytogenetics.

- CNS RELAPSE: Positive cytomorphology and WBC ≥ 5/μL OR clinical signs of CNS leukemia such as facial nerve palsy, brain/eye involvement, or hypothalamic syndrome that are, in the opinion of the investigator, more likely due to recurrent CNS leukemia than to alternative causes (e.g., viral infection or chemotherapy toxicity). If any CSF evaluation shows positive cytomorphology and WBC < 5/μL, a second CSF evaluation is recommended within 2 4 weeks. While identification of a leukemic clone in CSF by flow cytometry (TdT, CD19, CD10, etc.) or FISH for diagnostic karyotypic abnormality may be useful, definitive evidence of CNS involvement (i.e. WBC ≥ 5/μL OR clinical signs of CNS leukemia) is required for the diagnosis of a CNS relapse. Note that AALL1331 excludes patients with known optic nerve and/or retinal involvement (Section 3.2.6.5).
- <u>TESTICULAR RELAPSE</u>: Must be documented by testicular biopsy, if not associated with a marrow relapse.
- <u>ISOLATED EXTRAMEDULLARY (IEM) RELAPSE:</u> CNS and/or testicular relapse with an M1 marrow. The presence of MRD in the bone marrow does NOT exclude IEM.
- <u>COMBINED RELAPSE</u>: M2 or M3 marrow at any point after achieving remission with concomitant CNS and/or testicular relapse.

#### **CNS Status:**

<u>NOTE:</u> in this protocol "CNS-positive" means meeting the criteria for CNS Relapse (whether isolated CNS or combined relapse) at the time of AALL1331 study entry as listed in the Definitions of Relapse above. CNS 2 status first noted at the time of enrollment for concurrent relapse at another site (i.e. bone marrow) will not be considered 'CNS-positive'.

| CNS 1: | In cerebral spinal fluid (CSF), absence of blasts on cytospin preparation, | , |
|---|---|---|
| | magandless of the number of white blood calls (WDCs) | |

regardless of the number of white blood cells (WBCs).

CNS 2: In CSF, presence  $< 5/\mu$ L WBCs and cytospin positive for blasts, or  $\ge 5/\mu$ L

WBCs but negative by Steinherz/Bleyer algorithm:

CNS 2a:  $< 10/\mu L$  RBCs;  $< 5/\mu L$  WBCs and cytospin positive for blasts;

CNS 2b:  $\geq 10/\mu L$  RBCs;  $< 5/\mu L$  WBCs and cytospin positive for blasts; and

CNS 2c: > 10/µL RBCs; > 5/µL WBCs and cytospin positive for blasts but negative

by Steinherz/Bleyer algorithm (see below).

CNS3: In CSF, presence of  $\geq 5/\mu L$  WBCs and cytospin positive for blasts and/or

clinical signs of CNS leukemia:

CNS 3a:  $< 10/\mu L RBCs; \ge 5/\mu L WBCs$  and cytospin positive for blasts;

CNS 3b:  $\geq 10/\mu L$  RBCs,  $\geq 5/\mu L$  WBCs and positive by Steinherz/Bleyer algorithm

(see below);

CNS 3c: Clinical signs of CNS leukemia (such as facial nerve palsy, brain/eye

involvement or hypothalamic syndrome).



### Method of Evaluating Initial Traumatic Lumbar Punctures:

If the patient has leukemic cells in the peripheral blood and the lumbar puncture is traumatic and contains  $\geq 5$  WBC/ $\mu$ L and blasts, the following algorithm should be used to distinguish between CNS 2 and CNS 3 disease:

A patient with CSF WBC  $\geq$  5/ $\mu$ L blasts, whose CSF WBC/RBC is 2X greater than the blood WBC/RBC ratio, has CNS disease at diagnosis. Example: CSF WBC =  $60/\mu$ L; CSF RBC =  $1500/\mu$ L; blood WBC =  $46000/\mu$ L; blood RBC =  $3.0 \times 10^6/\mu$ L:

$$\frac{60}{1,500} = 0.04 > 2X \quad \frac{46,000}{3.0 \times 10^6} = 0.015$$

# **Bone Marrow Status:**

M1 Marrow: < 5% blasts in a bone marrow aspirate with at least 200 cells counted.

M2 Marrow: 5% - 25% blasts in a bone marrow aspirate with at least 200 cells counted.

M3 Marrow: > 25% blasts in a bone marrow aspirate with at least 200 cells counted.

For **initial remission** an M1 marrow must be achieved.

**Treatment Failure:** Failure to achieve the following:

| | Marrow | CNS | Testicular |
|---|---|---|---|
| End-Block 1 (All patients) | M2 or better | Remission<br>(clearance of CSF<br>blasts, i.e. CNS1) | None; patients with persistent testicular disease will receive testicular radiation in Block 2 (LR and HR/IR randomized to the control arm) or during Blinatumomab Block: Cycle 1 (HR/IR randomized to the experimental arm) |
| End-Block 2, or<br>End Blinatumomab<br>Block, Cycle 1<br>(HR/IR only) | M1 | Continued remission | Remission (clearance of testicular disease) |

**NOTE:** Patients who achieve remission (M1 marrow and clearance of extramedullary disease) at end-Block 1 or Block 2 but are no longer in remission on a subsequent evaluation will be removed from protocol therapy for relapse.

#### **Risk Assessment-End Block 1\*:**

#### Low Risk

- Late marrow ( $\geq$  36 months), end-Block 1 MRD < 0.1%
- Late (≥ 18 months) Isolated Extramedullary (IEM), end-Block 1 MRD < 0.1% (or indeterminate MRD)



# Intermediate Risk

- Late ( $\geq$  36 months) marrow, end-Block 1 MRD  $\geq$  0.1%
- Late ( $\geq$  18 months) IEM, end-Block 1 MRD  $\geq$  0.1%

# High Risk

- Early (< 36 months) marrow
- Early (< 18 months) IEM
- \* The timing of relapse (duration of first remission) is measured from the date of initial diagnosis to the date of relapse.

# **Complete Remission**

Complete remission (CR) is defined as an M1 marrow (< 5% blasts) with no evidence of circulating blasts or extramedullary disease and with peripheral count recovery, defined as absolute neutrophil count higher than or equal to  $500/\mu L$  and platelet count higher than or equal to  $50,000/\mu L$ .



#### 4.0 TREATMENT PLAN

Timing of protocol therapy administration, response assessment studies, and surgical interventions are based on schedules derived from the experimental design or on established standards of care. Minor unavoidable departures (up to 72 hours) from protocol directed therapy and/or disease evaluations (and up to 1 week for surgery) for valid clinical, patient and family logistical, or facility, procedure and/or anesthesia scheduling issues are acceptable per COG administrative Policy 5.14 (except where explicitly prohibited within the protocol).

# 4.1 **Overview of Treatment Plan**

All eligible patients with first relapse B-ALL who are enrolled on AALL1331 will receive standard chemotherapy during Block 1. All patients will then be risk assessed at the end of Block 1 as either HR, IR, LR or TF. Risk assessment is based on site of relapse, time to relapse, end Block 1 bone marrow morphology and MRD levels. Effective September 18, 2019, HR and IR patients are no longer eligible for post-Induction therapy on AALL1331 due to closure of the HR/IR randomization and will be removed from protocol therapy following completion of Block 1. LR patients will be eligible to participate in LR Randomization. See summary table below. Treatment failures are those patients whose disease status fails to meet pre-defined response criteria at end-Block 1 or end-Block 2. These patients are eligible to receive up to 2 blocks of blinatumomab if they have not previously received it on study and have no evidence of persistent CNS disease. These patients will also be eligible to continue on to HSCT if they achieve a CR. Otherwise, they will be removed from protocol therapy. See Section 3.3 for response definitions of TF CR.

Risk Stratification at end Block 1

| | Definition | Randomization | Treatment Arms |
|---|---|---|---|
| Risk Group | Definition | Eligibility | |
| High | <ul><li>Early (&lt; 36 months) marrow</li><li>Early (&lt; 18 months) IEM</li></ul> | HR/IR<br><i>Closed 09/18/2019</i> | <ul><li>Arm A (Control)</li><li>Arm B (Experimental)</li></ul> |
| Intermediate | <ul> <li>Late (≥ 36 months) marrow, end-Block 1 MRD ≥ 0.1%</li> <li>Late (≥ 18 months) IEM, end-Block 1 MRD ≥ 0.1%</li> </ul> | HR/IR<br>Closed 09/18/2019 | Arm A (Control) Arm B (Experimental) |
| Low | <ul> <li>Late (≥ 36 months) marrow, end-Block 1 MRD &lt; 0.1%</li> <li>Late (≥ 18 months) IEM, End-Block 1 MRD &lt; 0.1%</li> </ul> | LR | Arm C (Control) Arm D (Experimental) |
| Treatment Failure at end Block 1 | Failure to achieve the following: • M2 or better • CNS remission (clearance of CSF blasts, i.e. CNS1) | None (treatment assignment) | Salvage therapy (Blinatumomab-S) |

# **CNS Leukemia**

All patients with CNS3 involvement at the time of relapse will receive intrathecal triples (ITT) instead of IT MTX beginning on Day 8. During Block 1 these patients will receive two additional ITT doses (Days 15 and 22) and during Block 2 they will receive one additional ITT dose (Day 22). For LR patients with CNS3 involvement, AALL1331 will



further intensify CNS-directed therapy by replacing lower dose oral MTX (25 mg/m² every 6 hours x 4 doses) with intermediate dose IV MTX (1 g/m² over 24 hours) during the each of the 2 continuation phases. All of these patients will then receive 1800 cGy cranial radiation and concurrent chemotherapy (including high dose dexamethasone) between and the first and second 12 week blocks of Maintenance. IR and HR patients will proceed to TBI-based HSCT and these patients will also receive a protocol-specified cranial radiation boost as part of their HSCT preparative regimen.

### **Testicular Leukemia**

Patients with suspected isolated testicular relapse or equivocal testicular enlargement with concurrent bone marrow/CNS relapse must have a testicular biopsy performed at baseline. Patients with persistent or equivocal testicular enlargement at the end of Block 1 must have a testicular biopsy. Patients with persistent testicular leukemia at the end of Block 1 are eligible to continue on study and will receive 2400 cGy of testicular radiation during either Block 2 chemotherapy (for LR patients and HR/IR patients randomized to the control arm) or during blinatumomab (for HR/IR patients randomized to the experimental arm and TF.) Patients with extramedullary testicular leukemia that has resolved by end Block 1 will NOT receive testicular irradiation, with the exception of that which may be used in the HSCT preparative regimen for HR/IR patients.

#### **HSCT**

All patients enrolled on this protocol, their parents and full siblings should undergo HLA tissue typing as soon as possible after diagnosis of relapse, and should have transplantation consultation and initiation of a donor search. For HR/IR patients, and for TF patients who achieve CR with Salvage Therapy (Blinatumomab-S), the goal of this protocol is to move to transplant within 2 weeks of recovery from the last block/cycle of therapy prior to transplant. Because unrelated donor acquisition can take 8 - 12 weeks, centers must expedite the donor search process to meet this deadline.

# Patient Pill Diary

It is recommended that patients use a Patient Pill Diary to keep track of oral medications.

# 4.1.1 TREATMENT ASSIGNMENTS

# **IMPORTANT NOTE:**

In order to continue to receive protocol therapy, patients will need to begin post-Block 1 therapy within a specified time frame (see Section 4.2.7). If a patient has residual severe non-hematologic toxicities from Block 1 that are likely to preclude beginning post-Block 1 therapy within this time frame, please DO NOT complete end-Block 1 Callback for the patient. This is important to minimize the number of patients who are randomized/assigned but are unable to receive post-callback treatment.

#### 4.1.1.1 HR/IR Randomization

Effective 09/18/2019, HR/IR patients are not eligible for post-Induction therapy on AALL1331 and will be removed from protocol therapy. Patients receiving therapy on Arm A prior to Amendment #10 who have not yet received Day 22 treatment on Block 3 will be offered the opportunity to cross over to Arm B to receive blinatumomab.



- **Arm A (Control Arm)**: Patients receive Block 2 and Block 3 of standard therapy followed by HSCT. *Closed effective September 18, 2019.*
- **Arm B (Experimental Arm)**: Patients receive two 5 week blocks of Blinatumomab, followed by HSCT.

# 4.1.1.2 LR Randomization

Following submission of the end-Block 1 callback form LR patients will be randomized to receive treatment on either of 2 treatment arms (see Experimental Design Schema and Section 3.1.6):

- Arm C (Control): Patients receive Block 2 and Block 3 of standard therapy followed by Continuation 1, Continuation 2, and Maintenance.
- **Arm D (Experimental)**: Patients receive Block 2 of standard therapy followed by a 5 week Blinatumomab Block, Continuation 1, a 5 week Blinatumomab Block, Continuation 2, a 5 week Blinatumomab Block, and Maintenance.

# 4.1.1.3 Salvage Therapy (Blinatumomab-S)

Following submission of the end-Block 1 or End-Block 2 callback form, eligible Treatment Failure patients will be assigned to Salvage Therapy (see Experimental Design Schema and Section 3.1.6).

# 4.1.2 Concomitant Therapy Restrictions

#### 4.1.2.1 Cytochrome P450 Interactions with Antileukemic Drugs.

Since concurrent use of enzyme inducing anticonvulsants (e.g., phenytoin, phenobarbital, and carbamazepine) with anti-leukemic therapy has recently been associated with inferior EFS, every effort should be made to avoid these agents, as well as rifampin, which also induces many drug metabolizing enzymes. Neither gabapentin nor levetiracetam induce hepatic drug metabolizing enzymes and may be suitable alternative anticonvulsants. Azole antifungals (listed in the table below) and the macrolide group of antibiotics (listed in the table below) may have potent inhibitory effects on drug-metabolizing enzymes. Patients receiving some anti-leukemic drugs (e.g., vincristine, anthracyclines, etoposide) may experience excess toxicity when these agents are given concomitantly; alternate antifungal and antibacterial therapy should be used where possible (see table below).

| DRUGS | POTENTIAL | ACTION TO BE TAKEN |
|-----------------|----------------------|------------------------------|
| | INTERACTION | |
| Anticonvulsants | Induction of drug | AVOID phenytoin, |
| | metabolizing enzymes | phenobarbital, carbamazepine |
| | Lowered EFS | Consider gabapentin or |
| | | levetiracetam as alternative |
| Rifampin | Induction of drug | DO NOT USE |
| | metabolizing enzymes | |



| Azole Antifungals (fluconazole, itraconazole*, posaconazole voriconazole, ketoconazole) | Inhibition of drug<br>metabolizing enzymes | CONSIDER ALTERNATIVE MEDICATIONS May need dose reductions of vincristine*, anthracyclines, etoposide, steroids |
|---|---|---|
| Macrolide Antibiotics<br>(erythromycin,<br>clarithromycin,<br>azithromycin,<br>roxithromycin,<br>telithromycin) | Inhibition of drug<br>metabolizing enzymes | CONSIDER ALTERNATIVE MEDICATIONS May need dose reductions of vincristine, anthracyclines, etoposide, steroids |

<sup>\*</sup> Itraconazole should NOT be used in patients who are receiving vincristine due to a serious drug-drug interaction leading to severe neurotoxicity. 39.40

This is not an inclusive list. Because the lists of these agents are constantly changing, it is important to regularly consult frequently updated medical references.

# 4.1.2.2 Possible Drug Interactions with Intermediate Dose Methotrexate:

Avoid non-steroidal anti-inflammatory drugs (NSAIDs), trimethoprim/sulfamethoxazole (TMP/SMX), penicillins, probenecid, IV contrast media, proton pump inhibitors, phenytoin and fosphenytoin. Urinary acidifiers can cause methotrexate to precipitate in the urinary tract.

For COG Supportive Care Guidelines see <a href="https://cogmembers.org/\_files/disc/Pharmacy/ChemoAdminGuidelines.p">https://cogmembers.org/\_files/disc/Pharmacy/ChemoAdminGuidelines.p</a> df

# 4.1.3 Supportive Care for Patients 15 Years and Older

It is recommended that adolescent and young adult (AYA) patients enrolled on this protocol (defined as patients between the ages of 15 and 31 years) be monitored in the hospital during Block 1, Block 2 and Block 3 of chemotherapy until they show signs of bone marrow recovery (specifically until they show evidence that the absolute neutrophil count (ANC) is rising for 2 successive days) and the patient is afebrile and clinically stable. If a patient should experience profound myelosuppression at any other time, there should also be a very low threshold to hospitalize AYA patients, and to continue inpatient management until there is evidence of bone marrow recovery. Antibiotic prophylaxis against Gram-positive and Gram-negative organisms (e.g. levofloxacin) may be considered during these hospitalizations until patients meet the criteria for discharge. If the patient should develop febrile neutropenia while on antibiotic prophylaxis, the patient should be broad-spectrum intravenous antibiotics per guidelines. Antifungal prophylaxis may also be considered during periods of myelosuppression. Options include an echinocandin such as caspofungin or micafungin, or an azole. Azole antifungal agents (i.e., fluconazole, itraconazole, posaconazol, voriconazole) given concurrently with vincristine may increase the risk of neurotoxicity. Investigator caution is advised if azole antifungals are used. If antibiotic and/or antifungal prophylaxis is utilized, consultation with Infectious Disease may be considered.



# 4.2 Block 1 (All patients) - 4 Weeks Duration

Block 1 therapy is common to all patients on study. See <u>Experimental Design Schema</u>. The therapy delivery map (TDM) for Block 1 is in <u>APPENDIX II-A</u>.

NOTE: The risks of significant morbidity and mortality, including sudden death in patients with relapsed leukemia, are sufficient to strongly recommend hospitalization during remission Induction, until patients show consistent neutrophil recovery and transfusion needs that are deemed to be manageable in the outpatient setting. Please see <a href="#">Appendix I</a> for additional details.

#### 4.2.1 Disease Evaluation Pre-Treatment

See Section 7.0, Evaluations/Material and Data to be Accessioned

# 4.2.2 General Chemotherapy Guidelines

See Section 6.0, Drug Information, and the Parenteral and Oral Chemotherapy Administration Guidelines (CAGs) on the COG website at: <a href="https://members.childrensoncologygroup.org/files/disc/Pharmacy/ChemoAdminGuidelines.pdf">https://members.childrensoncologygroup.org/files/disc/Pharmacy/ChemoAdminGuidelines.pdf</a> for special precautions associated with chemotherapy administration. As applicable, also see the CAGs for suggestions on hydration, or hydrate according to institutional guidelines.

See <u>Section 5.0</u> for Dose Modifications based on Toxicities and <u>Appendix I</u> for Supportive Care Guidelines.

#### Dosing should be based on actual BSA.

#### 4.2.3 Block 1 Chemotherapy

# Dexamethasone: PO (may be given IV)

Days: 1 - 5, 15 - 19

Dose: 10 mg/m²/dose (Total daily dose: 20 mg/m²/day, divided BID; dose capped

at 40 mg per day)

If using tablets, adjust dose upward to the nearest 0.25 mg. Oral solutions are acceptable and intravenous preparations may be used on a temporary

basis, if needed.

# <u>VinCRIStine:</u> IV push over 1 minute or infusion via minibag as per institutional policy

Days: 1, 8, 15, 22

Dose: 1.5 mg/m<sup>2</sup>/dose (maximum dose: 2 mg)

# Special precautions: FOR INTRAVENOUS USE ONLY.

The container or the syringe containing vinCRIStine must be enclosed in an overwrap bearing the statement "Do not remove covering until moment of injection. For intravenous use only - Fatal if given by other routes."

Medication errors have occurred due to confusion between vinCRIStine and vinBLAStine. VinCRIStine is available in a liposomal formulation (vinCRIStine sulfate liposomal injection, VSLI, Marqibo®). Use conventional vinCRIStine only; the conventional and liposomal formulations are NOT interchangeable.



# Pegaspargase: IV over 1 - 2 hours

Days: 3, 17

Dose: 2,500 International Units/m²/dose

Administer through the tubing of a rapidly infusing solution of D<sub>5</sub>W or

0.9% NaCl

# **Special precautions:**

- 1. Pegaspargase is contraindicated with a history of severe pancreatitis with any prior asparaginase therapy. Caution should be used if serious thrombosis or hemorrhagic events have occurred with any prior asparaginase therapy (see Section 5.1)
- 2. Pegaspargase may affect coagulation factors and predispose to bleeding and/or thrombosis. Caution should be used when administering any concurrent anticoagulant therapy.
- 3. Suggested monitoring during and after administration: Because pegaspargase is long acting, hypersensitivity reactions may not appear for hours after drug administration. Monitor vital signs, for signs of fever, chills, or acute allergic reactions including anaphylaxis. Have medications to treat hypersensitivity reactions readily available at each administration (e.g., epinephrine, IV corticosteroids, antihistamines). Consider prescribing an EpiPen® for home use.

MitoXANTRONE: IV over 15 - 30 minutes, administered through the tubing of a rapidly infusing solution of D<sub>5</sub>W or 0.9% NaCl.

Days: 1, 2 Dose: 10 mg/m<sup>2</sup>

# **Methotrexate: Intrathecal (IT) - ALL PATIENTS**

Days: 1

Note: If intrathecal chemotherapy (methotrexate strongly preferred; cytarabine permissible) was given at the time of the diagnostic lumbar puncture, and if the treatment was given less than 7 days prior to the beginning of Day 1 systemic therapy, then the Day 1 IT treatment can be omitted at the discretion of the investigator. Otherwise, Day 1 intrathecal methotrexate must be given.

# Age-based dosing:

| Age (yrs) | Dose (mg) |
|-----------|-----------|
| 1 - 1.99 | 8 |
| 2 - 2.99 | 10 |
| 3 - 8.99 | 12 |
| ≥ 9 | 15 |

# Methotrexate: Intrathecal (IT) - CNS 1/2 PATIENTS ONLY

Days: 8

Note: For CNS2 patients continue weekly IT until 2 clear CSF samples (CNS1) are obtained.



#### Age-based dosing:

| Age (yrs) | Dose (mg) |
|-----------|-----------|
| 1 - 1.99 | 8 |
| 2 - 2.99 | 10 |
| 3 - 8.99 | 12 |
| $\geq$ 9 | 15 |

# <u>Intrathecal Triple Therapy (ITT)</u> - ANY PATIENT WITH CNS3 AT THE TIME OF RELAPSE

Days 8, 15, and 22.

# Age-based dosing:

| Age (yrs) | Dose (mg) | | |
|-----------|-----------|--------|----------|
| 1 - 1.99 | MTX: 8 | HC: 8 | ARAC: 16 |
| 2 - 2.99 | MTX: 10 | HC: 10 | ARAC: 20 |
| 3 - 8.99 | MTX: 12 | HC: 12 | ARAC: 24 |
| > 9 | MTX: 15 | HC: 15 | ARAC: 30 |

#### 4.2.4 Disease Evaluation End Block 1

- The end-Induction evaluation should occur no earlier than Day 29 ( $\pm$  1 day).
- The evaluation may be delayed no later than Day 36 ( $\pm$  1 day) if ANC <  $500/\mu$ L and platelets <  $50,000/\mu$ L on Day 29.
- The evaluation includes a bone marrow aspirate for all patients, a diagnostic lumbar puncture should be performed for CNS2 or CNS3 patients for whom clearance of CSF blasts has not yet been documented, and a testicular biopsy for patients with definite or equivocal residual testiculomegaly at end of Block 1.
- See <u>Sections 7.1</u> and <u>13.0</u> for details on specimen acquisition, handling and shipping.

#### 4.2.5 Research Studies Block 1

See Section 7.2 for a full list of research studies.

# 4.2.6 HLA Tissue Typing for Hematopoietic Stem Cell Transplant

All patients enrolled on this protocol, their parents and full siblings should undergo HLA tissue typing as soon as possible after diagnosis of relapse, and should have transplantation consultation and initiation of a donor search. The goal of this protocol is to initiate transplantation within 2 weeks of recovery from Block 3. Since unrelated donor acquisition can take 8 - 12 weeks, centers must expedite the search process to meet this timeframe.

# 4.2.7 Evaluation 1 (Risk Assessment following Block 1)

Following completion of Block 1, patients will be risk assessed based on end-Block 1 criteria outlined in <u>Section 3.3</u>, and according to procedures in <u>Section 3.1.6</u>, as HR, IR, LR, or TF.



# **IMPORTANT NOTE:**

In order to continue to receive protocol therapy, patients will need to begin post-Block 1 therapy within a specified time frame (see below). If a patient has residual severe non-hematologic toxicities from Block 1 that are likely to preclude beginning post-Block 1 therapy within this time frame, please DO NOT complete end-Block 1 Callback for the patient. This is important to minimize the number of patients who are randomized/assigned but are unable to receive post-callback treatment.

Post-Block 1 treatment should begin after submission of end-Block 1 Callback and receipt of treatment assignment as soon as clinically acceptable to the treating institution. Patients should have time for full or partial recovery (judged by the treating institution) from any toxicities experienced in the prior course(s) of therapy before proceeding to the next course. However, treatment must begin according to time frames below for patients to continue to receive protocol therapy.

#### HR B-ALL or IR B-ALL patients

Effective 09/18/2019, HR/IR patients are not eligible for post-Induction therapy on AALL1331 and will be removed from protocol therapy.

# LR B-ALL Eligible for the LR Randomization

• All LR B-ALL patients (**Arm C and Arm D**) will receive Block 2 therapy (<u>Section 4.3</u>, <u>APPENDIX II-B</u>) and should proceed with Day 1 vincristine and dexamethasone without awaiting count recovery (no later than 5 calendar days after callback). It is recommended, but not required, that proceeding with Day 8 IV methotrexate treatment await count recovery to ANC ≥ 500/μL and platelets ≥ 50,000/μL. Day 8 treatment must begin no later than <u>14 calendar days</u> after giving the Day 1 vincristine and dexamethasone to continue to receive protocol therapy.

**Treatment failures Post-Block 1** (see Section 3.3 for definition) have the option to receive up to two 5 week cycles of Blinatumomab (Sections 4.7, 4.8 and APPENDIX II-F, and II-G respectively) and continue on to HSCT after achieving CR.

- TF patients with residual CNS disease (CNS2/3) regardless of marrow status should be <u>removed from protocol therapy</u>.
- TF patients with M3 marrow disease and <u>no</u> residual CNS disease (CNS1) should proceed to <u>Blinatumomab-S Cycle 1</u> without awaiting count recovery (no later than <u>5 calendar days</u> after callback).

<u>NOTE</u>: If residual non-hematologic toxicities prevent a patient from beginning post Block-1 treatment within the time frames noted above, then the patient should be removed from protocol therapy.



# 4.3 Block 2 (LR Patients: Post-randomization) – 4 weeks duration

Block 2 therapy is for all LR patients post LR randomization (**Arm C and Arm D**). See Experimental Design Schema.

The Therapy Delivery Map (TDM) for Block 2 is in APPENDIX II-B.

END-BLOCK 1 CALLBACK OCCURS PRIOR TO STARTING BLOCK 2 THERAPY. PLEASE SEE SUMMARY TABLE IN <u>SECTION 3.1.5</u> FOR DETAILS ON STAGED CONSENT, AND APPROPRIATE TIMING TO OBTAIN INFORMED CONSENT.

# 4.3.1 Criteria to Begin Block 2 Therapy

Block 2 should begin after submission of the appropriate end-Block 1 Callback and receipt of treatment assignment as soon as clinically acceptable to the treating institution. Patients should have time for full or partial recovery (judged by the treating institution) from any toxicities experienced in the prior course(s) of therapy before proceeding to the next course. To continue to receive protocol therapy, however, Block 2 must begin no later than 5 calendar days after callback. Count recovery is not required to proceed to Block 2.

# 4.3.2 <u>Testicular Radiation Therapy (TRT)</u>

Patients with persistent testicular leukemia at the end of Block 1 are eligible to continue on study and will receive 2400 cGy of testicular radiation during either Block 2 chemotherapy (all LR patients) or during the first cycle of Blinatumomab (for HR/IR patients).

- Patients with extramedullary testicular leukemia that has resolved by end Block 1 will NOT receive testicular irradiation with the exception of that which may be used in the HSCT preparative regimen.
- See Section 14.2 for detailed testicular radiation guidelines

# 4.3.3 General Chemotherapy Guidelines

See Section 6.0, Drug Information, and the Parenteral and Oral Chemotherapy Administration Guidelines (CAGs) on the COG website at: <a href="https://members.childrensoncologygroup.org/files/disc/Pharmacy/ChemoAdminGuidelines.pdf">https://members.childrensoncologygroup.org/files/disc/Pharmacy/ChemoAdminGuidelines.pdf</a> for special precautions associated with chemotherapy administration. As applicable, also see the CAGs for suggestions on hydration, or hydrate according to institutional guidelines.

See Section 5.0 for Dose Modifications based on Toxicities and Appendix I for Supportive Care Guidelines.

Dosing should be based on actual BSA.



#### 4.3.4 Block 2 Chemotherapy

# **Dexamethasone:** PO (may be given IV)

Days: 1-5

Dose: 3 mg/m<sup>2</sup>/dose (Total daily dose: 6 mg/m<sup>2</sup>/day, divided BID)

If using tablets, adjust dose upward to the nearest 0.25 mg. Oral solutions are acceptable and intravenous preparations may be used on a temporary

basis, if needed.

# <u>VinCRIStine:</u> IV push over 1 minute or infusion via minibag as per institutional policy

Day: 1

Dose: 1.5 mg/m<sup>2</sup>/dose (maximum dose: 2 mg)

# Special precautions: FOR INTRAVENOUS USE ONLY.

The container or the syringe containing vinCRIStine must be enclosed in an overwrap bearing the statement "Do not remove covering until moment of injection. For intravenous use only - Fatal if given by other routes."

Medication errors have occurred due to confusion between vinCRIStine and vinBLAStine. VinCRIStine is available in a liposomal formulation (vinCRIStine sulfate liposomal injection, VSLI, Marqibo®). Use conventional vinCRIStine only; the conventional and liposomal formulations are NOT interchangeable.

# Intermediate Dose Methotrexate (ID MTX): IV over 36 hours

Day: 8

Dose:  $1,000 \text{ mg/m}^2/\text{dose}$ 

Given as a 100 mg/m<sup>2</sup> bolus over 30 minutes followed by 900 mg/m<sup>2</sup> over

35.5 hours.

Be certain that the ID MTX infusion is completed in the 36 hour period. Even if the infusion is not complete at this time point, it must be stopped.

Leucovorin rescue: See below.

Suggested hydration and alkalinization for IDMTX: Prehydrate with D5  $\frac{1}{4}$  NS with 30 mEq NaHCO3/L at 125 mL/m²/hour to achieve a urine specific gravity  $\leq 1.010$  and pH between 7 and 8. Ringers Lactate may be used as the initial fluid if a bicarbonate containing solution is unavailable. Adjust fluid volume and sodium bicarbonate to maintain urine specific gravity  $\leq 1.010$  and pH between 7 and 8. A bicarbonate bolus (25 mEq/m² over 15 min) may be given to raise the urine pH relatively quickly; a normal saline bolus may also be helpful in facilitating hydration. Continue hydration using D 5  $\frac{1}{4}$  NS with 30 mEq NaHCO3/L at 125 mL/m²/hour throughout IDMTX infusion after its completion until the last dose of leucovorin has been given.

#### **Timing of ID MTX:**

• For patients beginning Block 2 with **M1** marrow, it is recommended to await count recovery to an ANC  $\geq 500/\mu L$  and platelets  $\geq 50,000/\mu L$  prior to beginning Day 8 IV methotrexate.



• Patients beginning Block 2 with **M2** marrow should proceed without awaiting count recovery.

# Leucovorin: PO/IV

Day: 10, 11

Dose: 15 mg/m²/dose every 6 hours beginning **48 hrs** after the **START** of ID MTX infusion.

- If 48 hr methotrexate level is  $\leq 0.5 \,\mu\text{M}$ , do not give more than two doses of leucovorin (48 and 54 hours).
- If MTX level at 48 hours is  $> 0.5~\mu M$ , then continue hydration and leucovorin rescue at 15 mg/m²/dose po/IV every 6 hours until MTX levels are  $< 0.1~\mu M$ .

See Section 5.8 for ID MTX/LCV rescue and infusion guidelines.

# Methotrexate: Intrathecal (IT) - CNS1/2 PATIENTS ONLY

Day: 8

# Age-based dosing:

| Age (yrs) | <u>Dose</u> |
|-----------|-------------|
| 1 - 1.99 | 8 mg |
| 2 - 2.99 | 10 mg |
| 3 - 8.99 | 12 mg |
| $\geq$ 9 | 15 mg |

When IT therapy and ID MTX are scheduled for the same day, deliver the IT therapy within 6 hours of the beginning of the IV MTX infusion (hour -6 to +6, with 0 being the start of the MTX bolus).

# Triple Intrathecal Therapy (ITT) - CNS3 PATIENTS ONLY

Days: 8, 22

# Age-based dosing:

| Age (yrs) | <u>Dose</u> |
|-----------|------------------------------------|
| 1 - 1.99 | MTX: 8 mg, HC: 8 mg, ARAC: 16 mg |
| 2 - 2.99 | MTX: 10 mg, HC: 10 mg, ARAC: 20 mg |
| 3 - 8.99 | MTX: 12 mg, HC: 12 mg, ARAC: 24 mg |
| $\geq$ 9 | MTX: 15 mg, HC: 15 mg, ARAC: 30 mg |

When ITT therapy and ID MTX are scheduled for the same day, deliver the ITT therapy within 6 hours of the beginning of the IV MTX infusion (hour -6 to +6, with 0 being the start of the MTX bolus).

# Pegaspargase: IV over 1-2 hours

Administer 4 hours after completion of Day 8 IV MTX. (Day 9 or 10)

Dose: 2,500 International Units/m<sup>2</sup>/dose



#### **Special precautions:**

- 1. Pegaspargase is contraindicated with a history of severe pancreatitis with any prior asparaginase therapy. Caution should be used if serious thrombosis or hemorrhagic events have occurred with any prior asparaginase therapy (see Section 5.1)
- 2. Pegaspargase may affect coagulation factors and predispose to bleeding and/or thrombosis. Caution should be used when administering any concurrent anticoagulant therapy.
- 3. Suggested monitoring during and after administration: Because pegaspargase is long acting, hypersensitivity reactions may not appear for hours after drug administration. Monitor vital signs, for signs of fever, chills, or acute allergic reactions including anaphylaxis. Have medications to treat hypersensitivity reactions readily available at each administration (e.g., epinephrine, IV corticosteroids, antihistamines). Consider prescribing an EpiPen® for home use.

# Cyclophosphamide: IV over 15-30 minutes (see note below)

Days: 15-19

Dose: 440 mg/m<sup>2</sup>/dose

**Etoposide:** IV over 1-2 hours (see note below)

Days: 15-19

Dose: 100 mg/m<sup>2</sup>/dose

**NOTE:** Await count recovery to ANC  $\geq 500/\mu$ L and platelets  $\geq 50,000/\mu$ L prior to beginning Day 15 IV cyclophosphamide and etoposide.

#### 4.3.5 Evaluation 2 (Disease Evaluation End Block 2)

- Evaluation 2 should not be done earlier than Day 29 ( $\pm$  1 day);
- The evaluation may be delayed no later than Day 36 ( $\pm$  1 day) if ANC  $< 500/\mu$ L and platelets  $< 50,000/\mu$ L on Day 29.
- See Sections <u>7.1</u> and <u>13.0</u> for details on specimen acquisition, handling and shipping.

# 4.3.6 Following Completion of Block 2:

For LR B-ALL patients post-Block 2:

- Arm C, Block 3 (Section 4.4, APPENDIX II-C) starts when ANC  $\geq$  500/ $\mu$ L and platelets  $\geq$  50,000/ $\mu$ L.
- **Arm D**, therapy with Blinatumomab Block Cycle 1 (Section 4.15, APPENDIX II-M) starts when ANC  $\geq 500/\mu L$  and platelets  $\geq 50,000/\mu L$ .



# 4.4 Block 3 (LR Patients on Arm C) - 4 weeks

Block 3 therapy is for LR patients randomized to the control arm (Arm C). See Experimental Design Schema.

The Therapy Delivery Map (TDM) for Block 3 is in APPENDIX II-C.

#### 4.4.1 Criteria to Begin Block 3 Therapy

Start when ANC  $\geq 500/\mu L$  and platelets  $\geq 50,000/\mu L$ 

# 4.4.2 <u>General Chemotherapy Guidelines</u>

See <u>Section 6.0</u>, Drug Information, and the Parenteral and Oral Chemotherapy Administration Guidelines (CAGs) on the COG website at: <a href="https://members.childrensoncologygroup.org/files/disc/Pharmacy/ChemoAdminGuidelines.pdf">https://members.childrensoncologygroup.org/files/disc/Pharmacy/ChemoAdminGuidelines.pdf</a> for special precautions associated with chemotherapy administration. As applicable, also see the CAGs for suggestions on hydration, or hydrate according to institutional guidelines.

See <u>Section 5.0</u> for Dose Modifications based on Toxicities and <u>Appendix I</u> for Supportive Care Guidelines.

Dosing should be based on actual BSA.

# 4.4.3 <u>Block 3 Chemotherapy</u>

# Dexamethasone: PO (may be given IV)

Days: 1-5

Dose: 3 mg/m<sup>2</sup>/dose (Total daily dose: 6 mg/m<sup>2</sup>/day, divided BID)

If using tablets, adjust dose upward to the nearest 0.25 mg. Oral solutions are acceptable and intravenous preparations may be used on a temporary basis, if needed.

# <u>VinCRIStine:</u> IV push over 1 minute or infusion via minibag as per institutional policy

Day: 1

Dose: 1.5 mg/m<sup>2</sup>/dose (maximum dose: 2 mg)

# Special precautions: FOR INTRAVENOUS USE ONLY.

The container or the syringe containing vinCRIStine must be enclosed in an overwrap bearing the statement "Do not remove covering until moment of injection. For intravenous use only - Fatal if given by other routes."

Medication errors have occurred due to confusion between vinCRIStine and vinBLAStine. VinCRIStine is available in a liposomal formulation (vinCRIStine sulfate liposomal injection, VSLI, Marqibo®). Use conventional vinCRIStine only; the conventional and liposomal formulations are NOT interchangeable.



# Cytarabine: IV over 3 hours

Days: 1, 2, 8, 9

Dose: 3000 mg/m<sup>2</sup>/dose every 12 hours

Administer steroid eye drops (0.1% dexamethasone or 1% prednisolone ophthalmic solution), 2 drops to each eye every 6 hours, beginning immediately before the first dose of cytarabine and continuing for 24 hours after the last dose. If patient does not tolerate steroid eye drops, may administer artificial tears on an every 2-4 hour schedule.

# Asparaginase (Erwinia): IM (may be given IV over 1 hour)

Day: 2, 4, 9, 11, 23

Dose: 25, 000 International Units/m<sup>2</sup>/dose

- Asparaginase (Erwinia) should be given 4 hours after the completion of the last cytarabine infusion on Days 2 and 9.
- Asparaginase (Erwinia) should be given 4 hours after the MTX infusion is complete on Day 23.
- If Asparaginase (Erwinia) is not available, a single dose of Pegaspargase should be substituted 4 hours after the last cytarabine dose is complete on Day 9, and no asparaginase is given on Day 23.

# Methotrexate: Intrathecal (IT) Day: 1 FOR ALL PATIENTS

Day 22: CNS1/2 PATIENTS ONLY

# Age-based dosing:

| Age (yrs) | <u>Dose</u> |
|-----------|-------------|
| 1 - 1.99 | 8 mg |
| 2 - 2.99 | 10 mg |
| 3 - 8.99 | 12 mg |
| $\geq$ 9 | 15 mg |

When IT therapy and ID MTX are scheduled for the same day, deliver the IT therapy within 6 hours of the beginning of the IV MTX infusion (hour -6 to +6, with 0 being the start of the MTX bolus).

**<u>NOTE:</u>** Await count recovery to ANC  $\geq 500/\mu L$  and platelets  $\geq 50,000/\mu L$  prior to beginning Day 22 IV Methotrexate and intrathecal chemotherapy.

#### <u>Triple Intrathecal Therapy (ITT)</u> -

# **CNS3 PATIENTS ONLY**

Day: 22

# Age-based dosing:

| Age (yrs) | <u>Dose</u> | | |
|--------------|-------------|-----------|-------------|
| 1 to < 1.99 | MTX: 8 mg | HC: 8 mg | ARAC: 16 mg |
| 2 to < 2.99 | MTX: 10 mg | HC: 10 mg | ARAC: 20 mg |
| 3 to < 8.99 | MTX: 12 mg | HC: 12 mg | ARAC: 24 mg |
| $\geq 9$ | MTX: 15 mg | HC: 15 mg | ARAC: 30 mg |



When IT therapy and ID MTX are scheduled for the same day, deliver the IT therapy within 6 hours of the beginning of the IV MTX infusion (hour -6 to +6, with 0 being the start of the MTX bolus).

# **Intermediate Dose Methotrexate: IV over 36 hours**

Day: 22

Dose 1000 mg/m<sup>2</sup>/dose

See <u>Sections 4.3.4</u> and <u>5.8</u> for ID MTX/LCV rescue and infusion guidelines

#### Leucovorin: PO/IV

Days: 24, 25

Dose: 15 mg/m<sup>2</sup>/dose beginning **48 hrs** after the **START** of ID MTX infusion.

- If 48 hr methotrexate level is  $\leq 0.5 \mu M$ , do not give more than two doses of leucovorin (48 and 54 hours).
- If MTX level at 48 hours is  $> 0.5 \mu M$ , then continue hydration and leucovorin rescue at 15 mg/m<sup>2</sup>/dose po/IV every 6 hours until MTX levels are  $< 0.1 \mu M$ .

See <u>Section 5.8</u> for ID MTX/LCV rescue and infusion guidelines.

# 4.4.4 Disease Evaluation End Block 3 (HR/IR Patients ONLY):

- The End Block 3 disease evaluation should not be done earlier than Day 29 (± 1 day);
- The evaluation may be delayed no later than Day 36 ( $\pm$  1 day) if ANC  $< 500/\mu L$  and platelets  $< 50,000/\mu L$  on Day 29.
- See Sections <u>7.1</u> and <u>13.0</u> for details on specimen acquisition, handling and shipping.

#### **Notes regarding End Block 3 Disease Assessment:**

- BM assessment should be coordinated so that patients begin their preparative regimens no later than 2 weeks from BM documentation of M1.
- If delays > 14 days are required for donor timing or other reasons, patients may receive up to 6 weeks of bridging maintenance therapy as described in Section 4.10.
- For patients who receive bridging therapy, a repeat BM assessment is required to document remission and MRD status within 14 days of starting the HSCT preparative regimen.
- Patients who are unable to begin the transplant preparative regimen within 8 weeks of initial BM assessment are off protocol therapy.

#### 4.4.5 Following completion of Block 3:

#### For LR B-ALL patients:

**Arm C**, Continuation 1 (Section 4.11, APPENDIX II-I) starts when ANC  $\geq 500/\mu L$  and platelets  $\geq 50,000/\mu L$ .



# 4.5 Blinatumomab Block: Cycle 1 (HR/IR Patients in Arm B) - 5 weeks

With Amendment #10, HR/IR patients already assigned to Arm A (standard chemotherapy) who are at an appropriate point in their treatment program (prior to receiving Day 22 treatment on Block 3) will be offered the opportunity to cross over to Arm B to receive blinatumomab.

The therapy described in this section is for the 1<sup>st</sup> cycle of therapy with Blinatumomab for HR/IR patients. See Experimental Design Schema.

The Therapy Delivery Map (TDM) for the Blinatumomab Block: Cycle 1 (**Arm B**) is in APPENDIX II-D.

**NOTE:** Hospitalization is STRONGLY recommended during the first 9 days of this cycle in case of a cytokine reaction. Manifestations of cytokine release syndrome include fever, headache, nausea, asthenia, hypotension, increased alanine aminotransferase, increased aspartate aminotransferase, increased total bilirubin, and disseminated intravascular coagulation (DIC). Corticosteroids should be administered for severe or life threatening cytokine release syndrome.

# Blinatumomab infusion interruptions for technical reasons:

The drug administration should not be interrupted, if possible. In case of infusion interruption due to any technical or logistic reason the interruption should be as short as possible and the infusion continued at the earliest time possible. Every interruption longer than one hour should be documented. If the interruption is longer than four hours, re-start of the infusion should be performed in the hospital, under supervision of the investigator. The patient should be observed overnight for possible side effects after the re-start in the hospital and can be discharged the following day if no difficulties arise. Administration of the premedication (dexamethasone) described in Section 4.5.4, is recommended. If possible, the infusion time before and after a break should sum up to 28 days treatment per cycle.

END BLOCK 1 CALLBACK OCCURS PRIOR TO STARTING BLINATUMOMAB BLOCK: CYCLE 1 THERAPY. PLEASE SEE SUMMARY TABLE IN <u>SECTION 3.1.5</u> FOR DETAILS ON STAGED CONSENT, AND APPROPRIATE TIMING TO OBTAIN INFORMED CONSENT.

# 4.5.1 Criteria to Begin Blinatumomab Block: Cycle 1

Blinatumomab Cycle 1 should begin after submission of end- Block 1 Callback and receipt of treatment assignment and as soon as clinically acceptable to the treating institution. Patients should have time for full or partial recovery (judged by the treating institution) from any toxicities experienced in the prior course(s) of therapy before proceeding to the next course.

For patients beginning Blinatumomab Cycle 1 with M1 marrow, it is recommended to await count recovery to ANC  $\geq 500/\mu L$  and platelets  $\geq 50,000/\mu L$ . To continue to receive protocol therapy, M1 patients must begin Blinatumomab Cycle 1 no later than 14 calendar days after callback.



For patients beginning Blinatumomab Cycle 1 with M2 marrow, it is recommended to proceed without awaiting count recovery. To continue to receive protocol therapy, M2 patients must begin Blinatumomab Cycle 1 no later than 5 calendar days after Callback.

# 4.5.2 Testicular Radiation Therapy (TRT)

- Patients with persistent testicular leukemia at the end of Block 1 are eligible to continue on study and will receive 2400 cGy of testicular radiation during the 1<sup>st</sup> cycle of Blinatumomab (for HR/IR patients).
- Patients with extramedullary testicular leukemia that has resolved by end-Block 1 will NOT receive testicular irradiation with the exception of that which may be used in the HSCT preparative regimen.
- See Section 14.2 for detailed testicular radiation guidelines.

#### 4.5.3 General Chemotherapy Guidelines

See Section 6.0, DRUG INFORMATION, and the Parenteral and Oral Chemotherapy Administration Guidelines (CAGs) on the COG website at: <a href="https://members.childrensoncologygroup.org/files/disc/Pharmacy/ChemoAdminGuidelines.pdf">https://members.childrensoncologygroup.org/files/disc/Pharmacy/ChemoAdminGuidelines.pdf</a> for special precautions associated with chemotherapy administration. As applicable, also see the CAGs for suggestions on hydration, or hydrate according to institutional guidelines.

See <u>Section 5.0</u> for Dose Modifications based on Toxicities and <u>Appendix I</u> for Supportive Care Guidelines.

See <u>Appendix VII-A</u> for the management options of blinatumomab in the outpatient setting.

#### Dosing should be based on actual BSA. There is no maximum dosing

# 4.5.4 Blinatumomab Block: Cycle 1 Chemotherapy

# Blinatumomab: IV; Continuous Infusion over 28 days\*

Days: 1-28

Dose: 15 micrograms/m<sup>2</sup>/day

\*IV bag will be changed every 24 - 96 hours or every 168 hours (7 days), depending on the details of the infusion preparation

# Dexamethasone: PO/IV

Day:

Dose: Prior to day 1 therapy -

 A single dose of 5 mg/m²/dose (maximum 20 mg/dose) will be administered 30 to 60 minutes prior to the start of the blinatumomab infusion and when restarting an infusion after an interruption of 4 or more hours in the first cycle.



If using tablets, adjust dose upward to the nearest 0.25 mg. Oral solutions are acceptable and intravenous preparations may be used on a temporary basis, if needed.

# Methotrexate: Intrathecal (IT) - CNS1/2 PATIENTS ONLY

Day: 15, 29

#### Age-based dosing:

| Age (yrs) | Dose |
|-----------|-------|
| 1 - 1.99 | 8 mg |
| 2 - 2.99 | 10 mg |
| 3 - 8.99 | 12 mg |
| $\geq$ 9 | 15 mg |

# **Triple Intrathecal Therapy (ITT) - CNS3 PATIENTS ONLY**

Days: 15, 29

# Age-based dosing:

| Age (yrs) | <u>Dose</u> |
|-----------|------------------------------------|
| 1 - 1.99 | MTX: 8 mg, HC: 8 mg, ARAC: 16 mg |
| 2 - 2.99 | MTX: 10 mg, HC: 10 mg, ARAC: 20 mg |
| 3 - 8.99 | MTX: 12 mg, HC: 12 mg, ARAC: 24 mg |
| $\geq$ 9 | MTX: 15 mg, HC: 15 mg, ARAC: 30 mg |

# 4.5.5 <u>Disease Evaluation End-Blinatumomab Block: Cycle 1</u>

- The end block disease staging should be performed no earlier than Day 29 (± 1 day);
- The evaluation may be delayed to no later than Day 36 ( $\pm$  1 day) if ANC <  $500/\mu$ L and platelets <  $50,000/\mu$ L on Day 29.
- Two (2 mL) of bone marrow will be collected and shipped to the flow cytometry laboratory for MRD determination
- See Sections <u>7.1</u> and <u>13.0</u> for details on specimen handling and shipping.

#### 4.5.6 Following completion of Blinatumomab Block: Cycle 1 (Arm B)

# a. For HR/IR B-ALL patients assigned to Arm B:

Blinatumomab Block Cycle 2 (Section 4.6, APPENDIX II-E) starts when ANC  $\geq 500/\mu L$  and platelets  $\geq 50,000/\mu L$ .

#### b. Treatment Failures post-Blinatumomab Block:

Patients with a TF post Blinatumomab Block: Cycle 1 (see <u>Section 3.3</u> for definition) will be taken off protocol therapy.



# 4.6 Blinatumomab Block: Cycle 2 (HR/IR Patients in Arm B) - 5 weeks

With Amendment #10, HR/IR patients already assigned to Arm A (standard chemotherapy) who are at an appropriate point in their treatment program (prior to receiving Day 22 treatment on Block 3) will be offered the opportunity to cross over to Arm B to receive blinatumomab.

The therapy described in this section is for the 2<sup>nd</sup> cycle of therapy with blinatumomab on Arm B. See Experimental Design Schema.

The Therapy Delivery Map (TDM) for the Blinatumomab Block: Cycle 2 (Arm B) is in APPENDIX II-E.

**NOTE:** Hospitalization is STRONGLY recommended during the first 2 days of this cycle in case of a cytokine reaction. Manifestations of cytokine release syndrome include fever, headache, nausea, asthenia, hypotension, increased alanine aminotransferase, increased aspartate aminotransferase, increased total bilirubin, and disseminated intravascular coagulation (DIC). Corticosteroids should be administered for severe or life threatening cytokine release syndrome.

# Blinatumomab infusion interruptions for technical reasons:

The drug administration should not be interrupted, if possible. In case of infusion interruption due to any technical or logistic reason the interruption should be as short as possible and the infusion continued at the earliest time possible. Every interruption longer than one hour should be documented. If the interruption is longer than four hours, re-start of the infusion should be performed in the hospital, under supervision of the investigator. The patient should be observed overnight for possible side effects after the re-start in the hospital and can be discharged the following day if no difficulties arise. (NOTE: Administration of the premedication (dexamethasone) is NOT RECOMMENDED for the second cycle of blinatumomab.) If possible, the infusion time before and after a break should sum up to 28 days treatment per cycle.

# 4.6.1 Criteria to Begin Blinatumomab Block: Cycle 2

- Do not start Blinatumomab Cycle 2 before Day 36 after beginning of Cycle 1.
- Begin Blinatumomab Block: Cycle 2 therapy when ANC  $\geq 500/\mu L$  and platelets  $\geq 50,000/\mu L$ .

# 4.6.2 General Chemotherapy Guidelines

See Section 6.0, Drug Information, and the Parenteral and Oral Chemotherapy Administration Guidelines (CAGs) on the COG website at: <a href="https://members.childrensoncologygroup.org/files/disc/Pharmacy/ChemoAdminGuidelines.pdf">https://members.childrensoncologygroup.org/files/disc/Pharmacy/ChemoAdminGuidelines.pdf</a> for special precautions associated with chemotherapy administration. As applicable, also see the CAGs for suggestions on hydration, or hydrate according to institutional guidelines.

See <u>Section 5.0</u> for Dose Modifications based on Toxicities and <u>Appendix I</u> for Supportive Care Guidelines.

See <u>Appendix VII-A</u> for the management options of blinatumomab in the outpatient setting.



# Dosing should be based on actual BSA.

# 4.6.3 <u>Blinatumomab Block: Cycle 2 Administration Guidelines</u>

Blinatumomab: IV; Continuous Infusion over 28 days\*

Days: 1-28

Dose: 15 micrograms/m<sup>2</sup>/day

\*IV bag will be changed every 24 - 96 hours or every 168 hours (7 days), depending on the details of the infusion preparation

(<u>NOTE</u>: Administration of the premedication (dexamethasone) is NOT RECOMMENDED for the second cycle of blinatumomab.)

# **Methotrexate: Intrathecal (IT) - CNS1/2 PATIENTS ONLY**

Days: 8, 29

# Age-based dosing:

| Age (yrs) | <u>Dose</u> |
|-----------|-------------|
| 1 - 1.99 | 8 mg |
| 2 - 2.99 | 10 mg |
| 3 - 8.99 | 12 mg |
| $\geq$ 9 | 15 mg |

# Triple Intrathecal Therapy (ITT) - CNS3 PATIENTS ONLY

Days: 8, 29

# Age-based dosing:

| Age (yrs) | <u>Dose</u> | | |
|-----------|-------------|-----------|-------------|
| 1 - 1.99 | MTX: 8 mg | HC: 8 mg | ARAC: 16 mg |
| 2 - 2.99 | MTX: 10 mg | HC: 10 mg | ARAC: 20 mg |
| 3 - 8.99 | MTX: 12 mg | HC: 12 mg | ARAC: 24 mg |
| $\geq$ 9 | MTX: 15 mg | HC: 15 mg | ARAC: 30 mg |

### 4.6.4 Disease Evaluation End-Blinatumomab Block: Cycle 2

- The end block disease staging should be performed no earlier than Day 29 (± 1 day);
- The evaluation may be delayed to no later than Day 36 ( $\pm$  1 day) if ANC  $< 500/\mu$ L and platelets  $< 50,000/\mu$ L on Day 29.
- Two (2 mL) of bone marrow will be collected and shipped to the flow cytometry laboratory for MRD determination
- See Sections <u>7.1</u> and <u>13.0</u> for details on specimen handling and shipping.



# Notes regarding End-Blinatumomab Block: Cycle 2 Disease Assessment:

- BM assessment should be coordinated so that patients begin their preparative regimens no later than 2 weeks from BM documentation of M1.
- If delays > 14 days are required for donor timing or other reasons, patients may receive up to 6 weeks of bridging maintenance therapy as described in Section 4.10.
- For patients who receive bridging therapy, a repeat BM assessment is required to document remission and MRD status within 14 days of starting the HSCT preparative regimen.
- Patients who are unable to begin the transplant preparative regimen within 8 weeks of initial BM assessment are off protocol therapy.

# 4.6.5 Following completion of Blinatumomab Block: Cycle 2 (Arm B):

- Patients will continue on to HSCT (See <u>Section 4.9</u>). Patients may receive up to 6 weeks of bridging maintenance therapy prior to HSCT as described in <u>Section 4.10</u>.
- Treatment Failures post-Blinatumomab Block: Cycle 2 (see <u>Section 3.3</u> for definition) will be taken off protocol therapy.



# 4.7 Blinatumomab-S: Cycle 1 (Salvage Therapy) - 5 weeks

Patients classified as treatment failures after Block 1 or Block 2 treatment (see Section 3.3 for definitions) who have not previously received blinatumomab on study and who are without evidence of CNS disease will have the option to be non-randomly assigned treatment with up to 2 blocks of salvage blinatumomab (Blinatumomab-S), and continue on study with HSCT therapy if a CR is achieved. Eligible patients should complete the appropriate callback (Section 3.1.7) before initiating Salvage Therapy treatment. Note that blinatumomab dosing in Blinatumomab-S cycles differs from dosing in Blinatumomab Block cycles (See Section 4.7.4.) The schedule below describes treatment for the 1st cycle only. See Experimental Design Schema.

The Therapy Delivery Map (TDM) for the Blinatumomab-S: Cycle 1 is in <u>APPENDIX II-F</u>.

**NOTE:** Hospitalization is STRONGLY recommended during the first 9 days of this cycle in case of a cytokine reaction. Manifestations of cytokine release syndrome include fever, headache, nausea, asthenia, hypotension, increased alanine aminotransferase, increased aspartate aminotransferase, increased total bilirubin, and disseminated intravascular coagulation (DIC). Corticosteroids should be administered for severe or life threatening cytokine release syndrome.

# Blinatumomab infusion interruptions for technical reasons:

The drug administration should not be interrupted, if possible. In case of infusion interruption due to any technical or logistic reason the interruption should be as short as possible and the infusion continued at the earliest time possible. Every interruption longer than one hour should be documented. If the interruption is longer than four hours, re-start of the infusion should be performed in the hospital, under supervision of the investigator. The patient should be observed overnight for possible side effects after the re-start in the hospital and can be discharged the following day if no difficulties arise. Administration of the premedication (dexamethasone) described in Section 4.5.4, is recommended. If possible, the infusion time before and after a break should sum up to 28 days treatment per cycle.

OBTAIN INFORMED CONSENT PRIOR TO INITIATING THE FIRST CYCLE OF SALVAGE THERAPY. PLEASE SEE THE SUMMARY TABLE IN <u>SECTION 3.1.5</u> FOR DETAILS ON TIMING TO OBTAIN INFORMED CONSENT. CALLBACK OCCURS PRIOR TO STARTING BLINATUMOMAB-S: CYCLE 1 THERAPY (See <u>Section 3.1.7</u> for appropriate callback).

# 4.7.1 Criteria to Begin Blinatumomab-S: Cycle 1

• None

# 4.7.2 Testicular Radiation Therapy (TRT)

- All Treatment Failures on the basis of M3 marrow at the end of Block 1 who also have persistent testicular leukemia will receive 2400 cGy of testicular radiation during the 1<sup>st</sup> cycle of Salvage Therapy (Blinatumomab-S: Cycle 1).
- Patients with extramedullary testicular leukemia that has resolved by end Block 1 will NOT receive testicular irradiation with the exception of that which may be used in the HSCT preparative regimen for HR/IR patients.



• See Section 14.2 for detailed radiation guidelines.

# 4.7.3 General Chemotherapy Guidelines

See <u>Section 6.0</u>, Drug Information, and the Parenteral and Oral Chemotherapy Administration Guidelines (CAGs) on the COG website at: <a href="https://members.childrensoncologygroup.org/files/disc/Pharmacy/ChemoAdminGuidelines.pdf">https://members.childrensoncologygroup.org/files/disc/Pharmacy/ChemoAdminGuidelines.pdf</a> for special precautions associated with chemotherapy administration. As applicable, also see the CAGs for suggestions on hydration, or hydrate according to institutional guidelines.

See <u>Section 5.0</u> for Dose Modifications based on Toxicities and <u>Appendix I</u> for Supportive Care Guidelines.

See <u>Appendix VII-A</u> for the management options of blinatumomab in the outpatient setting.

Dosing should be based on actual BSA.

# 4.7.4 Blinatumomab-S: Cycle 1 Chemotherapy Guidelines

# Blinatumomab: IV; Continuous Infusion over 28 days\*

Days: 1-28

Dose: 5 micrograms/m²/day (Days 1-7) followed by 15 micrograms/m²/day

(Days 8-28)

# \*IV bag will be changed every 24 - 96 hours or every 168 hours (7 days), depending on the details of the infusion preparation

# **Dexamethasone: PO/IV**

Dose: Prior to day 1 and day 8 of therapy -

• A single dose of 5 mg/m²/dose (maximum 20 mg/dose) will be administered 30 to 60 minutes prior to the start of the blinatumomab infusion on Day 1, prior to a step dose (such as Cycle 1 Day 8), and when restarting an infusion after an interruption of 4 or more hours in the first cycle.

If using tablets, adjust dose upward to the nearest 0.25 mg. Oral solutions are acceptable and intravenous preparations may be used on a temporary basis, if needed.

#### **Methotrexate: Intrathecal (IT)**

Day: 15

# Age-based dosing:

| Age (yrs) | <u>Dose</u> |
|-----------|-------------|
| 1 - 1.99 | 8 mg |
| 2 - 2.99 | 10 mg |
| 3 - 8.99 | 12 mg |
| ≥9 | 15 mg |



# 4.7.5 <u>Disease Evaluation End Blinatumomab-S Cycle 1:</u>

- The end block disease staging should be performed no earlier than Day 29 (± 1 day);
- The evaluation may be delayed to no later than Day 36 ( $\pm$  1 day) if ANC  $< 500/\mu$ L and platelets  $< 50,000/\mu$ L on Day 29.
- Two (2 mL) of bone marrow will be collected and shipped to the flow cytometry laboratory for MRD determination
- See Sections <u>7.1</u> and <u>13.0</u> for details on specimen handling and shipping.

#### 4.7.6 Following completion of Blinatumomab-S: Cycle 1:

# a. Patients with M1 marrow after Blinatumomab-S Cycle 1:

- If patient has recovered counts to ANC ≥ 500/μL and platelets ≥ 50,000/μL (i.e., have achieved a CR), then proceed to HSCT on study as soon as possible. See Section 4.9.
- If patient has NOT recovered counts to ANC  $\geq 500/\mu L$  and platelets  $\geq 50,000/\mu L$  at the time of the marrow evaluation, but recovers counts within 1 week of the marrow evaluation, then this will be considered a CR and the patient should proceed to HSCT as soon as possible.
- If patient has NOT recovered counts to ANC ≥ 500/μL and platelets ≥ 50,000/μL at the time of the marrow evaluation, and does NOT recover counts within 1 week of the marrow evaluation, a repeat marrow every 1 2 weeks until either patient meets definition of CR (in which case the patient may proceed to HSCT) or develops an M2/M3 marrow (in which case proceed as detailed in Section 4.7.6.b).
- Patients should begin their preparative regimens no later than 2 weeks from BM documentation of M1.
- If patient achieves a CR but delays > 14 days are required for donor timing or other reasons, patients may receive Blinatumomab-S Cycle 2 as described in <u>Section 4.8</u> or up to 6 weeks of bridging maintenance therapy as described in <u>Section 4.10</u>.
- For patients who receive bridging therapy, a repeat BM assessment will be needed to document remission and MRD status within 14 days of starting the HSCT preparative regimen.
- Patients who are unable to begin the transplant preparative regimen within 8 weeks of initial BM assessment are off protocol therapy.

# b. Patients with M2/M3 marrow after Blinatumomab-S: Cycle 1

Such patients proceed to Blinatumomab-S: Cycle 2 (Section 4.8, APPENDIX II-G) without awaiting count recovery.



# 4.8 Blinatumomab-S: Cycle 2 (Salvage Therapy) - 5 weeks

Blinatumomab-S: Cycle 2 is for patients with M2/M3 marrow after completion of Blinatumomab-S: Cycle 1. Patients who are M1 after completion of Blinatumomab-S: Cycle 1 and have delays >14 days before initiating HSCT may also receive treatment on Blinatumomab-S: Cycle 2 (See Section 4.7.6). Note that blinatumomab dosing in Blinatumomab-S cycles differs from dosing in Blinatumomab Block cycles (See Section 4.8.3.)

The schedule below describes treatment for the 2nd cycle only. See <u>Experimental Design</u> Schema.

The Therapy Delivery Map (TDM) for the Blinatumomab-S: Cycle 2 is in APPENDIX II - G.

**NOTE:** Hospitalization is STRONGLY recommended during the first 2 days of this cycle in case of a cytokine reaction. Manifestations of cytokine release syndrome include fever, headache, nausea, asthenia, hypotension, increased alanine aminotransferase, increased aspartate aminotransferase, increased total bilirubin, and disseminated intravascular coagulation (DIC). Corticosteroids should be administered for severe or life threatening cytokine release syndrome.

# Blinatumomab infusion interruptions for technical reasons:

The drug administration should not be interrupted, if possible. In case of infusion interruption due to any technical or logistic reason the interruption should be as short as possible and the infusion continued at the earliest time possible. Every interruption longer than one hour should be documented. If the interruption is longer than four hours, re-start of the infusion should be performed in the hospital, under supervision of the investigator. The patient should be observed overnight for possible side effects after the re-start in the hospital and can be discharged the following day if no difficulties arise. NOTE: Administration of the premedication (dexamethasone) is NOT RECOMMENDED for the second cycle of blinatumomab.) If possible, the infusion time before and after a break should sum up to 28 days treatment per cycle.

# 4.8.1 Criteria to Begin Blinatumomab-S: Cycle 2

Do not start Blinatumomab-S: Cycle 2 before Day 36 after beginning of Cycle 1.

# 4.8.2 <u>General Chemotherapy Guidelines</u>

See <u>Section 6.0</u>, Drug Information, and the Parenteral and Oral Chemotherapy Administration Guidelines (CAGs) on the COG website at: <a href="https://members.childrensoncologygroup.org/files/disc/Pharmacy/ChemoAdminGuidelines.pdf">https://members.childrensoncologygroup.org/files/disc/Pharmacy/ChemoAdminGuidelines.pdf</a> for special precautions associated with chemotherapy administration. As applicable, also see the CAGs for suggestions on hydration, or hydrate according to institutional guidelines.

See <u>Section 5.0</u> for Dose Modifications based on Toxicities and <u>Appendix I</u> for Supportive Care Guidelines.

See <u>Appendix VII-A</u> for the management options of blinatumomab in the outpatient setting.



# Dosing should be based on actual BSA.

# 4.8.3 Blinatumomab-S: Cycle 2 Chemotherapy

Blinatumomab: IV; Continuous Infusion over 28 days\*

Days: 1-28

Dose: 15 micrograms/m<sup>2</sup>/day (Days 1-28)

\*IV bag will be changed every 24-96 hours or every 168 hours (7 days), depending on the details of the infusion preparation

(<u>NOTE</u>: Administration of the premedication (dexamethasone) is NOT RECOMMENDED for the second cycle of blinatumomab.)

# **Methotrexate: Intrathecal (IT)**

Day: 8 & 29

# Age-based dosing:

| Age (yrs) | <u>Dose</u> |
|-----------|-------------|
| 1 - 1.99 | 8 mg |
| 2 - 2.99 | 10 mg |
| 3 - 8.99 | 12 mg |
| ≥ 9 | 15 mg |

# 4.8.4 Disease Evaluation End-Blinatumomab-S: Cycle 2

- The end block disease staging should be performed no earlier than Day 29 (± 1 day);
- The evaluation may be delayed to no later than Day 36 ( $\pm$  1 day) if ANC  $< 500/\mu$ L and platelets  $< 50,000/\mu$ L on Day 29.
- Two (2 mL) of bone marrow will be collected and shipped to the flow cytometry laboratory for MRD determination
- See Sections 7.1 and 13.0 for details on specimen handling and shipping.

#### 4.8.5 Following completion of Blinatumomab-S: Cycle 2:

# a. Patients with M1 marrow after Blinatumomab-S Cycle 2:

- If patient has recovered counts to ANC  $\geq 500/\mu L$  and platelets  $\geq 50,000/\mu L$  (i.e., have achieved a CR), then proceed to HSCT on study as soon as possible. See Section 4.9.
- If patient has NOT recovered counts to ANC  $\geq 500/\mu L$  and platelets  $\geq 50,000/\mu L$  at the time of the marrow evaluation, but recovers counts within 1 week of the marrow evaluation, then this will be considered a CR and the patient should proceed to HSCT as soon as possible.
- If patient has NOT recovered counts to ANC  $\geq 500/\mu L$  and platelets  $\geq 50,000/\mu L$  at the time of the marrow evaluation, and does NOT recover counts within 1 week of the marrow evaluation, a repeat marrow



- every 1-2 weeks until either patient meets definition of CR (in which case the patient may proceed to HSCT) or develops an M2/M3 marrow (in which case proceed as detailed in Section 4.8.5.b).
- Patients should begin their preparative regimens no later than 2 weeks from BM documentation of M1.
- If patient achieves CR but delays > 14 days are required for donor timing or other reasons, patients may receive up to 6 weeks of bridging maintenance therapy as described in Section 4.10.
- For patients who receive bridging therapy, a repeat BM assessment will be needed to document remission and MRD status within 14 days of starting the HSCT preparative regimen.
- Patients who are unable to begin the transplant preparative regimen within 8 weeks of initial BM assessment are off protocol therapy.
- **b.** Patients with M2/M3 marrow after Blinatumomab-S Cycle 2 Remove from protocol therapy.



# 4.9 Hematopoietic Stem Cell Transplant

All transplants performed on COG trials must occur at FACT-accredited HSCT programs with the exception of adolescents/adults being treated on COG trials who are referred to an adult transplant facility. See the COG Administrative Policy 3.3 regarding the agreement requirements for these cases.

# 4.9.1 Overview

Stem cell transplantation in this study will be utilized in patients with HR/IR relapse ALL (see Section 3.3 for risk definitions).

All patients enrolled on this protocol and their full siblings should undergo HLA tissue typing as soon as possible after diagnosis of relapse. All high-risk patients should have transplantation consultation and initiation of a donor search early while undergoing their initial Block 1 therapy. It is recommended that all intermediate-risk patients also undergo transplantation consultation as soon as possible after Block 1 therapy, so that a donor search can be initiated immediately if they are noted to be MRD+ after initial induction. The goal of this protocol is to move to transplantation within 2 weeks of recovery from the final consolidation cycle or completion of Salvage Therapy (Blinatumomab-S). As unrelated donor acquisition can take 8 - 12 weeks, to meet this deadline centers must expedite the search process. Please see Section 7.1c for details of required evaluations.

Patients going on to HSCT will undergo an extensive pre-transplant evaluation to assess remission status, assure adequate organ system function, and document freedom from active viral, bacterial, and fungal infection. Patients should begin their preparative regimen no later than 2 weeks after obtaining the BM aspiration scheduled after recovery from their final consolidation cycle or completion of Salvage Therapy (Blinatumomab-S). If transplantation is delayed by 14 days for donor timing or other reasons, patients may receive up to 6 weeks of bridging maintenance therapy as described in Section 4.10, Appendix II-H. For patients who receive bridging therapy, a repeat BM assessment will be needed to document remission and MRD status within 14 days of starting the HSCT preparative regimen. Patients who are unable to begin the transplant preparative regimen within 8 weeks of initial BM assessment are off protocol therapy.

Patients will receive 1 of 3 designated preparative regimens (cyclophosphamide/total body irradiation (TBI) [cy/TBI] alone or with thiotepa or etoposide). Fludarabine will be added to cy/TBI for cord blood recipients. GVHD prophylaxis varies slightly according to stem cell source.

Patients who are high risk for relapse (MRD+ pre-HSCT with no evidence of GVHD by Day +55, or with + MRD post BMT) are eligible for early taper of immune suppression. The intent of the protocol will be for patients to undergo TBI-based myeloablative conditioning. If patients are not eligible for a myeloablative regimen and either do not undergo HSCT or undergo a reduced intensity procedure, limited data will be collected regarding post transplant survival and relapse.



In the recent COG ASCT0431 trial some variability was allowed in lung shielding with total body irradition. Review of ASCT0431 data showed that lung irradiation doses above 800 cGy were significantly associated with an increased risk of treatment-related mortality and relapse, largely due to toxicity (Pulsipher and Lu, unpublished data November 2014). Accordingly, AALL1331 mandates lung shielding with total body irradiation to limit the lung dose to less than 800 cGy (See Section 14.0 for Radiation Therapy Guidelines).

# 4.9.1.1 Eligibility Criteria for Hematopoietic Stem Cell Transplant (HSCT) Patients who have an appropriately matched stem cell source (see

Section 4.9.1.5) and who meet one of the following criteria:

- 1. Patients with HR relapse:
  - Early (< 36 months) marrow
  - Early (< 18 months) IEM
- 2. Patients with IR relapse with persistent MRD:
  - Late ( $\geq$  36 months) marrow, end-Block 1 MRD  $\geq$  0.1%
  - Late ( $\geq$  18 months) IEM, end-Block 1 MRD  $\geq$  0.1%
- 3. Patients with treatment failure (TF) who achieve a CR after receiving blinatumomab.

NOTE: Patients must maintain an M1 marrow (< 5% blasts) through the BM assessment prior to transplant. (Patients who achieve a remission and relapse prior to HSCT can go to HSCT later, but as they have met a study endpoint (relapse), this procedure will be as per center preference and the patient will only be followed for survival.)

# 4.9.1.2 Exclusion Criteria for Hematopoietic Stem Cell Transplant (HSCT)

Interval development of significant pathology that would preclude HSCT including the following infectious and organ system pathologies:

# 1. <u>Infections</u>

Patients with uncontrolled fungal, bacterial or viral infections are excluded.

Patients acquiring fungal disease during Induction therapy may proceed if they have a significant response to antifungal therapy with no or minimal evidence of active disease remaining by CT evaluation.

# 2. Organ Function Requirements for HSCT

Must meet the criteria for renal, biliary and cardiac function as outlined in Section 3.2.4. In addition, must have adequate pulmonary function defined as an FEV<sub>1</sub>, FVC, and DLCO (corrected for Hgb)  $\geq$  60% by pulmonary function tests (PFTs).

For children who are unable to cooperate for PFTs, the criteria are: no evidence of dyspnea at rest, no exercise intolerance, and not requiring supplemental oxygen therapy.



# 3. Performance Status

Patients must have a performance status corresponding to ECOG scores of 0, 1, or 2. Use Karnofsky for patients > 16 years of age and Lansky for patients  $\le$  16 years of age. Please refer to performance status scale at:

https://members.childrensoncologygroup.org/\_files/protocol/Standard/PerformanceStatusScalesScoring.pdf

### 4.9.1.3 Eligibility for Accelerated Taper of Immune Suppression

- a. Patients who are MRD+ ( $\geq 0.01\%$ ) within 2 weeks of beginning HSCT preparative regimen who do not have any evidence of aGVHD by Day +55 post HSCT (pre-MRD+ group)
- b. Patients who are MRD- (< 0.01%) within 2 weeks of beginning HSCT preparative regimen but are found to be MRD+ ( $\ge 0.01\%$ ) on periengraftment (Day +28-55) or Day +100 marrow who do not have any evidence of aGVHD by Day +55 (peri-engraftment group) or Day +100 (Day +100 group)

# 4.9.1.3.1 Adjustment of TBI/chemotherapy During the Preparative Regimen

The full dose of preparative regimen TBI and chemotherapy agents will be administered unless patients have a life threatening reaction thought likely to occur again with continued administration and an appropriate substitution cannot be made (i.e. etopophos for etoposide).

# 4.9.1.4 Dose Adjustment of Chemotherapy for Patients Whose Weight Exceeds > 125% Ideal Body Weight (IBW)

Chemotherapy given during the preparative regimen (thiotepa, cyclophosphamide, and etoposide) will be dosed based on actual weight for patients  $\leq$  125% IBW. Those > 125% IBW will be dosed based upon adjusted ideal body weight as follows:

Adjusted ideal body weight = IBW + 0.25 (Actual weight – IBW).

The following formulas for pediatric and adult IBW calculations are recommended, but IBW may be calculated according to institutional standard operating procedures (SOPs).

Recommended Ideal Body Weight Calculation for Children Age 1 - 17 years

$$IBW = \underline{Height (cm)^2 \times 1.65}$$

$$1000$$

Recommended Ideal Body Weight Calculation for Adults (Height > 5 feet/60 inches)

IBW (females) =  $(cm \div 2.54 - 60) \times 2.3 \text{ kg} + 45.5 \text{ kg}$ 



IBW (males) = 
$$(cm \div 2.54 - 60) \times 2.3 \text{ kg} + 50 \text{ kg}$$

# 4.9.1.5 Stem Cell Source Requirements

Molecular typing at high resolution of HLA A, B, C, and DRB1 is required, and DQB1 suggested, for all bone marrow or peripheral blood stem cell (PBSC) donors who are either unrelated or related but not matched siblings (i.e. matched parent, partially mismatched sibling, etc.). For matched sibling donors and cord blood units, intermediate level matching of class I antigens is acceptable, but allele level typing is required for DRB1 and encouraged for class I antigens and DQB1.

Hierarchy of stem cell choices is as follows:

- 1) Preferred: Genotypically HLA matched siblings
- 2) If genotypically matched sibling is not available, the following are equally acceptable:
  - a) Unrelated or "other" related (non-genotypically matched) donors must be matched at 8/8 or 7/8 alleles (HLA-A, B, C and DRB1 at high resolution).
  - b) Unrelated cord blood units must be matched at 4/6, 5/6, or 6/6 antigens (HLA A, B [intermediate), and DRB1 [high resolution]). Published data show lower non-relapse mortality when patients receive units matched at 8/8, 7/8, or 6/8 alleles (HLA-A, B, C and DRB1 at high resolution), therefore allele-level typing is strongly encouraged. Use of cords matched at 5/8 or 4/8 alleles leads to more TRM, but are acceptable if better matches are not available. It is recommended that units matching at the 3/8 allele level be avoided if possible. Minimum pre-thaw cell dose of 3x10<sup>7</sup> nucleated cells/kg recipient weight is required. Two cords may be used if this cell dose is not achieved with a single unit. The two units must each match the recipient at a minimum of 4/6 antigens and must match each other at a minimum of 3/6 antigens.

**NOTE:** Centers using unlicensed cord blood must consent the patient on the NMDP cord blood IND protocol or other cord blood IND protocols as appropriate in order to use such units on this study

3) Use of Peripheral Blood Stem Cells (PBSC)

Bone marrow should be requested from allogeneic donors. PBSC is allowed only if the donor is unable or unwilling to give marrow.

4.9.1.5.1 Recommended minimum cell doses:

HPC-M cell dose should be at least 1 x 10<sup>8</sup> TNC/kg HPC-A cell dose should be at least 2 x 10<sup>6</sup> CD34/kg



# 4.9.1.6 Preparative Regimens

Preparative regimens allowed on this protocol are standard regimens used in ASCT0431 for related and unrelated BM/PBSC recipients and BMT CTN 0501 for cord blood recipients. ASCT0431 designated TBI 1200cGy/thiotepa/cyclophosphamide, but also allowed a variation substituting etoposide for thiotepa and a second variation substituting a slightly higher TBI dose (1320cGy) for thiotepa. BMT CTN 0501 used TBI 1320/cyclophosphamide/fludarabine for all patients.

# 4.9.2 Preparative Regimen Administration

# 4.9.2.1 TBI Administration

Fractionated TBI will be administered according to protocol guidelines (see <u>Section 14.5</u> for radiotherapy guidelines). TBI may be delivered from either linear accelerator or Cobalt sources.

# 4.9.2.2 **Thiotepa Administration** (for centers choosing the thiotepa-containing regimen).

- Thiotepa will be administered intravenously over 3 hours. To minimize skin toxicity, frequent bathing (minimum 2 3x daily) is required on the days of thiotepa administration as per center standard.
- See above for dose modification if weight exceeds 125% of IBW

### 4.9.2.3 Cyclophosphamide Administration

- Cyclophosphamide will be administered intravenously over 1-6 hours.
- Hyperhydration, maintenance of significant urine output after administration, and the use of Mesna is required.
- Recommended mesna dosing: 360 mg/m<sup>2</sup> during cyclophosphamide followed by 120 mg/m<sup>2</sup>/hour for 12 hours after each dose. Institutional standards or protocols for mesna administration may also be used.
- See above for dose modification if weight exceeds 125% of IBW

# 4.9.2.4 Etoposide Administration (for centers choosing etoposide regimen)

- Etoposide will be administered intravenously at a maximum infusion rate of 300 mg/m²/hour for a minimum of 5 hours or per institutional standard.
- Patients should be given 1.5X maintenance fluids during etoposide administration to minimize the risk of hypotension.
- Etopophos substitution is allowed.
- See above for dose modification if weight exceeds 125% of IBW

# 4.9.2.5 Fludarabine Administration

- Fludarabine will be administered intravenously over 30 60 minutes each day.
- Fludarabine will not be adjusted for body weight.

# 4.9.3 <u>Preparative Regimen Administration Tables</u>

4.9.3.1 TBI 1200/thiotepa/cyclophosphamide Regimen (related and unrelated BM/PBSC)


| Treatment | Route | Dose | Days | Notes |
|------------------|-------------|-----------|-----------|-------------------|
| TBI | | 200 cGy | Day -8, - | May deliver |
| | | BID | 7, & -6 | 1200 cGy |
| | | | | fractionated TBI |
| | | | | over 4 days per |
| | | | | center preference |
| Thiotepa | IV over 3 | 5 | Day -5 & | |
| | hours daily | mg/kg/day | -4 | |
| Cyclophosphamide | IV over 1-6 | 60 | Day -3 & | |
| | hours daily | mg/kg/day | -2 | |
| Rest | | | Day -1 | |
| Infusion of | | | Day 0 | |
| allogeneic HSCT | | | - | |

# 4.9.3.2 TBI 1200/etoposide/cyclophosphamide Regimen (related and unrelated BM/PBSC)

| Drug/Treatment | Route | Dose | Days | Notes |
|---|---|---|---|---|
| TBI | | 200 cGy | Day -7, - | May deliver |
| | | BID | 6, & -5 | 1200 cGy |
| | | | | fractionated TBI |
| | | | | over 4 days per |
| | | | | center |
| E. 11 | TX 7 | 1500 / 2 | D 4 | preference |
| Etoposide | IV over a | $1500 \text{ mg/m}^2$ | Day -4 | maximum rate |
| | minimum | | | of infusion is |
| | of 5 hours | | | 300 mg/m <sup>2</sup> /hour |
| | or per | | | or per |
| | institutional | | | institutional |
| | standard | | | standard |
| Cyclophosphamide | IV over 1-6 | 60 | Day -3 & | |
| Cyclophosphamide | hours daily | mg/kg/day | -2 | |
| Rest | nours dairy | mg/kg/day | Day -1 | |
| | | | Day -1 | |
| Infusion of | | | Day 0 | |
| allogeneic HSCT | | | | |

# 4.9.3.3 TBI 1320/cyclophosphamide Regimen (related and unrelated BM/PBSC)

| Treatment | Route | Dose | Days | Notes |
|---|---|---|---|---|
| TBI | | 165 cGy | Day -7, -6, -5, & -4 | Total dose must |
| | | BID | -5, & -4 | be |
| | | | | 1320 cCy |
| Cyclophosphamide | IV over | 60 | Day -3 & | |
| | 1-6 | mg/kg/day | - 2 | |
| | hours | | | |
| | daily | | | |
| Rest | | | Day -1 | |
| Infusion of | | | Day 0 | |
| allogeneic HSCT | | | | |



| 4.9.3.4 | TBI 1320/fludarabin | e/cyclophos <sub>l</sub> | phamide Reg | gimen (relateo | d and unrelated |
|---|---|---|---|---|---|
| | cord blood) | | | | |

| Treatment | Route | Dose | Days | Notes |
|---|---|---|---|---|
| Fludarabine | IV over | 25 mg/m <sup>2</sup> /day | Day -10, -9, -8 | |
| | 30 - 60 | | - | |
| | minutes | | | |
| | daily | | | |
| TBI | | 165 cGy BID | Day -7, -6, -5, | Total dose |
| | | | & -4 | must be |
| | | | | 1320 сСу |
| Cyclophosphamide | IV over | 60 mg/kg/day | Day -3 & -2 | |
| | 1-6 | | | |
| | hours | | | |
| | daily | | | |
| Rest | | | Day -1 | |
| Infusion of | | | Day 0 | |
| allogeneic HSCT | | | - | |

## 4.9.4 <u>Sanctuary Site Therapy</u> (see <u>Section 14.0</u>)

Prior to transplant, designated patients with extramedullary relapse must receive cranial or testicular radiotherapy boosting in addition to the doses of TBI associated with the preparative regimen. The cranial boost and/or testicular boosts should be given over 3 days prior to the beginning of TBI.

# 4.9.4.1 Radiotherapy boost for patients with CNS leukemia (CNS3) at relapse:

Patients with CNS3 involvement at the time relapse with or without a history of prior CNS leukemia and/or radiotherapy will receive a cranial radiotherapy boost just prior to TBI (3 doses, maximum 200 cGy daily: total dose to cranial axis = 1800 cGy (unless alternative TBI dose given in which case the dose will be 1920 cGy). If the patient is  $\leq$  3 years at the time of transplant, centers may elect not to give a boost because of developmental concerns. If the patient has CNS1 or CNS2 status at relapse, no boost will be given.

#### 4.9.4.2 Testicular boost for patients with testicular leukemia at relapse:

The only patients that will receive a testicular boost prior to TBI (3 daily doses, 200 cGy fractions, total 600 cGy) are IR/HR/TF patients with extramedullary testicular leukemia at the time of relapse that DID resolve by end Block 1, since those without resolution have already received 2400 cGy of testicular radiation.

# 4.9.4.3 **Prophylactic testicular boosting**:

Prophylactic testicular boosting of 400 cGy for patients without testicular relapse is allowed, but not part of the designated therapy.

## 4.9.5 Growth Factor Administration

Filgrastim (G-CSF) at a dose of 5 micrograms/kg/day given IV or subcutaneously is required for recipients of cord blood starting at Day +1 and continuing until



patients are fully engrafted. G-CSF is generally not necessary for BM/PBSC recipients and is not recommended, unless engraftment is delayed.

#### 4.9.6 GVHD Prophylaxis

GVHD prophylaxis will consist of tacrolimus/methotrexate (TAC/MTX) for recipients of related and unrelated donor BM/PBSC and cyclosporine and mycophenolate mofetil (CYA/MMF) for cord blood recipients. Substitution of CYA for TAC or TAC for CYA according to center preference is allowed.

| Drug | Route* | Dose | Days | Important Notes |
|---|---|---|---|---|
| Drug | Koute | Dosc | Days | important Notes |
| BM Recipient | | | | |
| Tacrolimus | IV | 0.02 mg/kg/day | Begin Day -3 | Target |
| (TAC) | | cont infusion | | concentration |
| | | | | 8 - 12 ng/mL |
| Methotrexate | IV | 5 mg/m <sup>2</sup> sib donor | +1, +3, &+6 | |
| (MTX) | | $10 \text{ mg/m}^2 \text{ URD}^{\wedge}$ | sibs | |
| | | | +1, +3, +6, | |
| | | | +11 URD | |
| Cord Recipient | | | | |
| Cyclosporine A | IV | Varies by age, | Begin Day -3 | Target |
| (CYA) | | adjusted to target | | concentration |
| | | | | 200 - 400 ng/mL |
| Mycophenolate | IV | $\geq$ 50 kg: 1000 mg | Begin Day -3 | |
| mofetil (MMF) | | q8h | | |
| | | < 50kg: 15 mg/kg | | |
| | | q8h | | |

<sup>\*</sup> All drugs may be switched to PO after engraftment when patients are able to tolerate and absorb PO medications.

# 4.9.6.1 Tacrolimus Administration, Monitoring and Dose Adjustments (related or unrelated BM/PBSC)

Tacrolimus should be administered by continuous IV infusion until patients are able to take PO. Serum tacrolimus troughs and serum magnesium, potassium, and creatinine should be drawn at least twice per week while hospitalized, then as per good clinical practice thereafter unless a change in medication (e.g. use of concomitant CYP3A4 inhibitors) or renal function might result in an acute change in level.

At that point, concentrations will be measured as clinically indicated. Concentrations sent when dosing by continuous infusion are not true trough concentrations, however, the same target range of drug concentration will be used for both continuous IV and bolus PO routes of administration.

When converting patients at a therapeutic tacrolimus level from IV to PO formulation, multiply total daily IV dose times 4 and administer in 2 divided oral doses per day, every 12 hours (e.g., 1 mg of IV tacrolimus per

<sup>^</sup> URD, unrelated donor



day equates to 4 mg of PO tacrolimus per day). Younger children (eg. < 6 years of age) may require more frequent PO tacrolimus dosing (every 8 hours) to maintain target trough concentrations. The oral dose should be administered 8 - 12 hours after the end of the tacrolimus continuous infusion. 41

The target serum trough concentration for tacrolimus is 8 - 12 ng/mL. Dose adjustments are based on clinical judgment of the treating physician after considering clinical toxicity, serum levels, GVHD, concomitant drug use and the rate of rise or decline of the serum level.

# 4.9.6.2 Methotrexate Administration, Monitoring and Dose Adjustments (related or unrelated BM/PBSC)

For patients receiving sibling donors, methotrexate should be given at a dose of 5 mg/m<sup>2</sup> on Days +1, 3, and 6 after transplant. For patients receiving unrelated BM or PBSC, methotrexate should be given at a dose of 10 mg/m<sup>2</sup> on Days +1, 3, and 6, and 11. All doses of methotrexate should be administered as scheduled if possible, but centers may modify or hold methotrexate for significant toxicity (see Section 5.8 for methotrexate dose modification guidelines).

#### 4.9.6.3 Leucovorin Administration

Leucovorin may be given at the physician's discretion for patients at risk for methotrexate toxicity. Patients at risk for methotrexate toxicity include those with extravascular fluid collections (ascites, pleural effusions) or with decreased renal function (see Section 5.8).

# 4.9.6.4 Cyclosporine Administration, Monitoring and Dose Adjustments (related and unrelated cord blood)

Cyclosporine should be administered by IV infusion until patients are able to take PO. Cyclosporine levels as well as serum magnesium, potassium, and creatinine levels should be drawn at least twice per week while hospitalized, then weekly or monthly thereafter unless a change in medication (e.g. use of concomitant CYP3A4 inhibitors) or renal function might result in an acute change in level. At that point, levels will be measured as clinically indicated. When converting patients at a therapeutic tacrolimus level from IV to PO formulation, multiply the IV dose times 2.5 if using the modified formulation (i.e., Neoral or Gengraf) or times 3 if using the non-modified formulation (i.e., SandIMMUNE).

The target serum trough concentration for cyclosporine is 200 – 400 ng/mL. Variations in dosing levels based upon laboratory methodology (e.g. tandem mass-spec analysis) allowed. Dose adjustments are based on clinical judgment of the treating physician after considering clinical toxicity, serum levels, GVHD, concomitant drug use and the rate of rise or decline of the serum level.

# 4.9.6.5 Mycophenolate Mofetil (MMF) Administration and Dose Adjustments (related and unrelated cord blood)



MMF should be given at a dose of 1 gram IV q8 hours for patients  $\geq$  50kg or 15 mg/kg IV q8 hours for patients < 50 kg beginning the morning of Day -3. MMF should be given IV until patient can tolerate oral medications. MMF should be dosed upon actual body weight.

The FDA has determined that a REMS (Risk Evaluation and Mitigation Strategy) program is necessary to ensure the benefits of mycophenolate outweigh the risks of first trimester pregnancy loss and congenital malformations associated with mycophenolate use during pregnancy. Mycophenolate REMS is a program to tell doctors, nurses, pharmacists and patients about the risks of taking mycophenolate during pregnancy. The program also contains important information about patient education and reporting details for pregnancy. Please refer to the website for additional information (https://www.mycophenolaterems.com/). If ≤ Grade 1 acute GVHD, MMF will be discontinued by Day +30. For patients with > Grade 1 acute GVHD, the MMF taper will be per institutional protocols. Patients may transition to PO formulations at a 1:1 IV to PO conversion when clinically appropriate. Refer to Section 5.13 for dose adjustments based upon clinical and laboratory findings.

## 4.9.7 Standard Taper of Immune Suppression

This applies to all patients who are MRD negative pre- and at all times post-transplant who have not developed aGVHD requiring systemic therapy. (Patients who develop significant aGVHD will be tapered at the discretion of the transplant center.)

| Drug | Stem Cell Source | Taper Schedule |
|---------------|------------------|----------------------------------------|
| Tacrolimus | Matched Sibling | Start Day +42 over 8 weeks, off by |
| | BM/PBSC | Day +98 |
| Tacrolimus | Unrelated Donor | Start Day +100 off by Day +180 |
| | BM/PBSC | |
| Cyclosporine | Unrelated Cord | Start Day +100 off by Day +180 |
| Mycophenolate | Unrelated Cord | Continue until Day +45 or 7 days after |
| Mofetil | | engraftment, whichever day is later. |
| | | Stop without a taper. |

# 4.9.8 <u>Accelerated Taper of Immune Suppression</u>

See Section 4.9.1 for eligibility requirements.

4.9.8.1 Taper for patients who are MRD positive pre-HSCT with no aGVHD by Day +55 and for patients who are MRD positive > 0.01% by flow cytometry at their peri-engraftment BM test (approx Day +30)

| eytometry at the | n pen engranament | Biti test (approx. Bay 190) |
|------------------|-------------------|--------------------------------------|
| Drug | Stem Cell Source | Taper Schedule |
| Tacrolimus | Matched Sibling | Taper already started by Day +42. At |
| | BM/PBSC | Day +55 increase rate of taper to |
| | | complete taper by Day +70 |
| Tacrolimus | Unrelated Donor | Start Day+55 off by Day +100 |
| | BM/PBSC | |
| Cyclosporine | Unrelated Cord | Start Dav+55 off by Day +100 |



| Mycophenolate | Unrelated Cord | Continue until Day +45 or 7 days after |
|---------------|----------------|----------------------------------------|
| Mofetil | | engraftment, whichever day is later. |
| | | Stop without a taper. |

4.9.8.2 Taper for patients who are MRD negative pre- HSCT with no aGVHD by Day +55 who are MRD positive > 0.01% by flow cytometry at their Day +100 test.

| Drug | Stem Cell Source | Taper Schedule |
|---|---|---|
| Tacrolimus | Matched Sibling<br>BM/PBSC | Taper already started by Day +42 and pt should be off immune suppression. |
| | DW/T BSC | Stop tacrolimus without taper if still on medication. |
| Tacrolimus | Unrelated Donor | Taper over 2-3 weeks as soon as MRD |
| | BM/PBSC | report is received. |
| Cyclosporine | Unrelated Cord | Taper over 2-3 weeks as soon as MRD |
| | | report is received. |
| Mycophenolate | Unrelated Cord | |
| Mofetil | | Should be off this medication. |

# 4.10 Bridging Maintenance Therapy (All HR/IR Patients, as required) – up to 6 weeks

This therapy is for all HR/IR patients who have completed either Blocks 2 and 3 of chemotherapy or both cycles of blinatumomab and due to stem cell source or facility scheduling issues have a lag time > 2 weeks after count recovery prior to starting HSCT therapy. Patients should start bridging therapy when clinically able after meeting count requirements and continue until approximately one week prior to beginning the transplant preparative regimen.

The Therapy Delivery Map (TDM) for Bridging therapy is in Appendix II-H.

## 4.10.1 Criteria to Begin Bridging Maintenance Therapy

Start when peripheral counts recover to ANC  $\geq 500/\mu L$  and platelets  $\geq 50,000/\mu L$ .

## 4.10.2 General Chemotherapy Guidelines

See <u>Section 6.0</u>, Drug Information, and the Parenteral and Oral Chemotherapy Administration Guidelines (CAGs) on the COG website at: <a href="https://members.childrensoncologygroup.org/files/disc/Pharmacy/ChemoAdminGuidelines.pdf">https://members.childrensoncologygroup.org/files/disc/Pharmacy/ChemoAdminGuidelines.pdf</a> for special precautions associated with chemotherapy administration. As applicable, also see the CAGs for suggestions on hydration, or hydrate according to institutional guidelines.

See  $\underline{\text{Section 5.0}}$  for Dose Modifications based on Toxicities and  $\underline{\text{Appendix I}}$  for Supportive Care Guidelines.

Dosing should be based on actual BSA.

## 4.10.3 Bridging Maintenance Chemotherapy Guidelines

<u>VinCRIStine:</u> IV push over 1 minute or infusion via minibag as per institutional policy

Days: 1, 22



Dose: 1.5 mg/m<sup>2</sup>/dose (maximum dose: 2 mg)

# Special precautions: FOR INTRAVENOUS USE ONLY.

The container or the syringe containing vinCRIStine must be enclosed in an overwrap bearing the statement "Do not remove covering until moment of injection. For intravenous use only - Fatal if given by other routes."

Medication errors have occurred due to confusion between vinCRIStine and vinBLAStine. VinCRIStine is available in a liposomal formulation (vinCRIStine sulfate liposomal injection, VSLI, Marqibo®). Use conventional vinCRIStine only; the conventional and liposomal formulations are NOT interchangeable.

## **Mercaptopurine: PO**

Days: 1 - 42

Dose: 75 mg/m²/dose\* once daily

#### Other Considerations:

- \*See <u>Section 5.9</u> for suggested starting dose based on TPMT status (if status is known)
- Mercaptopurine should be taken consistently at the same time every day.
- The liquid or tablet formulation may be used. If using tablets, adjust daily
  dose using the dosing nomogram in <u>Appendix III</u> to attain a weekly
  cumulative dose as close to 525 mg/m²/week as possible

## **Methotrexate: PO**

Days: 1, 8, 15, 22, 29, 36 Dose: 20 mg/m<sup>2</sup>/dose

Administer on an empty stomach (at least 1 hour before or 2 hours after food or drink except water).

## 4.11 Continuation 1/Continuation 2 (All LR Patients) - 8 weeks

The therapy described in this section is for all LR patients in either **Arm C** or **Arm D** and represents therapy given during Continuation 1 and Continuation 2. See <u>Experimental Design Schema</u>.

The therapy delivery map for Continuation 1 and Continuation 2 is in <u>APPENDIX II-I</u>.

#### 4.11.1 Criteria to Begin and During Continuation Therapy

- a. Begin Continuation when ANC  $\geq 500/\mu L$  and platelets  $\geq 50,000/\mu L$ .
- **b.** All Patients should have ANC  $\geq 500/\mu L$  and platelets  $\geq 50,000/\mu L$  prior to starting therapy on Days 22 and 43.
  - If at Day 22 the ANC is  $< 500/\mu L$  and platelets  $< 50,000/\mu L$ , it is permissible to delay the divided dose oral methotrexate (ddMTX) (25 mg/m²/dose for CNS1/2) or ID MTX (for CNS3) by until counts recover.



• If counts are not recovered after one (1) week, then omit the Day 22 ddMTX or ID MTX for this cycle. After counts recover, resume with the Day 29 standard dose MTX.

## 4.11.2 General Chemotherapy Guidelines

See <u>Section 6.0</u>, Drug Information, and the Parenteral and Oral Chemotherapy Administration Guidelines (CAGs) on the COG website at: <a href="https://members.childrensoncologygroup.org/files/disc/Pharmacy/ChemoAdminGuidelines.pdf">https://members.childrensoncologygroup.org/files/disc/Pharmacy/ChemoAdminGuidelines.pdf</a> for special precautions associated with chemotherapy administration. As applicable, also see the CAGs for suggestions on hydration, or hydrate according to institutional guidelines.

See <u>Section 5.0</u> for Dose Modifications based on Toxicities and <u>Appendix I</u> for Supportive Care Guidelines.

Dosing should be based on actual BSA.

## 4.11.3 Continuation 1/Continuation 2 Chemotherapy Guidelines

# Dexamethasone: PO (may be given IV)

Days: 1 - 5

Dose: 3 mg/m²/dose (Total daily dose: 6 mg/m²/day, divided BID)

If using tablets, adjust dose upward to the nearest 0.25 mg. Oral solutions are acceptable and intravenous preparations may be used on a temporary

basis, if needed.

# <u>VinCRIStine:</u> IV push over 1 minute or infusion via minibag as per institutional policy

Day: 1

Dose: 1.5 mg/m<sup>2</sup>/dose (maximum dose: 2 mg)

## Special precautions: FOR INTRAVENOUS USE ONLY.

The container or the syringe containing vinCRIStine must be enclosed in an overwrap bearing the statement "Do not remove covering until moment of injection. For intravenous use only - Fatal if given by other routes."

Medication errors have occurred due to confusion between vinCRIStine and vinBLAStine. VinCRIStine is available in a liposomal formulation (vinCRIStine sulfate liposomal injection, VSLI, Marqibo®). Use conventional vinCRIStine only; the conventional and liposomal formulations are NOT interchangeable.

## Methotrexate: Intrathecal (IT) -CNS1/2 PATIENTS ONLY

Days: 1, 43

#### Age-based dosing:

| Age (yrs) | Dose |
|-----------|-------|
| 1 - 1.99 | 8 mg |
| 2 - 2.99 | 10 mg |
| 3 - 8.99 | 12 mg |
| ≥9 | 15 mg |



When IT therapy and ID MTX are scheduled for the same day, deliver the IT therapy within 6 hours of the beginning of the IV MTX infusion (hour -6 to +6, with 0 being the start of the MTX bolus).

## Triple Intrathecal Therapy (ITT) - CNS3 PATIENTS ONLY

Days: 1, 43

## Age-based dosing:

| Age (yrs) | <u>Dose</u> |
|-----------|------------------------------------|
| 1 - 1.99 | MTX: 8 mg, HC: 8 mg, ARAC: 16 mg |
| 2 - 2.99 | MTX: 10 mg, HC: 10 mg, ARAC: 20 mg |
| 3 - 8.99 | MTX: 12 mg, HC: 12 mg, ARAC: 24 mg |
| ≥ 9 | MTX: 15 mg, HC: 15 mg, ARAC: 30 mg |

When ITT therapy and ID MTX are scheduled for the same day, deliver the ITT therapy within 6 hours of the beginning of the IV MTX infusion (hour -6 to +6, with 0 being the start of the MTX bolus).

# **Mercaptopurine: PO**

Days: 1 - 42

Dose: 75 mg/m<sup>2</sup>/dose\* once daily

#### Other Considerations:

- \*See <u>Section 5.9</u> for suggested starting dose based on TPMT status, if known
- Mercaptopurine should be taken consistently at the same time every day.
- The liquid or tablet formulation may be used. If using tablets, adjust daily dose using the dosing nomogram in <u>Appendix III</u> to attain a weekly cumulative dose as close to 525 mg/m<sup>2</sup>/week as possible

#### Methotrexate: PO

Days: 8, 15, 29, 36 Dose: 20 mg/m²/dose

Administer on an empty stomach (at least 1 hour before or 2 hours after

food or drink except water).

## Divided Dose Methotrexate (dd MTX): PO - CNS1/2 PATIENTS ONLY

Day: 22

Dose:  $25 \text{ mg/m}^2/\text{dose Q6H x 4 doses}$ 

#### Other Considerations:

- ANC must be  $\geq 500/\mu L$  and platelets must be  $\geq 50,000/\mu L$  prior to Day 22 therapy.
- Administer on an empty stomach (at least 1 hour before or 2 hours after food or drink except water).

#### **Leucovorin: PO CNS 1 AND 2 PATIENTS ONLY**

Day: 24

81



Dose: 10 mg/m<sup>2</sup>/dose for 2 doses 6 hours apart beginning 48 hrs after the

START of Day 22 Methotrexate

# **Intermediate Dose Methotrexate (ID MTX):** IV over 36 hours - CNS3 PATIENTS ONLY

Day: 22

Dose: 1000 mg/m<sup>2</sup>/dose

Given as a 100 mg/m<sup>2</sup> bolus over 30 minutes followed by 900 mg/m<sup>2</sup> over

35.5 hours.

Be certain that the ID MTX infusion is completed in the 36 hour period. Even if the infusion is not complete at this time point, it must be stopped.

Leucovorin rescue: See below.

**Suggested hydration and alkalinization for IDMTX:** Prehydrate with D5 ¼ NS with 30 mEq NaHCO3/L at 125 mL/m²/hour to achieve a urine specific gravity  $\leq$  1.010 and pH between 7 and 8. Ringers Lactate may be used as the initial fluid if a bicarbonate containing solution is unavailable. Adjust fluid volume and sodium bicarbonate to maintain urine specific gravity  $\leq$  1.010 and pH between 7 and 8. A bicarbonate bolus (25 mEq/m² over 15 min) may be given to raise the urine pH relatively quickly; a normal saline bolus may also be helpful in facilitating hydration. Continue hydration using D 5 ¼ NS with 30 mEq NaHCO<sub>3</sub>/L at 125 mL/m²/hour throughout IDMTX infusion, and until the last dose of leucovorin has been given. In patients with delayed MTX clearance, continue hydration until the plasma MTX concentration is  $\leq$  0.1 μM.

#### **Timing of ID MTX**

ANC must be  $\geq 500/\mu L$  and platelets must be  $\geq 50~000/\mu L$  prior to ID MTX.

#### Leucovorin: PO/IV CNS 3 PATIENTS ONLY

Days: 24, 25

Dose: 15 mg/m²/dose every 6 hours beginning 48 hrs after the START of ID

MTX infusion.

- If 48 hr methotrexate level is  $\leq 0.5 \mu M$ , do not give more than two doses of leucovorin (48 and 54 hours).
- If MTX level at 48 hours is  $> 0.5~\mu M$ , then continue hydration and leucovorin rescue at 15 mg/m²/dose po/IV every 6 hours until MTX levels are  $< 0.1~\mu M$ .

See Section 5.8 for ID MTX/LCV rescue and infusion guidelines.

Cyclophosphamide: IV over 15 - 30 minutes

Days: 43, 50

Dose: 300 mg/m<sup>2</sup>/dose (see note below)

**Etoposide: IV over 1 - 2 hours** 

Days: 43, 50

Dose: 150 mg/m<sup>2</sup>/dose

82



<u>Note</u>: ANC must be  $\geq 500/\mu L$  and platelets must be  $\geq 50,000/\mu L$  prior to Day 43 therapy. Once the Day 43 cyclophosphamide/etoposide is given, the Day 50 cyclophosphamide/etoposide doses should be given regardless of blood counts (hold only for presumed or proven significant infection).

# **Thioguanine: PO**

Days: 43 - 49.

Dose: 40 mg/m<sup>2</sup>/dose once daily

#### Other Considerations:

- Administer consistently at the same time every day.
- Adjust daily dose using the dosing nomogram in <u>Appendix IV</u> to attain a weekly cumulative dose as close to 280 mg/m<sup>2</sup>/week as possible.
- An oral suspension can also be compounded for patients who cannot swallow pills. The compounded oral suspension is recommended for patients with a BSA between 0.27 and 0.48 m<sup>2</sup>. (see Section 6.18)

# Cytarabine: IV over 1 - 30 minutes or SQ

Days: 44 - 47, 51 -54

Dose: 50 mg/m<sup>2</sup>/dose once daily

## 4.11.4 Following Continuation 1:

- a. LR B-ALL patients randomized to the control arm (**Arm C**) will receive Continuation 2 (<u>Section 4.11</u>, <u>APPENDIX II-I</u>) when ANC  $\geq$  500/ $\mu$ L and platelets  $\geq$ 50,000/ $\mu$ L.
- b. LR B-ALL patients randomized to the experimental arm (**Arm D**) will receive Blinatumomab Block: Cycle 2 (**Arm D**) (<u>Section 4.16</u>, <u>APPENDIX II-N</u>) when ANC  $\geq 500/\mu$ L and platelets  $\geq 50,000/\mu$ L.

## 4.11.5 Following Continuation 2:

- a. LR B-ALL patients randomized to the control arm (Arm C) will receive Maintenance Cycle 1 therapy (Section 4.12, Appendix II-J) when ANC  $\geq 500/\mu L$  and platelets  $\geq 50,000/\mu L$ .
- b. LR B-ALL patients randomized to the experimental arm (**Arm D**) will receive Blinatumomab Block: Cycle 3 (**Arm D**) (Section 4.16, APPENDIX II-N) when ANC  $\geq 500/\mu L$  and platelets  $\geq 50,000/\mu L$ .



#### 4.12 Maintenance Cycle 1 (All LR patients) – 12 weeks

Maintenance Cycle 1 therapy is for common for all LR B-ALL patients randomized to either **Arm C** or **Arm D**. See Experimental Design Schema.

The Therapy Delivery Map (TDM) for Maintenance Cycle 1 is in Appendix II-J.

CNS3 patients ONLY are to be given Chemoradiation (<u>Section 4.13</u>, <u>Appendix II-K</u>) BETWEEN Maintenance Cycle 1 and subsequent Maintenance cycles (Maintenance Post Cycle 1, <u>Section 4.14</u>, <u>Appendix II-L</u>).

All other patients receive **Maintenance-Post Cycle 1 treatment** (Section 4.14, Appendix II-L) immediately following Maintenance Cycle 1.

#### 4.12.1 Criteria to Begin Maintenance Therapy

- Maintenance begins when peripheral counts recover to ANC  $\geq 500/\mu L$  and platelets  $\geq 50,000/\mu L$ , whichever occurs later. This count recovery applies to Maintenance Cycle 1 only.
- For subsequent Maintenance cycles, please follow the dose modifications for low ANC or low platelets (Section 5.9).
- Only oral mercaptopurine and methotrexate will be interrupted for myelosuppression as outlined in <u>Section 5.9</u>. Triple Intrathecal therapy (ITT), vincristine and prednisone will be delivered as scheduled, despite myelosuppression.

#### 4.12.2 Duration of Cycles in Maintenance Therapy

- Maintenance consists of 12 week cycles repeated until total duration of therapy is 2 years from start of Block 1 therapy for both male and female patients.
- Therapy may be stopped on anniversary date if the 5-day dexamethasone is completed for the cycle (i.e. complete all 5 days of dexamethasone before ending therapy). Otherwise continue current cycle through dexamethasone administration.

## 4.12.3 General Chemotherapy Guidelines

See <u>Section 6.0</u>, Drug Information, and the Parenteral and Oral Chemotherapy Administration Guidelines (CAGs) on the COG website at: <a href="https://members.childrensoncologygroup.org/files/disc/Pharmacy/ChemoAdminGuidelines.pdf">https://members.childrensoncologygroup.org/files/disc/Pharmacy/ChemoAdminGuidelines.pdf</a> for special precautions associated with chemotherapy administration. As applicable, also see the CAGs for suggestions on hydration, or hydrate according to institutional guidelines.

See <u>Section 5.0</u> for Dose Modifications based on Toxicities and <u>Appendix I</u> for Supportive Care Guidelines.

Dosing should be based on actual BSA.



#### 4.12.4 <u>Maintenance Chemotherapy Cycle 1</u>

# **Dexamethasone:** PO (may be given IV)

Days: 1 - 5, 29 - 33, & 57 - 61

Dose: 3 mg/m<sup>2</sup>/dose (Total daily dose: 6 mg/m<sup>2</sup>/day, divided BID)

If using tablets, adjust dose upward to the nearest 0.25 mg. Oral solutions are acceptable and intravenous preparations may be used on a temporary

basis, if needed.

# <u>VinCRIStine:</u> IV push over 1 minute or infusion via minibag as per institutional policy

Days: 1, 29, 57

Dose: 1.5 mg/m<sup>2</sup>/dose (maximum dose: 2 mg)

## Special precautions: FOR INTRAVENOUS USE ONLY.

The container or the syringe containing vinCRIStine must be enclosed in an overwrap bearing the statement "Do not remove covering until moment of injection. For intravenous use only - Fatal if given by other routes."

Medication errors have occurred due to confusion between vinCRIStine and vinBLAStine. VinCRIStine is available in a liposomal formulation (vinCRIStine sulfate liposomal injection, VSLI, Marqibo®). Use conventional vinCRIStine only; the conventional and liposomal formulations are NOT interchangeable.

# **Mercaptopurine: PO**

Days: 1 - 84

Dose: 75 mg/m<sup>2</sup>/dose\* once daily

Other Considerations:

- \*See <u>Section 5.9</u> for suggested starting dose based on TPMT status, if known
- Mercaptopurine should be taken consistently at the same time every day.
- The liquid or tablet formulation may be used. If using tablets, adjust daily dose using the dosing nomogram in <u>Appendix III</u> to attain a weekly cumulative dose as close to 525 mg/m²/week as possible

# **Triple Intrathecal Therapy (ITT)** - CNS3 PATIENTS ONLY

Day: 1

Age-based dosing:

| Age (yrs) | <u>Dose</u> |
|-----------|------------------------------------|
| 1 - 1.99 | MTX: 8 mg, HC: 8 mg, ARAC: 16 mg |
| 2 - 2.99 | MTX: 10 mg, HC: 10 mg, ARAC: 20 mg |
| 3 - 8.99 | MTX: 12 mg, HC: 12 mg, ARAC: 24 mg |
| $\geq 9$ | MTX: 15 mg, HC: 15 mg, ARAC: 30 mg |

## Methotrexate: Intrathecal (IT) - CNS1/2 PATIENTS ONLY

Day: 1

Age-based dosing:

| Age (yrs) | Dose |
|-----------|-------|
| 1 - 1.99 | 8 mg |
| 2 - 2.99 | 10 mg |



3 - 8.99 12 mg  $\ge 9$  15 mg

**Methotrexate: PO** 

Days: 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, 78

Dose: 20 mg/m<sup>2</sup>/dose

# 4.12.5 Following Maintenance Cycle 1:

• ONLY CNS3 will receive Chemoradiation (see <u>Section 4.13</u>, <u>APPENDIX II-K</u>) prior to moving on to subsequent Maintenance cycles (Maintenance-Post Cycle 1, <u>Section 4.14</u>, <u>APPENDIX II-L</u>).

• All other patients in both Arm C and Arm D will continue on to **Maintenance-Post Cycle 1** (Section 4.14, APPENDIX II-L).



#### 4.13 Maintenance Chemoradiation - 3 weeks

The CNS-directed therapy described in this section is for LR B-ALL CNS3 Patients ONLY (Patients with late B-ALL isolated CNS3 or CNS3 combined relapse).

The Therapy Delivery Map for this additional CNS-directed therapy during Maintenance is in APPENDIX II-K.

#### 4.13.1 Criteria to Begin Maintenance Chemoradiation

Start when ANC  $\geq 500/\mu L$  and platelets  $\geq 50,000/\mu L$ .

## 4.13.2 <u>Cranial Radiation Therapy</u>

Cranial radiation will be administered during this phase of therapy, which is between the 1<sup>st</sup> and 2<sup>nd</sup> cycles of Maintenance therapy. Patients with CNS3 and isolated CNS relapse will receive 1800 cGy cranial radiation to the brain in 10 daily fractions along with concurrent chemotherapy. See <u>Section 14.1</u> for details on cranial irradiation.

## 4.13.3 General Chemotherapy Guidelines

See <u>Section 6.0</u>, Drug Information, and the Parenteral and Oral Chemotherapy Administration Guidelines (CAGs) on the COG website at: <a href="https://members.childrensoncologygroup.org/files/disc/Pharmacy/ChemoAdminGuidelines.pdf">https://members.childrensoncologygroup.org/files/disc/Pharmacy/ChemoAdminGuidelines.pdf</a> for special precautions associated with chemotherapy administration. As applicable, also see the CAGs for suggestions on hydration, or hydrate according to institutional guidelines.

See <u>Section 5.0</u> for Dose Modifications based on Toxicities and <u>Appendix I</u> for Supportive Care Guidelines.

Dosing should be based on actual BSA.

## 4.13.4 Chemotherapy Guidelines for Maintenance Chemoradiation

# **Dexamethasone:** PO (may be given IV)

Days: 1 - 7, 15 - 21

Dose: 5 mg/m²/dose (Total daily dose: 10 mg/m²/day, divided BID; dose capped

at 40 mg per day)

If using tablets, adjust dose upward to the nearest 0.25 mg. Oral solutions are acceptable and intravenous preparations may be used on a temporary

basis, if needed.

# <u>VinCRIStine:</u> IV push over 1 minute or infusion via minibag as per institutional policy

Days: 1, 8, and 15

Dose: 1.5 mg/m<sup>2</sup>/dose (maximum dose: 2 mg)

#### Special precautions: FOR INTRAVENOUS USE ONLY.

The container or the syringe containing vinCRIStine must be enclosed in an overwrap bearing the statement "Do not remove covering until moment of injection. For intravenous use only - Fatal if given by other routes."



Medication errors have occurred due to confusion between vinCRIStine and vinBLAStine. VinCRIStine is available in a liposomal formulation (vinCRIStine sulfate liposomal injection, VSLI, Marqibo®). Use conventional vinCRIStine only; the conventional and liposomal formulations are NOT interchangeable.

## Pegaspargase: IV over 1-2 hours

Day:

Dose: 2,500 International Units/m<sup>2</sup>/dose

## **Special precautions:**

- 1. Pegaspargase is contraindicated with a history of severe pancreatitis with any prior asparaginase therapy. Caution should be used if serious thrombosis or hemorrhagic events have occurred with any prior asparaginase therapy (see Section 5.1)
- 2. Pegaspargase may affect coagulation factors and predispose to bleeding and/or thrombosis. Caution should be used when administering any concurrent anticoagulant therapy.
- 3. Suggested monitoring during and after administration: Because pegaspargase is long acting, hypersensitivity reactions may not appear for hours after drug administration. Monitor vital signs, for signs of fever, chills, or acute allergic reactions including anaphylaxis. Have medications to treat hypersensitivity reactions readily available at each administration (e.g., epinephrine, IV corticosteroids, antihistamines). Consider prescribing an EpiPen® for home use.

## 4.13.5 Following Maintenance Chemoradiation:

 All patients will continue on to Maintenance-Post Cycle 1 (see Section 4.14, APPENDIX II-L).



## 4.14 Maintenance-Post Cycle 1 (All LR patients)

Maintenance-Post Cycle 1 therapy is common for all LR B-ALL patients randomized to either **Arm C** or **Arm D**. See Experimental Design Schema.

NOTE: CNS3 and Isolated CNS Relapse ONLY are to be given Chemoradiation (see Section 4.13, APPENDIX II-K) between Maintenance Cycle 1 and subsequent Maintenance cycles (Maintenance-Post Cycle 1). All other patients receive Maintenance-Post Cycle 1 immediately following Maintenance Cycle 1.

## 4.14.1 <u>Criteria to Continue Maintenance Therapy</u>

Maintenance continues based on the dose modifications for low ANC or low platelets (see <u>Section 5.9</u>). Only oral mercaptopurine and methotrexate will be interrupted for myelosuppression as outlined in <u>Section 5.9</u>. Triple Intrathecal therapy, vincristine and prednisone will be delivered as scheduled, despite myelosuppression.

# 4.14.2 <u>Duration of Cycles in Maintenance Chemotherapy</u>

- Maintenance consists of 12 week cycles repeated until total duration of therapy is 2 years from start of Block 1 therapy for both male and female patients.
- Therapy may be stopped on anniversary date if the 5 day dexamethasone is completed for the cycle (i.e. complete all 5 days of dexamethasone before ending therapy). Otherwise continue current cycle through dexamethasone administration.

# 4.14.3 General Chemotherapy Guidelines

See <u>Section 6.0</u>, Drug Information, and the Parenteral and Oral Chemotherapy Administration Guidelines (CAGs) on the COG website at: <a href="https://members.childrensoncologygroup.org/files/disc/Pharmacy/ChemoAdminGuidelines.pdf">https://members.childrensoncologygroup.org/files/disc/Pharmacy/ChemoAdminGuidelines.pdf</a> for special precautions associated with chemotherapy administration. As applicable, also see the CAGs for suggestions on hydration, or hydrate according to institutional guidelines.

See <u>Section 5.0</u> for Dose Modifications based on Toxicities and <u>Appendix I</u> for Supportive Care Guidelines.

Dosing should be based on actual BSA.

#### 4.14.4 Chemotherapy Guidelines for Maintenance-Post Cycle 1

Dexamethasone: PO (may be given IV)

Days: 1 - 5, 29 - 33, & 57 - 61

Dose: 3 mg/m<sup>2</sup>/dose (Total daily dose: 6 mg/m<sup>2</sup>/day, divided BID)

If using tablets, adjust dose upward to the nearest 0.25 mg. Oral solutions are acceptable and intravenous preparations may be used on a temporary basis, if needed.



# <u>VinCRIStine:</u> IV push over 1 minute or infusion via minibag as per institutional policy

Days: 1, 29, 57

Dose: 1.5 mg/m<sup>2</sup>/dose (maximum dose: 2 mg)

## Special precautions: FOR INTRAVENOUS USE ONLY.

The container or the syringe containing vinCRIStine must be enclosed in an overwrap bearing the statement "Do not remove covering until moment of injection. For intravenous use only - Fatal if given by other routes."

Medication errors have occurred due to confusion between vinCRIStine and vinBLAStine. VinCRIStine is available in a liposomal formulation (vinCRIStine sulfate liposomal injection, VSLI, Marqibo®). Use conventional vinCRIStine only; the conventional and liposomal formulations are NOT interchangeable.

## Mercaptopurine: PO

Days: 1 - 84

Dose: 75 mg/m<sup>2</sup>/dose\* once daily

#### Other Considerations:

- \*See <u>Section 5.9</u> for suggested starting dose based on TPMT status (if status is known)
- Mercaptopurine should be taken consistently at the same time every day.
- The liquid or tablet formulation may be used. If using tablets, adjust daily dose using the dosing nomogram in <u>Appendix III</u> to attain a weekly cumulative dose as close to 525 mg/m²/week as possible

## **Methotrexate: PO - CNS3 PATIENTS ONLY**

Day:

Dose: 20 mg/m<sup>2</sup>/dose

#### **Methotrexate: Intrathecal (IT) - CNS1/2 PATIENTS ONLY**

Day:

Age-based dosing:

| <u>Dose</u> |
|-------------|
| 8 mg |
| 10 mg |
| 12 mg |
| 15 mg |

#### **Methotrexate: PO**

Days: 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, 78

Dose:  $20 \text{ mg/m}^2/\text{dose}$ 



## 4.15 Blinatumomab Block: Cycle 1 (Patients in Arm D) - 5 weeks

The therapy described in this section is for the 1<sup>st</sup> cycle of therapy with Blinatumomab on **Arm D**. See Experimental Design Schema.

The Therapy Delivery Map (TDM) for the Blinatumomab Block: Cycle 1 (Arm D) is in APPENDIX II-M.

**NOTE:** Hospitalization is STRONGLY recommended during the first 9 days of this cycle in case of a cytokine reaction. Manifestations of cytokine release syndrome include fever, headache, nausea, asthenia, hypotension, increased alanine aminotransferase, increased aspartate aminotransferase, increased total bilirubin, and disseminated intravascular coagulation (DIC). Corticosteroids should be administered for severe or life threatening cytokine release syndrome.

## Blinatumomab infusion interruptions for technical reasons:

The drug administration should not be interrupted, if possible. In case of infusion interruption due to any technical or logistic reason the interruption should be as short as possible and the infusion continued at the earliest time possible. Every interruption longer than one hour should be documented. If the interruption is longer than four hours, re-start of the infusion should be performed in the hospital, under supervision of the investigator. The patient should be observed overnight for possible side effects after the re-start in the hospital and can be discharged the following day if no difficulties arise. Administration of the premedication (dexamethasone) described in Section 4.5.4, is recommended. If possible, the infusion time before and after a break should sum up to 28 days treatment per cycle.

#### 4.15.1 Criteria to Begin Blinatumomab

Start when ANC  $\geq 500/\mu L$  and platelets  $\geq 50,000/\mu L$ 

# 4.15.2 General Chemotherapy Guidelines

See <u>Section 6.0</u>, Drug Information, and the Parenteral and Oral Chemotherapy Administration Guidelines (CAGs) on the COG website at: <a href="https://members.childrensoncologygroup.org/files/disc/Pharmacy/ChemoAdminGuidelines.pdf">https://members.childrensoncologygroup.org/files/disc/Pharmacy/ChemoAdminGuidelines.pdf</a> for special precautions associated with chemotherapy administration. As applicable, also see the CAGs for suggestions on hydration, or hydrate according to institutional guidelines.

See <u>Appendix VII-A</u> for the management options of blinatumomab in the outpatient setting.

See <u>Section 5.0</u> for Dose Modifications based on Toxicities and <u>Appendix I</u> for Supportive Care Guidelines.

Dosing should be based on actual BSA. There is no maximum dosing.



## 4.15.3 Blinatumomab Block: Cycle 1 (Patients in Arm D) Chemotherapy

# Blinatumomab: IV; Continuous Infusion over 28 days\*

Days: 1 - 28

Dose: 15 micrograms/m<sup>2</sup>/day

# \*IV bag will be changed every 24 - 96 hours or every 168 hours (7 days), depending on the details of the infusion preparation

# Dexamethasone: PO/IV

Day:

Dose: Prior to day 1 therapy -

• A single dose of 5 mg/m²/dose (maximum 20 mg/dose) will be administered 30 to 60 minutes prior to the start of the blinatumomab infusion and when restarting an infusion after an interruption of 4 or more hours in the first cycle.

If using tablets, adjust dose upward to the nearest 0.25 mg. Oral solutions are acceptable and intravenous preparations may be used on a temporary basis, if needed

# **Methotrexate: Intrathecal (IT)** - CNS1/2 PATIENTS ONLY

Day: 8, 29 Age-based dosing:

| Age (yrs) | <u>Dose</u> |
|-----------|-------------|
| 1 - 1.99 | 8 mg |
| 2 - 2.99 | 10 mg |
| 3 - 8.99 | 12 mg |
| $\geq$ 9 | 15 mg |

# Triple Intrathecal Therapy (ITT) - CNS3 PATIENTS ONLY

Days: 8, 29

Age-based dosing:

| Age (yis) | Dose |
|-----------|------------------------------------|
| 1 - 1.99 | MTX: 8 mg, HC: 8 mg, ARAC: 16 mg |
| 2 - 2.99 | MTX: 10 mg, HC: 10 mg, ARAC: 20 mg |
| 3 - 8.99 | MTX: 12 mg, HC: 12 mg, ARAC: 24 mg |
| ≥9 | MTX: 15 mg, HC: 15 mg, ARAC: 30 mg |

#### 4.15.4 Following Blinatumomab Block: Cycle 1 (Arm D)

The next phase of therapy is Continuation 1 (Section 4.11, APPENDIX II-I).



## 4.16 Blinatumomab Block: Cycle 2/3 (LR Patients in Arm D) - 5 weeks

The therapy described in this section is therapy given during Blinatumomab Block Cycle 2 and Blinatumomab Block Cycle 3. Do not start Blinatumomab Cycle 2 before Day 56 after beginning of Continuation 1. Do not start Blinatumomab Cycle 3 before Day 56 after beginning of Continuation 2. See Experimental Design Schema.

**NOTE:** Hospitalization is STRONGLY recommended during the first 2 days of these cycles in case of a cytokine reaction. Manifestations of cytokine release syndrome include fever, headache, nausea, asthenia, hypotension, increased alanine aminotransferase, increased aspartate aminotransferase, increased total bilirubin, and disseminated intravascular coagulation (DIC). Corticosteroids should be administered for severe or life threatening cytokine release syndrome.

The Therapy Delivery Map (TDM) for the Blinatumomab Block: Cycle 2/3 (Arm D) is in APPENDIX II-N.

#### Blinatumomab infusion interruptions for technical reasons:

The drug administration should not be interrupted, if possible. In case of infusion interruption due to any technical or logistic reason the interruption should be as short as possible and the infusion continued at the earliest time possible. Every interruption longer than one hour should be documented. If the interruption is longer than four hours, re-start of the infusion should be performed in the hospital, under supervision of the investigator. The patient should be observed overnight for possible side effects after the re-start in the hospital and can be discharged the following day if no difficulties arise. If possible, the infusion time before and after a break should sum up to 28 days treatment per cycle.

# 4.16.1 <u>Criteria to Begin Blinatumomab Block: Cycle 2/3</u> Start when ANC > 500/μL and platelets > 50,000/μL

#### 4.16.2 General Chemotherapy Guidelines

See Section 6.0, Drug Information, and the Parenteral and Oral Chemotherapy Administration Guidelines (CAGs) on the COG website at: <a href="https://members.childrensoncologygroup.org/files/disc/Pharmacy/ChemoAdminGuidelines.pdf">https://members.childrensoncologygroup.org/files/disc/Pharmacy/ChemoAdminGuidelines.pdf</a> for special precautions associated with chemotherapy administration. As applicable, also see the CAGs for suggestions on hydration, or hydrate according to institutional guidelines.

See <u>Appendix VII-A</u> for the management options of blinatumomab in the outpatient setting.

See <u>Section 5.0</u> for Dose Modifications based on Toxicities and <u>Appendix I</u> for Supportive Care Guidelines.

Dosing should be based on actual BSA. There is no maximum dosing.

## 4.16.3 Blinatumomab Block: Cycle 2/3: Chemotherapy Guidelines

<u>Blinatumomab</u>: IV; Continuous Infusion over 28 days\* Days: 1 - 28



Dose: 15 micrograms/m<sup>2</sup>/day

\*IV bag will be changed every 24 - 96 hours or every 168 hours (7 days), depending on the details of the infusion preparation (<u>NOTE</u>: Administration of the premedication (dexamethasone) is NOT RECOMMENDED for the second or third cycle of blinatumomab.)

# 4.16.4 Following Blinatumomab Block Cycle 2:

LR B-ALL patients randomized to the experimental arm (**Arm D**) will receive Continuation 2- (Section 4.11, APPENDIX II-I)

# 4.16.5 Following Blinatumomab Block Cycle 3:

LR B-ALL patients randomized to the experimental arm (**Arm D**) will receive Maintenance Cycle 1 therapy- (Section 4.12, Appendix II-J.)



#### 5.0 DOSE MODIFICATIONS FOR TOXICITIES

Notify the Study Chair at the time of removing a patient from protocol therapy for toxicity. The drugs are listed in alphabetical order.

# 5.1 Asparaginase [Pegaspargase (PEG-Asparaginase) or Erwinia]

## Systemic Allergic Reactions/Anaphylaxis:

For severe allergic reaction, discontinue pegaspargase and substitute *Erwinia*. Erwinia therapy should begin within 72 hours of the pegaspargase reaction or as soon as possible. Erwinia dosing: 25,000 international units (IU)/m² IM M-W-F for six doses substituted for each dose of pegaspargase. If Erwinia is given IV it should be given as a 1-2 hour infusion. Note that the M-W-F schedule documenting acceptable activity was established using IM not IV Erwinia; thus consideration should be given to administer IV Erwinia at the above dose every other day for 2 weeks (7 total doses).

For mild-moderate reversible reaction:

1. If the infusion was completed, consider sending an asparaginase activity level. Note that a therapeutic level of asparaginase of at least 0.1 IU/mL 14 days after administration is considered therapeutic. Please see the table below for guidance on using levels to switch to Erwinia asparaginase. Management decisions for levels obtained on other days are up to the treating physician.

| Time point after completion of pegaspargase infusion | Asparaginase activity level | Action |
|---|---|---|
| 1 hour – 1 day | < 0.5 IU/mL | Substitute <i>Erwinia</i> asparaginase |
| 7 days | < 0.3 IU/mL | Substitute <i>Erwinia</i> asparaginase |
| 14 days | < 0.1 IU/mL | Substitute Erwinia asparaginase |

2. If the infusion was discontinued early, consider re-challenging with pegaspargase after premedication and send asparaginase levels as above.

Premedication with antihistamines in the absence of prior hypersensitivity has been discouraged in the past since antihistamine use may mask the appearance of systemic allergy and fail to alert the provider of the presence of asparaginase neutralizing antibodies. The use of asparaginase activity assays, as described above, are commercially available and may help determine if neutralizing antibodies are present.

If there is a question of silent inactivation, check levels as described above between 1 hour and 7 days after the dose. Change to Erwinia based on activity levels described above. Of note, Erwinia asparaginase is recommended only for pegaspargase hypersensitivity reactions and/or in the presence of silent antibody. It is not recommended as a substitute for pancreatitis, hepatitis, coagulation abnormalities, or other non-hypersensitivity toxicities associated with pegaspargase. To best suit the needs of each individual patient, additional modifications to these recommendations may be made at the discretion of the treating physician.

<u>Coagulopathy</u>: If symptomatic, hold asparaginase until symptoms resolve, then resume with the next scheduled dose. Consider factor replacement (FFP, cryoprecipitate, factor VIIa). Do not withhold dose for abnormal laboratory findings without clinical symptoms.

<u>Hyperbilirubinemia</u>: asparaginase may need to be withheld in patients with an elevated direct bilirubin, since asparaginase has been associated with hepatic toxicity. No specific



dose adjustment guidelines are provided in the manufacturer's labeling. Below are proposed dose adjustment guidelines from published literature:  $\frac{42}{3}$ 

| Direct Bilirubin | Dose Modification |
|---|---|
| $\leq$ 3.0 mg/dl | Full dose |
| 3.1 - 5.0 mg/dl | Hold pegaspargase and resume when direct bilirubin is < 2 mg/dl; consider |
| | switching to alternate asparaginase product |
| >5.0 mg/dl | Hold the dose of pegasparagase; do not substitute other asparaginase products; |
| | do not make up the missed dose |

Hyperglycemia: Do not modify dose. Treat hyperglycemia as medically indicated.

Hyperlipidemia: Do not modify dose

<u>Ketoacidosis</u>: Hold asparaginase until blood glucose can be regulated with insulin.

<u>Pancreatitis</u>: Discontinue asparaginase in the presence of Grade 3 or 4 pancreatitis. In the case of asymptomatic Grade 2 pancreatitis (enzyme elevation or radiologic findings only), asparaginase should be held until symptoms and signs subside, and amylase/lipase levels return to normal and then resumed.

<u>Thrombosis (including CNS and non-CNS events)</u>: Withhold asparaginase until resolved, and treat with appropriate antithrombotic therapy and consider repletion of AT-III, as indicated. Upon resolution of symptoms consider resuming asparaginase, while continuing low molecular weight heparin (LMWH) or antithrombotic therapy. Do not withhold dose for abnormal laboratory findings without clinical correlate. Consider measurement and repletion of AT-III during subsequent courses of asparaginase if unable to achieve therapeutic Anti-Xa levels. For significant thrombosis, which is not catheter-related, consider evaluation for inherited predisposition to thrombosis.

#### 5.2 Blinatumomab

The most frequent serious adverse events noted in patients treated with blinatumomab to date are disorders of the nervous system, both peripheral and central, and systemic cytokine release syndrome (CRS), though both are less likely to occur in patients with lower burden of disease at the time of administration. Both categories of events are more likely to occur within the first week of treatment with blinatumomab, and both categories of events are usually reversible and able to be managed with attentive supportive care.

AEs related to blinatumomab that require treatment interruption (according to table below) and do not resolve to CTCAE  $\leq$  Grade 1 within 14 days will require permanent discontinuation of blinatumomab treatment. If the patient is otherwise eligible to continue protocol therapy (standard chemotherapy and/or HSCT), then the patient may, at the discretion of the investigator and family, continue to receive protocol therapy.

In the case that the AE(s) **DO resolve within 14 days**, blinatumomab treatment may resume at a **reduced dose of 5 mcg/m<sup>2</sup>/day** to complete the 28 day course (not counting the duration of treatment interruption). **NOTE**: **For Grade 4 Central Nervous** 



# System/Psychiatric, Grade 4 thromboembolic or Grade 4 CRS AEs, blinatumomab must be permanently discontinued.

For patients who had experienced a  $\geq$  Grade 2 Neurologic Systems and Psychiatric AE related to blinatumomab, no dose escalation beyond 5 mcg/m²/day will be permitted for subsequent cycles. For patients who experienced other AEs related to blinatumomab, subsequent cycles will begin at the reduced dose of 5 mcg/m²/day, but may escalate to 15 mcg/m²/day after 7 days if there are no significant blinatumomab-related AEs.

A second occurrence of the same AE that requires interruption will require permanent discontinuation of blinatumomab. If the patient is otherwise eligible to continue protocol therapy (standard chemotherapy, and or HSCT), then the patient may, at the discretion of the investigator and family, continue to receive protocol therapy.

The resumption of the infusion at the reduced dose should be accompanied by **dexamethasone premedication** as indicated in the relevant subsection of <u>Section 4.0</u>, and should be performed in the hospital under supervision of the investigator. Patients should be observed for at least 72 hours after the start of the next infusion at the reduced dose before considering discharge to the outpatient setting.

**Table: Dose modifications for Adverse Events (AE) Possibly, Probably or Definitely Related to Blinatumomab:** 

| Category: AE<br>(CTCAE v4.03) | AE<br>Grade | Stop<br>Infusion? | Supportive<br>Care (in<br>addition to<br>institutional<br>guidelines)* | Restart<br>allowed (with<br>dex premeds)<br>if<br>Gr 1 within<br>14 days? | Restarting<br>dose<br>(mcg/m²/day) | Escalation to 15 mcg/m2/day after 7 days (with dex premed) in subsequent cycle allowed? |
|---|---|---|---|---|---|---|
| Nervous system/ | 1 | N | CNS | - | - | - |
| Psychiatric <sup>1</sup> : (Confusion, Hallucination, Delerium, | 2 | N | CNS | - | - | - |
| Psychosis), Dysarthria, | 3 | Y | CNS, DEX | Y | 5 | N |
| Tremor | 4 | Y | CNS, DEX | N | - | - |
| Central Nervous system: | 1, 2, 3 | Y | SZ, CNS, DEX | Y | 5 | N |
| Seizure | 4 | Y | SZ, CNS, DEX | N | - | - |
| | 1 | N | - | - | - | - |
| Immune system: Cytokine release syndrome- NOTE that it is NOT recommended to use the CTCAE grading <sup>3</sup> | 2 | N, unless<br>patient is<br>unable to<br>tolerate<br>symptoms<br>(e.g. due<br>to other<br>comorbidi<br>ties) | TOCI,DEX<br>only if patient is<br>unable to<br>tolerate<br>symptoms (e.g.<br>due to other<br>comorbidities) | Y | 5 | Y |
| | 3 | Y | TOCI, DEX | Y | 5 | Y |
| | 4 | Y | DEX | N | - | - |



| Blood and lymphatic<br>system <sup>4</sup> : Disseminated<br>intravascular | 1, 2 | N | - | - | - | - |
|---|---|---|---|---|---|---|
| coagulation, hemolysis, hemolytic uremic syndrome, thrombotic thrombocytopenic purpura | 3, 4 | Y | - | Y | 5 | Y |
| Blood and lymphatic<br>system <sup>5</sup> : All others<br>(lymphopenia,<br>neutropenia, anemia,<br>thrombocytopenia, etc.) | 1, 2, 3, 4 | N | - | | - | - |
| 77 1 | 1 | N | - | - | - | - |
| Vascular: Thromboembolic event | 2, 3 | Y | - | Y | 5 | Y |
| i momocemoone event | 4 | Y | - | N | - | - |
| Investigations <sup>6,7</sup> Metabolism and Nutrition: All (if not considered clinically relevant or responding to routine medical management) | 1, 2, 3, 4 | N | - | - | - | - |
| Investigations <sup>6,7</sup> Metabolism and Nutrition: All | 1,2 | N | 1 | 1 | 1 | - |
| (if clinically relevant<br>and not responding to<br>routine medical<br>management) | 3,4 | Y | - | Y | 5 | Y |
| | 1,2 | N | - | - | - | - |
| All other AE | 3,4 | Y | - | Y | 5 | Y |

## **Table Footnotes:**

- Most neurologic AEs associated with blinatumomab are central in nature (e.g. dysarthria, encephalopathy, tremor). Peripheral neurologic AEs are very unlikely to be secondary to blinatumomab, and are far more likely to be secondary to other causes such as vincristine. Discontinuation of blinatumomab secondary to peripheral neurologic AEs should be avoided when possible. Most AEs in the psychiatric disorders category are unlikely to be caused by blinatumomab and generally require supportive care rather than dose modification or discontinuation of blinatumomab (e.g., Insomnia, Depression, Anxiety). Psychiatric AEs that may reflect underlying central nervous system toxicity (e.g., Confusion, Delirium, Hallucinations, Psychosis) are of greater interest, particularly if accompanied by other AEs in the nervous system disorders category.
- <sup>2</sup> Close monitoring of fluid status by intake and output should be undertaken for the first 48 hours of blinatumomab infusion. Efforts to keep patients balanced between intake and output should be maintained, even if diuretic therapy (furosemide or similar) is needed to do this. Careful attention to fluid status may prevent deterioration from capillary leak, however even with meticulous attention some patients may experience pulmonary edema and require more aggressive respiratory support. Treating physicians should use their clinical judgment and institutional standards for whatever supportive care measures are needed during this period of time.



Grading of cytokine release syndrome (CRS) severity should be performed according to that of Lee et al (see below table). As many of the symptoms of CRS overlap with those of other medical complications such as infection, attribution should be carefully considered. Accurate application of this grading system requires clinical judgment to confirm that the symptoms are most likely due to CRS rather than to another medical condition. In all grades of CRS, aggressive supportive care is required. In grade 2 or 3 CRS, careful monitoring of cardiac function is strongly suggested.

| Grade 1 | Symptoms are not life threatening and require symptomatic treatment only, eg. fever, nausea, fatigue, headache |
|---|---|
| Grade 2 | Symptoms require and respond to moderate intervention |
| | Oxygen requirement <40%, or |
| | Hypotension responsive to fluids or low dose of one vasopressor, or |
| | Grade 2 organ toxicity |
| Grade 3 | Symptoms require and respond to aggressive intervention |
| | Oxygen requirement >=40%, or |
| | Hypotension requiring high dose of one vasopressor or multiple vasopressors, or |
| | Grade 3 organ toxicity or grade 4 transaminitis |
| Grade 4 | Life-threatening symptoms |
| | Requirement for ventilator support, or |
| | Grade 4 organ toxicity (excluding transaminitis) |

- <sup>4</sup> In the first days of treatment, transient DIC-like pictures may develop. Because patients are at risk for capillary leak syndrome and cytokine release syndrome, appropriate supportive care with dexamethasone (described above), blood products and factors (packed red cells, platelets, cryoprecipitate, fresh frozen plasma), vitamin K, and/or albumin should be considered according to institutional standards of care. Particularly in the first week of infusion, when the risk of capillary leak and cytokine release is more prominent, appropriate use of blood products and factors is preferred if laboratory indications suggest the need for replacement, as large volumes of crystalloid fluids tend to exacerbate the capillary leak.
- <sup>5</sup> In the first days of treatment, a rapid transient drop in platelets, neutrophils and/or hemoglobin may be observed. These effects are not necessarily cytokine-mediated. Counts typically recover to baseline during treatment, and usually within two weeks of starting blinatumomab. Transfusion of blood and platelets should be performed according to appropriate institutional standards.
- <sup>6</sup> In the first days of treatment, transient increases in transaminases up to over 1000 U/L may develop. These have generally returned to baseline in the 1st week of treatment.
- Decrease in serum immunoglobulins have been observed in patients treated with blinatumomab. Intravenous immunoglobulin should be administered according to institutional standards, but is recommended for any patient with a total IgG level below 400. Immunoglobulin must not be administered through the line through which blinatumomab is actively being infused.
- \* Definitions of supportive care abbreviations:

**DEX**: Given its potential to interfere with the efficacy of blinatumomab, the use of dexamethasone should be reserved for serious side effects that are unresponsive to other treatments (supportive care, discontinuation of blinatumomab infusion, tocilizumab) and for clinically significant neurologic toxicity. If required, dexamethasone should be administered at a total daily dose of at least 0.2 - 0.4 mg/kg/day (maximum 24 mg per day) administered preferably intravenous divided 3 - 4 times daily for at least 1 day but no more than 4 days. The dose should then be stopped or tapered as clinically indicated.

99



**SZ**: Appropriate imaging should be performed to evaluate for possible hemorrhage or thrombosis, and other diagnostic procedures should be performed as clinically appropriate. Prophylactic anticonvulsant treatment with a therapeutic dose of institutional standard agents (e.g., lorazepam, phenytoin, levetiracetam) should be administered if seizures develop, and continued throughout the blinatumomab infusion. Anti-convulsant therapy should be considered starting at least 24 - 48 hours prior to any subsequent blinatumomab infusions, and continuing for the remainder of those treatment cycles. Diagnostic measures to exclude potential infectious causes should be conducted once the patient has stabilized (i.e., a lumbar puncture to evaluate for bacterial, viral or fungal sources should be performed). Any identified pathology should be treated as clinically appropriate.

CNS: A daily finger-nose-finger or writing sample test is recommended according to age-appropriate activities for patients. In adults treated with blinatumomab, it has been found that a daily handwriting sample can often predict future nervous system toxicity before the clinical toxicity develops. Dexamethasone should be used for clinically significant neurologic toxicity. In case of a change in finger-nose-finger or handwriting test it is recommended to start dexamethasone on the schedule above to prevent possible deterioration of nervous system toxicity. Patients who experience nervous system toxicity in the first cycle typically do not experience it again in subsequent cycles, although it is possible.

**TOCI**: In patients with CRS who respond to tocilizumab, fever and hypotension often resolve within 6 hours, and pressors and other supportive care measures can be weaned quickly thereafter. In some cases, however, symptoms may not completely resolve, and continued aggressive support may be necessary for several days. If the patient's condition does not improve or stabilize within 24 hours of the tocilizumab dose, administration of a second dose of tocilizumab and/or a second immunosuppressive agent, such as dexamethasone, should be considered. Tocilizumab is generally not used in the management of CNS symptoms without significant hemodynamic instability or other life-threatening symptomatology.

# **TOCI Suggested Dosing:**

<30 kg: 12 mg/kg</li>≥30 kg: 8 mg/kg

## 5.3 Cyclophosphamide

Gross Hematuria: Omit in the presence of macroscopic hematuria.

Microscopic hematuria: Begin pre-hydration as in the treatment section of the protocol. Increasing the rate and duration of post-hydration should be considered (eg., 200 mL/m²/hr x 12-24 hours). Give IV mesna at a total dose that is 100% of the cyclophosphamide dose divided to 5 doses. Give the first mesna dose 15 minutes before or at the same time as the cyclophosphamide dose and repeat at Hours 3, 6, 9 and 12 after the start of cyclophosphamide. This total daily dose of mesna can also be administered as IV continuous infusion. The continuous infusion should be started 15 - 30 minutes before or at the same time as cyclophosphamide and finished no sooner than 12 hours after the start of cyclophosphamide infusion. If the child develops gross hematuria, continue mesna infusion for 24 hours from the start of the cyclophosphamide infusion.

<u>Renal Dysfunction</u>: If creatinine clearance or radioisotope GFR is < 10 mL/min/1.73 m<sup>2</sup>, reduce dose of cyclophosphamide by 50%. Prior to dose adjustment of cyclophosphamide, the creatinine clearance should be repeated with good hydration.



# 5.4 Cytarabine (ARAC)

<u>Cytarabine Syndrome</u>: Do not withhold cytarabine for fever if it is likely to have been caused by the cytarabine. Obtain blood cultures if a central line is present.

For rash or conjunctivitis, withhold for Grade 3 - 4 toxicity until resolved. Make up missed doses and consider concurrent treatment with hydrocortisone or dexamethasone, and/or with dexamethasone ophthalmic drops for conjunctivitis.

<u>Myelosuppression:</u> Do not interrupt high dose (3,000 mg/m²/dose) cytarabine, once started, for uncomplicated myelosuppression; do hold for proven or presumed serious infection and do not make up missed doses during Block 3.

Once Continuation 1 and 2 have started, do not interrupt for uncomplicated myelosuppression; do hold for proven or presumed serious infection.

<u>Stipulations for High Dose Cytarabine</u>: Adequate renal function (defined as creatinine within normal range) is required for the administration of high dose (3,000 mg/m²/dose) cytarabine. Creatinine clearance (CrCl) should be measured for patients with elevated creatinine or suspected renal insufficiency. For CrCl < 60 mL/min/1.73 m², hold pending recovery and omit if CrCl < 30 mL/min/1.73 m² or if recovery requires > 3 weeks.

<u>Neurotoxicity</u>: Discontinue cytarabine immediately for  $\geq$  Grade 2 CNS toxicity, (e.g., ataxia, nystagmus, dysarthria, dysmetria, seizures and/or encephalopathy).

#### 5.5 Anthracycline-Mitoxantrone

Consider Dexrazoxane prior to each dose for patients with:

- Anticipated cumulative anthracycline dose >150 mg/m<sup>2</sup>.
- Past or anticipated radiotherapy including the myocardium (including whole-abdomen or left flank irradiation).
- Recommended dose of dexrazoxane is 10 x the DAUNOrubicin/DOXOrubicin dose or 30 x the mitoXANtrone dose, given over 5-15 minutes immediately before the chemotherapeutic agent.

#### Monitoring Cardiac Echocardiogram:

At baseline and then recommended after cumulative dose of 175, 300, 375, and 450 mg/m<sup>2</sup>.

## Dose modification for cardiac toxicity:

If left ventricular ejection fraction (EF) < 50% (as determined by the Biplane Simpson method), or if EF inevaluable shortening fraction (SF) < 24%, hold the anthracycline or anthracenedione and repeat the echocardiogram in one week. If EF remains < 50% (or if EF inevaluable, SF < 24%), discontinue the anthracycline or anthracenedione and deliver alternate therapy as per the protocol or provider decision. Resuming cardiotoxic therapy depends on the cause of the cardiac dysfunction and the results of further cardiac evaluation.

#### Myelosuppression (beyond Induction):

If patient has severe infection or severe mucositis, consider modifying or omitting



anthracycline.

Hyperbilirubinemia:

| Direct Bilirubin | Dose Adjustment |
|---|---|
| $\leq$ 3.0 mg/dl | Full dose |
| 3.1 - 5.0 mg/dl | Administer 50% of calculated dose |
| 5.1 - 6.0 mg/dl | Administer 25% of calculated dose |
| > 6.0 mg/dl | Withhold dose and administer next scheduled dose if toxicity has resolved. Do |
| | not make up missed doses. |

#### **Extravasation:**

In the event of an extravasation, discontinue the IV administration of the drug and institute appropriate measures to prevent further extravasation and damage according to institutional guidelines. Also, see <a href="https://cogmembers.org/files/disc/pharmacy/ExtravasationReference.pdf">https://cogmembers.org/files/disc/pharmacy/ExtravasationReference.pdf</a> for COG reference.

## 5.6 **Etoposide**

Allergic Reaction: Premedicate with diphenhydramine (1-2 mg/kg slow IV push, maximum dose is 50 mg). If symptoms persist, add hydrocortisone 100-300 mg/m². Continue to use premedication before etoposide in future. Also consider substituting an equimolar amount of etoposide phosphate, in the face of significant allergy and/or hypotension. Etoposide phosphate is a water soluble prodrug that does not contain polysorbate 80 and polyethyleneglycol, the solubilizing agent in etoposide that may induce allergic reactions and hypotension. Etoposide phosphate is rapidly converted to etoposide *in vivo* and provides total drug exposure, as represented by AUC (0-infinity), that is statistically indistinguishable from that measured for etoposide at equimolar doses.

<u>Hypotension</u>: If diastolic or systolic blood pressure (BP) falls 20 mm Hg during infusion, reduce infusion rate by 50%. Start a simultaneous infusion of NS 10 mL/kg if BP fails to recover or falls further. Stop infusion if BP does not recover, continue NS. If the patient has had any episode of hypotension, prehydrate with 0.9% NaCl at 10 mL/kg/hr for 2 hours prior to any subsequent infusion.

<u>Renal Insufficiency</u>: If renal function decreases, adjust etoposide as follows: CrCl 10-50 mL/min/1.73 m<sup>2</sup>, decrease dose by 25%; if CrCl < 10 mL/min/1.73 m<sup>2</sup>, decrease dose by 50%.

<u>Hyperbilirubinemia</u>: If direct bilirubin is > 2 mg/dL, decrease dose by 50%. If direct bilirubin is > 5 mg/dL, hold etoposide.

## 5.7 Intrathecal Methotrexate/Triple Intrathecal Therapy

<u>Systemic toxicity</u>: The dosage for IT methotrexate will not be reduced for systemic toxicity (myelosuppression, mucositis, etc.). Instead, leucovorin may be used at a dose of 5 mg/m²/dose every 6 hours x 2 doses, beginning 24 hours after the IT therapy may be administered in an attempt to reduce the risk of worsening already existent myelosuppression (ANC  $< 500/\mu L$ ) or mucositis. Do not administer leucovorin solely to prevent myelosuppression.



# Dose modifications following an episode of acute neurotoxicity:

Neurotoxicity has extremely protean manifestations, ranging from transient events, seizures or episodes of acute hemiparesis, to severe necrotizing encephalopathies. 44-46

The following guidelines are offered for consideration following an acute event, but it must be recognized that there are little data to support these approaches or any others. Many acute events, seizures or episodes of transient hemiparesis, are temporally related to the administration of intrathecal therapy, commonly 9 to 11 days after the IT administration.<sup>47</sup>

Complete clinical evaluation including imaging of the brain is strongly recommended. For patients who return to their baseline pre-event neurological status, clinicians may:

- 1. hold the next dose planned dose of IT therapy, or
- 2. substitute IT cytarabine or IT cytarabine/hydrocortisone for 1 dose of IT methotrexate or
- 3. proceed with IT methotrexate and include leucovorin rescue at a dose of 5 mg/m<sup>2</sup> IV/PO q 6 hrs x 2 doses beginning 24 hours after the LP.

If the event does not recur, resumption of standard therapy should be considered for subsequent intrathecal therapy.

For patients who do not return to baseline pre event neurological status or for those with recurrent events, or evidence of progressive encephalopathy, additional evaluations may be warranted and the treating physician may consider a more prolonged or definitive change in therapy upon discussion with the Study Chair.

## Leucovorin rescue of IT MTX without acute neurotoxicity

Prevention of neurotoxicity by using leucovorin after IT MTX has not been studied in a randomized fashion. Neither the BFM, DFCI, nor COG have routinely introduced leucovorin rescue to prevent acute neurotoxicity, however SJCRH protocols use leucovorin rescue during remission induction and consolidation phases. The cumulative incidence of all neurotoxicities among non-DS patients enrolled on AALL0932 and AALL1131 indicate a less than 1% incidence of acute neurotoxicity during induction. For non-DS patients enrolled on AALL0932, the incidence during consolidation was 0.3%. For non-DS patients receiving consolidation therapy on AALL1131, the incidence was 3.3%.

For the reasons above, it is permissible for patients receiving augmented consolidation such as that prescribed for NCI-SR-High (AALL1731) or NCI-HR (AALL1732) patients to receive leucovorin during consolidation therapy after the 4 doses of weekly IT MTX on the following schedule:

1. Leucovorin, 5 mg/m2 IV/PO at hours 24 and 30 after IT MTX.

It is not known if providing leucovorin rescue after IT MTX during consolidation as a measure to reduce acute neurotoxicity will reduce therapeutic efficacy in the context of



COG protocols.

Hydrocephalus, microcephaly or known abnormality of CSF flow precluding intrathecal chemotherapy via lumbar puncture:

Intraventricular chemotherapy via Ommaya catheter may be used in place of intrathecal therapy delivered by LP. Intraventricular chemotherapy should be given according to the same schedule, but at 50% of the corresponding age-based doses that would be given by LP. NOTE: Obstruction to CSF flow may be a contraindication to intrathecal and/or intraventricular therapy.

Viral, bacterial, or fungal meningitis: Omit until resolved.

5.8 Intermediate-Dose Methotrexate (ID MTX) and Leucovorin Rescue [Please note that IDMTX refers to IV MTX 1000 mg/m² given over 36 hrs]

#### 5.8.1 ID MTX Infusion Guidelines and dose modifications for toxicity

When IT therapy and ID MTX are scheduled for the same day, deliver the IT therapy within 6 hours of the beginning of the IV MTX infusion (hour -6 to +6, with 0 being the start of the MTX bolus).

Hold trimethoprim/sulfamethoxazole (TMP-SMX), any nonsteroidal anti-inflammatory medications, penicillins, proton pump inhibitors or aspirin-containing medications on the day of ID MTX infusion and for at least 72 hours after the start of the ID MTX infusion and until the MTX level is less than 0.5  $\mu$ M for ID MTX. In the presence of delayed clearance continue to hold these medications until MTX level is less than 0.1  $\mu$ M.

**Recommended Prehydration:** to start at least 6 hours prior to commencement of intravenous methotrexate. **Fluid:** D5  $\frac{1}{4}$  NS with 30 - 50 mEq NaHCO<sub>3</sub>/L at 125 mL/m<sup>2</sup>/hour. Ringers Lactate may be used as the initial fluid if a bicarbonate containing solution is unavailable. Adjust fluid volume and sodium bicarbonate to maintain urine specific gravity  $\leq 1.010$  and pH between 7 and 8. A bicarbonate bolus (25 mEq/m<sup>2</sup> over 15 min) may be given to raise the urine pH relatively quickly; a normal saline bolus may also be helpful in facilitating hydration.

**Hour 0**: MTX 100 mg/m<sup>2</sup> IV infused over 30 minutes. This is followed, immediately, by MTX 900 mg/m<sup>2</sup> given by continuous IV infusion over 35.5 hours. Be certain that the ID MTX infusion is completed in the 36 hour period. **Note, even if the infusion is not complete at this time point, it must be stopped.** 

**Recommended Posthydration**: Continue hydration using D 5  $^{1}$ /4 NS with 30-50 mEq NaHCO<sub>3</sub>/L at 125 mL/m²/hour (3 L/m²/day) throughout IDMTX infusion until the last dose of leucovorin has been given. In patients with delayed MTX clearance, continue hydration until the plasma MTX concentration is below 0.1  $\mu$ M.

<u>Leucovorin rescue</u>: 15 mg/m<sup>2</sup> PO/IV at 48 and 54 **hrs** after the start of the MTX infusion. If 48 hr methotrexate level is  $\leq$  0.5  $\mu$ M, then only two doses of leucovorin are administered (at 48 and 54 hours). If MTX level at 48 hours is > 0.5  $\mu$ M, then



continue hydration and leucovorin rescue at 15 mg/m²/dose po/IV every 6 hours until MTX levels are  $< 0.1 \ \mu M$ .

**Hour 48**: Check plasma methotrexate level at 48 hours after start of the methotrexate infusion. If the level is  $\leq 0.5~\mu M$ , then do not give more than two doses of leucovorin (48 and 54 hours). If MTX level at 48 hours is  $> 0.5~\mu M$ , then continue hydration and leucovorin rescue at 15 mg/m²/dose po/IV every 6 hours until MTX levels are  $< 0.1~\mu M$ .

For MTX levels that exceed these expected values modify the rescue regimen as noted below and increase hydration to 200 mL/m²/hr. Monitor urine pH to assure a value  $\geq 7.0$  and monitor urine output to determine if volume is  $\geq 80\%$  of the fluid intake, measured every 4 hours. If serum creatinine rises significantly, at any time point (> 100% in 24 hours), assure appropriate urine pH and urine volume as above and consider glucarpidase If urine output fails to continue at 80% of the fluid intake, consider furosemide or acetazolamide. Regardless of urine output, also consider glucarpidase (carboxypeptidase  $G_2$ ) (see below).

| 48 hr MTX | Leucovorin Rescue |
|---|---|
| level | |
| $\leq 0.5~\mu M$ | Continue 15 mg/m <sup>2</sup> IV/PO q 6hrs for 2 doses. |
| $0.5 - 1 \mu M$ | Increase to 15 mg/m $^2$ q 6 hrs until MTX level < 0.1 $\mu$ M (draw q 6-24 hrs). |
| $1-5 \mu M$ | Increase to 15 mg/m $^2$ q 3 hrs until MTX level < 0.1 $\mu$ M (draw q 6-24 hrs). |
| $5-10~\mu M$ | Increase to $100 \text{ mg/m}^2 \text{ q}$ 6hrs until MTX level $< 0.1 \mu\text{M}$ (draw q 6-24 hrs). |
| > 10 μM | Increase to 1000 mg/m² q 6hrs until MTX level $<$ 0.1 $\mu$ M (draw q 6-24 hrs). Consider glucarpidase. |

Nephrotoxicity: Postpone course if pre-treatment (MTX) serum creatinine is > 1.5 x baseline or GFR creatinine clearance < 65 mL/minute/1.73m². If there is a rising creatinine (> 100% in 24 hours) or the 48 hour methotrexate level is > 10  $\mu$ /L consider using glucarpidase. If renal function does not recover, omit MTX. Do not give ID MTX to a patient with this degree or renal impairment, assuming that prolonged excretion can be managed with glucarpidase.

NOTE: For patients who have markedly delayed MTX clearance secondary to renal dysfunction, consider using glucarpidase (carboxypeptidase G<sub>2</sub>, Voraxaze<sup>TM</sup>). To obtain supplies of glucarpidase in the US contact the Voraxaze 24-hour Customer Service line at 855-786-7292. Additional information can be found at <a href="https://www.voraxaze.com/Order-Voraxaze">https://www.voraxaze.com/Order-Voraxaze</a> regarding product availability through ASD Healthcare, Cardinal, and McKesson. Canadian sites should contact McKesson at (877) 384-7425 for further information. Sites in Australia and New Zealand should contact Hospira at 1300 – 046 – 774 (local) or medicalinformationAUS@hospira.com. Patients requiring glucarpidase rescue will remain on study.

Stop leucovorin 2 hours before administering glucarpidase as it is a competitive substrate and may compete with MTX for glucarpidase binding sites.



Dose of glucarpidase: 50 units/kg administered by intravenous bolus over 5 minutes. Reconstitute each vial with 1 mL sodium chloride 0.9% (do not further dilute). Each vial contains 1,000 units/mL (after reconstitution) and round dose up to vial size. No further dose is required.

Maintaining alkalinization of urine with sodium bicarbonate is essential to maintain urinary pH > 7.

It is essential that patients are NOT co-prescribed the following medicines which reduce MTX excretion: NSAIDS, aspirin, ciprofloxacin, co-trimoxazole, penicillins, probenecid, omeprazole (or other proton pump inhibitors).

Two hours after administration of glucarpidase, leucovorin should be administered at a dose of 250 mg/m² every 6 hours by IV bolus (maximum rate: 160 mg/min) for up to 48 hours and then decreased based on plasma MTX concentrations to  $15 \text{ mg/m}^2$  intravenously or orally every 6 hours until the plasma MTX concentration is  $< 0.2 \ \mu M$ .

<u>Liver Dysfunction</u>: Samples for the determination of ALT value must be drawn within 72 hours, PRIOR to a course of intravenous MTX. Blood samples for ALT should not be drawn following the start of MTX infusions as MTX causes significant short term elevation in ALT levels.

| ALT | IV MTX |
|----------------------------|-------------------------------------------------|
| < 10 X ULN | Continue with therapy as scheduled |
| 10 – 20 X ULN | Continue with therapy as scheduled for 1 cycle |
| 10 – 20 X ULN for 2 | Discontinue TMP/SMX* |
| consecutive cycles | Hold therapy until ALT < 10 X ULN, then |
| | resume at full doses at point of interruption. |
| | Do not skip doses. |
| > 20 X ULN | Hold therapy until ALT < 10 X ULN, then |
| | resume at full doses at point of interruption. |
| | Do not skip doses. |
| > 20 X ULN for > 2 weeks | Evaluate with AST, Bili, Alkaline phosphatase, |
| | PT, albumin, total protein, and hepatitis A, B, |
| | C, CMV, and EBV serologies. |
| | Consider liver biopsy before additional therapy |
| | given. Notify Study Chair. |

<sup>\*</sup> Please see COG Supportive Care Guidelines in <u>Appendix I</u> for trimethoprim-sulfamethoxazole (TMP/SMX) substitutions.

Hold IV MTX for direct hyperbilirubinemia of > 2.0 mg/dL.

<u>Mucositis</u>: For Grade 3 - 4 mucositis, withhold IV MTX until resolved. Increase leucovorin rescue following the next course from 2 to 4 doses on a q6 hr schedule. If subsequent course is not associated with Grade 3 - 4 mucositis, attempt to decrease the number of leucovorin doses to 2. If mucositis recurs despite the extended leucovorin, decrease the dose of MTX by 25%, increase hydration to 200 mL/m²/hr and continue increased leucovorin as above. Should subsequent courses be well



tolerated, use a stepwise approach to resuming a standard approach to drug delivery. Consider culturing lesions for herpes simplex if mucositis persists or recurs.

See <u>Section 5.13</u> for dose modifications when MTX is used post HSCT.

# 5.9 PO Methotrexate (MTX) and 6-Mercaptopurine (MP)

## **During Continuation:**

ANC  $< 500/\mu$ L and/or platelets  $< 50,000/\mu$ L:

Discontinue dose until ANC is  $\geq 750/\mu L$  and platelets are  $\geq 75,000/\mu L$ . Restart mercaptopurine and/or MTX at 50% of the original dose on the same day the counts recover. Increase to 75% and then 100% of the original dose at 2-week intervals provided ANC remains  $\geq 750/\mu L$  and platelets remain  $\geq 75,000/\mu L$ . Consider a marrow evaluation in the face of persistent or prolonged neutropenia.

Prolonged cytopenia is defined as ANC <  $750/\mu L$  and/or platelets <  $75,000/\mu L$  after withholding therapy for > 2 weeks. Perform a bone marrow examination after 2 weeks of withholding chemotherapy, if no recovery is apparent. If monocyte count is increasing or viral myelosuppression is clinically suspected, the bone marrow examination may be postponed for 1 - 2 weeks and omitted if ANC and platelets fully recover by the 4<sup>th</sup> week after therapy is withheld.

If patient develops severe or unexpected myelosuppression, i.e., doesn't tolerate at least half dose MP, see section below on thiopurine pharmacology testing.

#### **During Maintenance:**

<u>Myelosuppression:</u> If absolute neutrophil count (ANC) falls below  $500/\mu L$  or if platelet count falls below  $50,000/\mu L$  during Maintenance, mercaptopurine and methotrexate should be held until recovery above these levels.

- 1. For the first drop below  $500/\mu L$  ANC or platelet count  $< 50,000/\mu L$ , resume mercaptopurine and methotrexate at the same dose the patient was taking prior to the episode of myelosuppression when ANC  $\geq 500/\mu L$  and platelet count  $\geq 50,000/\mu L$ .
- 2. If ANC falls below  $500/\mu L$  or if platelet count falls below  $50,000/\mu L$  for a second (or greater) time, hold mercaptopurine and methotrexate until ANC is  $\geq 750/\mu L$  and platelets are  $\geq 75,000/\mu L$ . Consider discontinuing trimethoprim/sulfamethoxazole (TMP/SMX) in favor of an alternative approach to Pneumocystis prophylaxis.
  - a. When ANC  $\geq$  750/ $\mu$ L and platelet count  $\geq$  75,000/ $\mu$ L, restart mercaptopurine and methotrexate at 50% of the dose prescribed at the time that the medications were stopped.
  - b. Increase doses of mercaptopurine and methotrexate to 75% and then 100% of dose prescribed prior to stopping the medications at 2-4 week intervals provided ANC remains > 750 / $\mu$ L and platelets remain > 75,000/ $\mu$ L. May increase both mercaptopurine and methotrexate simultaneously.
  - c. Once at 100% of the dose prescribed prior to stopping, see below for instructions regarding further dose escalation.



Continue to follow ANC q 2-4 weeks with target ranges ANC 500 – 1,500/ $\mu$ L and platelet count  $\geq 50,000/\mu$ L

If patient develops severe or unexpected myelosuppression, i.e., doesn't tolerate at least half dose mercaptopurine, in the absence of TMP/SMZ or other myelosuppressive agents, strongly consider evaluation of TPMT and/or NUDT15 status if not already done)

Prolonged cytopenia is defined as ANC <  $500/\mu L$  and/or platelets <  $50,000/\mu L$  after withholding therapy for > 2 - 4 weeks. Consider a marrow evaluation in the face of persistent or prolonged neutropenia if no recovery is apparent. If monocyte count is increasing or viral myelosuppression is clinically suspected, the bone marrow examination may be postponed for 1-2 weeks and omitted if ANC and platelets fully recover by the 4th week after therapy is withheld.

<u>Inadequate Myelosuppression:</u> For persistent ANC  $\geq 1,500/\mu L$ , no dose escalations are recommended during the first cycle of Maintenance.

- For ANC ≥ 1,500/µL on 3 CBC(s) done over 6 weeks or 2 successive monthly CBC(s), alternately increase doses of methotrexate or mercaptopurine by 25%. Always wait at least 4 weeks before making another dose adjustment.
- If both methotrexate and mercaptopurine are increased once without a fall in ANC, consider noncompliance as a possibility. Noncompliance can be assessed by obtaining a sample for thiopurine metabolites. Although there are no specific values to use to indicate non-adherence, low concentrations of TGN and methylated derivatives in a sample taken after at least three weeks after continuous dosing may indicate non-adherence. Also consider observing the administration of an oral dose of methotrexate and checking plasma methotrexate concentration 2-4 hours later; this value should be ≥ 0.2 μM.
- If ANC remains high after intervention for possible noncompliance.
  - o For patients who are heterozygous or homozygous deficient for TPMT/NUDT15 and have high ANCs as described above, increase methotrexate alone by 25% and repeat evaluation. Unless noncompliance is suspected, increase methotrexate preferentially over mercaptopurine Consider carefully increasing mercaptopurine doses as well, if high ANCs persist. Increase the mercaptopurine dose in 25% increments until ANC is in target. Always wait at least 4 weeks before making another dose adjustment or re-measuring TGN. If ANC remains high, alternate mercaptopurine dose increases with methotrexate dose increases.
  - o If the methylated derivatives are significantly elevated, in concert with abdominal symptoms or Grade 4 SGPT/ALT, SGOT/AST and or direct bilirubin ≥ 2 mg/dl, and ANC indicates that the 6-MP should be increased, consider adding allopurinol at a dose of 50 mg/m² with a dose of 6-MP that has been decreased by 50-75%. 50

#### Mucositis Grade 3 - 4:

MTX should be reduced to 50% if Grade 3 toxicity develops; withhold in the presence of Grade 4 toxicity until there is a resolution, then resume at 50% of original dose with gradual


dose escalation. If mucositis persists or recurs, consider culturing for herpes simplex.

#### Liver Dysfunction:

- For Grade 3 toxicity, increase in hepatic transaminases (SGPT/ALT or SGOT/AST to greater than >5.0 20.0 x ULN), obtain total direct bilirubin. Monitor SGPT/ALT or SGOT/AST and total direct bilirubin weekly during Consolidation as long as transaminases remain over 5x ULN.
- Continue full dose therapy unless either of the following occurs:
- Direct bilirubin > 2 mg/dL
- Grade 4 SGPT/ALT or SGOT/AST > 20x ULN (consistent with Grade 4 toxicity) elevation on 2 determinations at least 1 week apart.
- If either of these occurs, hold mercaptopurine and monitor labs as above, weekly. Restart at full dose therapy when the transaminase elevation is < Grade 3 (are less than 5x ULN), as long as direct bilirubin is < 2 mg/dL
- Exclude infectious hepatitis for persistent (> 1 month) Grade 3 elevations in SGPT/ALT or SGOT/AST(above 5x ULN). Consider discontinuing trimethoprim/sulfamethoxazole (TMP/SMX) in favor of an alternative approach to Pneumocystis prophylaxis

For dose modifications when MTX is given for GVHD prophylaxis see Section 5.13.3.

#### **Thiopurine Pharmacology Testing and Dosage Adjustments:**

Mercaptopurine and thioguanine are methylated directly by thiopurine methyltransferase (TPMT) to an inactive metabolite. TPMT activity varies tremendously among patients, because of a common inherited genetic defect in TPMT. One in 300 patients is completely deficient (homozygous defective) and 10% of the population are moderately deficient in TPMT activity because they have inherited one variant (non-functional) TPMT allele (i.e., heterozygotes). Patients with low TPMT form higher concentrations of the 6-thioguanine nucleotides (6-TGN) and are more susceptible to acute thiopurine toxicity (primarily myelosuppression, involving neutropenia, thrombocytopenia, and anemia). Patients with the complete deficiency of TPMT tolerate less than 10% of protocol doses of 6 MP (10 to 30 mg/m²/day 3 days per week). About 35% of heterozygotes require a lower dose of 6-MP to avoid dose-limiting myelosuppression. 54

There are now CLIA certified tests for TPMT genotype and phenotype, and for thiopurine metabolites (6-methyl mercaptopurine [6-MMP] and 6-TGN) measurements. Only 3 SNPs constitute well over 90% of the inactivating mutations in the gene, based on studies in numerous racial and ethnic groups worldwide. 51,55-58 Thus, the genotyping test has a low false negative rate, and may be preferable to TPMT phenotype testing in cases where a history of red cell transfusions would potentially confound assessments of RBC TPMT activity. When the genotyping result is coupled with a phenotyping test for TPMT or with thiopurine metabolite concentrations in erythrocytes, the reliability of the tests will be even greater. Moreover, metabolite levels can provide an index of patient compliance with thiopurine therapy.

#### Recommendations for Thiopurine Monitoring and Dosage Adjustments:

When myelosuppression has led to significant delays in therapy (> 2 weeks) or is disproportionate to the therapy, thiopurine testing should be performed:



- For patients who have received full dose thiopurine therapy during the 2 weeks immediately preceding the test, RBC thiopurine metabolites will likely predict TPMT status and actual thiopurine exposure.
- In the absence of RBC transfusions for 3 months prior, TPMT activity will accurately reflect TPMT status
- TPMT genotyping will be informative in all patients, if at least 1 mutant allele is identified. If not, and myelosuppression continues, send samples for TPMT activity and/or metabolites since TPMT genotyping will miss 5% 10% of mutants. NOTE: Genotyping can be done despite recent transfusions.

#### Suggested Dose Adjustments in Patients With Unacceptable Myelosuppression:

- If the patient is <u>homozygous deficient</u> for TPMT, the thiopurine dose should be <u>reduced to</u> 10 20 mg/m²/day 3 days per week. If the patient is <u>heterozygous for TPMT and</u> has experienced significant myelosuppression, the thiopurine dose should be reduced by 30% 50%. Do not increase the dose in response to a high ANC for 4 weeks to allow for achievement of steady state. All other myelosuppressive medications should be delivered at full dose, and the thiopurine dose should be titrated based on blood counts. Further thiopurine pharmacologic measures are not often necessary.
- If the patient is homozygous wild-type (high activity) for TPMT, then discontinue TMP/SMX and use pentamidine or dapsone. For modifications of the oral MP and MTX see the beginning of this section.

#### 5.10 Steroids (Dexamethasone)

<u>Hypertension</u>: Dose should not be reduced. Sodium restriction and anti-hypertensives should be employed in an effort to control hypertension.

Hyperglycemia: Dose should not be reduced for hyperglycemia.

<u>Pancreatitis</u>: Do not modify dose for asymptomatic elevations of amylase and/or lipase. Discontinue steroids, except for stress doses, in the presence of Grade 3 or 4 pancreatitis. In the case of asymptomatic Grade 2 pancreatitis (enzyme elevation or radiographic findings only), steroids should be held until symptoms and signs subside, and amylase/lipase levels return to normal and then consider resuming steroids.

Osteonecrosis (ON): Do not modify corticosteroid therapy for osteonecrosis (also referred to as avascular necrosis) prior to Maintenance therapy. Consider omitting Maintenance steroid for osteonecrosis Grade 1 (clinically asymptomatic, radiographic finding only). Omit Maintenance steroid for osteonecrosis Grade 2 or greater, and notify study chair. Consider resuming Maintenance steroid after 6 months if joint symptoms have resolved and if MRI findings have significantly improved or normalized.

<u>Varicella</u>: Steroids should be held during active infection except during Induction. Do not hold during incubation period following exposure.

#### Inability to use oral doses:

For dexamethasone, substitute the IV preparation mg for mg.

<u>Severe infection</u>: Do not hold or discontinue steroids during Induction without serious consideration, as this is a critical period in the treatment of ALL. Later in therapy, one may



consider holding steroid until patient achieves cardiovascular stability, except for "stress doses."

#### 5.11 **PO 6-Thioguanine (TG)**

#### Continuation:

Infection: Oral TG will be held for suspected or proven serious infection.

For severe and/or unexpected myelosuppression, evaluate for TPMT activity as described in Section 5.9.

#### 5.12 Vincristine

## PLEASE USE "BALIS" SCALE FOR GRADING NEUROPATHY (See text box below)

#### Severe neuropathic pain (Grade 3 or greater):

Hold dose(s). When symptoms subside, resume at 50% previous <u>calculated</u> dose (<u>maximum dose: 1 mg</u>), then escalate to full dose as tolerated. NOTE: neuropathic pain can be not only severe but difficult to treat. However, because vincristine is an important component of curative therapy and the majority of neuropathies are ultimately reversible, vincristine therapy may be given at full dose at investigator discretion. Severe peripheral neuropathies, with or without a positive family history might suggest the need for a molecular diagnostic evaluation to rule out Charcot Marie Tooth Disease (CMT), Type 1A or Hereditary neuropathy with liability to pressure palsies. Drugs such as gabapentin may be of value.

#### Vocal Cord paralysis:

Hold dose(s). When symptoms subside, resume at 50% previous <u>calculated</u> dose <u>(maximum dose: 1 mg)</u>, then escalate to full dose as tolerated. See above for comment on CMT.

#### Foot Drop, paresis:

Should be Grade 3 to consider holding or decreasing dose. These toxicities are largely reversible but over months to years. Accordingly, holding doses of vincristine and/or lowering the dose may not result in rapid resolution of symptoms and may compromise cure. See above for comment on CMT. Physical therapy may be beneficial to maintain range of motion and provide AFO's and other forms of support. Drugs such as gabapentin may be of value.

Jaw pain: Treat with analgesics; do not modify vincristine dose.

#### <u>Hyperbilirubinemia<sup>59</sup>,60</u>:

| Direct Bili | Dose reduction |
|---|---|
| < 3.1 mg/dL | Full dose (maximum dose: 2 mg), |
| 3.1-5.0 mg/dL | 50% of calculated dose (maximum dose: 1 mg), |
| 5.1-6.0 mg/dL | 75% of calculated dose (maximum dose: 0.5 mg), |
| > 6.0 mg/dL | Withhold dose and administer next scheduled dose if toxicity has |
| · · | resolved. |
| | Do not make up missed doses. |



<u>Constipation or ileus (≥ Grade 3) or typhlitis</u>: Hold dose(s); institute aggressive regimen to treat constipation if present. When symptoms abate resume at 50% <u>of calculated</u> dose (<u>maximum dose</u>: 1 mg) and escalate to full dose as tolerated.

#### Extravasation:

In the event of an extravasation, discontinue the IV administration of the drug and institute appropriate measures to prevent further extravasation and damage according to institutional guidelines. Also see <a href="https://cogmembers.org/\_files/disc/pharmacy/ExtravasationReference.pdf">https://cogmembers.org/\_files/disc/pharmacy/ExtravasationReference.pdf</a> for COG reference.

#### Modified ("Balis") Pediatric Scale of Peripheral Neuropathies

#### **Peripheral Motor Neuropathy:**

- <u>Grade 1</u>: Subjective weakness, but no deficits detected on neurological exam, other than abnormal deep tendon reflexes.
- <u>Grade 2</u>: Weakness that alters fine motor skills (buttoning shirt, coloring, writing or drawing, using eating utensils) or gait without abrogating ability to perform these tasks.
- <u>Grade 3</u>: Unable to perform fine motor tasks (buttoning shirt, coloring, writing or drawing, using eating utensils) or unable to ambulate without assistance.
- Grade 4: Paralysis.

#### **Peripheral Sensory Neuropathy:**

- <u>Grade 1</u>: Paresthesias, pain, or numbness that do not require treatment or interfere with extremity function.
- <u>Grade 2</u>: Paresthesias, pain, or numbness that are controlled by non-narcotic medications (without causing loss of function), or alteration of fine motor skills (buttoning shirt, writing or drawing, using eating utensils) or gait, without abrogating ability to perform these tasks.
- <u>Grade 3</u>: Paresthesias or pain that are controlled by narcotics, or interfere with extremity function (gait, fine motor skills as outlined above), or quality of life (loss of sleep, ability to perform normal activities severely impaired).
- Grade 4: Complete loss of sensation, or pain that is not controlled by narcotics.

#### 5.13 Stem Cell Transplant Regimen Agents

#### 5.13.1 Tacrolimus

Tacrolimus commonly causes mild/moderate hypertension and alopecia and less commonly kidney or liver dysfunction, transplant associated microangiopathy (TAM), and neurological changes associated with significant hypertension. When trough levels are kept in the therapeutic range and patients receive adequate hydration and magnesium replacement, most of these side effects can be minimized. Hypertension should be managed with single or combination antihypertensive therapy. Tacrolimus should be held for severe toxicities thought



to be related to its administration (significant neurological changes/malignant hypertension, TAM, kidney failure, etc.). Other immune suppressive medications may be substituted if tacrolimus is not tolerated (MMF, cyclosporine, etc.).

#### 5.13.2 Cyclosporine

Cyclosporine commonly causes mild/moderate hypertension and less commonly kidney or liver dysfunction, TAM, and neurological changes associated with significant hypertension. When trough levels are kept in the therapeutic range and patients receive adequate hydration and magnesium replacement, most of these side effects can be minimized. Hypertension should be managed with single or combination antihypertensive therapy. Cyclosporine should be held for severe toxicities thought to be related to its administration (significant neurological changes/malignant hypertension, TAM, kidney failure, etc.). Other immune suppressive medications may be substituted if cyclosporine is not tolerated

#### 5.13.3 Methotrexate

The most common acute side-effects of methotrexate include delay of count recovery, worsened mucositis, and kidney and liver damage (can contribute to VOD). Toxicity is directly related to the length of exposure to the drug. While methotrexate is generally excreted rapidly, delayed excretion of methotrexate occurs with decreased renal function and in circumstances where patients have third-space fluid collections (pulmonary effusions, ascites, joint effusions, etc.). The attending transplant physician should assess each patient prior to delivery of each dose and decide whether full dose methotrexate should be administered. Guidelines for modification of methotrexate dosing are listed in the tables below.

Table 5.13.3.1: Methotrexate Dose Modification for Renal Impairment

| | Mild | Moderate | Severe | <b>Life-Threatening</b> |
|---|---|---|---|---|
| Serum creatinine | > 1.5 - 2x baseline | > 2 - 2.5x | > 2.5 - 3x | > 3x baseline or |
| | | baseline | baseline | dialysis |
| % Methotrexate | 0 - 50% | 50 - 100% | 100% | 100% |
| Dose reduction | | | (no drug) | (no drug) |
| (Day +1, 3, 6, 11) | | | | |



| Stomatitis, | Painless ulcers, | Painful | Cannot eat | Complete |
|---|---|---|---|---|
| mucositis | erythema, mild | erythema, | solids or | obstruction or |
| | soreness or | edema, | requires | perforation |
| | mild dysphagia | ulcers or | narcotics to | |
| | | moderate | eat, requires | |
| | | dysphagia, | parenteral | |
| | | but can eat | or enteral | |
| | | without | support. | |
| | | narcotics | | |
| % Methotrexate | 0% | 0% | 0 - 50% | 50 - 100% |
| Dose reduction | | | | |
| (Day +1, 3, 6, 11) | | | | |

Table 5.13.3.2: Methotrexate Dose Modification for Significant Mucositis

For significant third spacing (ascites, effusions, significant edema or weight gain > 5 - 10% above baseline) consider dose reductions of 50% and leucovorin rescue.

#### 5.13.4 Guidelines for Leucovorin Rescue

Dose: Patients at risk for methotrexate toxicity should receive leucovorin at a dose of 5 - 10 mg/m<sup>2</sup> IV Q6H x 4 doses beginning 24 hours after administration of methotrexate. While most patients will need only 4 doses of leucovorin, if methotrexate levels are elevated due to renal dysfunction or other problems, leucovorin doses should be continued until serum methotrexate concentration is  $< 1 \text{x} 10^{-7} \text{M}$ . If serum methotrexate concentration is  $> 5 \text{x} 10^{-6} \text{M}$ , increase dose to  $100 \text{ mg/m}^2/\text{dose IV Q3H}$  until the serum methotrexate level is  $< 1 \text{x} 10^{-8} \text{M}$ .

#### 5.13.5 Mycophenolate Mofetil (MMF)

MMF can cause decreased counts, nausea, vomiting, diarrhea, hypertension, dizziness, insomnia, hyperglycemia, electrolyte imbalances, rash, leg cramps, and bone pain. For significant diarrhea or low counts (neutropenia, etc.), a decrease of MMF by approximately 20% is usually sufficient to decrease the toxicity. Further dose modifications for significant toxicity likely caused by MMF are allowed.

#### 5.13.6 Adjustment of TBI/chemotherapy During the Preparative Regimen.

The full dose of preparative regimen TBI and chemotherapy agents will be administered unless patients have a life threatening reaction thought likely to occur again with continued administration and an appropriate substitution cannot be made (i.e. etopophos for etoposide).

## 5.13.7 <u>Dose Adjustment of Chemotherapy for Patients Whose Weight Exceeds > 125%</u> Ideal Body Weight (IBW)

Chemotherapy given during the preparative regimen (thiotepa, cyclophosphamide, and etoposide) will be dosed based on actual weight for patients  $\leq$  125% IBW. Those > 125% IBW will be dosed based upon adjusted ideal body weight as follows:

Adjusted ideal body weight = IBW + 0.25 (Actual weight – IBW).



The following formulas for pediatric and adult IBW calculations are recommended, but IBW may be calculated according to institutional standard operating procedures (SOPs).

Recommended Ideal Body Weight Calculation for Children Age 1- 17 years IBW =  $\frac{\text{Height (cm)}^2 \times 1.65}{1000}$ 

Recommended Ideal Body Weight Calculation for Adults (Height > 5 feet/60 inches)

IBW (females) = 
$$(cm \div 2.54 - 60) \times 2.3 \text{ kg} + 45.5 \text{ kg}$$

IBW (males) = 
$$(cm \div 2.54 - 60) \times 2.3 \text{ kg} + 50 \text{ kg}$$



#### 6.0 DRUG INFORMATION

#### 6.1 **BLINATUMOMAB**

(11/18/2019)

(Blincynto®, AMG103, MT103, recombinant bispecific antibody derivative, NSC# 765986)

Source and Pharmacology

Blinatumomab is a fusion protein composed of two single-chain antibodies (scFv), murine anti-CD19 scFv and murine anti-CD3 scFv. Through CD3 binding, blinatumomab recruits and engages T cells for redirected lysis of CD19-positive B cells, including those expressed with B-cell malignancies. T cells are bound by its anti-CD3 moiety, whereas B cells are bound by the anti-CD19 moiety. The subsequent serial lysis of multiple malignant cells by a single blinatumomab-activated T cell closely resembles a natural cytotoxic T cell reaction. Treatment with blinatumomab is associated with a rapid depletion of peripheral B cells, accompanied by T cell activation and a transient increase in cytokines.

Blinatumomab consists of a single chain of 504 amino acids with a molecular weight of approximately 54 kDa. The pharmacokinetics of blinatumomab was assessed over a dose range from 5 to 90 mcg/m²/day (approximately equivalent to 9-162 mcg/day). Following continuous intravenous infusion, the steady state serum concentration (Css) was achieved within a day and remained stable over time. The estimated mean (SD) volume of distribution based on terminal phase (Vz) was 4.52 (2.89) L. The estimated mean (SD) systemic clearance was 2.92 (2.83) L/hour and the estimated mean (SD) half-life was 2.11(1.42) hours. Negligible amounts of blinatumomab were excreted in the urine at the tested clinical doses. Like other protein therapeutics, blinatumomab is expected to be degraded into small peptides and amino acids via catabolic pathways. At the clinical doses of 9 mcg/day and 28 mcg/day for the treatment of adult relapsed/refractory ALL, the mean (SD) Css was 211 (258) pg/mL and 621 (502) pg/mL, respectively.

At this time there are no known drug interactions with blinatumomab.

#### **Toxicity:**

## Comprehensive Adverse Events and Potential Risks list (CAEPR) for Blinatumomab (AMG 103, NSC 765986)

The Comprehensive Adverse Events and Potential Risks list (CAEPR) provides a single list of reported and/or potential adverse events (AE) associated with an agent using a uniform presentation of events by body system. In addition to the comprehensive list, a subset, the Specific Protocol Exceptions to Expedited Reporting (SPEER), appears in a separate column and is identified with bold and italicized text. This subset of AEs (SPEER) is a list of events that are protocol specific exceptions to expedited reporting to NCI (except as noted below). Refer to the 'CTEP, NCI Guidelines: Adverse Event Reporting Requirements'

http://ctep.cancer.gov/protocolDevelopment/electronic\_applications/docs/aeguidelines.pdf for further clarification. *Frequency is provided based on 1276 patients*. Below is the CAEPR for Blinatumomab.

**NOTE**: Report AEs on the SPEER <u>ONLY IF</u> they exceed the grade noted in parentheses next to the AE in the SPEER. If this CAEPR is part of a combination protocol using multiple investigational agents and has an AE listed on different SPEERs, use the lower of the grades to determine if expedited reporting is required.

Version 2.5, September 4, 2019<sup>1</sup>



| Adverse Events with Possible Relationship to Blinatumomab (AMG 103) (CTCAE 5.0 Term) [n= 1276] | | Specific Protocol Exceptions to<br>Expedited Reporting<br>(SPEER) | |
|---|---|---|---|
| Likely (>20%) | Less Likely (<=20%) | Rare but Serious (<3%) | |
| BLOOD AND LYMPHAT | TIC SYSTEM DISORDERS | | |
| Anemia | | | Anemia (Gr 2) |
| | Blood and lymphatic system disorders - Other (coagulopathy) <sup>2</sup> | | Blood and lymphatic system disorders -<br>Other (coagulopathy) <sup>2</sup> (Gr 2) |
| | | Blood and lymphatic system disorders - Other (hematophagic histiocytosis) | |
| | | Blood and lymphatic system disorders - Other (lymphadenitis) | |
| | | Blood and lymphatic system disorders - Other (lymphadenopathy) | |
| | | Blood and lymphatic system disorders - Other (pancytopenia) | |
| | Disseminated intravascular coagulation <sup>2,3</sup> | | Disseminated intravascular coagulation <sup>2,3</sup> (Gr 2) |
| | Febrile neutropenia | | Febrile neutropenia (Gr 3) |
| CARDIAC DISORDERS | | | |
| | Sinus tachycardia | | Sinus tachycardia (Gr 2) |
| GASTROINTESTINAL D | ISORDERS | | |
| | Abdominal pain | | Abdominal pain (Gr 2) |
| | Constipation | | Constipation (Gr 2) |
| | Diarrhea | | Diarrhea (Gr 2) |
| | | Gastric hemorrhage | |
| | | Gastrointestinal disorders - Other (pneumoperitoneum) | |
| | Mucositis oral | | |
| Nausea | | | Nausea (Gr 2) |
| | | Oral hemorrhage | |
| | | Pancreatitis | · |
| GENERAL DIGORDERG | Vomiting | NIDITIONE | Vomiting (Gr 2) |
| GENERAL DISORDERS | AND ADMINISTRATION SITE CO | DNDITIONS | grun 2 (g. A) |
| | Chills <sup>3</sup> | | Chills <sup>3</sup> (Gr 2) |
| Г 3 | Edema limbs | | Edema limbs (Gr 2) |
| Fatigue <sup>3</sup> Fever <sup>3</sup> | | | Fatigue <sup>3</sup> (Gr 2) |
| rever | Conoralizad adams | | Fever <sup>3</sup> (Gr 2) |
| | Generalized edema | | |
| | Non-cardiac chest pain Pain | | |
| HEPATOBILIARY DISOR | | | |
| HEI ATOBILIART DISOR | Hepatobiliary disorders - Other (hepatic function abnormal) <sup>4</sup> | | Hepatobiliary disorders - Other (hepatic function abnormal) <sup>4</sup> (Gr 2) |
| IMMUNE SYSTEM DISO | | | janetton uonormusj (Gr 2) |
| INTROCKE STOTEM DISC | | Allergic reaction <sup>3</sup> | |
| | Cytokine release syndrome <sup>3</sup> | zmorgie reaction | Cytokine release syndrome <sup>3</sup> (Gr 3) |
| | Immune system disorders - Other (immunodeficiency [immunoglobulin decreased]) <sup>5</sup> | | Immune system disorders - Other (immunodeficiency [immunoglobulin decreased]) <sup>5</sup> (Gr 2) |



| Adverse Events with Possible Relationship to Blinatumomab (AMG 103) (CTCAE 5.0 Term) [n= 1276] | | | Specific Protocol Exceptions to<br>Expedited Reporting<br>(SPEER) |
|---|---|---|---|
| Likely (>20%) | Less Likely (<=20%) | Rare but Serious (<3%) | |
| INFECTIONS AND INFESTA | ATIONS | | |
| Infection <sup>6</sup> | | | Infection <sup>6</sup> (Gr 4) |
| INJURY, POISONING AND | PROCEDURAL COMPLICATION | ONS | |
| | Infusion related reaction | | |
| | | Injury, poisoning and procedural complications - Other (overdose) <sup>7</sup> | |
| INVESTIGATIONS | | | |
| | | Activated partial thromboplastin time prolonged <sup>2</sup> | |
| | Alanine aminotransferase increased <sup>4</sup> | | Alanine aminotransferase increased <sup>4</sup> (Gr 3) |
| | Alkaline phosphatase increased <sup>4</sup> | | Alkaline phosphatase increased <sup>4</sup><br>(Gr 2) |
| | Aspartate aminotransferase increased <sup>4</sup> | | Aspartate aminotransferase increased <sup>4</sup><br>(Gr 4) |
| | Blood bilirubin increased <sup>4</sup> | | Blood bilirubin increased <sup>4</sup> (Gr 2) |
| | Blood lactate dehydrogenase | | |
| | increased | Creatinine increased <sup>8</sup> | |
| | GGT increased <sup>4</sup> | Creatinine increased* | GGT increased <sup>4</sup> (Gr 2) |
| | GG1 mereased | Investigations - Other (blood fibrinogen increased) <sup>2</sup> | oor mercuscu (or 2) |
| | Investigations - Other (C-reactive protein increased) Investigations - Other (fibrin D | , | Investigations - Other (C-reactive protein increased) (Gr 2) |
| | dimer increased) <sup>2</sup> | | |
| Lymphocyte count decreased | | | Lymphocyte count decreased (Gr 4) |
| Neutrophil count decreased Platelet count decreased <sup>2</sup> | | | Neutrophil count decreased (Gr 4) Platelet count decreased <sup>2</sup> (Gr 2) |
| Platelet count decreased | Weight gain | | Weight gain (Gr 2) |
| | Weight loss | | meight guin (Gr 2) |
| | White blood cell decreased | | White blood cell decreased (Gr 4) |
| METABOLISM AND NUTRI | • | <u> </u> | |
| | Anorexia | | |
| | Hyperglycemia | | Hyperglycemia (Gr 2) |
| | Hyperuricemia | | |
| | Hypoalbuminemia | | |
| | Hypocalcemia | | |
| Hypokalemia | | | Hypokalemia (Gr 2) |
| | Hypomagnesemia | | |
| | Hypophosphatemia | T 1 : 1 0 | |
| MUCCIII OCKELETAL AND CO | ONNECTIVE TICCLE DICORDERG | Tumor lysis syndrome <sup>9</sup> | |
| MOSCULUSKELETAL AND CO | ONNECTIVE TISSUE DISORDERS Arthralgia | | |
| | Back pain | | Back pain (Gr 2) |
| | Bone pain | | Buck puin (Or 2) |
| | Generalized muscle weakness | | |
| | Myalgia Myalgia | | |



| Adverse Events with Possible Relationship to Blinatumomab (AMG 103) (CTCAE 5.0 Term) [n= 1276] | | | Specific Protocol Exceptions to<br>Expedited Reporting<br>(SPEER) |
|---|---|---|---|
| Likely (>20%) | Less Likely (<=20%) | Rare but Serious (<3%) | |
| | Pain in extremity | | Pain in extremity (Gr 2) |
| NERVOUS SYSTEM DISC | | | |
| | Ataxia <sup>10</sup> | | |
| | Cognitive disturbance <sup>10</sup> | | |
| | Dizziness <sup>10</sup> | | Dizziness <sup>10</sup> (Gr 2) |
| | | Dysarthria <sup>10</sup> | ( ) |
| | Dysphasia <sup>10</sup> | | |
| | Encephalopathy <sup>10</sup> | | |
| | 1 1 3 | Facial nerve disorder <sup>10</sup> | |
| Headache <sup>10</sup> | | | Headache <sup>10</sup> (Gr 2) |
| | | Intracranial hemorrhage | |
| | | Leukoencephalopathy | |
| | Memory impairment <sup>10</sup> Nervous system disorders - Other (apraxia) | | |
| | Nervous system disorders - Other (cerebellar syndrome) <sup>10</sup> | | |
| | | Nervous system disorders -<br>Other <sup>10</sup> | |
| | Paresthesia <sup>10</sup> | | |
| | | Reversible posterior leukoencephalopathy syndrome | |
| | Seizure <sup>10</sup> | | |
| | Somnolence <sup>10</sup> | | |
| | | Transient ischemic attacks <sup>10</sup> | |
| | Tremor <sup>10</sup> | | Tremor <sup>10</sup> (Gr 2) |
| PSYCHIATRIC DISORDE | RS | | |
| | | Agitation <sup>10</sup> | |
| | Anxiety <sup>10</sup> | | |
| | Confusion <sup>10</sup> | | |
| | | Hallucinations <sup>10</sup> | |
| | Insomnia | | Insomnia (Gr 2) |
| | | Personality change <sup>10</sup> | |
| | | Psychosis <sup>10</sup> | |
| RESPIRATORY, THORAC | CIC AND MEDIASTINAL DISORI | DERS | |
| | Cough | | Cough (Gr 2) |
| | Dyspnea | | |
| | Epistaxis | | |
| | | Hypoxia | |
| | Oropharyngeal pain | | |
| | | Pneumonitis | |
| | Voice alteration <sup>10</sup> | | |
| SKIN AND SUBCUTANE | OUS TISSUE DISORDERS | | |
| | Hyperhidrosis | | |
| | Pruritus | | |
| - | Skin and subcutaneous tissue disorders - Other (rash) <sup>11</sup> | | Skin and subcutaneous tissue disorders - Other (rash) $^{11}$ (Gr 2) |
| VASCULAR DISORDERS | | | |



| Adverse Events with Possible Relationship to Blinatumomab (AMG 103) (CTCAE 5.0 Term) [n= 1276] | | | Specific Protocol Exceptions to<br>Expedited Reporting<br>(SPEER) |
|---|---|---|---|
| Likely (>20%) | Less Likely (<=20%) | Rare but Serious (<3%) | |
| | | Capillary leak syndrome <sup>3</sup> | |
| | Flushing <sup>3</sup> | | |
| | Hypertension <sup>3</sup> | | Hypertension <sup>3</sup> (Gr 2) |
| | Hypotension <sup>3</sup> | | Hypotension <sup>3</sup> (Gr 2) |
| | Thromboembolic event <sup>2</sup> | | Thromboembolic event <sup>2</sup> (Gr 2) |

<sup>1</sup>This table will be updated as the toxicity profile of the agent is revised. Updates will be distributed to all Principal Investigators at the time of revision. The current version can be obtained by contacting <a href="PIO@CTEP.NCI.NIH.GOV">PIO@CTEP.NCI.NIH.GOV</a>. Your name, the name of the investigator, the protocol and the agent should be included in the e-mail.

<sup>2</sup>Blinatumomab (AMG 103) is known to cause a variety of adverse events associated with coagulopathy which may include: Activated partial thromboplastin time prolonged, Disseminated intravascular coagulation, Fibrinogen decreased, INR increased, Investigations - Other (blood fibrinogen increased), Investigations - Other (fibrin D dimer increased), Investigations - Other (activated partial thromboplastin time shortened), Investigations - Other (antithrombin III decreased), Investigations - Other (coagulation factor XIII level increased), Investigations - Other (haptoglobin decreased), Investigations - Other (protein S decreased), Platelet count decreased, and Thromboembolic events.

<sup>3</sup>Symptoms of cytokine release syndrome (CRS) and/or allergic reaction may include chills, fever, fatigue, flushing, bronchospasm, and hypotension. In some cases, disseminated intravascular coagulation (DIC), capillary leak syndrome (CLS), and hemophagocytic lymphohistiocytosis/macrophage activation syndrome (HLH/MAS) have been reported in the setting of CRS.

<sup>4</sup>Symptoms of hepatic dysfunction may include Alanine aminotransferase increased, Alkaline phosphatase increased, Aspartate aminotransferase increased, Blood bilirubin increased, and GGT increased under the INVESTIGATIONS SOC.

<sup>5</sup>Immunodeficiency (immunoglobulin decreased) includes immunoglobulins decreased, blood immunoglobulin G decreased, blood immunoglobulin M decreased, and blood immunoglobulin A decreased.

<sup>6</sup>Infection includes all 75 sites of infection under the INFECTIONS AND INFESTATIONS SOC.

<sup>7</sup>Overdoses have been observed. Overdoses resulted in adverse reactions, which were consistent with the reactions observed at the recommended therapeutic dose and included fever, tremors, and headache. In the event of overdose, interrupt the infusion, monitor the patient for signs of toxicity, and provide supportive care. Consider re-initiation of blinatumomab at the correct therapeutic dose when all toxicities have resolved and no earlier than 12 hours after interruption of the infusion.

<sup>8</sup>Acute kidney injury (acute renal failure) is associated with increased creatinine levels.

<sup>9</sup>Tumor lysis syndrome is defined as a massive overload of potassium, phosphate, uric acid, plus hypocalcemia, potentially causing lethal cardiac arrhythmias and/or renal failure.

<sup>10</sup>Blinatumomab (AMG103) is known to cause a variety of nervous system disorders which may include: Ataxia, Cognitive disturbance, Concentration impairment, Depressed level of consciousness, Dizziness, Dysphagia, Dysarthria, Dysesthesia, Dysphasia, Encephalopathy, Facial nerve disorder, Headache,



Lethargy, Memory impairment, Paresthesia, Peripheral sensory neuropathy, Seizure, Somnolence, Syncope, Transient ischemic attacks, Tremor, Voice alteration, Nervous system disorders - Other (allodynia), Nervous Systems disorders - Other (cerebellar syndrome), Nervous system disorders - Other (dysgraphia), Nervous system disorders - Other (facial palsy), Nervous system disorders - Other (hemiparesis), Nervous system disorders - Other (hypertonia), Nervous system disorders - Other (hypotonia), Nervous system disorders - Other (pleocytosis), and Nervous system disorders - Other (polyneuropathy). Additionally, symptoms of some nervous system disorders are adverse events under the PSYCHIATRIC DISORDERS SOC and may include: Agitation, Anxiety, Confusion, Hallucinations, Personality change, and Psychosis.

<sup>11</sup>Rash includes rash, rash maculo-papular, erythema, local erythema, erythematous rash, generalized rash, exanthema, allergic dermatitis, and palmar-plantar erythrodysesthesia syndrome.

Adverse events reported on blinatumomab (AMG 103) trials, but for which there is insufficient evidence to suggest that there was a reasonable possibility that blinatumomab (AMG 103) caused the adverse event:

#### **BLOOD AND LYMPHATIC SYSTEM DISORDERS** - Leukocytosis

CARDIAC DISORDERS - Atrial fibrillation; Cardiac arrest; Heart failure; Left ventricular systolic dysfunction; Myocardial infarction; Pericardial effusion; Sinus bradycardia; Supraventricular tachycardia CONGENITAL, FAMILIAL AND GENETIC DISORDERS - Congenital, familial and genetic disorders - Other (aplasia)

EAR AND LABYRINTH DISORDERS - Vertigo

**EYE DISORDERS** - Blurred vision; Optic nerve disorder; Papilledema; Periorbital edema; Photophobia **GASTROINTESTINAL DISORDERS** - Abdominal distension; Anal mucositis; Dyspepsia; Dysphagia **GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS** - Edema face; Gait disturbance; General disorders and administration site conditions - Other (thrombosis in device); Hypothermia; Malaise; Multi-organ failure

INJURY, POISONING AND PROCEDURAL COMPLICATIONS - Fall; Vascular access complication

**INVESTIGATIONS** - Cardiac troponin I increased; Electrocardiogram QT corrected interval prolonged; INR increased; Investigations - Other (hypoproteinemia); Investigations - Other (lipase decreased); Lipase increased; Lymphocyte count increased

**METABOLISM AND NUTRITION DISORDERS** - Acidosis; Dehydration; Hypercalcemia; Hyperkalemia; Hyperphosphatemia; Hyponatremia; Metabolism and nutrition disorders - Other (fluid overload)

MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS - Muscle cramp; Neck pain NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED (INCL CYSTS AND POLYPS) - Leukemia secondary to oncology chemotherapy; Treatment related secondary malignancy

**NERVOUS SYSTEM DISORDERS** - Amnesia; Facial muscle weakness; Muscle weakness left-sided; Nervous system disorders - Other (difficulty following commands); Neuralgia

**PSYCHIATRIC DISORDERS** - Delirium; Depression; Psychiatric disorders - Other (altered mental status); Psychiatric disorders - Other (sleep disorder); Restlessness

**RENAL AND URINARY DISORDERS** - Acute kidney injury<sup>7</sup>; Hematuria; Proteinuria; Urinary incontinence

REPRODUCTIVE SYSTEM AND BREAST DISORDERS - Genital edema

**RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS** - Adult respiratory distress syndrome; Bronchospasm<sup>3</sup>; Pleural effusion; Productive cough; Pulmonary edema; Respiratory failure; Respiratory, thoracic and mediastinal disorders - Other (chronic obstructive pulmonary disease)

**SKIN AND SUBCUTANEOUS TISSUE DISORDERS** - Dry skin; Purpura; Skin and subcutaneous tissue disorders - Other (skin irritation)

VASCULAR DISORDERS - Hematoma



**Note**: Blinatumomab (AMG 103) in combination with other agents could cause an exacerbation of any adverse event currently known to be caused by the other agent, or the combination may result in events never previously associated with either agent.

#### **Pregnancy and lactation**

<u>Pregnancy Category Unknown</u>: The effect of blinatumomab on fertility has not been evaluated. Blinatumomab is not recommended in pregnant women and in women of childbearing potential not using contraception. It is not known whether blinatumomab or its metabolites are excreted in human milk. Women are not allowed to breastfeed while receiving blinatumomab and for at least 48 hours after the last dose.

#### Formulation and Stability

Blinatumomab is available as a 38.5 mcg preservative-free, white to off-white lyophilized powder for injection in 4 mL single-use vial. The agent is formulated with 3.68 mg citric acid monohydrate, 105 mg trehalose dihydrate, and 25.55 mg lysine hydrochloride, and 0.7 mg polysorbate 80, pH 7. The stopper of the vial is latex free.

IV solution stabilizer for blinatumomab (NSC 773150) is **not for reconstitution of blinatumomab**; it is a component of the final intravenous product. The stabilizer is available as a 10 mL single-use vial of a preservative-free, clear, colorless-to-slightly yellow liquid solution. Each solution consists of 25 mM citric acid monohydrate, 1.25 M L-lysine hydrochloride, and 0.1% (w/v) polysorbate 80, pH 7. The stopper of the vial is latex free.

Store intact vials of blinatumomab and the IV solution stabilizer of blinatumomab refrigerated at  $2^{\circ} - 8^{\circ}$ C ( $36^{\circ} - 46^{\circ}$ F). Protect from light. Shelf life stability studies of the intact vials of blinatumomab and stabilizer solution are on-going.

The stability of the prepared IV solution in **preservative-free 0.9% NaCl** is 8 days when stored refrigerated at  $2^{\circ} - 8^{\circ}$ C ( $36^{\circ} - 46^{\circ}$ F). For storage prior to administration, the prepared infusion solution must be kept at  $2^{\circ}$  C to  $8^{\circ}$  C ( $36^{\circ}$ F to  $46^{\circ}$ F). The total storage and administration time must not exceed 8 days. Once at room temperature, discard the IV bag after 96 hours (4 days).

The stability of the prepared IV solution in **Bacteriostatic 0.9% NaCl** is 14 days when stored refrigerated at  $2^{\circ} - 8^{\circ}$ C ( $36^{\circ} - 46^{\circ}$ F). For storage prior to administration, the prepared infusion solution must be kept at  $2^{\circ}$  C to  $8^{\circ}$  C ( $36^{\circ}$ F to  $46^{\circ}$ F). The total storage and administration time must not exceed 14 days. Once at room temperature, discard the IV bag after 168 hours (7 days). **The 7-day infusion with Bacteriostatic 0.9% NaCl preserved with benzyl alcohol is not allowed in patients weighing less than 22 Kg.** 

#### Preparation

Only trained staff may prepare the blinatumomab IV solution. Blinatumomab must be prepared in an ISO Class 5 containment device, ideally in an ISO Class 7 room as described in USP <797>, but ISO Class 7 is not required. Use aseptic technique and prepare blinatumomab IV solution under a qualified biological safety cabinet.

The label on the IV bag must include the following:

- Patient name and number
- Name of the drug
- Dose (mcg/day and volume/day)
- Infusion rate
- Expiration date and time
- CAUTION: NEW DRUG Limited by United States law to investigational use.



Additional information as required by state, local, and country pharmacy regulations.

Blinatumomab must be dispensed in an acceptable IV bag. Acceptable bags include those made of polyolefin/polyethylene, ethylene vinyl acetate (EVA), or PVC non-DEHP.

The final IV solution <u>must</u> be prepared in the following sequential order (do not deviate from this order; refer to the table below for volume details):

#### 1. Reconstitute blinatumomab lyophilized powder

# Blinatumomab 38.5 mcg/vial Add 3 mL of Sterile Water for Injection (SWFI) to the vial to yield 3.08 mL of blinatumomab at a final concentration of 12.5 mcg/mL.

- a. Rotate the vial to dissolve all powder. Do not shake.
- b. The stability of the reconstituted vial is 4 hours at room temperature  $(22^{\circ}C 27^{\circ}C)$  or 24 hours refrigerated at  $2^{\circ} 8^{\circ}C$ .
- 2. Add the appropriate amount of 0.9% NaCl into the IV bag
- 3. Add the IV solution stabilizer for blinatumomab to the IV bag
  - a. Gently mix the contents of the bag to avoid foaming.
  - b. Discard remaining IV solution stabilizer vial.
- 4. Add the calculated dose (mL) of blinatumomab into the solution in the IV bag
  - a. Rotate the IV bag to mix the solution thoroughly. Do not shake. Avoid foaming the IV bag.
  - b. Visually inspect for floating particles or discoloration of the IV solution. If floaters or discoloration is present, do not use the prepared solution.
  - c. The total volume of blinatumomab IV solution will account for the volume of the IV infusion set for the inpatient or outpatient setting.

**Note:** Overfill volume depends on the volume of **the IV set** used at each institution. See Volume Calculation Table below for details.

#### **VOLUME CALCULATION TABLE**

| | Volume to be prepared | Volume to be infused (rate) |
|---|---|---|
| 24-hour IV bag<br>(includes 30 mL<br>overfill) | <ol> <li>Add mL NaCl (calculated volume of 0.9% NaCl)¹ into approved IV bag*</li> <li>Add 3 mL IV solution stabilizer for blinatumomab²</li> <li>Add mL blinatumomab (calculated dose volume per 150 mL bag)³</li> <li>150 mL total volume⁴</li> </ol> | 120 mL<br>(5 mL/hr) |

123



<sup>1</sup>0.9% NaCl (mL) = total volume to be prepared (150 mL) – stabilizer solution volume (3 mL) – blinatumomab calculated dose volume (mL) per 150 mL bag

 $^{2}$ Stabilizer solution (3 mL) = 0.02 x total volume to be prepared (150 mL)

<sup>3</sup>Blinatumomab calculated dose volume per 150 mL bag (mL) = **24 hour dose** (mcg)  $\div$  24 hour infusion volume (120 mL) x total volume to be prepared (150 mL)  $\div$  blinatumomab concentration (12.5 mcg/mL)

<sup>4</sup>Total volume (150 mL) = Volume to be infused (120 mL) + IV infusion set volume (30 mL)

| | Volume to be prepared | Volume to be infused (rate) |
|---|---|---|
| ALTERNATE 24-hour IV bag (includes 30 mL overfill) | Add mL NaCl (calculated volume of 0.9% NaCl)¹ into approved IV bag* Add 5.4 mL IV solution stabilizer for blinatumomab² Add mL blinatumomab (calculated dose volume per 270 mL bag)³ 270 mL total volume⁴ | 240 mL<br>(10 mL/hr)<br>Note rate difference |

<sup>1</sup>0.9% NaCl (mL) = total volume to be prepared (270 mL) – stabilizer solution volume (5.4 mL) – blinatumomab calculated dose volume (mL) per 270 mL bag

<sup>2</sup>Stabilizer solution (5.4 mL) = 0.02 x total volume to be prepared (270 mL)

<sup>3</sup>Blinatumomab calculated dose volume per 270 mL bag (mL) = 24 hour dose (mcg) ÷ 24 hour infusion volume (240 mL) x total volume to be prepared (270 mL) ÷ blinatumomab concentration (12.5 mcg/mL)

<sup>4</sup>Total volume (270 mL) = Volume to be infused (240 mL) + IV infusion set volume (30 mL)

| | Volume to be prepared | Volume to be infused (rate) |
|---|---|---|
| 48-hour IV bag<br>(includes 30 mL<br>overfill) | <ul> <li>4. Add mL NaCl (calculated volume of 0.9% NaCl)¹ into approved IV bag*</li> <li>5. Add 5.4 mL IV solution stabilizer for blinatumomab²</li> <li>6. Add mL blinatumomab (calculated dose volume per 270 mL bag)³</li> <li>270 mL total volume⁴</li> </ul> | 240 mL<br>(5 mL/hr) |



<sup>1</sup>0.9% NaCl (mL) = total volume to be prepared (270 mL) – stabilizer solution volume (5.4 mL) – blinatumomab calculated dose volume (mL) per 270 mL bag

<sup>2</sup>Stabilizer solution (5.4 mL) = 0.02 x total volume to be prepared (270 mL)

<sup>3</sup>Blinatumomab calculated dose volume per 270 mL bag (mL) = **48 hour dose** (mcg) ÷ 48 hour infusion volume (240 mL) x total volume to be prepared (270 mL) ÷ blinatumomab concentration (12.5 mcg/mL)

<sup>4</sup>Total volume (270 mL) = Volume to be infused (240 mL) + IV infusion set volume (30 mL)

| | Volume to be prepared | Volume to be infused (rate) |
|---|---|---|
| 72-hour IV bag<br>(includes 30 mL<br>overfill) | <ol> <li>Add mL NaCl (calculated volume of 0.9% NaCl)¹ into approved IV bag*</li> <li>Add 7.8 mL IV solution stabilizer for blinatumomab²</li> <li>Add mL blinatumomab (calculated dose volume per 390 mL bag)³</li> <li>390 mL total volume⁴</li> </ol> | 360 mL<br>(5 mL/hr) |

<sup>1</sup>0.9% NaCl (mL) = total volume to be prepared (390 mL) – stabilizer solution volume (7.8 mL) – blinatumomab calculated dose volume (mL) per 390 mL bag

<sup>2</sup>Stabilizer solution (7.8 mL) = 0.02 x total volume to be prepared (390 mL)

<sup>3</sup>Blinatumomab calculated dose volume per 390 mL bag (mL) = **72 hour dose** (mcg) ÷ 72 hour infusion volume (360 mL) x total volume to be prepared (390 mL) ÷ blinatumomab concentration (12.5 mcg/mL)

<sup>4</sup>Total volume (390 mL) = Volume to be infused (360 mL) + IV infusion set volume (30 mL)

| | Volume to be prepared | Volume to be infused (rate) |
|---|---|---|
| 96-hour IV bag<br>(includes 30 mL<br>overfill) | <ol> <li>Add mL NaCl (calculated volume of 0.9% NaCl)¹ into approved IV bag*</li> <li>Add 10.2 mL IV solution stabilizer for blinatumomab²</li> <li>Add mL blinatumomab (calculated dose volume per 510 mL bag)³</li> <li>510 mL total volume⁴</li> </ol> | 480 mL<br>(5 mL/hr) |

<sup>1</sup>0.9% NaCl (mL) = total volume to be prepared (510 mL) – stabilizer solution volume (10.2 mL) – blinatumomab calculated dose volume (mL) per 510 mL bag

<sup>2</sup>Stabilizer solution (10.2 mL) = 0.02 x total volume to be prepared (510 mL)

<sup>3</sup>Blinatumomab calculated dose volume per 510 mL bag (mL) = **96 hour dose** (mcg)  $\div$  96 hour infusion volume (480 mL) x total volume to be prepared (510 mL)  $\div$  blinatumomab concentration (12.5 mcg/mL)

<sup>4</sup>Total volume (510 mL) = Volume to be infused (480 mL) + IV infusion set volume (30 mL)

<sup>\*</sup> Approved bags include those made of polyolefin/polyethylene, ethylene vinyl acetate (EVA), or PVC non-DEHP.



**VOLUME CALCULATION TABLE: 168 hour (7 day) bags (for patients ≥ 22 Kg)** 

| | Volume to be prepared | Volume to be infused (rate) |
|---|---|---|
| 168-hour IV bag<br>(includes 10 mL<br>overfill) | <ol> <li>Add 90 mL Bacteriostatic Sodium<br/>Chloride preserved with 0.9% benzyl<br/>alcohol into compatible empty IV bag.<sup>1</sup></li> <li>Add 2.2 mL IV Solution Stabilizer into<br/>90 mL Bacteriostatic Sodium Chloride<br/>IV bag<sup>2</sup></li> <li>Add the calculated dose volume of<br/>blinatumomab into solution.<sup>3</sup></li> <li>Q.S. with preservative-free 0.9% NaCl<br/>to final volume of 110 mL.<sup>4</sup></li> </ol> | 100.8 mL<br>(0.6 mL/hr) |

<sup>&</sup>lt;sup>1</sup>Approved bags include those made of polyolefin/polyethylene, ethylene vinyl acetate (EVA), or PVC non-DEHP.

[Total volume to be prepared (110 mL)] – [Bacteriostatic Sodium Chloride volume (90 mL)] – [IV stabilizer solution volume (2.2 mL)] – [blinatumomab calculated dose volume (mL)] = mL preservative-free NS

Guidelines for Administration: See Treatment and Dose Modifications sections of the protocol.

Premedication with dexamethasone is required prior to the first dose of blinatumomab in the first cycle, prior to a step dose and when restarting an infusion after an interruption of 4 or more hours in the first cycle.

#### IV infusion and infusion set details:

Blinatumomab must be administered as an infusion through an acceptable central line at rates described in the tables above to deliver the intended daily dose. Only non-DEHP PVC, polyolefin, or EVA tubing/lines with a 0.2 µm inline filter are acceptable for bags prepared for 24 to 96 hour infusions (i.e., prepared with preservative-free normal saline).

For 168 hour (7-day) infusions prepared with bacteriostatic sodium chloride, use non-DEHP PVC, polyolefin, or EVA tubing/lines; an in-line filter is NOT required during the administration of blinatumomab 7-day IV bag. This is to alleviate the IV pressure or backflow into the IV line during the IV infusion of 7-day bag.

Avoid flushing the line during the Blinatumomab infusion to avoid bolus dosing. There are some times when there will be unavoidable flushing for central line care. It is also unavoidable to flush the line at completion of the Blinatumomab 28 day cycle. For outpatient administration, use FDA approved pumps. Only the exact volume should be administered; any remaining overfill should be discarded appropriately.

<sup>&</sup>lt;sup>2</sup>Stabilizer solution (2.2 mL) = 0.02 x total volume to be prepared (110 mL)

 $<sup>^3</sup>$ Blinatumomab calculated dose volume per 110 mL bag (mL) = 168-hour dose (mcg)  $\div$  volume to be infused (100.8 mL) x total volume to be prepared (110 mL)  $\div$  12.5 mcg/mL of blinatumomab

<sup>&</sup>lt;sup>4</sup>Calculated volume of preservative-free 0.9% NaCl (mL):



#### <u>Infusion pump requirements:</u>

Use a programmable pump that is approved by the appropriate regulatory authority for the country in which the subject is undergoing treatment. The pump alarm must be visual and auditory. **The pump must be lockable. Elastomeric pumps are NOT allowed.** CADD pumps are allowed; however, the cassettes used in CADD pumps are not compatible with blinatumomab and thus, **not** allowed.

Should blinatumomab need to be administered through a pharmacy satellite or home health care service center, refer to the outpatient administration guidelines in <u>Appendix VII-A</u>.

**Record all infusion interruptions.** Blinatumomab continuous infusion administration should not be interrupted, if possible. In case of infusion interruption due to any technical or logistical reasons (e.g. routine PORT needle changes, procedural sedation), the interruption should be as short as possible and the infusion restarted as soon as possible.

For interruptions lasting longer than four hours, the re-initiation of the infusion must take place in the hospital under supervision of the investigator for at least 12 hours after re-initiation of the infusion to evaluate for possible side effects. Monitor patients for potential adverse events as described in the protocol and the Investigator Brochure.

Monitor patients for cytokine release syndrome, tumor lysis syndrome, and infusion reaction. Refer to protocol for specific recommendation. Monitor patients for psychiatric events such as confusion, disorientation, and cognitive attention disturbances. Patients should not drive or operate dangerous machinery while receiving blinatumomab.

#### **Supplier**

Blinatumomab and the solution stabilizer for blinatumomab is supplied by Amgen, Inc and distributed by the Division of Cancer Treatment and Diagnosis (DCTD), NCI. **Do not use commercial supply.** 

#### **Obtaining the Agent**

#### Agent Ordering:

NCI supplied agent may be requested by the eligible participating investigator (or their authorized designee) at each participating institution. The CTEP assigned protocol number must be used for ordering all CTEP supplied investigational agents. The responsible investigator at each participating institution must be registered with CTEP, DCTD through an annual submission of FDA form 1572 (Statement of Investigator), NIH Biosketch, Agent Shipment Form, and Financial Disclosure Form (FDF). If there are several participating investigators at one institution, CTEP supplied investigational agents for the study should be ordered under the name of one lead participating investigator at that institution. This study does not need a starter supply. Confirmation of patient enrollment to an arm with blinatumomab is required for initial drug shipment.

Submit agent requests through the PMB Online Agent Order Processing (OAOP) application. Access to OAOP requires the establishment of a CTEP Identity and Access Management (IAM) account and the maintenance of an "active" account status, and a "current" password, and active person registration status. For questions about drug orders, transfers, returns, or accountability, call or email PMB any time. Refer to the PMB's website for specific policies and guidelines related to agent management.

#### **Agent Accountability**

#### **Agent Inventory Records:**

The investigator, or a responsible party designated by the investigator, must maintain a careful record of



the receipt, dispensing and final disposition of all agents received from the PMB using the appropriate NCI Investigational Agent (Drug) Accountability Record (DARF) available on the CTEP forms page. Store and maintain separate NCI Investigational Agent Accountability Records for each agent, strength, formulation and ordering investigator on this protocol.

#### **Investigator Brochure Availability**

The current version(s) of the IB(s) for the agent will be accessible to site investigators and research staff through the PMB Online Agent Order Processing (OAOP) application. Access to OAOP requires the establishment of a CTEP IAM account and the maintenance of an "active" account status, a "current" password, and active person registration status. Questions about IB access may be directed to the PMB IB coordinator via email.

#### **Useful Links and Contacts**

- CTEP Forms, Templates, Documents: http://ctep.cancer.gov/forms/
- NCI CTEP Investigator Registration: <u>RCRHelpDesk@nih.gov</u>
- PMB policies and guidelines: http://ctep.cancer.gov/branches/pmb/agent management.htm
- PMB Online Agent Order Processing (OAOP) application: <a href="https://ctepcore.nci.nih.gov/OAOP/">https://ctepcore.nci.nih.gov/OAOP/</a>
- CTEP Identity and Access Management (IAM) account: <a href="https://ctepcore.nci.nih.gov/iam/">https://ctepcore.nci.nih.gov/iam/</a>
- CTEP IAM account help: <a href="mailto:ctepreghelp@ctep.nci.nih.gov">ctepreghelp@ctep.nci.nih.gov</a>
- PMB email: PMBAfterHours@mail.nih.gov
- IB Coordinator: IBCoordinator@mail.nih.gov
- PMB phone and hours of service: (240) 276-6575 Monday through Friday between 8:30 am and 4:30 pm (ET)



#### 6.2 ASPARAGINASE Erwinia chrysanthemi

(05-07-19)

(Erwinia *chrysanthemi*, Erwinase<sup>®</sup>, Erwinaze<sup>TM</sup>, Crisantaspase) NSC #106977

#### Source and Pharmacology:

L-asparagine is a nonessential amino acid synthesized by the transamination of L-aspartic acid by a reaction catalyzed by the enzyme L-asparagine synthetase. Neoplastic cells associated with acute lymphoblastic leukemia, acute myeloid leukemia and lymphoblastic lymphosarcoma are asparagine-dependent but lack asparagine synthetase activity. The administration of L-asparaginase produces an anti-neoplastic effect by catalyzing asparagine into aspartic acid and ammonia. As a result, these cells lack the ability to produce the asparagine necessary for protein metabolism and survival. Deamination of glutamine may also play a role in the antineoplastic activity of asparaginase.

Asparaginase Erwinia chrysanthemi (Erwinaze®) is asparaginase derived from cultures of Erwinia chrysanthemi. L-asparaginase is a tetrameric enzyme; each of the four identical subunits has a molecular weight of approximately 35 kDa. Asparaginase Erwinia chrysanthemi is immunologically distinct from E. coli L-asparaginase and may allow continued asparaginase therapy when a hypersensitivity reaction occurs to Escherichia coli-derived asparaginase. The package labeling states that there is insufficient information to characterize the incidence of antibodies to asparaginase Erwinia chrysanthemi. Several factors are involved in immunogenicity assay results and the assessment of antibodies, including assay methodology, assay sensitivity and specificity, sample handling, timing of sample collection, concomitant medications, and the underlying disease state. The following data have been reported on each of the three preparations of asparaginase:

| Clinical Pharmacology<br>of Asparaginase<br>Formulation | Elimination half-life (IM) | % Anti-Asparaginase<br>Antibody positive<br>patients |
|---|---|---|
| Native Escherichia Coli | 26-30 hours | 45-75 |
| Pegylated-asparaginase | 5.5-7 days | 5-18 |
| Erwinia Asparaginase | 16 hours (7-13 hrs package insert) | 30-50 |

From: Avramis, V; Panosyan, E; Pharmacokinetic/Pharmacodynamic Relationships of Asparaginase Formulations: The Past, the Present and Recommendations for the Future. Clin Pharmacokinet 2005; 44 (4): 367-393.

Effective asparaginase levels have been defined as activity of  $\geq 0.1$  International Units per mL. Clinical trials with asparaginase *Erwinia chrysanthemi* demonstrated that 100% of patients achieved effective asparaginase levels at 48 and 72 hours (n=35 and n=13, respectively) following the third total dose when given on a Monday, Wednesday, Friday schedule using the IM route of administration. In a multicenter study characterizing the pharmacokinetic profile of 25,000 International Units/m<sup>2</sup> Erwinaze® given intravenously over one hour on the same dosing schedule of Monday, Wednesday, Friday for 2 consecutive weeks, 83% (20/24) and 43% (9/21) of evaluable patients achieved an asparaginase activity level of  $\geq 0.1$  International Units/mL at 48 post-dose 5 and 72 hours post-dose 6, respectively. No formal drug interaction studies have been performed with asparaginase *Erwinia chrysanthemi*.

129



| | • | • , | |
|-----|-----|--------------|----|
| To | 711 | <b>11</b> 11 | 7. |
| 104 | 71/ | JΙU | ٧. |

| - | Common | Occasional | Rare |
|---|---|---|---|
| | Happens to 21-100 | Happens to 5-20 children | Happens to < 5 children out of |
| | children out of every 100 | out of every 100 | every 100 |
| Immediate: | | Allergic reactions, | Local injection site reactions, |
| Within 1-2 days of | | anaphylaxis, urticaria | fever |
| receiving drug | | | |
| Prompt: | | | Pancreatitis, glucose |
| Within 2-3 weeks, | | | intolerance, |
| prior to the next | | | thrombosis, hemorrhage, |
| course | | | transient ischemic attack, |
| | | | disseminated intravascular |
| | | | coagulation, |
| | | | hyperbilirubinemia, alanine |
| | | | aminotransferase increased, |
| | | | aspartate aminotransferase |
| | | | increased, hyperglycemia, |
| | | | hyperammonemia, vomiting, |
| | | | nausea, abdominal pain, |
| | | | headache, diarrhea, seizure |
| Unknown | Fetal toxicities and terato | genic effects of L-asparag | ginase have been noted in |
| Frequency and | animals. Adequate, well- | controlled studies of aspar | aginase <i>Erwinia</i> |
| Timing: | chrysanthemi have NOT | been conducted. It is not l | known whether asparaginase |
| | | | ct the ability to reproduce. It |
| | | | is excreted into breast milk. |
| | | | uld be avoided in pregnant or |
| | lactating patients. | <b>,</b> | 1 8 |
| (I) T | | | |

(L) Toxicity may also occur later.

#### Formulation and Stability:

Asparaginase *Erwinia chrysanthemi* is supplied as a sterile, white lyophilized powder for reconstitution in a clear glass vial with a 3 mL capacity. Each vial contains 10,000 International Units of asparaginase *Erwinia chrysanthemi* and the following inactive ingredients: glucose monohydrate (5.0 mg), sodium chloride (0.5 mg). Store intact vials between 2°C and 8°C (36° to 46°F). Protect from light.

Guidelines for Administration: See Treatment and Dose Modifications sections of the protocol.

*Erwinia* asparaginase can be administered by intramuscular injection or by intravenous infusion. Use appropriate precautions for preparation of a hazardous agent. Visually inspect the powder in vial for foreign particles or discoloration prior to reconstitution.

For intramuscular administration, the contents of each vial should be reconstituted by slowly adding 1 mL or 2 mL of sterile, preservative-free NS to the inner vial wall. The final concentration is 10,000 International Units per mL when using 1 mL for reconstitution or 5,000 International Units per mL when using 2 mL for reconstitution. Gently mix or swirl the contents to dissolve the contents of the vial. Do not shake or invert the vial. The resulting solution should be clear and colorless. Discard if any particulate matter or protein aggregates are visible. Withdraw the appropriate dosing volume into a polypropylene syringe within 15 minutes of reconstitution. Polycarbonate luerlok syringes from B-D (1 mL) are also acceptable (personal communication, EUSA Pharma). Discard any unused drug; do not save or use any unused drug remaining in the vial. No more than 2 mL should be given at any one injection site. Doses larger than 2 mL should be divided and given in separate administration sites.



For intravenous use, slowly inject the appropriate volume of reconstituted solution into a Normal Saline 100 mL infusion bag; do not shake or squeeze the bag. Infuse *Erwinia* asparaginase over 1 hour. Do not infuse other intravenous drugs through the same intravenous line while infusing *Erwinia* asparaginase. Please see <a href="http://www.erwinazesupply.com">http://www.erwinazesupply.com</a> to check which batches may require the use a 0.2-micron, low protein binding, in-line filter for IV administration.

Administer the dose within a 4 hour time period from reconstitution. If the dose is not used within this time period, discard the dose. Do not freeze or refrigerate the reconstituted solution.

The product used in Australia has an 8 hour expiry (from Porton Biopharma, Salisbury, UK).

Have available during and after the infusion: antihistamine, epinephrine, oxygen, and IV corticosteroids. Observe patient for ONE hour after administration for signs of hypersensitivity reactions.

#### **Drug Ordering:**

In the United States, asparaginase *Erwinia chrysanthemi* (Erwinaze®) is McKesson Plasma and Biologics. Verify your institution has a contract with McKesson Plasma and Biologics before ordering. If not, contact McKesson at 877-625-2566 for assistance setting up an account.

Orders may be placed online or via phone, fax, or email. Orders placed by 7:30 pm EST will ship the next day.

Orders may be placed online via http://Connect.McKesson.com

Orders may be submitted via fax to 888-752-7626

Orders may be submitted via email or MPBOrders@McKesson.com

Email all other information requests to MPB@McKesson.com

Regular order hours: M-F 9:00 am – 7:30 pm EST;

Emergency order after hours services (24/7/365): 877-625-2566

#### **CANADIAN SITES**

Asparaginase *Erwinia chrysanthemi* is commercially available in Canada. Canadian sites may purchase the Canadian commercial supply from Jazz Pharmaceuticals via CGF Pharmatech, Montreal, Quebec, (order desk phone: 1-514-343-0344 or 1-866-343-0344, fax: 1-514-343-0340). CGF requests that a site fax a Purchase Order number. There is no special fax order form. Shipments are sent Monday to Wednesday only and usually arrive at the site within 48-72 hours.

#### 6.3 CYCLOPHOSPHAMIDE INJECTION

(03/13/13)

(Cytoxan) NSC #26271

#### Source and Pharmacology:

Cyclophosphamide is an alkylating agent related to nitrogen mustard. Cyclophosphamide is inactive until it is metabolized by P450 isoenzymes (CYP2B6, CYP2C9, and CYP3A4) in the liver to active compounds. The initial product is 4-hydroxycyclophosphamide (4-HC), which is in equilibrium with aldophosphamide, which spontaneously releases acrolein to produce phosphoramide mustard. Phosphoramide mustard, which is an active bifunctional alkylating species, is 10 times more potent *in vitro* than is 4-HC and has been shown to produce interstrand DNA cross-link analogous to those produced by mechlorethamine. Approximately 70% of a dose of cyclophosphamide is excreted in the urine as the inactive carboxyphosphamide and 5-25% as unchanged drug. The plasma half-life ranges from 4.1 to 16 hours after IV administration.



**Toxicity:** 

| | Common | Occasional | Rare |
|---|---|---|---|
| | Happens to 21-100 | Happens to 5-20 children | Happens to < 5 children |
| | children out of every 100 | out of every 100 | out of every 100 |
| Immediate: | Anorexia, nausea & | Abdominal discomfort, | Transient blurred vision, |
| Within 1-2 | vomiting | diarrhea | nasal stuffiness with |
| days of | (acute and delayed) | | rapid administration, |
| receiving drug | | | arrhythmias (rapid |
| | | | infusion), skin rash, |
| | | | anaphylaxis, SIADH |
| Prompt: | Leukopenia, alopecia, | Thrombocytopenia, | Cardiac toxicity with |
| Within 2-3 | immune suppression | anemia, hemorrhagic | high dose (acute – CHF |
| weeks, prior to | | cystitis (L) | hemorrhagic myocarditis, |
| the next course | | | myocardial necrosis) (L), |
| | | | hyperpigmentation, nail |
| | | | changes, impaired wound |
| | | | healing, infection |
| | | | secondary to immune |
| | | | suppression |
| Delayed: | Gonadal dysfunction: | Amenorrhea <sup>1</sup> | Gonadal dysfunction: |
| Any time later | azoospermia or | | ovarian failure <sup>1</sup> (L), |
| during therapy | oligospermia (prolonged | | interstitial pneumonitis, |
| | or permanent) <sup>1</sup> (L) | | pulmonary fibrosis <sup>2</sup> (L) |
| Late: | | | Secondary malignancy |
| Any time after | | | (ALL, ANLL, AML), |
| completion of | | | bladder carcinoma (long |
| treatment | | | term use > 2 years), |
| | | | bladder fibrosis |
| Unknown | | ogenic effects of cycloph | |
| Frequency | | intineoplastic agents) have | |
| and Timing: | | somal abnormalities, multipl | |
| | | Cyclophosphamide is exc | |
| | | raindicated during breastfe | |
| | | east fed infants and the po | tential for serious adverse |
| | effects. | | |

Dependent on dose, age, gender, and degree of pubertal development at time of treatment.

#### Formulation and Stability:

Cyclophosphamide for injection is available as powder for injection or lyophilized powder for injection in 500 mg, 1 g, and 2 g vials. The powder for injection contains 82 mg sodium bicarbonate/100 mg cyclophosphamide and the lyophilized powder for injection contains 75 mg mannitol/100 mg cyclophosphamide. Storage at or below 25°C (77°F) is recommended. The product will withstand brief exposures to temperatures up to 30°C (86°F).

Guidelines for Administration: See Treatment and Dose Modifications sections of the protocol.

#### Cyclophosphamide for Injection:

If the drug will be administered as undiluted drug at the 20 mg/mL concentration, then reconstitute to 20 mg/mL with NS ONLY to avoid a hypotonic solution. If the drug will be further diluted prior

<sup>&</sup>lt;sup>2</sup> Risk increased with pulmonary chest irradiation and higher doses.

<sup>(</sup>L) Toxicity may also occur later.



to administration, then first reconstitute with NS, SWFI, or Bacteriostatic Water for Injection (paraben preserved only) to a concentration of 20 mg/mL. Following reconstitution further dilute in dextrose or saline containing solutions for IV use.

**Supplier:** Commercially available from various manufacturers. See package insert for further information.

#### 6.4 CYCLOSPORINE A

(11/16/17)

132

(Cyclosporine, CYA, Sandimmune®, Neoral®, Gengraf®) NSC #290193

#### Source and Pharmacology:

Cyclosporine (CSA) is a lipophilic fungal peptide consisting of 11 amino acids. CSA is a potent immunosuppressive agent which prolongs survival of allogeneic transplants involving skin, heart, kidney, pancreas, bone marrow, small intestine, and lung. Current evidence suggests that cyclosporine selectively inhibits the transcription of IL-2, the action of which stimulates the proliferation of activated T-lymphocytes. CSA has been shown in vitro to be a potent inhibitor of P-glycoprotein, which has been postulated to be a factor in multi-drug resistance to various antineoplastic agents. The terminal half-life of CSA is approximately 19 hours (range 10 to 27 hours). Ninety-nine percent of CSA is metabolized. Elimination is primarily biliary with approximately 6% excreted in the urine. In the circulation, CSA is mainly bound to high, low, or very low density lipoproteins and to chylomicrons. Only a small fraction circulates unbound. The volume of distribution varies from 3.5 L/kg to 13 L/kg with higher concentrations of drug found in the liver, lymphocytes, kidney, heart, lung, pancreas, fat, neural, and muscle cells. CSA clearance rates have been shown to be higher in pediatric patients and for patients < 25 years old. The absorption of cyclosporine from the gastrointestinal tract is incomplete and variable exhibiting large intra- and inter-patient variability. Drugs that stimulate or inhibit hepatic P450 enzymes will alter clearance of CSA and close attention to potential drug interactions is crucial.

**Toxicity:** 

| | Common | Occasional | Rare |
|---|---|---|---|
| | Happens to 21-100 | Happens to 5-20 | Happens to < 5 children |
| | children out of every 100 | children out of every 100 | out of every 100 |
| Immediate: | Hypertension (L), | Headache (L), nausea | Anaphylaxis, |
| Within 1-2 days | immunosuppression (L) | and vomiting, diarrhea | angioedema, seizure (L), |
| of receiving drug | | | arrhythmia, chest pain, fever, facial flushing |
| Prompt: | Tremor (L), renal | Hypomagnesemia (L), | Confusion (L), |
| Within 2-3 | dysfunction (acute with | hyperlipidemia (L) | somnolence (L), |
| weeks, prior to | decrease in GFR, | | insomnia, depression (L), |
| the next course | impaired urinary | | anxiety, dizziness, rash, |
| | concentrating ability, and | | urticaria, acne, |
| | sodium retention) | | hyperkalemia, |
| | | | encephalopathy, |
| | | | hemolytic-uremic |
| | | | syndrome, cardiac failure, |
| | | | MI, leukopenia (L), |
| | | | anemia, |
| | | | thrombocytopenia, |
| | | | increased creatinine, |
| | | | infections, |
| | | | hyperbilirubinemia (L), |
| | | | hepatic insufficiency |

133



| Delayed: | Hirsutism (L) | Gingival hyperplasia (L) | Tinnitus, vestibular |
|---|---|---|---|
| Any time later | | | disorder, cholelithiasis, |
| during therapy, | | | cataracts (L), |
| excluding the | | | gynecomastia, chronic |
| above conditions | | | renal dysfunction |
| Late: | | | Lymphoproliferative |
| Any time after | | | disorders, skin |
| completion of | | | malignancies |
| treatment | | | |
| Unknown | Fetal toxic effects of cycle | osporine have been noted | in animals. Of the reported |
| Frequency and | outcomes of 116 pregn | ancies in women recei | ving cyclosporine during |
| Timing: | pregnancy, 90% of whom | were transplant patients, a | and most of whom received |
| | cyclosporine throughout | the entire gestational pe | eriod, the only consistent |
| | | | ational period of 28 to 36 |
| | | | Cyclosporine is excreted in |
| | human milk; nursing shou | ld be avoided. | |

(L) Toxicity may also occur later.

#### Formulation and Stability:

#### IV formulation:

Cyclosporine (non-modifiedSandIMMUNE®) is available as a (50 mg/mL) 5 mL ampule use containing 650 mg polyoxyethylated castor oil (cremophor) and 32.9% alcohol. Store at temperatures below 30°C (86°F) and protected from light.

#### Oral formulations:

#### 1. Non-modified:

Cyclosporine (SandIMMUNE®) 25 mg and 100 mg capsule, 100 mg/mL oral solution. Inactive ingredients include: Sandimmune® Capsule = dehydrated alcohol, sorbitol, glycerol, corn oil, gelatin, polyoxyethylated glycolysed glycerides. Sandimmune® Solution = olive oil, dehydrated alcohol, polyoxyethylated glycolysed glycerides.

#### 2. Modified:

Cyclosporine (modified, Neoral®, Gengraf®) is available as a 25 mg capsule, 100 mg capsule, and 100 mg/mL oral solution. Inactive ingredients include: Neoral® capsule and solution = dehydrated alcohol, corn oil, polyoxyl 40 hydrogenated castor oil, α tocopherol, gelatin, and propylene glycol. Gengraf® Capsule and solution = dehydrated alcohol, gelatin, polyethylene glycol, polyoxyl 35 castor oil, polysorbate 80, propylene glycol, and sorbitan monooleate.

Store capsules in the original unit-dose container at controlled room temperature, 15°-30°C (59°-86°F). Store oral solutions in the original container at controlled room temperature, 68°-77°F (20°-25°C). Do not store in the refrigerator. Once opened, the contents must be used within two months. At temperatures below 68°F (20°C) the solution may gel; light flocculation or the formation of a light sediment may also occur. There is no impact on product performance or dosing using the syringe provided. Allow to warm to room temperature, 77°F (25°C), to reverse these changes.

NOTE: Sandimmune®, Neoral®, and Gengraf® ARE NOT BIOEQUIVALENT. Liquid formulations of each trade name are equivalent to capsules of that same trade name. Conversion from one trade name product to another is generally done at a 1:1 ratio, but requires close monitoring. Conversions from IV to PO are usually done at a 1:3 ratio, but should be monitored closely. Adjusting emulsion products to the same trough concentration as other oral products results in greater total exposure to the drug.



Guidelines for Administration: See Treatment and Dose Modifications sections of the protocol.

#### Injection:

Dilute 1 mL (50 mg) of cyclosporine injection IV concentrate (non-modified, SandIMMUNE®) in 20 mL-100 mL NS or D5W (0.5-2.5 mg/mL). Diluted infusion solutions are stable for 24 hours at room temperature under fluorescent light.

Cyclosporine injection was physically and chemically stable for at least 14 days when diluted in NS or D5W to a concentration of 0.2 and 2.5 mg/mL and stored at 25°C in polypropylene–polyolefin bags (Li M, et al. Am J Health-Syst Pharm. 2011; 68:1646-50).

Cyclosporine injection was stable for at least two weeks when diluted in NS or D5W to a 2.5 mg/mL concentration and stored at 25°C in EVA containers. Cyclosporine injection is stable for up to 1 week when diluted in NS or D5W to a 0.2 mg/mL concentration and stored in EVA containers at 25°C (Li M, et al. Am J Health-Syst Pharm 2013; 70:1970-1972).

The Cremophor® EL (polyoxyethylated castor oil) contained in the concentrate for intravenous infusion can cause phthalate stripping from PVC. It is strongly recommended that glass bottles and non-PVC tubing be used to minimize patient exposure to DEHP.

Monitor closely for an acute allergic reaction for the first 30 minutes and at frequent intervals thereafter. Note: cyclosporine absorbs into plastics and can give falsely high serum or blood concentrations if blood samples are collected from the same line through which cyclosporine was administered.

#### Oral:

Administer at a consistent time of day and at consistent intervals with regard to meals. Do not use plastic or styrofoam cups. If diluted with juice or milk, use a glass container and rinse with additional diluent, and then consume to ensure that complete dose has been taken. Do not use water or cleaning agents on the dosing syringe. To improve palatability, mix Sandimmune® with milk, chocolate milk or orange juice; mix Neoral® or Gengraf® with orange juice or apple juice but NOT milk. After mixed, have patient consume immediately. **DO NOT MIX GRAPEFRUIT JUICE with any cyclosporine-containing product.** Grapefruit juice consumption should be avoided during therapy with cyclosporine.

**Supplier:** Commercially available. See package insert for further information.

#### 6.5 **CYTARABINE - ALL ROUTES**

(07/13/15)

(Cytosine arabinoside, Ara-C, Cytosar®) NSC #63878

#### Source and Pharmacology:

Cytarabine appears to act through the inhibition of DNA polymerase. A limited, but significant, incorporation of cytarabine into both DNA and RNA has also been reported. It exhibits cell Phase specificity, primarily killing cells undergoing DNA synthesis (S-Phase) and under certain conditions blocking the progression of cells from the G1 Phase to the S-Phase. Cytarabine is metabolized by deoxycytidine kinase and other nucleotide kinases to the nucleotide triphosphate (Ara-CTP), an effective inhibitor of DNA polymerase. Ara-CTP is inactivated by a pyrimidine nucleoside deaminase, which converts it to the nontoxic uracil derivative (Ara-U). It appears that the balance of kinase and deaminase levels may be an important factor in determining sensitivity



or resistance of the cell to cytarabine. It has an initial distributive Phase  $t_{1/2}$  of about 10 minutes, with a secondary elimination Phase  $t_{1/2}$  of about 1 to 3 hours. Peak levels after intramuscular or subcutaneous administration of cytarabine occur about 20 to 60 minutes after injection and are lower than IV administration. Intrathecally administered doses are metabolized and eliminated more slowly with a  $t_{1/2}$  of about 2 hours.

Toxicity: (Intravenous, SubQ, IM)

| Toxicity: (Intravend | | Occasional | Dan. |
|---|---|---|---|
| | Common Happens to 21-100 children | Happens to 5-20 children | Rare Happens to < 5 children |
| | out of every 100 | out of every 100 | * * |
| T | | | out of every 100 |
| Immediate:<br>Within 1-2 days of<br>receiving drug | Nausea, vomiting, anorexia With High Dose: conjunctivitis | Flu-like symptoms with fever, rash | Ara-C syndrome (fever, myalgia, bone pain, occasionally chest pain, maculopapular rash, malaise, conjunctivitis), anaphylaxis, swelling, pain and redness at the site of the medication injection (SubQ or IM injection) |
| | | | With High Dose: cardiomyopathies (vasculitis, and pericarditis), cerebral and cerebellar dysfunction including: encephalopathy, aseptic meningitis, ataxia, dysphasia, nystagmus, a decreased level of consciousness, personality changes, somnolence, seizures |
| Prompt: | Myelosuppression (anemia, | Diarrhea, hypokalemia, | Hepatotoxicity, sinusoidal |
| Within 2-3 weeks, | thrombocytopenia, | hypocalcemia, | obstruction syndrome |
| prior to the next course | leukopenia, megaloblastosis,<br>reticulocytopenia),<br>stomatitis, alopecia | hyperuricemia With High Dose: capillary pulmonary leak syndrome (RDS, pulmonary edema) | (SOS, formerly VOD),<br>urinary retention, renal<br>dysfunction, pain and<br>erythema of the palms<br>and soles |
| Delayed:<br>Any time later during<br>therapy, excluding the<br>above conditions | | | Asymptomatic<br>nonoliguric<br>rhabdomyolysis |
| Unknown Frequency and Timing: | Fetal toxicities and teratogen is unknown whether the drug | | e been noted in humans. It |

**Toxicity: (Intrathecal)** 

| * | Common | Occasional | Rare |
|---|---|---|---|
| | Happens to 21-100 | Happens to 5-20 children | Happens to < 5 children |
| | children out of every 100 | out of every 100 | out of every 100 |
| Immediate: | Nausea, vomiting, fever, | Arachnoiditis | Rash, somnolence, |
| Within 1-2 days of | headache | | meningismus, |
| receiving drug | | | convulsions, paresis |
| Prompt: | | | Myelosuppression, |
| Within 2-3 weeks, | | | ataxia |
| prior to the next | | | |
| course | | | |



| Delayed: | Necrotizing |
|---------------------|---------------------------|
| Any time later | leukoencephalopathy, |
| during therapy, | paraplegia, blindness (in |
| excluding the above | combination with XRT |
| condition | & systemic therapy) |

#### Formulation:

Cytarabine for Injection is available in vials of 100 mg, 500 mg, 1 g, and 2 g containing a sterile powder for reconstitution. It is also available at a 20 mg/mL concentration with benzyl alcohol (25 mL per vial) or as a preservative free solution (5 mL, 50 mL per vial), and at a 100 mg/mL concentration with benzyl alcohol (20 mL vial) or as preservative free solution (20 mL vial). Hydrochloric acid and/or sodium hydroxide may be added to adjust the pH. Store at 25°C (77°F); excursions permitted to 15°-30°C (59°-86°F). Cytarabine solutions should be protected from light.

Guidelines for Administration: See <u>Treatment</u> and <u>Dose Modifications</u> sections of the protocol.

#### IV Infusion:

Reconstitute the lyophilized powder with Bacteriostatic Water for Injection or NS injection. Solution containing bacteriostatic agent should not be used for the preparation of doses > 200 mg/m². May be further diluted with dextrose or sodium chloride containing solutions. May give by IV push injection, by IV infusion, or by continuous infusion.

**Low Dose** ( $\leq$  200 mg/m<sup>2</sup>/dose): For administration by IV push, reconstitute to a concentration of 20-100 mg/mL.

**High Dose** (≥ 1000 mg/m²/dose): Administer steroid eye drops (dexamethasone or prednisolone), 2 drops each eye q6h beginning immediately before the first dose and continuing 24 hours after the last dose. If patient does not tolerate steroid eye drops, administer artificial tears on a q2-4 hour schedule.

Stability: When reconstituted with Bacteriostatic Water for Injection, cytarabine is stable for 48 hours at room temperature. Solutions reconstituted without a preservative should be used immediately. Discard if solution appears hazy. Diluted solutions in D5W or NS are stable for 8 days at room temperature; however, the diluted cytarabine should be used within 24 hours for sterility concerns.

<u>Subcutaneous or IM:</u> Dilute with Bacteriostatic Water for Injection or NS to a concentration not to exceed 100 mg/mL. Rotate injection sites for subcutaneous/IM administration.

Supplier: Commercially available from various manufacturers. See package insert for further information.

#### 6.6 **DEXAMETHASONE**

(05/07/19)

(Decadron®, Hexadrol®, Dexone®, Dexameth®) NSC #34521

#### Source and Pharmacology:

Dexamethasone is a synthetic fluorinated glucocorticoid devoid of mineralocorticoid effects. Dexamethasone, 0.75 mg, has potent anti-inflammatory activity equivalent to approximately 5 mg of prednisone. Glucocorticoids produce widespread and diverse physiologic effects on carbohydrate, protein, and lipid metabolism, electrolyte and water balance, functions of the cardiovascular system, kidney, skeletal muscle, and the nervous systems. Glucocorticoids reduce the concentration of thymus-dependent lymphocytes (T-lymphocytes), monocytes, and eosinophils. Glucocorticoids



selectively bind to the cortisol receptors on human lymphoid cells which are found in larger numbers on leukemic lymphoblasts. They also decrease binding of immunoglobulin to cell surface receptors and inhibit the synthesis and/or release of interleukins, thereby decreasing T-lymphocyte blastogenesis and reducing expansion of the primary immune response. The specific cellular mechanisms that act to halt DNA synthesis are thought to be related to inhibition of glucose transport or phosphorylation, retardation of mitosis, and inhibition of protein synthesis. Elimination half-lives for the following age groups have been reported to be: infants and children under 2 years of age: 2.3 to 9.5 hours, 8 to 16 years: 2.82 to 7.5 hours, and adults (age not specified): 3 to 6 hours. The biologic half-life is 36-72 hours. It is primarily metabolized in the liver and excreted by the kidneys.

**Toxicity:** 

| | Common | Occasional | Rare |
|---|---|---|---|
| | Happens to 21-100 | Happens to 5-20 children | Happens to < 5 children |
| | children out of every 100 | out of every 100 | out of every 100 |
| Immediate:<br>Within 1-2 days<br>of receiving<br>drug | Insomnia, hyperphagia | Gastritis | Hyperuricemia |
| Prompt: Within 2-3 weeks, prior to the next course | Immunosuppression,<br>personality changes (mood<br>swings, euphoria, anxiety,<br>depression), pituitary-<br>adrenal axis suppression,<br>acne (L) | Hyperglycemia, facial<br>erythema, poor wound<br>healing, infections<br>(bacterial, fungal, parasitic,<br>viral), edema | Pancreatitis (L),<br>increased intraocular<br>pressure (L),<br>hypertension, psychosis,<br>vertigo, headache |
| Delayed:<br>Any time later<br>during therapy | Cushing's syndrome<br>(moon facies, truncal<br>obesity) | Striae and thinning of the<br>skin, easy bruising, muscle<br>weakness, osteopenia | Spontaneous fractures (L), growth suppression, peptic ulcer and GI bleeding, pseudotumor cerebri (increased intracranial pressure with papilledema, headache), aseptic necrosis of the femoral and humeral heads (L), urolithiasis¹ (L) |
| Late:<br>Any time after<br>completion of<br>treatment | | Cataracts (which may be reversible on discontinuation of dexamethasone in children) | |
| Unknown<br>Frequency and<br>Timing: | <b>Fetal and teratogenic toxicities</b> : dexamethasone crosses the placenta with 54% metabolized by enzymes in the placenta. In animal studies, large doses of cortisol administered early in pregnancy produced cleft palate, stillborn fetuses, and decreased fetal size. Chronic maternal ingestion during the first trimester | | |
| | has shown a 1% incidence of cleft palate in humans. There are no reports of dexamethasone excretion into breast milk in humans; however, it is expected due to its low molecular weight that it would partition into breast milk. | | |

<sup>&</sup>lt;sup>1</sup> Mainly reported in pediatric patients with ALL. Howard SC et al. Urolithiasis in pediatric patients with acute lymphoblastic leukemia. Leukemia 2003; 17: 541-6.

<sup>(</sup>L) Toxicity may also occur later.



#### Formulation and Stability:

#### Oral:

Available in 0.5 mg, 0.75 mg, 1 mg, 1.5 mg, 2 mg, 4 mg, and 6 mg tablets; liquid formulations are available in 0.5 mg/5 mL and 1 mg/1 mL concentrations. Inactive ingredients vary depending on manufacturer but tablet formulations may include: calcium or magnesium stearate, corn starch, lactose, and various dyes. Liquid formulations may include: 5%-30% alcohol, benzoic acid, sorbitol, sodium saccharin, glycerin, purified water, and various dyes.

Australia – only 0.5 mg and 4 mg tablets available.

#### Injection:

Dexamethasone Sodium Phosphate Solution for Injection is available as 4 mg/mL (1 mL, 5 mL, and 30 mL vials) and 10 mg/mL (1 mL and 10 mL vial sizes). Vials are available in multi-dose vials as well as unit of use vials and syringes. Inactive ingredients vary depending on manufacturer but include creatinine, sodium citrate, sodium hydroxide to adjust pH, Water for Injection, sodium sulfite, bisulfite and metabisulfite, methyl and propyl paraben, benzyl alcohol, and EDTA.

Australia – 1 mg/mL solution for injection available.

Guidelines for Administration: See Treatment and Dose Modifications section of the protocol.

Dexamethasone Sodium Phosphate for Injection may be given IV, or IM undiluted. For IV use, it may be further diluted in dextrose or saline containing solutions. Avoid using benzyl alcohol-containing dexamethasone solutions in neonates. Diluted solutions that contain no preservatives should be used within 24 hours, but maintain stability for at least 14 days in PVC bags at room temperature protected from light.

#### **Supplier:**

Commercially available from various manufacturers. See package insert for further information.

#### 6.7 ETOPOSIDE – INJECTION

(11/15/2016)

(Toposar®, Etopophos®, VP-16) NSC #141540

#### Source and Pharmacology:

A semisynthetic derivative of podophyllotoxin that forms a complex with topoisomerase II and DNA which results in single and double strand DNA breaks. Its main effect appears to be in the S and  $G_2$  Phase of the cell cycle. The initial  $t_{1/2}$  is 1.5 hours and the mean terminal half-life is 4 to 11 hours. It is primarily excreted in the urine. In children, approximately 55% of the dose is excreted in the urine as etoposide in 24 hours. The mean renal clearance of etoposide is 7 to  $10 \text{ mL/min/m}^2$  or about 35% of the total body clearance over a dose range of 80 to 600 mg/m². Etoposide, therefore, is cleared by both renal and non renal processes, i.e., metabolism and biliary excretion. The effect of renal disease on plasma etoposide clearance is not known. Biliary excretion appears to be a minor route of etoposide elimination. Only 6% or less of an intravenous dose is recovered in the bile as etoposide. Metabolism accounts for most of the non renal clearance of etoposide.

The maximum plasma concentration and area under the concentration time curve (AUC) exhibit a high degree of patient variability. Etoposide is highly bound to plasma proteins (~94%), primarily serum albumin. Pharmacodynamic studies have shown that etoposide systemic exposure is related



to toxicity. Preliminary data suggests that systemic exposure for unbound etoposide correlates better than total (bound and unbound) etoposide. There is poor diffusion into the CSF < 5%.

Etoposide phosphate is a water soluble ester of etoposide which is rapidly and completely converted to etoposide in plasma. Pharmacokinetic and pharmacodynamic data indicate that etoposide phosphate is bioequivalent to etoposide when it is administered in molar equivalent doses.

**Toxicity:** 

| children<br>100<br>nsion |
|---|
| nsion |
| nsion |
| ls, fever, |
| nea, |
| oathy, |
| toxicity, |
| , |
| failure, |
| ative |
| failure, |
| ulatory |
| orrhea, |
| ils |
| nancy |
| eukemic |
| Fetal toxicities and teratogenic effects of etoposide have been noted in animals |
| in breast |
| , f |

#### Formulation and Stability:

Etoposide for Injection is available as a 20 mg/mL solution in sterile multiple dose vials (5 mL, 25 mL, or 50 mL each). The pH of the clear, nearly colorless to yellow liquid is 3 to 4. Each mL contains 20 mg etoposide, 2 mg citric acid, 30 mg benzyl alcohol, 80 mg modified polysorbate 80/tween 80, 650 mg polyethylene glycol 300, and 30.5 percent (v/v) alcohol. Vial headspace contains nitrogen. Unopened vials of etoposide are stable until expiration date on package at controlled room temperature (20°-25°C or 68°-77°F).

Etoposide phosphate for injection is available for intravenous infusion as a sterile lyophilized powder in single-dose vials containing etoposide phosphate equivalent to 100 mg etoposide, 32.7 mg sodium citrate *USP*, and 300 mg dextran 40. Etoposide phosphate must be stored under refrigeration (2°-8°C or 36°-46°F). Unopened vials of etoposide phosphate are stable until the expiration date on the package.

Guidelines for Administration: See Treatment and Dose Modifications sections of the protocol.



#### **Etoposide**:

Dilute etoposide to a final concentration  $\leq 0.4$  mg/mL in D5W or NS. Etoposide infusions are stable at room temperature for 96 hours when diluted to concentrations of 0.2 mg/mL; stability is 24 hours at room temperature with concentrations of 0.4 mg/mL. The time to precipitation is highly unpredictable at concentrations > 0.4 mg/mL. Use in-line filter during infusion secondary to the risk of precipitate formation. However, the use of an in-line filter is not mandatory since etoposide precipitation is unlikely at concentrations of 0.1-0.4 mg/mL. **Do not administer etoposide by rapid intravenous injection.** Slow rate of administration if hypotension occurs.

Leaching of diethylhexyl phthalate (DEHP) from polyvinyl chloride (PVC) bags occurred with etoposide 0.4 mg/mL in NS. To avoid leaching, prepare the etoposide solution as close as possible, preferably within 4 hours, to the time of administration or alternatively as per institutional policy; glass or polyethylene-lined (non-PVC) containers and polyethylene-lined tubing may be used to minimize exposure to DEHP.

#### **Etoposide Phosphate:**

Reconstitute the 100 mg vial with 5 or 10 mL of Sterile Water for Injection, D5W, NS, Bacteriostatic Water for Injection with Benzyl Alcohol, or Bacteriostatic Sodium Chloride for Injection with Benzyl Alcohol for a concentration equivalent to 20 mg/mL or 10 mg/mL etoposide equivalent (22.7 mg/mL or 11.4 mg/mL etoposide phosphate), respectively. Use diluents without benzyl alcohol for neonates and infants < 2 years of age or patients with hypersensitivity to benzyl alcohol.

When reconstituted as directed, etoposide phosphate solutions can be stored in glass or plastic containers under refrigeration for 7 days. When reconstituted with a diluent containing a bacteriostat, store at controlled room temperature for up to 48 hours. Following reconstitution with SWFI, D5W, or NS store at controlled room temperature for up to 24 hours.

Following reconstitution, etoposide phosphate may be further diluted to a concentration as low as 0.1 mg/mL of etoposide with D5W or NS. The diluted solution can be stored under refrigeration or at controlled room temperature for 24 hours.

#### Supplier:

Commercially available from various manufacturers. See package insert for more detailed information.

#### CANADIAN SITES

Etoposide for Injection is available as a 20mg/mL solution.

Etopophos® (etoposide phosphate) is not commercially available in Canada. Sites may purchase and import the USA commercial supply from Bristol Laboratories via an International Distributor (Pharma Exports LLC, phone: 1-412-885-3700, fax: 1-412-885-8022, email: <a href="mailto:pharexp@aol.com">pharexp@aol.com</a>) under the authority of the protocol's No Objection Letter (NOL). Drug Accountability Log (DAL) must record Lot #'s and expiry dates of shipments received and doses dispensed. Sites may use their own DAL as long as it complies with all elements of ICH GCP and Division 5 of the Food and Drugs Act. Each site is responsible for the procurement (import +/- purchase) of Etoposide Phosphate (Etopophos). Sites may import and manage a single clinical trial supply for multiple protocols as long as each protocol has an NOL and the protocol the patient is registered on is recorded on the DAL.



#### 6.8 FILGRASTIM, TBO-FILGRATIM, FILGRATIM-SNDZ

(05/13/2019)

(Granulocyte Colony-Stimulating Factor, r-metHuG-CSF, G-CSF, Neupogen®, Granix®, Zarxio®, Grastofil®) NSC #614629

#### Source and Pharmacology:

Filgrastim is a human granulocyte colony-stimulating factor (G-CSF), produced by recombinant DNA technology. Filgrastim is a 175 amino acid protein with a molecular weight of 18,800 daltons manufactured by recombinant DNA technology utilizing E coli bacteria into which has been inserted the human granulocyte colony stimulating factor gene. It differs from the natural protein in that the N- amino acid is methionine and the protein is not glycosylated. G-CSF is a lineage specific colony-stimulating factor which regulates the production of neutrophils within the bone marrow and affects neutrophil progenitor proliferation, differentiation, and selected end-cell functional activation (including enhanced phagocytic ability, priming of the cellular metabolism associated with respiratory burst, antibody dependent killing, and the increased expression of some functions associated with cell surface antigens). Filgrastim exhibits nonlinear pharmacokinetics with clearance dependent on filgrastim concentration and neutrophil count. Filgrastim is cleared by the kidney. The elimination half-life is similar for subcutaneous and intravenous administration, approximately 3.5 hours. The time to peak concentration when administered subcutaneously is 2-8 hours

**Toxicity:** 

| | Common | Occasional | Rare |
|---|---|---|---|
| | Happens to 21-100 | Happens to 5-20 children | Happens to < 5 children out |
| | children out of every 100 | out of every 100 | of every 100 |
| Immediate: | | Local irritation at the | Allergic reactions (more |
| Within 1-2 days of | | injection site, headache | common with IV |
| receiving drug | | | administration than |
| | | | subq):skin (rash, urticaria, |
| | | | facial edema), respiratory |
| | | | (wheezing, dyspnea) and |
| | | | cardiovascular (hypotension, |
| | | | tachycardia), low grade fever |
| Prompt: | Mild to moderate | Increased: alkaline | Splenomegaly, splenic |
| Within 2-3 weeks, | medullary bone pain | phosphatase, lactate | rupture, rash or exacerbation |
| prior to the next | | dehydrogenase and uric | of pre-existing skin rashes, |
| course | | acid, thrombocytopenia | sickle cell crises in patients |
| | | | with SCD, excessive |
| | | | leukocytosis, Sweet's |
| | | | syndrome (acute febrile |
| | | | neutrophilic dermatosis) |
| Delayed: | | | Cutaneous vasculitis, ARDS |
| Anytime later | | | |
| during therapy | | | |
| Late: | | | MDS or AML (confined to |
| Anytime after | | | patients with severe chronic |
| completion of | | | neutropenia and long term |
| treatment | | | administration) |
| Unknown | Fetal toxicities and teratogenic effects of filgrastim in humans are unknown. | | |
| Frequency and | Conflicting data exist in animal studies and filgrastim is known to pass the | | |
| Timing: | placental barrier. It is unknown whether the drug is excreted in breast milk. | | |



#### Formulation and Stability:

Neupogen® supplied as a clear solution of 300 mcg/mL in 1 mL or 1.6 mL vials. Neupogen® vials are preservative free single use vials. Discard unused portions of open vials.

Neupogen®, Granix® and Zarxio® are also available as single use prefilled syringes containing 300 mcg/0.5 mL or 480 mcg/0.8 mL of filgrastim for subcutaneous administration. Store refrigerated at 2°-8°C (36°-46°F). Protect from light. Do not shake. Prior to injection, filgrastim and filgrastim-sndz may be allowed to reach room temperature for a maximum of 24 hours (infusion must be completed within 24 hours of preparation). TBO-filgrastim may be removed from 2°C 8°C (36°F 46°F) storage for a single period of up to 5 days between 23°C to 27°C (73°F to 81°F). Avoid freezing and temperatures > 30°C.

For IV use, dilute filgrastim (Neupogen®) and tbo-filgrastim (Granix®) in D5W only to concentrations > 15 mcg/mL. Filgrastim-sndz (Zarxio®) may be diluted in D5W to concentrations between 5 mcg/mL and 15 mcg/mL. At concentrations below 15 mcg/mL, human serum albumin should be added to make a final albumin concentration of 0.2% (2 mg/mL) in order to minimize the adsorption of filgrastim to plastic infusion containers and equipment for all 3 products (communication on file from Teva Pharmaceuticals USA). Filgrastim or filgrastim-sndz dilutions of 5 mcg/mL or less are not recommended. Tbp-filgratim dilutions below 2 mcg/mL are not recommended. Diluted filgrastim biosimilar products should be stored at 2°-8°C (36°-46°F) and used within 24 hours. Do not shake.

Do not dilute with saline-containing solutions at any time; precipitation will occur.

#### **Guidelines for Administration:**

See Treatment, Dose Modifications and Supportive Care sections of the protocol.

Filgrastim or biosimilar products should not be administered within 24 hours of (before AND after) chemotherapy.

**Supplier:** Commercially available from various manufacturers. See package insert for further information

#### **CANADIAN SITES:**

Grastofil® brand of filgrastim biosimilar is available in Canada. See package insert for further information.

#### 6.9 FLUDARABINE (01/10/18)

(Fludara®, fludarabine phosphate, 2-fluoro-ara-AMP) NSC# 312887

#### Source and Pharmacology:

Fludarabine phosphate is a synthetic purine nucleoside. It differs from the physiologic nucleosides, adenosine, in that the sugar moiety is arabinose instead of ribose, and by the addition of a fluorine atom to the purine base adenine. Fludarabine is also a fluorinated nucleotide analog the antiviral agent vidarabine, (ara-A). The addition of fluorine results in increased aqueous solubility and resistance to enzymatic degradation by adenosine deaminase. Fludarabine (2-fluoro-ara-A) is commercially available as the monophosphate salt (2-fluoro-ara-AMP). The monophosphorylation increases the drug's aqueous solubility while maintaining pharmacologic activity. The chemical name for fludarabine phosphate is 9H-Purin-6-amine, 2-fluoro-9-(5- $\underline{0}$ -phosphono  $\beta$ -D-arabino-furanosyl) (2-fluoro-ara-AMP) and the molecular weight is 365.2.



Fludarabine is a purine antagonist antimetabolite. *In vivo*, fludarabine phosphate is rapidly dephosphorylated to 2-fluoro-ara-A and then it is phosphorylated intracellularly by deoxycytidine kinase to the active triphosphate, 2-fluoro-ara-ATP. This metabolite appears to act by inhibiting DNA polymerase alpha, ribonucleotide reductase and DNA primase, thus inhibiting DNA synthesis. The mechanism of action of this antimetabolite is not completely characterized and may be multi-faceted.

Phase I studies in humans have demonstrated that within several minutes after intravenous infusion, fludarabine phosphate is converted to the active metabolite, 2-fluoro-ara-A and becomes undetectable. Therefore, pharmacokinetics studies have focused on 2-fluoro-ara-A. Fludarabine phosphate 25 mg/m² infused intravenously over 30 minutes to adult cancer patients, showed a moderate accumulation of 2-fluoro-ara-A. During a 5-day treatment schedule, 2-fluoro-ara-A plasma trough levels increased by a factor of about 2.

Fludarabine is widely distributed. The volume of distribution at steady state ( $V_{ss}$ ) reported after daily administration of  $25 \text{mg/m}^2$  for 5 days to adults averaged at  $96\text{-}98 \text{ L/m}^2$ . Tissue distribution studies in animals indicate that the highest concentrations of the drug are in liver, kidney, and spleen. Although the extent to which fludarabine and/or its metabolites distribute into the CNS in humans has not been determined to date, severe neurologic toxicity (e.g., blindness, coma) has been reported in patients receiving the drug, particularly in high dosages. There is evidence from animal studies that fludarabine distributes into the CNS and that a toxic metabolite (2-fluoroadenine, possibly formed by bacteria in the GI tract), can be absorbed systematically via enterohepatic circulation and distributed into CSF. According to *in vitro* data, about 19-29% of fludarabine is bound to plasma proteins.

Following IV administration, fludarabine phosphate is dephosphorylated rapidly to fludarabine. Plasma concentrations of fludarabine decline in a linear, dose-independent manner. The elimination profile of fludarabine also has been reported to be either biphasic or triphasic; however, reported terminal elimination half-lives have been similar. In adult cancer patients receiving fludarabine 25 mg/m<sup>2</sup> as a 30-minute IV infusion daily for 5 days, a terminal half-life of about 20 hours was reported. In a limited number of pediatric patients, the plasma concentration profile of fludarabine exhibited both monoexponential and biexponential decay, with a mean  $t_{1/2}$  of 10.5 hours in patients with monoexponential elimination and a  $t_{1/2}$  of 1.2-1.4 and 12.4-19 hours, respectively, in patients with biexponential elimination.

Renal clearance accounts for about 40% of the total body clearance of fludarabine. Renal elimination appears to become more important at high dosages of the drug. The dose of fludarabine needs to be adjusted in patients with moderate renal impairment.

The use of fludarabine in combination with pentostatin is not recommended due to the risk of severe pulmonary toxicity.

**Toxicity:** 

| | _ | | _ |
|---|---|---|---|
| | Common | Occasional | Rare |
| | Happens to 21- | Happens to 5-20 subjects | Happens to < 5 subjects out of every |
| | 100 subjects out | out of every 100 | 100 |
| | of every 100 | | |
| Immediate: | Fever, fatigue, | Edema including | Anaphylaxis, tumor lysis syndrome, |
| | weakness, pain, | peripheral edema, chills, | dehydration* |
| | nausea, vomiting, | rash, diarrhea, rhinitis, | • |
144



| | Common | Occasional | Rare |
|---|---|---|---|
| | Happens to 21- | Happens to 5-20 subjects | Happens to < 5 subjects out of every |
| | 100 subjects out | out of every 100 | 100 |
| | of every 100 | 0.00 01 0 1 01 1 0 0 | 100 |
| Within 1-2 | anorexia, cough, | diaphoresis, malaise, | |
| days of | dyspnea | abdominal pain, | |
| receiving drug | , | headache, back pain, | |
| recorring arang | | myalgia, stomatitis, flu- | |
| | | like syndrome | |
| Prompt: | Myelosuppressio | Weight loss, | Sinusitis, dysuria, opportunistic |
| Within 2-3 | n (anemia, | gastrointestinal bleeding, | infections and reactivation of latent |
| weeks, prior to | neutropenia, | hemoptysis, paresthesia, | viral infections like Epstein-Barr virus |
| next course | thrombocytopeni | allergic pneumonitis, | (EBV), herpes zoster and John |
| | a), infection | bronchitis, pharyngitis, | Cunningham (JC) virus (progressive |
| | (urinary tract | visual disturbance, | multifocal leukoencephalopathy |
| | infection, herpes | hearing loss, | [PML]) <sup>L</sup> , EBV associated |
| | simplex infection, | hyperglycemia | lymphoproliferative disorder, |
| | pneumonia, upper | 71 07 | panycytopenia (can be prolonged), |
| | respiratory) | | pulmonary hypersensitivity <sup>a</sup> (dyspnea, |
| | , | | cough, hypoxia, interstitial pulmonary |
| | | | infiltrate), pulmonary toxicity (acute |
| | | | respiratory distress syndrome |
| | | | [ARDS], pulmonary fibrosis, |
| | | | pulmonary hemorrhage, respiratory |
| | | | distress, respiratory failure), |
| | | | pericardial effusion, skin toxicity |
| | | | (erythema multiforme, Stevens- |
| | | | Johnson syndrome, toxic epidermal |
| | | | necrolysis, pemphigus), liver failure, |
| | | | renal failure, hemorrhage, transfusion- |
| | | | associated graft-versus-host disease |
| | | | has occurred following transfusion of |
| | | | nonirradiated blood products, |
| | | | phlebitis*, sleep disorder*, cerebellar |
| | | | syndrome*, depression*, mentation |
| | | | impaired*, alopecia*, pruritus*, |
| | | | seborrhea*, esophagitis*, |
| | | | constipation*, mucositis*, dysphagia*, |
| | | | hesitancy*, cholelithiasis*, abnormal |
| | | | liver function tests *, osteoporosis*, |
| | | | arthralgia*, abnormal renal function |
| | | | test*, proteinuria*, epistaxis*, |
| | | | hemorrhagic cystitis*, eosinophilia* |
| Delayed: | | | Neurotoxicity (increased with high |
| Any time later | | | doses): seizures, agitation, confusion, |
| during therapy, | | | weakness, visual disturbances, optic |
| excluding the | | | neuritis, optic neuropathy, |
| above | | | photophobia, blindness, paralysis, |
| conditions | | | coma, death, peripheral neuropathy <sup>a</sup> ); |
| | | | autoimmune phenomena: |
| | | | thrombocytopenia/thrombocytopenic |
| | | | purpura (ITP), Evans syndrome, |
| | | | hemolytic anemia, acquired |
| | | | hemophilia |



| | Common | Occasional | Rare |
|---|---|---|---|
| | Happens to 21- | Happens to 5-20 subjects | Happens to < 5 subjects out of every |
| | 100 subjects out | out of every 100 | 100 |
| | of every 100 | | |
| Late: | | | Myelodysplastic syndrome/acute |
| Any time after | | | myeloid leukemia (mainly associated |
| completion of | | | with prior or concomitant or |
| treatment | | | subsequent treatment with other |
| | | | anticancer treatments), skin cancer |
| | | | (new onset or exacerbation) |
| Unknown | <b>Pregnancy Catego</b> | ory D | |
| Frequency and Timing: | Based on its mechanism of action, fludarabine phosphate can cause fetal harm when | | |
| | administered to a pregnant woman. Fludarabine phosphate was embryolethal and teratogenic in both rats and rabbits. | | |
| | teratogenic in both | rats and rabbits. | |

#### (L) Toxicity may also occur later.

#### Formulation and Stability:

Fludarabine phosphate injection is available as sterile lyophilized powder and in solution. Each single-dose vial of powder contains 50 mg of the active ingredient fludarabine phosphate, 50 mg of mannitol, and sodium hydroxide to adjust the pH to 7.7. After reconstitution, the pH range for the final product is 7.2-8.2. The single-dose solution vial contains 25 mg/mL, 2 mL of fludarabine phosphate. It may contain mannitol and is preservative-free.

Fludarabine phosphate vials should be stored refrigerated at 2-8°C (36-46°F).

Guidelines for Administration: See Treatment and Dose Modifications sections of the protocol.

Fludarabine phosphate powder should be reconstituted with 2 mL of Sterile Water for Injection. The solid cake should fully dissolve in 15 seconds or less. The resulting concentration is 25 mg/mL. When reconstituted to a final concentration of 25 mg/mL, the drug is stable for at least 16 days at room temperature and normal light conditions. The manufacturer recommends that the solution be used within 8 hours after reconstitution.

Prior to administration, fludarabine 25 mg/mL solution or the reconstituted 25 mg/mL solution should be further diluted in 100 mL or 125 mL of D5W or NS. Concentrations of 0.25 to 1 mg/mL have been used in clinical trials. When diluted to a final concentration of 1 mg/mL, fludarabine is stable for at least 16 days at room temperature and normal light conditions. The manufacturer recommends that the diluted solution be used within 8 hours after preparation. Parenteral drug products should be inspected visually for particulate matter and discoloration prior to administration.

**Supplier:** Commercially available from various manufacturers. See package insert for further information.

<sup>\*</sup> Reported in  $\leq$  3% of subjects. Since these are not considered life threatening they are not included in the consent.

<sup>&</sup>lt;sup>a</sup> These effects were not reported in children.



#### 6.10 INTRATHECAL TRIPLES

(05/08/12)

(Methotrexate/Hydrocortisone/Cytarabine, IT-3)

#### Source and Pharmacology:

The intrathecal route of administration of a drug produces more consistent CSF drug concentrations at relatively smaller doses because of the volume difference between the CSF and blood compartments (140 mL vs. 3500 mL in an adult). (The CSF volume of children after the first 3 years is equivalent to that of an adult). Drug half-lives are longer as well because clearance is related to flow rather than metabolism or protein binding. Intrathecal methotrexate has a biphasic elimination curve from the CSF with a  $t_{1/2}$  of 4.5 and 14 hours respectively. Following IT injection of cytarabine the elimination of the drug from the CSF is biphasic with a  $t_{1/2}$  of 1 and 3.4 hours respectively, which is 8-fold longer than the clearance from plasma. The elimination of hydrocortisone is similarly prolonged.

Intrathecal Triple Therapy (Methotrexate/ Hydrocortisone/Cytarabine) Toxicity:

| Intrathecal Tri | hecal Triple Therapy (Methotrexate/ Hydrocortisone/Cytarabine) Toxicity: | | |
|---|---|---|---|
| | Common | Occasional | Rare |
| | Happens to 21-100 | Happens to 5-20 children | Happens to < 5 children out of |
| | children out of every 100 | out of every 100 | every 100 |
| Immediate: | Nausea, vomiting, fever, | Arachnoditis: (headache, | Rash, anaphylaxis (L), paresis, |
| Within 1-2 | headache | fever, vomiting, | bleeding into subarachnoid or |
| days of | | meningismus and | subdural space (risk > with |
| receiving drug | | pleocytosis) | platelet counts < 20,000), |
| | | | confusion, fatigue, |
| | | | disorientation, seizures |
| Prompt: | | | Myelosuppression, |
| Within 2-3 | | | somnolence, ataxia, cranial |
| weeks, prior to | | | nerve palsy, transient and |
| the next course | | | rarely permanent paraplegia |
| | | | (L), speech disorders |
| Delayed: | | Cognitive | Demyelinating |
| Any time later | | disturbances (L), learning | leukoencephalopathy1 (L), |
| during therapy, | | disabilities (L) | blindness <sup>1</sup> |
| excluding the | | | |
| above condition | | | |
| Late: | | | Progressive CNS |
| Any time after | | | deterioration <sup>1</sup> |
| the completion | | | |
| of treatment | | | |

<sup>&</sup>lt;sup>1</sup> May be enhanced by systemic therapy such as high dose methotrexate or cytarabine and/or cranial irradiation.

#### Formulation and Stability:

Methotrexate 25 mg/mL **preservative free** 2 mL vial or methotrexate 20 mg preservative free sterile powder for injection vial. Cytarabine 100 mg preservative free sterile powder for injection. Hydrocortisone sodium succinate 100 mg vial sterile powder for injection.

Guidelines for Administration: See <u>Treatment</u> and <u>Dose Modifications</u> sections of the protocol.

For intrathecal administration, dilute each agent with 5-10 mL preservative free NS, lactated ringers or Elliot's B solution or as per institutional standard of practice. The volume of CSF removed should be equal to at least half the volume delivered.

<sup>(</sup>L) Toxicity may also occur later.



| Patient Age<br>(years) | Doses<br>(MTX/Hydrocortisone/Ara-C) | Recommended volume | 10% CSF<br>volume | CSF Volume * |
|---|---|---|---|---|
| 0 - 0.99 | 7.5 mg / 7.5 mg / 15 mg | 5-10 mL | 5 mL | 50 <u>+</u> 10 mL |
| | | | | (babies) |
| 1 - 1.99 | 8 mg / 8 mg / 16 mg | 5-10 mL | 5 mL | 50 <u>+</u> 10 mL |
| | | | | (babies) |
| 2 - 2.99 | 10 mg / 10 mg / 20 mg | 5-10 mL | 8 mL | 80 <u>+</u> 20 mL |
| | | | | (younger children) |
| 3 - 8.99 | 12 mg / 12 mg / 24 mg | 5-10 mL | 10 mL | 100 <u>+</u> 20 mL |
| | | | | (older children) |
| 9 or greater | 15 mg / 15 mg / 30 mg | 5-10 mL | 13 mL | 130 <u>+</u> 30 mL |
| | | | | (adults) |

<sup>\*</sup>Rieselbach, R.E. et.al. Subarachnoid distribution of drugs after lumbar injection. N Engl J Med 1962 Dec 20; 267:1273-8

Of note: Larger volumes approximating at least 10% of the CSF volume, isovolumetric delivery, with the patient remaining prone after the procedure may facilitate drug distribution. These procedures have not been validated in clinical trials. They are allowed but not mandated for patients on COG studies.

Intrathecal triples are stable in NS for 24 hours at 25°C but contain no preservative and should be administered as soon as possible after preparation.

**Supplier:** Commercially available from various manufacturers. See package insert for further information.

#### 6.11 **LEUCOVORIN CALCIUM**

(05/07/19)

147

(LCV, Wellcovorin®, citrovorum factor, folinic acid, Calcium folinate) NSC #003590

#### Source and Pharmacology:

Leucovorin is a mixture of the diastereoisomers of the 5-formyl derivative of tetrahydrofolic acid (THF). The biologically active compound of the mixture is the (-)- l-isomer, known as Citrovorum factor or (-)-folinic acid. Leucovorin does not require reduction by the enzyme dihydrofolate reductase in order to participate in reactions utilizing folates as a source of "one-carbon" moieties. Administration of leucovorin can counteract the therapeutic and toxic effects of folic acid antagonists such as methotrexate, which act by inhibiting dihydrofolate reductase. In contrast, leucovorin can enhance the therapeutic and toxic effects of fluoropyrimidines used in cancer therapy, such as 5-fluorouracil. Leucovorin is readily converted to another reduced folate, 5,10methylenetetrahydrofolate, which acts to stabilize the binding of fluorodeoxyuridylic acid (an active metabolite of 5-FU) to thymidylate synthase and thereby enhances the inhibition of this enzyme. Peak serum levels of 5-methyl THF (an active metabolite) were reached at approximately 1.3-1.5 hours (IV/IM) and 2.3 hours for the oral form. The terminal half-life of total reduced folates was approximately 6.2 hours. Following oral administration, leucovorin is rapidly absorbed and expands the serum pool of reduced folates. At a dose of 25 mg, almost 100% of the *l*-isomer (the biologically active form) but only 20% of the d-isomer is absorbed. Oral absorption of leucovorin is saturable at doses above 25 mg. The apparent bioavailability of leucovorin was 97% for 25 mg, 75% for 50 mg, and 37% for 100 mg doses. Both oral and parenteral leucovorin raise the CSF folate levels.



| | • | • 4 | |
|-------|-----|-----|------|
| Tox | 714 | "It | £7 • |
| 1 0 4 | 110 | ıι | y . |

| · | Common | Occasional | Rare |
|---|---|---|---|
| | Happens to 21-100 | Happens to 5-20 children | Happens to < 5 children out |
| | children out of every 100 | out of every 100 | of every 100 |
| Immediate: | | | Anaphylaxis, urticaria, |
| Within 1-2 days of | | | seizure |
| receiving drug | | | |
| Unknown | Fetal toxicities and terato | genic effects of leucovori | n in humans are unknown. |
| Frequency and | It is unknown whether the drug is excreted in breast milk. | | |
| timing: | | - | |

#### Formulation and Stability:

Leucovorin calcium for injection is supplied as a sterile ready to use liquid and a sterile powder for injection. The 10 mg/mL preservative free liquid is available in 50 mL vials containing sodium chloride 400 mg/vial. Store preservative free liquid in the refrigerator at 2°-8°C (36°-46°F) protected from light. The powder for injection is available in 50 mg, 100 mg, 200 mg, and 350 mg vials. Store at room temperature 15°-25°C (59°-77°F) protected from light. Reconstitute the sterile powder with sterile water for injection or bacteriostatic water for injection to a concentration of 10 mg/mL leucovorin calcium. **Do not use diluents containing benzyl alcohol for doses** > 10 mg/m² or in infants < 2 years of age or patients with allergy to benzyl alcohol. When Bacteriostatic Water is used, the reconstituted solution is good for 7 days. If reconstituted with SWFI, use solution immediately as it contains no preservative. One milligram of leucovorin calcium contains 0.004 mEq of leucovorin and 0.004 mEq of calcium.

The oral form of leucovorin is available as 5 mg, 10 mg, 15 mg, and 25 mg tablets. Inactive ingredients vary depending on manufacturer but tablet formulations may include: corn starch, dibasic calcium phosphate, magnesium stearate, pregelatinized starch, lactose, microcrystalline cellulose, and sodium starch glycolate.

Guidelines for Administration: See <u>Treatment</u> and <u>Dose Modifications</u> sections of the protocol.

#### Injection:

Because of the calcium content of the leucovorin solution, no more than 160 mg of leucovorin should be injected intravenously per minute (16 mL of a 10 mg/mL solution per minute). IV leucovorin and sodium bicarbonate are incompatible.

#### Oral:

Oral leucovorin should be spaced evenly (e.g., every six hours) throughout the day and may be taken without regard to meals. Doses > 25 mg should be given IV due to the saturation of absorption.

Leucovorin should not be administered < 24 hours after intrathecal injections which contain methotrexate unless there are special circumstances.

**Supplier:** Commercially available from various manufacturers. See package insert for further information.



#### 6.12 **MERCAPTOPURINE**

(11/27/17)

(6-MP, Purinethol®, Purixan<sup>TM</sup>, 6-mercaptopurine) NSC #000755

#### Source and Pharmacology:

Mercaptopurine is an analogue of the purine bases adenine and hypoxanthine. The main intracellular pathway for MP activation is catalyzed by the enzyme hypoxanthine-guanine phosphoribosyl transferase (HGPRT) which catalyzes the conversion of MP to several active nucleotide metabolites including thioinosinic acid, a ribonucleotide which can interfere with various metabolic reactions necessary for nucleic acid (RNA and DNA) biosynthesis. It can also cause pseudofeedback inhibition of the first step in de novo purine biosynthesis or convert to another ribonucleotide which can cause feedback inhibition. Mercaptopurine can be incorporated into DNA in the form of TG nucleotides as well and thus produce toxicity. The absorption of an oral dose of MP is incomplete and variable, with only about 16%-50% of an administered dose reaching the systemic circulation secondary to a first pass metabolism in the liver. Food intake and coadministration with cotrimoxazole (TMP/SMX) significantly reduces absorption of MP. After IV administration, MP has a plasma half-life of 21 minutes in children and 47 minutes in adults. Approximately 19% is bound to protein. Mercaptopurine is well distributed into most body compartments except the CSF. (With high dose IV MP the CSF to plasma ratio is 0.15.) MP is metabolized by xanthine oxidase in the liver to 6-Thiouric acid an inactive metabolite. In patients receiving both MP and allopurinol (a xanthine oxidase inhibitor) the dose of MP must be reduced by 50-75%. Since TPMT, 6-thiopurine methyltransferase, is also one of the enzymes involved in the metabolism of MP, those individuals who have an inherited deficiency of the enzyme may be unusually sensitive to the myelosuppressive effects of MP and prone to develop rapid bone marrow suppression following the initiation of treatment. Mercaptopurine is excreted in urine as metabolites and some unchanged drug; about half an oral dose has been recovered in 24 hours. A small proportion is excreted over several weeks.

#### **Toxicity:**

| Incidence | Toxicities |
|---|---|
| Common (>20% of patients) | Neutrophil count decreased, white blood cell decreased, anorexia, fatigue |
| Occasional<br>(4 - 20% of<br>patients) | Diarrhea, nausea, vomiting, malaise, oligospermia, infection, fever, platelet count decreased, anemia, mucositis, stomach pain, ulcerative bowel lesion, skin rash, alanine aminotransferase increased, aspartate aminotransferase increased |
| Rare<br>(≤3% of<br>patients) | Urticaria, skin hyperpigmentation, alopecia, hyperuricemia, hepatic failure, hepatic necrosis, blood bilirubin increased, pulmonary fibrosis, secondary malignant neoplasm, renal toxicity, uricosuria, pancreatitis |
| Pregnancy and<br>Lactation | Pregnancy Category D Mercaptopurine can cause fetal harm, including an increased incidence of abortion and stillbirth. Advise women to avoid becoming pregnant while receiving mercaptopurine. Mercaptopurine was embryo-lethal and teratogenic in several animal species (rat, mouse, rabbit, and hamster). It is not known whether mercaptopurine is excreted in human milk; breastfeeding should be avoided. |

#### Formulation and Stability:

Mercaptopurine is available as a 50 mg tablet containing mercaptopurine and the inactive ingredients corn and potato starch, lactose, magnesium stearate, and stearic acid. Store at 15°-25°C (59°-77°F) in a dry place. In the United States, mercaptopurine is also available as an oral



suspension in a concentration of 20 mg/mL (2000 mg/100 mL per bottle). The oral suspension is a pink to brown viscous liquid supplied in amber glass multiple-dose bottles with a child resistant closure. It should be stored at 15°-25°C (59°-77°F) in a dry place.

**NOTE**: the concentration of the commercially available suspension (20 mg/mL) and the compounded suspension (50 mg/mL) are NOT the same; doses should be prescribed in the milligrams required, not mL.

**Guidelines for Administration:** See <u>Treatment</u> and <u>Dose Modifications</u> sections of the protocol. Mercaptopurine should be taken consistently at the same time every day.

If allopurinol is also given, the oral dose of mercaptopurine should be reduced by 67-75%. Patients with severe myelosuppression should have their thiopurine S-methyltransferase (TPMT) status and/or their thiopurine metabolite concentrations evaluated, so that the dose of mercaptopurine can be reduced in patients with a TPMT defect. Patients with the rare homozygous deficient TPMT phenotype may tolerate only 1/10th to 1/20th the average mercaptopurine dose. TPMT testing and thiopurine metabolite measurements are commercially available.

### Suspension:

For children unable to swallow the tablets whole, a 50 mg/mL oral suspension can be compounded. The suspension is prepared by crushing 50 mercaptopurine 50 mg tablets in a mortar and adding 8.5 mL sterile water for irrigation. The mixture is triturated to form a smooth paste. Next, 16.5 mL simple syrup (pH=7) are added with continuous mixing and finally cherry syrup (pH=7.1) is added to a total volume of 50 mL. The suspension is stable in amber glass bottles at room temperature (19°C -23°C) for up to 5 weeks. The suspension should be shaken well before each use. Procedures for proper handling and disposal of cytotoxic drugs should be used when preparing the suspension. (Aliabadi HM, Romanick M, Desai S et al. Effect of buffer and antioxidant on stability of mercaptopurine suspension. *Am J Heath-Syst Pharm.* 65:441-7, 2008.)

Supplier: Commercially available from various manufacturers. See package insert for further information. PLEASE NOTE there is a difference in the concentration of the commercially available (20 mg/mL) and extemporaneously compounded (50 mg/mL) oral suspensions.

#### 6.13 **METHOTREXATE-ALL ROUTES**

(05/07/19)

(MTX, amethopterin, Trexall®, Xatmep®) NSC #000740

#### Source and Pharmacology:

A folate analogue which reversibly inhibits dihydrofolate reductase, the enzyme that reduces folic acid to tetrahydrofolic acid. Inhibition of tetrahydrofolate formation limits the availability of one carbon fragments necessary for the synthesis of purines and the conversion of deoxyuridylate to thymidylate in the synthesis of DNA and cell reproduction. The polyglutamated metabolites of MTX also contribute to the cytotoxic effect of MTX on DNA repair and/or strand breaks. MTX cytotoxicity is highly dependent on the absolute drug concentration and the duration of drug exposure. MTX is actively transported across cell membranes. At serum methotrexate concentrations exceeding 0.1 µmol/mL, passive diffusion becomes a major means of intracellular transport of MTX. The drug is widely distributed throughout the body with the highest concentration in the kidney, liver, spleen, gallbladder and skin. Plasma concentrations following high dose IV MTX decline in a biphasic manner with an initial half-life of 1.5-3.5 hours, and a terminal half life of 8-15 hours. About 50% is bound to protein. After oral administration, approximately 60% of a 30 mg/m² dose is rapidly



absorbed from the GI tract, with peak blood levels at 1 hour. At doses  $> 30 \text{ mg/m}^2$  absorption decreases significantly. Even at low doses absorption may be very erratic, varying between 23% and 95%. The elimination of MTX from the CSF after an intrathecal dose is characterized by a biphasic curve with half-lives of 4.5 and 14 hours. After intrathecal administration of 12 mg/m², the lumbar concentration of MTX is  $\sim 100$  times higher than in plasma. (Ventricular concentration is  $\sim 10\%$  of lumbar concentration). MTX is excreted primarily by the kidneys via glomerular filtration and active secretion into the proximal tubules. Renal clearance usually equals or exceeds creatinine clearance. Small amounts are excreted in the feces. There is significant entero-hepatic circulation of MTX. The distribution of MTX into third-space fluid collections, such as pleural effusions and ascitic fluid, can substantially alter MTX pharmacokinetics. The slow release of accumulated MTX from these third spaces over time prolongs the terminal half-life of the drug, leading to potentially increased clinical toxicity.

**Toxicity:** 

| | Common | Occasional | Rare |
|---|---|---|---|
| | Happens to 21-100 | Happens to 5-20 children | Happens to < 5 children out of |
| | children out of every 100 | out of every 100 | every 100 |
| Immediate:<br>Within 1-2 days of<br>receiving drug | Transaminase elevations | Nausea, vomiting, anorexia | Anaphylaxis, chills, fever, dizziness, malaise, drowsiness, blurred vision, acral erythema, urticaria, pruritus, toxic epidermal necrolysis, Stevens-Johnson Syndrome, tumor lysis syndrome, seizures <sup>1</sup> , |
| Prompt: Within 2-3 weeks, prior to the next course | | Myelosuppression,<br>stomatitis, gingivitis,<br>photosensitivity, fatigue | photosensitivity Alopecia, folliculitis, acne, renal toxicity (ATN, increased creatinine/BUN, hematuria), enteritis, GI ulceration and bleeding, acute neurotoxicity <sup>1</sup> (headache, drowsiness, aphasia, paresis, blurred vision, transient blindness, dysarthria, hemiparesis, decreased reflexes) diarrhea, conjunctivitis |
| <b>Delayed:</b> Any time later during therapy, excluding the above conditions | | Learning disability <sup>1</sup> (L) | Pneumonitis, pulmonary fibrosis (L), hepatic fibrosis (L), osteonecrosis (L), leukoencephalopathy¹ (L), pericarditis, pericardial effusions, hyperpigmentation of the nails |
| Late: Any time after the completion of therapy | | | Progressive CNS deterioration <sup>1</sup> |
| Unknown Frequency<br>and Timing: | Methotrexate crosses the placenta. Fetal toxicities and teratogenic effects of nethotrexate have been noted in humans. The toxicities include: congenital defects, hromosomal abnormalities, severe newborn myelosuppression, low birth weight, bortion, and fetal death. Methotrexate is excreted into breast milk in low oncentrations. | | |

May be enhanced by HDMTX and/or cranial irradiation.

<sup>(</sup>L) Toxicity may also occur later.



# **Intrathecal Therapy (Methotrexate Single Agent)**

#### **Toxicity:**

| | Common | Occasional | Rare |
|---|---|---|---|
| | Happens to 21-100 | Happens to 5-20 children | Happens to < 5 children |
| | children out of every 100 | out of every 100 | out of every 100 |
| Immediate:<br>Within 1-2<br>days of<br>receiving drug | Nausea, headache | Arachnoditis: (headache, fever, vomiting, meningismus, nuchal rigidity, and pleocytosis) | Anaphylaxis, vomiting, seizures(L), malaise, confusion, back pain, rash, bleeding into subarachnoid or subdural space (risk > with platelet counts < 20,000), |
| Prompt: Within 2-3 weeks, prior to the next course | | | Myelosuppression, ataxia, somnolence, cranial nerve palsy, subacute myelopathy (paraparesis/paraplegia), speech disorders, pain in the legs, bladder dysfunction |
| Delayed: Any time later during therapy, excluding the above condition | | Cognitive disturbances (L) <sup>1</sup> , learning disability (L) <sup>1</sup> | Leukoencephalopathy <sup>1</sup> (L) |
| Late: Any time after the completion of treatment | | | Progressive CNS<br>deterioration <sup>1</sup> |

<sup>&</sup>lt;sup>1</sup> May be enhanced by HDMTX and/or cranial irradiation.

#### Formulation & Stability:

Methotrexate tablets are available as 2.5 mg, 5 mg, 7.5 mg, 10 mg and 15 mg tablets. Inactive ingredients vary depending on manufacturer but tablet formulations may include: anhydrous lactose, crospovidone, hydroxypropyl methylcellulose, magnesium stearate, microcrystalline cellulose, polyethylene glycol, polysorbate 80, pregelatinized starch, sodium carbonate monohydrate, talc and titanium dioxide and various dyes. Store at controlled room temperature 15°-30°C (59°-86°F) and protect from light.

Australia/NZ – only 2.5 mg and 10 mg tablets available.

Methotrexate is also available as a clear yellow to orange oral solution (Xatmep®) that contains 2.5 mg of methotrexate per milliliter (equivalent to 2.74 mg of methotrexate sodium/mL) in a 120 mL bottle. Inactive ingredients include purified water, sodium citrate, citric acid, methylparaben sodium, propylparaben sodium, and sucralose. It may also contain sodium hydroxide or hydrochloric acid for pH adjustment. It is packaged in a high-density polyethylene (HDPE) bottle with a child-resistant cap and tamper-evident seal. Store oral solution under refrigeration (2°C to 8°C/36°F to 46°F) prior to dispensing. Avoid freezing and excessive heat. After dispensing, patients may store methotrexate oral solution at room temperature (20°C to 25°C/68°F to 77°F) for up to 60 days; excursions permitted to 15°C to 30°C (59°F to 86°F).

<sup>(</sup>L) Toxicity may also occur later.



Methotrexate for Injection is available as a lyophilized powder for injection in 1000 mg vials. The powder for injection contains approximately 7 mEq sodium in the 1000 mg vial. Methotrexate for Injection is also available as a 25 mg/mL solution in 2, 4, 8, 10, and 40 mL preservative free vials and 2 and 10 mL vials with preservative. The 2, 4, 8, 10, and 40 mL solutions contain approximately 0.43, 0.86, 1.72, 2.15, and 8.6 mEq sodium per vial, respectively. The preserved vials contain 0.9% benzyl alcohol as a preservative.

Sterile methotrexate powder or solution is stable at 20°-25°C (68°-77°F); excursions permitted to 15°-30°C (59°- 86 F°). Protect from light

**Guidelines for Administration:** See <u>Treatment</u> and <u>Dose Modifications</u> sections of protocol. Leucovorin rescue may be necessary with certain doses of methotrexate.

**Oral administration**: Food or milk delays absorption and reduces peak concentration. Methotrexate for oral use should preferentially be given on an empty stomach, 1 hour before or 2 hours after food or milk and at the same time each day. Methotrexate injection diluted in water can be used for oral administration, if an oral formulation is not readily available (Marshall PS, Gertner E. Oral administration of an easily prepared solution of injectable methotrexate diluted in water: a comparison of serum concentrations vs methotrexate tablets and clinical utility. *J Rheumatol* 23:455-8, 1996).

For IM/IV use: Powder for injection: Dilute 1000 mg vial with 19.4 mL of preservative free SWFI, D5W or NS to a 50 mg/mL concentration. The powder for injection may be further diluted in NS or dextrose containing solutions to a concentration of  $\leq 25$  mg/mL for IV use.

The 25 mg/mL solution may be given directly for IM administration or further diluted in Saline or Dextrose containing solutions for IV use. **Do not use the preserved solution for high dose methotrexate administration due to risk of benzyl alcohol toxicity.** Methotrexate dilutions are chemically stable for at least 7 days at room temperature but contain no preservative and should be used within 24 hours. Diluted solutions especially those containing bicarbonate exposed to direct sunlight for periods exceeding 4 hours should be protected from light.

High dose methotrexate requires alkalinization of the urine, adequate hydration and leucovorin rescue. Avoid sulfamethoxazole/trimethoprim, probenecid, penicillins, cephalosporins, aspirin, proton pump inhibitors, and NSAIDS as renal excretion of MTX is inhibited by these agents.

For Intrathecal use: Use preservative free 25 mg/mL solution.

For intrathecal administration, dilute with 5-10 mL preservative free NS, lactated Ringer's, or Elliot's B solution as per institutional standard of practice. The volume of CSF removed should be equal to at least half the volume delivered.

**Note:** When IT therapy and ID MTX are scheduled for the same day, deliver the IT therapy within 6 hours of the beginning of the IV MTX infusion (hour -6 to +6, with 0 being the start of the MTX bolus).

For IT administration, use the preservative free formulation. The volume to be given IT should be in the range of 5-10 mL. The volume of CSF removed should be equal to at least half the volume delivered (see <u>drug monograph</u>).



| Patient Age (years) | Methotrexate dose | Recommended volume | 10% CSF<br>volume | CSF Volume * |
|---|---|---|---|---|
| 1–1.99 | 8 mg | 5–10 mL | 5 mL | 50 <u>+</u> 10 mL<br>(babies) |
| 2–2.99 | 10 mg | 5-10 mL | 8 mL | 80 ± 20 mL<br>(younger children) |
| 3–8.99 | 12 mg | 5-10 mL | 10 mL | 100 <u>+</u> 20 mL<br>(older children) |
| 9 or greater | 15 mg | 5-10 mL | 13 mL | 130 <u>+</u> 30 mL<br>(adults) |

<sup>\*</sup> Rieselbach, R.E. et.al. Subarachnoid distribution of drugs after lumbar injection; N Engl J Med. 1962 Dec 20; 267:1273-8

Of Note: Larger volumes approximating at least 10% of the CSF volume, isovolumetric delivery, with the patient remaining prone after the procedure may facilitate drug distribution. These procedures have not been validated in clinical trials. They are allowed but not mandated for patients on COG studies.

Diluted methotrexate for intrathecal administration is stable for 24 hours at 25°C but contains no preservative and should be administered as soon as possible after preparation.

**Supplier:** Commercially available from various manufacturers. See package insert for further information.

#### 6.14 MITOXANTRONE

(11/27/17)

(Novantrone®, CL 232315, DAD, DHAD, Mitozantrone) NSC #301739

# Source and Pharmacology:

Mitoxantrone is a substituted alkylaminoanthraquinone and is a potent inhibitor of DNA and RNA synthesis *in vitro* and binds strongly to DNA. Mitoxantrone most likely acts through intercalation between base pairs of the DNA double helix causing crosslinks and strand breaks. In addition, it is a topoisomerase II inhibitor, an enzyme responsible for uncoiling and repairing damaged DNA. It has a cytocidal effect on both proliferating and non-proliferating cultured human cells, suggesting lack of cell cycle Phase specificity. The drug disappears rapidly from plasma (drug found only in the 3-minute sample) and <1% appears in the urine in 24 hours. The mean alpha half-life of mitoxantrone is 6 to 12 minutes, the mean beta half-life is 1.1 to 3.1 hours and the mean gamma (terminal or elimination) half-life is 23 to 215 hours (median approximately 75 hours). Primary excretion is biliary with 25% appearing in the feces; renal excretion accounting for only 11% of the total dose. Mitoxantrone clearance is reduced by hepatic impairment. Patients with severe hepatic dysfunction (bilirubin > 3.4 mg/dL) have an AUC more than three times greater than that of patients with normal hepatic function receiving the same dose. Mitoxantrone is approximately 95% protein bound.

| 1 | ( | X | ıc | Iţ | y | : |
|---|---|---|----|----|---|---|
|---|---|---|----|----|---|---|

| Common | Occasional | Rare |
|---------------------|--------------------|---------------------|
| Happens to 21- | Happens to 5- | Happens to |
| 100 children out of | 20 children out of | < 5 children out of |
| every 100 | every 100 | every 100 |



| Immediate: Within 1-2 days of receiving drug | Nausea, vomiting,<br>diarrhea, fever,<br>anorexia, green blue<br>discoloration of the<br>urine and/or sclera | Abdominal pain, back pain, headache, phlebitis, constipation | Anaphylaxis, angioedema, cardiac arrhythmias¹ (bradycardia), seizures, extravasation reactions rare but if occur can lead to: (erythema, swelling, pain, burning and/or blue discoloration of the |
|---|---|---|---|
| Prompt: Within 2-3 weeks, prior to the next course | Myelosuppression (L),<br>mucositis /stomatitis,<br>immunosuppression,<br>alopecia, fatigue | Transient elevation of LFTs, pruritus with desquamation of the skin due to progressive dryness | skin and rarely tissue<br>necrosis), tumor lysis<br>Rash, conjunctivitis,<br>(GI) hemorrhage,<br>interstitial pneumonitis |
| <b>Delayed:</b> Any time later during therapy | Amenorrhea, menstrual disorders, temporary reduction in sperm count | Cardiotoxicity<br>(decreased LVEF) <sup>2</sup> (L) | CHF, hepatotoxicity |
| Late: Any time after completion of treatment | | | Secondary malignancy |
| Unknown Frequency<br>and Timing: | in animals. Toxicities Mitoxantrone is excrete | togenic effects of mitoxa<br>include: low birth we<br>ed in human milk and sign<br>reported for 28 days after | eight and prematurity. gnificant concentrations |

<sup>&</sup>lt;sup>1</sup> Rarely clinically significant.

#### Formulation and Stability:

The concentrate is a sterile, non-pyrogenic, non-preserved, dark blue aqueous solution containing mitoxantrone hydrochloride equivalent to 2 mg/mL mitoxantrone free base, with sodium chloride (0.80% w/v), sodium acetate (0.005% w/v), and acetic acid (0.046% w/v) as inactive ingredients with 0.14 mEq of sodium per mL. Mitoxantrone is provided as 20 mg (10 mL), 25 mg (12.5 mL) and 30 mg (15 mL) vials. Store intact vials at 15°-25°C (59°-77°F). Undiluted mitoxantrone injection should be stored not longer than 7 days between 15°-25°C (59°-77°F) or 14 days under refrigeration. Refrigeration of the concentrate may result in a precipitate, which redissolves on warming to room temperature. DO NOT FREEZE.

Guidelines for Administration: See <u>Treatment</u> and <u>Dose Modifications</u> sections of the protocol.

Mitoxantrone must be diluted prior to injection. DO NOT GIVE IV PUSH. The dose of mitoxantrone should be diluted in at least 50 mL or to a concentration  $\leq 0.5$  mg/mL with either NS or D5W. The dilution is stable at room temperature for 48 hours with no loss of potency. Admixture with heparin may result in precipitation. Mitoxantrone is an irritant: Care should be taken to avoid extravasation; the use of a central line is suggested.

**Supplier:** Commercially available. See package insert for more detailed information.

<sup>&</sup>lt;sup>2</sup> Risk increases with chest radiation and prior anthracycline dosage

<sup>(</sup>L) Toxicity may also occur later.



**Special precautions:** Incompatible with heparin; precipitate may form.

#### 6.15 **MYCOPHENOLATE MOFETIL**

(12/06/18)

(CellCept®, MMF, RS-61443) NSC# 724229

#### Source and Pharmacology:

Mycophenolate (MMF) is the morpholinoethyl ester of mycophenolic acid (MPA), an antibiotic with immunosuppressant properties isolated from Penicillium spp. The chemical name for oral mycophenolate mofetil is 2-morpholinoethyl (E)-6-(1,3-dihydro-4-hydroxy-6-methoxy-7-methyl-3-oxo-5-isobenzofuranyl)-4-methyl-4-hexenoate. It has an empirical formula of  $C_{23}H_{31}NO_7$  and a molecular weight of 433.50. Mycophenolate mofetil is a white to off-white crystalline powder which is slightly soluble in water (43 µg/mL at pH 7.4); the solubility increases in acidic medium (4.27 mg/mL at pH 31 3.6). The intravenous product is the hydrochloride salt of mycophenolate mofetil. The chemical name for the hydrochloride salt of mycophenolate mofetil is 2-morpholinoethyl (E)-6-(1,3-dihydro-4-hydroxy-6-methoxy-7-methyl-3-oxo-5-isobenzofuranyl)-4-methyl-4-hexenoate hydrochloride. It has an empirical formula of  $C_{23}H_{31}NO_7$  HCl and a molecular weight of 469.96.

MMF has been used in a variety of solid organ and hematopoietic stem cell transplant settings for the prevention of acute rejection. MMF is a prodrug which, after oral administration, is rapidly and primarily hydrolyzed by the liver, to the biologically active metabolite mycophenolic acid. MPA is metabolized principally by glucuronyl transferase to form the pharmacologically inactive phenolic glucuronide of MPA (MPAG). In vivo, MPAG is converted to MPA via enterohepatic recirculation. Mycophenolic acid inhibits nucleic acid synthesis and produces a potent, noncompetitive, and reversible inhibition of inosine monophosphate dehydrogenase (IMPDH), blocking the de novo synthesis of guanosine nucleotides without being incorporated into DNA. Both T and B lymphocytes rely on this de novo pathway for purine synthesis. As a result, the proliferative responses of T and B lymphocytes to both mitogenic and allospecific stimulation are inhibited. Other rapidly dividing cell lines are capable of recycling purine nucleotides via the "salvage" pathway, which is not blocked by mycophenolic acid.

In vitro and in vivo studies have demonstrated the ability of mycophenolic acid to block proliferative responses of T and B lymphocytes, inhibit antibody formation and the generation of cytotoxic T-cells, and suppress antibody formation by B lymphocytes. Mycophenolic acid prevents the glycosylation of lymphocyte and monocyte glycoproteins that are involved in intercellular adhesion of these cells to endothelial cells, and may inhibit recruitment of leukocytes into sites of inflammation and graft rejection. Antirejection effects have been attributed to decreased recruitment of activated lymphocytes to the graft site.

The mean absolute bioavailability of oral mycophenolate mofetil relative to intravenous mycophenolate mofetil (based on MPA AUC) was 94% in a small sample of healthy, adult volunteers. In this group the mean (±SD) apparent volume of distribution of MPA was approximately 3.6 (±1.5) and 4.0 (±1.2) L/kg following intravenous and oral administration, respectively. At clinically relevant concentrations, MPA is 97% bound to plasma albumin. MPAG is 82% bound to plasma albumin at MPAG concentration ranges that are normally seen in stable renal transplant patients; however, at higher MPAG concentrations (e.g., patients with renal impairment), the binding of MPA may be reduced as a result of competition between MPAG and MPA for protein binding. A negligible amount of the agent (< 1% of dose) is excreted as MPA in the urine. Most of the administered dose (~87%) is excreted in the urine as MPAG. Bile acid



sequestrants (e.g., cholestyramine) reduce the AUC of MPA by interfering with the enterohepatic circulation of the drug.

Mycophenolate mofetil can cause fetal harm when administered to a pregnant woman. Use of MMF during pregnancy is associated with an increased risk of first trimester pregnancy loss and an increased risk of congenital malformations, especially external ear and other facial abnormalities including cleft lip and palate, and anomalies of the distal limbs, heart, esophagus, and kidney. According to the package labeling, the National Transplantation Pregnancy Registry (NTPR) presents data on 33 MMF-exposed pregnancies in 24 transplant patients. Of these, there were 15 spontaneous abortions and 18 live-born infants. Four of the 18 infants had structural malformations (22%). In postmarketing data (collected 1995-2007) of 77 women exposed to systemic MMF during pregnancy, 25 had spontaneous abortions and 14 had a malformed infant or fetus. Six of 14 malformed offspring had ear abnormalities. Because these postmarketing data are reported voluntarily, it is not always possible to reliably estimate the frequency of particular adverse outcomes. These malformations seen in offspring were similar to findings in animal reproductive toxicology studies. In animal reproductive toxicology studies, there were increased rates of fetal resorptions and malformations in the absence of maternal toxicity. Female rats and rabbits received MMF doses equivalent to 0.02 to 0.9 times the recommended human dose for renal and cardiac transplant patients, based on body surface area conversions. In rat offspring, malformations included anophthalmia, agnathia, and hydrocephaly. In rabbit offspring, malformations included ectopia cordis, ectopic kidneys, diaphragmatic hernia, and umbilical hernia. If this drug is used during pregnancy, or if the patient becomes pregnant while taking this drug, the patient should be apprised of the potential hazard to the fetus.

Women of childbearing potential should have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 1 week prior to beginning therapy (manufacturer's recommendation). MMF should not be initiated until a negative pregnancy test report is obtained. Women of childbearing potential taking MMF must receive contraceptive counseling and use effective contraception. It is recommended by the manufacturer that the patient begin using two chosen methods of contraception 4 weeks prior to starting MMF, unless abstinence is the chosen method. She should continue contraceptive use during therapy and for 6 weeks after stopping MMF. Patients should be aware that MMF reduces blood levels of the hormones in the oral contraceptive pill and could theoretically reduce its effectiveness.

An approved medication guide (<a href="https://www.mycophenolaterems.com/REMSMaterials.aspx">https://www.mycophenolaterems.com/REMSMaterials.aspx</a>) must be dispensed with each refill of mycophenolate mofetil.

The table below lists the toxicity profile of mycophenolate mofetil:

| Incidence | Toxicities |
|---|---|
| Common (> 20% of patients) | Hypertension, edema (face, limbs, trunk), rash maculo-papular, cholesterol high, hyperglycemia, hyperkalemia, hypocalcemia, hypokalemia, hypomagnesemia, abdominal pain, constipation, diarrhea, nausea, vomiting, anorexia, dyspepsia, anemia, white blood cell decreased, platelet count decreased, back pain, anxiety, generalized muscle weakness, dizziness, headache, insomnia, tremor, creatinine increased, dyspnea, cough, fever, pleural effusion, alanine aminotransferase increased, alkaline phosphatase increased, aspartate aminotransferase increased, blood bilirubin increased, GGT increased, pain, paresthesia, infection <sup>1</sup> |



| Occasional (4-20% of patients) | Sepsis, urinary tract pain, urinary frequency, phlebitis (IV only), thrombosis (IV only) |
|---|---|
| Rare (<3% of patients) | Phlebitis, Neoplasms benign, malignant and unspecified (including cysts and polyps) - Other, [Malignant epithelial neoplasm of skin, non-melanoma; lymphoproliferative disease or lymphoma], gastric ulcer, gastrointestinal hemorrhage, gastric perforation, mucositis oral, thromboembolic event, infective endocarditis, renal calculi, pulmonary fibrosis, pneumonitis, neutrophil count decreased, leukoencephalopathy, colitis, pancreatitis, pure red cell aplasia |
| | Pregnancy Category D |
| Pregnancy &<br>Lactation | Mycophenolate is associated with an increased risk of congenital malformations and spontaneous abortions when used during pregnancy. Adverse events have been reported in animal studies at doses less than the equivalent recommended human dose. Data from the National Transplantation Pregnancy Registry (NTPR) have observed an increase in structural malformations (including ear malformations) in infants born to mothers taking mycophenolate during pregnancy. Spontaneous abortions have also been noted. Females of childbearing potential should have a negative pregnancy test within 1 week prior to beginning therapy. Two reliable forms of contraception should be used beginning 4 weeks prior to, during, and for 6 weeks after therapy. The effectiveness of hormonal contraceptive agents may be affected by mycophenolate. It is unknown if mycophenolate is excreted in human milk. Due to potentially serious adverse reactions, the decision to discontinue the drug or discontinue breast-feeding should be considered. Breast- |
| | feeding is not recommended during therapy or for 6 weeks after treatment is complete. |

<sup>1</sup>Infection includes all 75 sites of infection under the INFECTIONS AND INFESTATIONS SOC.

#### Formulation and Stability:

Mycophenolate mofetil is available in the following preparations:

Capsule: 250 mgTablet: 500 mg

• Powder for suspension, oral: 200 mg/mL (following reconstitution)

• Powder for reconstitution, <u>injection</u>: 500 mg per vial

A delayed release tablet (mycophenolic acid, Myfortic) is also commercially available. This preparation is not interchangeable with mycophenolate mofetil (Cellcept®, MMF) due to differences in absorption. This tablet is not discussed in this monograph and should not be used by patients treated on this protocol.

Inactive ingredients in the 250 mg capsules include the following: croscarmellose sodium, magnesium stearate, povidone (K-90) and pregelatinized starch. The capsule shells contain black iron oxide, FD&C blue #2, gelatin, red iron oxide, silicon dioxide, sodium lauryl sulfate, titanium dioxide, and yellow iron oxide.

Inactive ingredients in the 500 mg tablets include black iron oxide, croscarmellose sodium, FD&C blue #2 aluminum lake, hydroxypropyl cellulose, hydroxypropyl methylcellulose, magnesium



stearate, microcrystalline cellulose, polyethylene glycol 400, povidone (K-90), red iron oxide, talc, and titanium dioxide; may also contain ammonium hydroxide, ethyl alcohol, methyl alcohol, n-butyl alcohol, propylene glycol, and shellac.

Inactive ingredients in the powder for oral suspension include aspartame, citric acid anhydrous, colloidal silicon dioxide, methylparaben, mixed fruit flavor, sodium citrate dihydrate, sorbitol, soybean lecithin, and xanthan gum.

The injectable product is available as a sterile, white to off-white, lyophilized powder in vials containing mycophenolate mofetil hydrochloride for administration by intravenous infusion only. Each vial contains the equivalent of 500 mg mycophenolate mofetil as the hydrochloride salt. Inactive ingredients include polysorbate 80 (25 mg), citric acid (5 mg), and sodium hydroxide to adjust the pH. Reconstitution and dilution with D5W yields a final solution of mycophenolate mofetil that is slightly yellow in color.

Guidelines for Administration: See <u>Treatment</u> and <u>Dose Modifications</u> sections of the protocol.

#### Preparation:

To prepare the oral suspension, add 47 mL of water to the bottle and shake well for approximately 1 minute. Add another 47 mL of water to the bottle and shake well for an additional minute. The final concentration is 200 mg/mL of mycophenolate mofetil. Avoid inhalation or direct contact with skin or mucous membranes of the dry powder or the constituted suspension. If such contact occurs, wash thoroughly with soap and water; rinse eyes with water.

To prepare the intravenous injection, reconstitute the contents of each vial with 14 mL of D5W. Dilute the contents of a vial with D5W to a final concentration of 6 mg/mL. Each vial is vacuum-sealed; if a lack of vacuum is noted during preparation, the vial should not be used.

#### Stability:

Oral formulations should be stored at 25°C (77°F); excursions are permitted to 15°C to 30°C (59°F to 86°F). Protect from moisture and light. Once reconstituted, the oral solution may be stored at room temperature or under refrigeration. Do not freeze. The mixed suspension is stable for 60 days.

Store intact vials and diluted solutions at 25°C (77°F); excursions permitted to 15°C to 30°C (59°F to 86°F). Do not freeze. Begin infusion within 4 hours of reconstitution.

#### Administration:

Oral formulations of MMF should be administered on an empty stomach to avoid variability in MPA absorption. The oral solution may be administered via a nasogastric tube (minimum 8 French, 1.7 mm interior diameter). Do not mix the oral suspension with other medications. Some products may contain phenylalanine; refer to the package labeling for additional details.

The intravenous solution should be given over at least 2 hours. Do not administer by rapid or bolus injection.

#### **Supplier:**

Commercially available from various manufacturers. See package insert for further information.

160



# 6.16 **PEGASPARGASE**

(06/05/17)

(PEG-asparaginase, PEGLA, PEG-L-asparaginase, polyethylene glycol-L-asparaginase, Oncaspar®) NSC #624239

# Source and Pharmacology:

Pegaspargase is a modified version of the enzyme L-asparaginase. L-asparaginase is modified by covalently conjugating units of monomethoxypolyethylene glycol (PEG), molecular weight of 5000, to the enzyme, forming the active ingredient PEG-L-asparaginase. The L-asparaginase (Lasparagine amidohydrolase, type EC-2, EC 3.5.1.1) used in the manufacture of Pegaspargase is derived from Escherichia coli which is purchased in bulk from Merck, Sharp and Dohme. Lasparagine is a nonessential amino acid synthesized by the transamination of L-aspartic acid by a reaction catalyzed by the enzyme L-asparagine synthetase. The ability to synthesize asparagine is notably lacking in malignancies of lymphoid origin. Asparaginase depletes L-asparagine from leukemic cells (especially lymphoblasts) by catalyzing the conversion of L-asparagine to aspartic acid and ammonia. In predominately L-asparaginase naive adult patients with leukemia and lymphoma, initial plasma levels of L-asparaginase following intravenous administration of pegaspargase were determined. Apparent volume of distribution was equal to estimated plasma volume. L-asparaginase was measurable for at least 15 days following the initial treatment with Pegaspargase. The approximate t<sub>1/2</sub> in adult patients is 5.73 days. The enzyme could not be detected in the urine. The half-life is independent of the dose administered, disease status, renal or hepatic function, age, or gender. In a study of newly diagnosed pediatric patients with ALL who received either a single intramuscular injection of pegaspargase (2500 IU/m²), E. coli L-asparaginase (25000 IU/m<sup>2</sup>), or Erwinia (25000 IU/m<sup>2</sup>), the plasma half-lives for the three forms of L-asparaginase were:  $5.73 \pm 3.24$  days,  $1.24 \pm 0.17$  days, and  $0.65 \pm 0.13$  days respectively. The plasma half-life of pegaspargase is shortened in patients who are previously hypersensitive to native L-asparaginase as compared to non-hypersensitive patients. L-asparaginase is cleared by the reticuloendothelial system and very little is excreted in the urine or bile. Cerebrospinal fluid levels are < 1% of plasma levels.

**Toxicity:** 

| | Common | Occasional | Rare |
|---|---|---|---|
| | Happens to 21-100 children | Happens to 5-20 children | Happens to < 5 children out |
| | out of every 100 | out of every 100 | of every 100 |
| Immediate: | Allergic reactions (total | Allergic reactions | Anaphylaxis, |
| Within 1- | likelihood of local, and or | (total likelihood of | hyper/hypotension, |
| 2 days of | systemic reaction | local, and or systemic | tachycardia, periorbital |
| receiving | especially if previous | reaction if <b>no</b> previous | edema, chills, fever, |
| drug | hypersensitivity reaction to | hypersensitivity | dizziness, dyspnea, |
| | native asparaginase), pain | reaction to native | bronchospasm, lip edema, |
| | at injection site, weakness, | asparaginase), rash | arthralgia, myalgia, urticaria, |
| | fatigue, diarrhea | | mild nausea/vomiting, |
| | | | abdominal pain, flatulence, |
| | | | somnolence, lethargy, |
| | | | headache, seizures (L), |
| | | | hyperuricemia |
| Prompt: | Hyperammonemia (L), | Hyperglycemia, | Hemorrhage (L), DIC, |
| Within 2- | coagulation abnormalities | abnormal liver | thrombosis, anorexia, weight |
| 3 weeks, | with prolonged PTT, PT | function tests, | loss, CNS ischemic attacks, |
| prior to the | and bleeding times | pancreatitis (L), | edema, azotemia and |
| next course | (secondary to decreased | | decreased renal function, |



| | Common | Occasional | Rare |
|---|---|---|---|
| | Happens to 21-100 children | Happens to 5-20 children | Happens to < 5 children out |
| | out of every 100 | out of every 100 | of every 100 |
| | synthesis of fibrinogen, | increased serum | mild leukopenia, |
| | AT-III & other clotting | lipase/amylase | granulocytopenia, |
| | factors) (L) | | thrombocytopenia, |
| | | | pancytopenia, hemolytic |
| | | | anemia, infections (sepsis |
| | | | with/without septic shock, |
| | | | subacute bacterial |
| | | | endocarditis [SBE], URI), |
| | | | CNS changes including |
| | | | irritability, depression, |
| | | | confusion, EEG changes, |
| | | | hallucinations, coma and |
| | | | stupor, paresthesias, |
| | | | hypertriglyceridemia, |
| | | | hyperlipidemia, Parkinson- |
| | | | like syndrome with tremor |
| | | | and increase in muscular |
| | | | tone, hyperbilirubinemia, |
| D. 1 | | | chest pain |
| Delayed: | | | Renal failure, urinary |
| Any time | | | frequency, hemorrhagic |
| later during | | | cystitis, elevated creatinine |
| therapy | | | and BUN, fatty liver deposits, |
| Unknown | Animal nameduation studies | harra not haan aandrists dee | hepatomegaly, liver failure |
| | | Animal reproduction studies have not been conducted with pegaspargase. It is not | |
| Frequency and | | known whether pegaspargase can cause fetal harm when administered to a pregnant | |
| Timing: | woman or can affect reproduction capacity. However, fetal toxicities and teratogenic effects of asparaginase have been noted in animals. It is unknown whether the drug is | | |
| i iiiiiig. | excreted in breast milk. | | |
| | exercica in oreast innik. | | |

(L)Toxicity may also occur later.

#### Formulation and Stability:

Each milliliter of pegaspargase contains: PEG-L-asparaginase 750 IU  $\pm$  20%, monobasic sodium phosphate, USP 1.20 mg  $\pm$  5% dibasic sodium phosphate, USP 5.58 mg  $\pm$  5%, sodium chloride, USP 8.50 mg  $\pm$  5%, Water for Injection, USP qs to 1 mL. The specific activity of pegaspargase is at least 85 IU per milligram protein. Available in 5 mL vials as Sterile Solution for Injection in ready to use single-use vials, preservative free. Keep refrigerated at 2°-8°C (36°-46°F). Do not use if stored at room temperature for more than 48 hours. **DO NOT FREEZE.** Do not use product if it is known to have been frozen. Freezing destroys activity, which cannot be detected visually.

Guidelines for Administration: See Treatment and Dose Modifications sections of the protocol.

For IM administration: the volume at a single injection site should be limited to 2 mL. If the volume to be administered is greater than 2 mL, multiple injection sites should be used.

For IV administration: dilute pegaspargase in 100 mL of NS or D5W and infuse over 1 to 2 hours through a NS or D5W running infusion line. Pegaspargase admixed in 100 mL of NS or D5W is stable for 48 hours at room temperature. Pegaspargase diluted in 100 mL of NS is stable for up to 72 hours refrigerated (4°C [39°F]) (refrigerated stability data on file with Sigma-Tau). Avoid excessive agitation. DO NOT SHAKE. Do not use if cloudy of if precipitate is present.



Have available during and after the infusion: antihistamine, epinephrine, oxygen, and IV corticosteroids. Observe patient for ONE hour after administration for signs of hypersensitivity reactions.

Supplier: Comercially available. See package insert for further information.

# 6.17 TACROLIMUS (11/27/17)

(FK-506, Prograf®) NSC #717865

#### Source and Pharmacology:

Tacrolimus is a macrolide immunosuppressant produced by Streptomyces tsukubaensis. Tacrolimus is a potent immunosuppressive agent which prolongs the survival of the host and transplanted grafts in animal transplant models of liver, kidney, heart, bone marrow, small bowel and pancreas, lung and trachea, skin, cornea, and limb. Tacrolimus inhibits T-lymphocyte activation, although the exact mechanism of action is not known. Experimental evidence suggests that tacrolimus binds to an intracellular protein, FKBP-12. A complex of tacrolimus-FKBP-12, calcium, calmodulin, and calcineurin is then formed and the phosphatase activity of calcineurin inhibited. This effect may prevent the dephosphorylation and translocation of nuclear factor of activated T-cells (NF-AT), a nuclear component thought to initiate gene transcription for the formation of lymphokines (such as interleukin-2, gamma interferon). The net result is the inhibition of T-lymphocyte activation (immunosuppression). Additionally, tacrolimus may inhibit cellular activities such as nitric oxide synthetase activation and apoptosis, and may potentiate the action of corticosteroids in these processes. Tacrolimus activity is primarily due to the parent drug. The plasma protein binding of tacrolimus is approximately 99% and is independent of concentration over a range of 5-50 ng/mL. Tacrolimus is bound mainly to albumin and alpha-1-acid glycoprotein, and has a high level of association with erythrocytes. The t<sub>1/2</sub> in adult patients ranges from 11-19 hours. The pharmacokinetics of tacrolimus have been studied in pediatric liver transplant patients (0.7 to 13.2 years of age). Following the IV administration of a 0.037 mg/kg/day dose to 12 pediatric patients, mean terminal half-life, volume of distribution and clearance were  $11.5 \pm 3.8$  hours,  $2.6 \pm 2.1$  L/kg and  $0.138 \pm 0.071$  L/hr/kg, respectively. Following oral administration to 9 pediatric patients, the absolute bioavailability was  $31 \pm 21\%$ . Whole blood trough concentrations from 31 patients less than 12 years old showed that pediatric patients needed higher doses than adults to achieve similar tacrolimus trough concentrations. Tacrolimus is extensively metabolized by the mixed-function oxidase system, primarily the cytochrome P-450 system (CYP3A) in the liver and to a lesser extent in the intestinal mucosa. The major metabolite identified in incubations with human liver microsomes is 13-demethyl tacrolimus. The main route of elimination is via the biliary tract and excretion in feces. The mean clearance in renal dysfunction and mild hepatic dysfunction is the same as normal volunteers. Severe hepatic dysfunction (Pugh score > 10) led to a substantially decreased clearance. A retrospective comparison of Black and Caucasian kidney transplant patients indicated that Black patients required higher tacrolimus doses to attain similar trough concentrations; there were no gender-based differences. The absorption of tacrolimus from the gastrointestinal tract is incomplete and variable exhibiting large intra- and inter-patient variability. Administration with food significantly decreases the rate and extent of absorption Drugs that stimulate or inhibit hepatic p-450 enzymes will alter clearance of tacrolimus and close attention to potential drug interactions is crucial.



# **Toxicity:**

| | Common | Occasional | Rare |
|---|---|---|---|
| | Happens to 21- | Happens to 5- | Happens to < 5 children out |
| | 100 children out of | 20 children out of | of every 100 |
| | every 100 | every 100 | · |
| Immediate: | Headache (L), | Chest pain | Anaphylaxis with the |
| Within 1-2 days | hypertension (L), nausea, | | injection, allergic reaction, |
| of receiving drug | vomiting, anorexia, | | hypotension, asthma, |
| | immunosuppression (L), | | dyspnea, increased cough, |
| | diarrhea, constipation, | | flu like syndrome, pleural |
| | fever | | effusion, seizure (L), |
| | | | tachycardia, angina |
| Prompt: | Tremor (L), ), renal | Alopecia, dizziness, | Dyspepsia, dysphagia, |
| Within 2- | dysfunction (acute with | elevated LFTs, UTI, | gastritis, esophagitis, |
| 3 weeks, prior to | decrease in GFR, | peripheral edema, | flatulence, CNS |
| the next course | impaired urinary | rash, pruritus, | abnormalities (confusion |
| | concentrating ability, and | hyperlipidemia, | (L), somnolence (L), |
| | sodium retention), | hypercholesteremia | depression (L), anxiety, |
| | elevated creatinine/BUN, | | anxiousness, abnormal |
| | anemia, insomnia, | | dreams, emotional labiality, |
| | asthenia, pain | | hallucinations, psychosis, |
| | (abdominal, back, pain), | | hypertonia, incoordination, |
| | hyperglycemia, | | neuropathy, nervousness |
| | hypomagnesemia (L), | | encephalopathy), |
| | hyper/hypokalemia (L), | | coagulation disorder, |
| | hypophosphatemia, | | leukopenia (L), |
| | paresthesia | | thrombocytopenia, |
| | | | polycythemia, anemia, |
| | | | leukocytosis, infections |
| | | | (bacterial, fungal, viral – |
| | | | sepsis, cellulites, fungal |
| | | | dermatitis, herpes simplex, |
| | | | sinusitis, pharyngitis, |
| | | | abscess, pneumonia, |
| | | | bronchitis, peritonitis), |
| | | | hyperbilirubinemia (L), |
| | | | thrombosis, phlebitis, |
| | | | arthralgia, myalgia, |
| | | | electrolyte abnormalities |
| Delayed: | | | Acne, exfoliative dermatitis, |
| Any time later | | | skin discoloration, |
| during therapy, | | | photosensitivity reaction, |
| excluding the | | | skin ulcer, delayed wound |
| above conditions | | | healing, hirsutism |
| | | | (hypertrichosis) (L), gingival |
| | | | hyperplasia, abnormal |
| | | | vision, amblyopia, ear pain, |
| | | | otitis, tinnitus, GI |
| | | | hemorrhage, GI perforation, |
| | | | cholelithiasis, cholestatic |
| | | | jaundice, chronic renal |
| | | | dysfunction, renal failure, |
| | | | post-transplant diabetes |
| | | | mellitus (L), myocardial |
| | | | hypertrophy, elevated liver |



| | Common | Occasional | Rare |
|---|---|---|---|
| | Happens to 21- | Happens to 5- | Happens to < 5 children out |
| | 100 children out of | 20 children out of | of every 100 |
| | every 100 | every 100 | |
| | | | function tests, liver damage, |
| | | | ascites |
| Late: | | | Lymphoproliferative |
| Any time after | | | disorders, skin malignancies |
| completion of | | | |
| treatment | | | |
| Unknown | Fetal toxic effects of tac | rolimus have been not | ed in animals. Tacrolimus is |
| Frequency and | transported across the placenta and its use during pregnancy has been associated | | |
| Timing: | with neonatal hyperkalemia and renal dysfunction. Tacrolimus is excreted in | | |
| - | human milk, nursing should be avoided. | | |

(L) Toxicity may also occur later.

#### Formulation and Stability:

# Injection:

Tacrolimus is available as a sterile solution (tacrolimus injection) containing the equivalent of 5 mg anhydrous tacrolimus per 1 mL. Each mL also contains polyoxyl 60 hydrogenated castor oil (HCO-60), 200 mg, and dehydrated alcohol, *USP*, 80% v/v. Store between 5°C and 25°C (41°F and 77°F).

#### Oral:

Tacrolimus is available for oral administration as capsules containing the equivalent of 0.5 mg, 1 mg or 5 mg of anhydrous tacrolimus. Inactive ingredients include lactose, hydroxypropyl methylcellulose, croscarmellose sodium, and magnesium stearate. The 0.5 mg capsule shell contains gelatin, titanium dioxide and ferric oxide, the 1 mg capsule shell contains gelatin and titanium dioxide, and the 5 mg capsule shell contains gelatin, titanium dioxide and ferric oxide. Store at 25°C (77°F); excursions permitted to 15°-30°C (59°-86°F).

Guidelines for Administration: See <u>Treatment</u> and <u>Dose Modifications</u> sections of the protocol.

#### Injection:

Tacrolimus Injection must be diluted with NS or D5W before use to a concentration between 0.004 mg/mL and 0.02 mg/mL. Diluted infusion solution should be stored in glass or polyethylene containers and should be discarded after 24 hours. The polyoxyethylated castor oil contained in the concentrate for intravenous infusion can cause phthalate stripping from PVC. It is strongly recommended that non-PVC tubing be used to minimize patient exposure to DEHP. Due to the chemical instability of tacrolimus in alkaline media, tacrolimus injection should not be mixed or co-infused with solutions of pH 9 or greater (e.g., ganciclovir or acyclovir).

Tacrolimus 0.001 mg/mL solution stored in polyolefin bags at room temperature (20–25°C) was stable for 24 hours when prepared in NS and for at least 48 hours when prepared in D5W. Solutions of 0.01 and 0.1 mg/mL prepared in either NS or D5W were stable for at least 48 hours at room temperature in polyolefin bags (Lee JH, et al. Am J Health-Syst Pharm. 2016;73:137-42).

Monitor closely for an acute allergic reaction for the first 30 minutes and at frequent intervals thereafter.

#### Oral:

Administer at a consistent time of day and at consistent intervals with regard to meals. Tacrolimus may be given with food as long as it is given the same way each time; however; administration with



food significantly decreases the rate and extent of absorption. Grapefruit or grapefruit juice should be avoided during the entire course of tacrolimus administration.

**Supplier:** Commercially available from various manufacturers. See package insert for further information.

## 6.18 THIOGUANINE (12/05/2016)

(6-thioguanine, thioguanine, 2-amino-1,7-dihydro-6H-purine-6-thione, WR-1141, Tabloid®, Lanvis®) NSC #752

# **Source and Pharmacology:**

Thioguanine is a purine analogue of the nucleic acid guanine with the substitution of a thiol group in place of the hydroxyl group on guanine. The main intracellular pathway for 6-TG activation is catalyzed by the enzyme hypoxanthine-guanine phosphoribosyl transferase (HGPRT) which catalyzes the conversion of 6-TG to the active nucleotide, 6-thioguanylic acid. The monophosphate nucleotide form of 6-TG inhibits *de novo* purine synthesis and purine interconversion reactions, whereas the nucleotide triphosphate metabolite is incorporated directly into nucleic acids. Incorporation of fraudulent nucleotides into DNA interferes with DNA replication and results in the formation of DNA strand breaks. The net consequence of its action is a sequential blockade of the synthesis and utilization of the purine nucleotides. The relative contribution of each of these actions to the mechanism of cytotoxicity of 6-TG is unclear. The absorption of an oral dose of 6-TG is incomplete and variable, averaging approximately 30% of the administered dose (range: 14% to 46%).

6-TG undergoes deamination by the enzyme guanine deaminase resulting in 6-thioxanthene, which is then oxidized by xanthine oxidase to 6-thiouric acid. In contrast to mercaptopurine, 6-TG is not a direct substrate for xanthine oxidase. Because the inhibition of xanthine oxidase results in the accumulation of 6-thioxanthene, an inactive metabolite, adjustments in 6-TG dosage are not required for patients receiving allopurinol. Since TPMT, 6-thiopurine methyltransferase, is one of the enzymes involved in the deactivation of 6-TG, those individuals who have an inherited deficiency of the enzyme may be unusually sensitive to the myelosuppressive effects of 6-TG and prone to developing rapid bone marrow suppression following the initiation of treatment.

Peak levels occur 2 to 4 hours after oral administration with a median half-life is about 90 minutes (range: 25-240 minutes). Very little unchanged drug is excreted renally.

**Toxicity:** 

| | Common Happens to 21- 100 children out of every 100 | Occasional Happens to 5- 20 children out of every 100 | Rare Happens to < 5 children out of every 100 |
|---|---|---|---|
| Immediate: Within 1-2 days of receiving drug | , | Anorexia, nausea,<br>vomiting, diarrhea,<br>malaise | Urticaria, rash, hyperuricemia |
| Prompt: Within 2-3 weeks, prior to next course | Myelosuppression | | Toxic hepatitis (L), increased SGOT (AST)/SGPT (ALT), ataxia, mucositis |
| Delayed:<br>Anytime later during<br>therapy | | | Hepatic fibrosis(L), sinusoidal obstruction syndrome (SOS, formerly VOD) (L), hyperbilirubinemia |



| | Common | Occasional | Rare |
|---|---|---|---|
| | Happens to 21- | Happens to 5- | Happens to < 5 children out of |
| | 100 children out of | 20 children out of | every 100 |
| | every 100 | every 100 | - |
| <b>Unknown Frequency</b> | Fetal toxicities and teratogenic effects of thioguanine have been noted in animals. | | |
| and Timing: | It is unknown whether the drug is excreted in breast milk. | | |

(L) Toxicity may also occur later.

# Formulation and Stability:

Each greenish-yellow, scored tablet contains 40 mg thioguanine. Store at 15°-25°C (59°-77°F) in a dry place.

For patients unable to swallow tablets, a 20 mg/mL oral suspension may be compounded. Crush fifteen (n=15) 40 mg tablets in a mortar and reduce to a fine powder. Add 10 mL methylcellulose 1% in incremental proportions and mix to a uniform paste. Transfer to a graduated cylinder, rinse mortar with simple syrup, and add quantity of simple syrup sufficient to make 30 mL. Dispense in an amber glass bottle and label "shake well" and "refrigerate". If methylcellulose is not available, substitute 15 mL of Ora-Plus in place of the methylcellulose and qs with Ora-Sweet (in place of simple syrup) to a final volume of 30 mL. Both preparations are stable for 63 days at 19° C – 23° C. (Aliabadi HM, Romanick M, Somayah V, et al. Stability of compounded thioguanine oral suspensions. *Am J Health Syst Pharm* 2011;68:1278.)

**Guidelines for Administration:** See <u>Treatment</u> and <u>Dose Modifications</u> sections of the protocol. Thioguanine should be taken consistently at the same time every day.

Substantial dosage reductions may be required in patients with an inherited deficiency of the enzyme thiopurine methyltransferase (TPMT) due to accumulation of active thioguanine metabolites resulting in a higher incidence of myelosuppression.

**Supplier:** Commercially available. See package insert for more detailed information.

#### 6.19 THIOTEPA (01/23/18)

(Tepadina, Tespa, Thiophosphamide, Triethylenethiophosphoramide Tspa, WR-45312) NSC #6396

# Source and Pharmacology:

Thiotepa is a cytotoxic agent of the polyfunctional type, related chemically and pharmacologically to nitrogen mustard. The radiomimetic action of thiotepa is believed to occur through the release of ethylenimine radicals which, like irradiation, disrupt the bonds of DNA. One of the principal bond disruptions is initiated by alkylation of guanine at the N-7 position, which severs the linkage between the purine base and the sugar and liberates alkylated guanines. Thiotepa is desulfurated by cytochrome P-450 enzymes such as 2B1 and 2C11 which catalyze the conversion of thiotepa to tepa. Tepa is less toxic than thiotepa and has been demonstrated to produce alkali-labile sites in DNA, rather than cross-links. These findings indicate that tepa reacts differently from thiotepa and produces monofunctional alkylation of DNA. A second metabolite of thiotepa, a mercapturic acid conjugate, is formed via glutathione conjugation. Monochloro tepa is the third metabolite found in the urine.

Following short intravenous infusion (less than 5 minutes), peak concentrations of thiotepa were measured within 5 minutes. At steady state, the volume of distribution was independent of dose and ranged from 0.3 to 1.6 liters per kilogram (L/kg).



Approximately 4.2% of the original dose is eliminated in the urine within 24 hours as tepa. The elimination half-life of thiotepa ranges from 2.3 to 2.4 hours. The half-life of tepa ranged from 3 to 21.1 hours in one study.

**Toxicity:** 

| | Common | Occasional | Rare |
|---|---|---|---|
| | Happens to 21-100 children<br>out of every 100 | Happens to 5-20 children out of every 100 | Happens to < 5 children<br>out of every 100 |
| Immediate:<br>Within 1-2 days<br>of receiving<br>drug | Nausea, vomiting, anorexia, fatigue, weakness | Pain at the injection site,<br>dizziness, headache,<br>blurred vision, abdominal<br>pain, contact dermatitis,<br>rash | Anaphylaxis, laryngeal edema, wheezing, hives |
| Prompt:<br>Within 2-<br>3 weeks, prior to<br>next course | Myelosuppression; at<br>higher doses in<br>conditioning regimens for<br>BMT: mucositis,<br>esophagitis | At higher doses in conditioning regimens for BMT: encephalopathy (inappropriate behavior, confusion, somnolence), increased liver transaminases, increased bilirubin, hyperpigmentation of the skin (bronzing effect) | Febrile reaction,<br>conjunctivitis, dysuria,<br>urinary retention |
| Delayed:<br>Anytime later<br>during therapy,<br>excluding the<br>above<br>conditions | Gonadal<br>dysfunction/infertility,<br>azoospermia, amenorrhea | | Alopecia, secondary malignancy |
| Unknown<br>Frequency and<br>Timing: | Fetal and teratogenic toxicities: Carcinogenic and teratogenic effects of thiotepa have been noted in animal models at doses ≤ to those used in humans. It is not known if thiotepa is excreted into human breast milk. | | |

(L) Toxicity may also occur later.

#### Formulation and Stability:

Thiotepa for Injection *USP*, for single use only, is available in vials containing 15 mg of nonpyrogenic, sterile lyophilized powder. Store in a refrigerator at 2°-8°C (36°-46°F). **PROTECT FROM LIGHT AT ALL TIMES.** 

**Note:** FDA is allowing temporary importation of a European product (Tepadina). Verify product, storage, and preparation instructions prior to dispensation and administration. Refer to specific product labeling for details.

Tepadina: Store intact vials under refrigeration at 2°C to 8°C (36°F to 46°F). Protect from light; do not freeze. Reconstituted solution (10 mg/mL) is stable for 8 hours when stored at 2°C to 8°C (36°F to 46°F). Solution further diluted for infusion is stable for 24 hours when stored at 2°C to 8°C (36°F to 46°F), or for 4 hours when stored at 25°C (77°F).

Guidelines for Administration: See <u>Treatment</u> and <u>Dose Modifications</u> sections of the protocol. Reconstitute Thiotepa for Injection with 1.5 mL of Sterile Water for Injection resulting in a drug concentration of approximately 10 mg/mL. (As per manufacturer's information: Actual content per vial 15.6 mg; withdrawable amount 14.7 mg/1.4 mL; approximate reconstituted concentration:



10.4 mg/mL). When reconstituted with Sterile Water for Injection, solutions of thiotepa should be stored at refrigerated temperatures 2°-8°C (36°-46°F) protected from light and used within 8 hours. The reconstituted solution is hypotonic and should be further diluted with Sodium Chloride Injection (0.9% NaCl) prior to use. Thiotepa at a concentration of 1-5mg/mL in 0.9% NaCl is stable for 24 hours at room temperature. At concentration of 0.5mg/mL it is stable for only one hour and stability decreases significantly at concentrations of less than 0.5mg/mL. Therefore, solutions diluted to 0.5mg/mL should be used immediately

In order to eliminate haze, filter solutions through a 0.22 micron filter [Polysulfone membrane (Gelman's Sterile Aerodisc®, Single Use) or triton-free mixed ester of cellulose/PVC (Millipore's MILLEX®-GSFilter Unit)] prior to administration. Filtering does not alter solution potency. Reconstituted solutions should be clear. Solutions that remain opaque or precipitate after filtration should not be used.

Tepadina: Reconstitute each 15 mg vial with 1.5 mL SWFI, or each 100 mg vial with 10 mL SWFI, to a concentration of 10 mg/mL. Gently mix by repeated inversions. Solution may be clear or opalescent; do not use if particulate matter is present. Further dilute reconstituted solution for IV infusion in 500 mL NS (1,000 mL NS if dose >500 mg). If dose is <250 mg, dilute in an appropriate volume of NS to achieve a final concentration of 0.5 to 1 mg/mL.

When thiotepa is given in bone marrow transplant doses, bath the patient and change linen frequently ( $\geq 2$  baths/day) to avoid the contact dermatitis and discoloration of the skin that is seen with high dose.

**Supplier:** Commercially available. See package insert for further information.

#### 6.20 VINCRISTINE SULFATE

(08/16/12)

168

(Oncovin®, VCR, LCR) NSC #67574

#### Source and Pharmacology:

Vincristine is an alkaloid isolated from Vinca rosea Linn (periwinkle). It binds to tubulin, disrupting microtubules and inducing metaphase arrest. Its serum decay pattern is triphasic. The initial, middle, and terminal half-lives are 5 minutes, 2.3 hours, and 85 hours respectively; however, the range of the terminal half-life in humans is from 19 to 155 hours. The liver is the major excretory organ in humans and animals; about 80% of an injected dose of vincristine sulfate appears in the feces and 10% to 20% can be found in the urine. The p450 cytochrome involved with vincristine metabolism is CYP3A4. Within 15 to 30 minutes after injection, over 90% of the drug is distributed from the blood into tissue, where it remains tightly, but not irreversibly bound. It is excreted in the bile and feces. There is poor CSF penetration.

**Toxicity:** 

| • | Common | Occasional | Rare |
|---|---|---|---|
| | Happens to 21-100 children | Happens to 5-20 children | Happens to < 5 children |
| | out of every 100 | out of every 100 | out of every 100 |
| Immediate: | | Jaw pain, headache | Extravasation (rare) but if |
| Within 1-2 days | | | occurs = local ulceration, |
| of receiving drug | | | shortness of breath, and |
| | | | bronchospasm |
| Prompt: | Alopecia, constipation | Weakness, abdominal | Paralytic ileus, ptosis, |
| • | - | pain, mild brief | diplopia, night blindness, |



| Within 2- | | myelosuppression | hoarseness, vocal cord |
|---|---|---|---|
| 3 weeks, prior to | | (leukopenia, | paralysis, SIADH, seizure, |
| the next course | | thrombocytopenia, | defective sweating |
| | | anemia) | _ |
| Delayed: | Loss of deep tendon | Peripheral paresthesias | Difficulty walking or |
| Any time later | reflexes | including numbness, | inability to walk; |
| during therapy | | tingling and pain; | sinusoidal obstruction |
| | | clumsiness; wrist drop, | syndrome (SOS, formerly |
| | | foot drop, abnormal gait | VOD) (in combination); |
| | | | blindness, optic atrophy; |
| | | | urinary tract disorders |
| | | | (including bladder atony, |
| | | | dysuria, polyuria, nocturia, |
| | | | and urinary retention); |
| | | | autonomic neuropathy |
| | | | with postural hypotension; |
| | | | 8 <sup>th</sup> cranial nerve damage |
| | | | with dizziness, nystagmus, |
| | | | vertigo and hearing loss |
| Unknown | Fetal toxicities and terate | ogenic effects of vincris | stine (either alone or in |
| Frequency and | combination with other ant | ineoplastic agents) have b | een noted in humans. The |
| Timing: | toxicities include: chromosome abnormalities, malformation, pancytopenia, | | |
| | and low birth weight. It is u | ınknown whether the drug | is excreted in breast milk. |

#### Formulation and Stability:

Vincristine is supplied in 1 mL and 2 mL vials in which each mL contains vincristine sulfate 1 mg (1.08  $\mu$ mol), mannitol 100 mg, SWFI; acetic acid and sodium acetate are added for pH control. The pH of vincristine sulfate injection, *USP* ranges from 3.5 to 5.5. This product is a sterile, preservative free solution. Store refrigerated at 2°-8°C or 36°-46°F. Protect from light and retain in carton until time of use.

Do not mix with any IV solutions other than those containing dextrose or saline.

Guidelines for Administration: See Treatment and Dose Modifications sections of protocol.

The World Health Organization, the Institute of Safe Medicine Practices (United States) and the Safety and Quality Council (Australia) all support the use of minibag rather than syringe for the infusion of vincristine. The delivery of vincristine via either IV slow push or minibag is acceptable for COG protocols. Vincristine should **NOT** be delivered to the patient at the same time with any medications intended for central nervous system administration. Vincristine is fatal if given intrathecally.

Injection of vincristine sulfate should be accomplished as per institutional policy. Vincristine sulfate must be administered via an intact, free-flowing intravenous needle or catheter. Care should be taken to ensure that the needle or catheter is securely within the vein to avoid extravasation during administration. The solution may be injected either directly into a vein or into the tubing of a running intravenous infusion.

#### **Special precautions:** FOR INTRAVENOUS USE ONLY.

The container or the syringe containing vinCRIStine must be enclosed in an overwrap bearing the statement: "Do not remove covering until moment of injection. For intravenous use only - Fatal if given by other routes."



**Supplier:** Commercially available from various manufacturers. See package insert for more detailed information.



#### 7.0 EVALUATIONS/MATERIAL AND DATA TO BE ACCESSIONED

Timing of protocol therapy administration, response assessment studies, and surgical interventions are based on schedules derived from the experimental design or on established standards of care. Minor unavoidable departures (up to 72 hours) from protocol directed therapy and/or disease evaluations (and up to 1 week for surgery) for valid clinical, patient and family logistical, or facility, procedure and/or anesthesia scheduling issues are acceptable per COG administrative Policy 5.14 (except where explicitly prohibited within the protocol).

# 7.1 Required and Optional Clinical, Laboratory and Disease Evaluations All baseline studies must be performed prior to starting protocol therapy unless otherwise indicated. Obtain other studies prior to start of phase unless otherwise indicated.

#### 7.1a **HR/IR Patients**

| STUDIES TO BE OBTAINED | Baseline | Block 1 | Block 2 | Block 3 | Blinatumomab Blocks |
|---|---|---|---|---|---|
| Hx/PE with VS/Wt (BSA) | X | | start of | start of | start of phase* |
| | | | phase | phase | |
| CBC/diff/plts | X | weekly | weekly | weekly | weekly |
| Bilirubin <sup>0</sup> , ALT, creatinine, BUN | X | weekly | weekly | weekly | weekly |
| Local Bone Marrow (BM) | $X^1$ | end of | end of | end of | end of phase |
| Evaluation | | phase | phase | phase | |
| Bone Marrow (BM) for central | | end of | end of | end of | end of Cycle 1++, |
| flow MRD <sup>2</sup> | | phase+ | phase++ | phase+++ | end of Cycle 2+++ |
| Bone Marrow (BM) for | $X^{2,7}$ | | | | |
| Immunophenotyping | | | | | |
| Bone Marrow (BM) for future | $X^8$ | X8 | | | |
| research banking | Λ | | | | |
| CSF cell count and cytospin | X | with | with each | with each | with each IT |
| | | each IT | IT | IT | |
| Peripheral Blood for | | | | | Cycle 1: Day 2 and Day |
| Pharmacokinetics (PK) | | | | | 14 <sup>6</sup> |
| Peripheral Blood for | | | | | • Prior to (Hour 0) start |
| Immunogenicity | | | | | of first blinatumomab |
| | | | | | infusion (Cycle 1) |
| | | | | | • End of Cycle 2 <sup>\$</sup> |
| Peripheral Blood for future | X8 | X8 | $X^8$ | | $X^8$ |
| research banking | | 21 | 21 | | A |
| Echocardiogram | X | | | | |
| Pregnancy test <sup>3</sup> | X | | | | |
| Testicular exam | X | end of | end of | | |
| | | phase | phase | | |
| Testicular biopsy | X <sup>4</sup> | $X^5$ | | | |

- Adequate liver function as defined by direct bilirubin is required for eligibility (see Section 3.2.5.2).
- <sup>1</sup> BM evaluation to confirm relapse and/or detect marrow disease in presumed isolated extramedullary relapse patients should include morphology, immunophenotyping & cytogenetics/FISH. Cytogenetic/FISH analysis must be performed at a COG approved cytogenetics lab and cases will be reviewed retrospectively by the COG Cytogenetics Committee. See <a href="Section 13.2">Section 13.2</a> for details.
- <sup>2</sup> See <u>Section 13.3</u> for details on shipping and handling
- <sup>3</sup> Female patients of childbearing potential require a negative pregnancy test prior to starting treatment; sexually active patients must use an acceptable method of birth control.
- <sup>4</sup> Patients with suspected testicular involvement at relapse (either isolated or with concurrent BM/CNS relapse) must have biopsy performed at baseline.
- <sup>5</sup> Patients with definite or equivocal residual testiculomegaly at end of Block 1 must have a biopsy to determine whether TRT is to be given during designated blocks of therapy (see <a href="Experimental Design Schema"><u>Experimental Design Schema</u></a>).
- <sup>6</sup> See lab manual on protocol webpage for sample collection and shipping details
- <sup>7</sup> Includes optional sample for CRLF2 expression for consenting patients (see Section 7.2 and Section 13.4).



- <sup>8</sup> Optional for future research (see Section 7.2 and Section 13.1).
- \* See recommended vital sign monitoring for Blinatumomab blocks in Section 7.1e
- § In cases where blinatumomab treatment will not continue to Cycle 2, collect sample at end of Cycle 1.
- + Evaluation 1 ++ Evaluation 2 +++ pre-HSCT evaluation

This table only includes evaluations necessary to answer the primary and secondary aims. Obtain other studies as indicated for good clinical care.

#### 7.1b LR Patients

| STUDIES TO BE<br>OBTAINED | Baseline | Block 1 | Block 2 | Block 3,<br>Blinatumomab<br>blocks, Continuation | Maintenance and post-therapy |
|---|---|---|---|---|---|
| Hx/PE with VS/Wt (BSA) | X | | start of<br>phase | start of phase* | every 28 days<br>during<br>maintenance |
| CBC/diff/plts | X | weekly | weekly | weekly | every 28 days<br>during<br>maintenance |
| Bilirubin <sup>0</sup> , ALT, creatinine, BUN | X | weekly | weekly | weekly | every 28 days<br>during<br>maintenance |
| Local Bone Marrow | $X^1$ | end of | end of | | |
| (BM) Evaluation | | phase | phase | | |
| Bone Marrow (BM) for | | end of | end of | | |
| central flow MRD <sup>2</sup> | | phase+ | phase++ | | |
| Bone Marrow (BM) for | $X^{2,7}$ | | | | |
| Immunophenotyping | | | | | |
| Bone Marrow (BM) for | $X^9$ | $X^9$ | | | |
| future research banking | | | | | |
| CSF cell count and | X | with | with | with each IT | with each IT |
| cytospin | | each IT | each IT | | |
| Absolute lymphocyte | | | | | At end of each 12 |
| count with T and B | | | | | week maintenance |
| subset quantification | | | | | cycle, and every 3 |
| | | | | | months after |
| | | | | | completion of therapy for 1 year |
| Peripheral Blood for | | | | Blinatumomab Cycle | therapy for 1 year |
| Pharmacokinetics (PK) | | | | 1:Day 2 and Day 14 <sup>6</sup> | |
| Peripheral Blood for | | | | •Prior to (Hour 0) start | Prior to start of |
| Immunogenicity | | | | of first blinatumomab | Maintenance |
| immunogementy | | | | infusion (Cycle 1) •End of Cycle 2 <sup>\$</sup> | Cycle 1 therapy <sup>8</sup> |
| Peripheral Blood for future research banking | X <sup>9</sup> | X <sup>9</sup> | X <sup>9</sup> | | X <sup>9</sup> |
| Echocardiogram | X | | | | |
| Pregnancy Test <sup>3</sup> | X | | | | |
| Testicular Biopsy | $X^4$ | X <sup>5</sup> | | | |

Adequate liver function as defined by direct bilirubin is required for eligibility (see <u>Section 3.2.5.2</u>).

BM evaluation to confirm relapse and/or detect marrow disease in presumed isolated extramedullary relapse patients should include morphology, immunophenotyping & cytogenetics/FISH. Cytogenetic/FISH analysis must be performed at a COG approved cytogenetics lab and cases will be reviewed retrospectively by the COG Cytogenetics Committee. See Section 13.2 for details.

<sup>&</sup>lt;sup>2</sup> See Section 13.3 for details on shipping and handling

Female patients of childbearing potential require a negative pregnancy test prior to starting treatment; sexually active patients must use an acceptable method of birth control.



- <sup>4</sup> Patients with suspected testicular involvement at relapse (either isolated or with concurrent BM/CNS relapse) must have biopsy performed at baseline.
- <sup>5</sup> Patients with definite or equivocal residual testiculomegaly at end of Block 1 must have a biopsy to determine whether TRT is to be given during designated blocks of therapy (see <a href="Experimental Design Schema">Experimental Design Schema</a>).
- <sup>6</sup> See lab manual on protocol webpage for sample collection and shipping details
- <sup>7</sup> Includes optional sample for CRLF2 expression for consenting patients (see Section 7.2 and Section 13.4).
- <sup>8</sup> **Arm D ONLY.** Prior to start of Maintenance therapy for eligible patients (see <u>Section 13.7</u> and lab manual for details)
- <sup>9</sup> Optional for future research (see <u>Section 7.2</u> and <u>Section 13.1</u>).
- \* See recommended vital sign monitoring for Blinatumomab blocks in Section 7.1e
- In cases where blinatumomab treatment will not continue to Cycle 2, collect sample at end of Cycle 1.
- + Evaluation 1 ++ Evaluation 2

This table only includes evaluations necessary to answer the primary and secondary aims. Obtain other studies as indicated for good clinical care.

#### 7.1c **HSCT**

| Observation | Prior to | 1-2 | 3 mo | 6 mo | 9 mo | 1 yr. | 2 | 3 | 4 | 5 | At |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | transplant | weeks | Post- | Post- | Post- | Post- | yrs. | yrs. | yrs. | yrs. | subsequent |
| | (Tx) | after | Tx | Tx | Tx | Tx | Post- | Post- | Post- | Post- | relapse |
| | | ANC> | | | | | Tx | Tx | Tx | Tx | |
| | | 500/μL | | | | | | | | | |
| Bone | X+++ | X* | X** | | | | | | | | |
| Marrow | | | | | | | | | | | |
| (BM) for | | | | | | | | | | | |
| central | | | | | | | | | | | |
| $MRD^1$ | | | | | | | | | | | |
| CSF cell | X | | | | | | | | | | X |
| count and | | | | | | | | | | | |
| cytospin | | | | | | | | | | | |
| CBC, | X | X | X | X | X | X | X | | | | X |
| differential, | | | | | | | | | | | |
| platelets | | | | | | | | | | | |
| BUN, | X | | | | | | | | | | |
| Creatinine | | | | | | | | | | | |
| LFT | X | X | X | X | X | X | X | | | | |
| Pulmonary | X | | | | | | | | | | |
| function test | | | | | | | | | | | |
| Performance | X | X | X | X | X | X | X | X | X | X | X |
| score | | | | | | | | | | | |

See Section 13.3 for details on shipping and handling; (see Section 7.2)

This table only includes evaluations necessary to answer the primary and secondary aims. Obtain other studies as indicated for good clinical care.

#### 7.1d Salvage Therapy (Blinatumomab-S)

| STUDIES TO BE | Blinatumomab Blocks |
|------------------|---------------------|
| OBTAINED | |
| Hx/PE with VS/Wt | Start of phase* |
| (BSA) | - |
| CBC/diff/plts | weekly |

<sup>+++</sup> pre-HSCT evaluation

<sup>\*</sup> Day 30 (25-30)

<sup>\*\*</sup> Day100 (+/- 3 weeks)



| Bilirubin, ALT, | weekly |
|---|---|
| creatinine, BUN | |
| Local Bone Marrow | end of phase |
| (BM) Evaluation | |
| Bone Marrow (BM) for | pre-HSCT |
| central flow MRD <sup>2</sup> | |
| CSF cell count and | with each IT |
| cytospin | |
| Peripheral Blood for | Cycle 1: Day 2 and Day 14** |
| Pharmacokinetics (PK) | |
| Peripheral Blood for | •Prior to (Hour 0) start of first blinatumomab infusion (Cycle 1) |
| Immunogenicity | •End of Cycle 2 <sup>§</sup> |

<sup>\*</sup> See recommended vital sign monitoring for Blinatumomab blocks in Section 7.1e

#### 7.1e Recommended Observations: Blinatumomab Blocks

The investigator is recommended to monitor the patient's vital signs (body temperature, heart rate and blood pressure) approximately every 4 hours during the first 12 hours after the start of a cycle, and upon resumption after suspension for adverse event. On Day 2 and 3 vital signs should be measured once daily.

#### 7.2 Research Studies

The following are correlative biology studies for which patient participation is optional. Please see Section 13.0 for details on volumes of specimen collection and shipping information. Note: Patient consent is required.

| Study | Summary of Sample and Timing |
|---|---|
| (see section for details) | |
| Banking for Future | Peripheral blood: |
| Research * | Baseline |
| ( <u>Section 13.1</u> ) | • End Block 1 |
| | • End Block 2 (Arm A, C or D, End of Blinatumomab<br>Cycle 1 (Arm B) |
| | Relapse |
| | Bone marrow: |
| | Baseline |
| | • End Block 1 |
| | Relapse |
| CRLF2 expression | No separate specimen required – cell pellet from required |
| ( <u>Section 13.4</u> ) | baseline central flow bone marrow will be used |
| Protein Cell Stress | Peripheral blood: |
| ( <u>Section 13.6</u> ) | Day 1 of Block 1 |
| | o Before chemotherapy (Hour 0) |
| | <ul> <li>After Chemotherapy (Hour 6 and Hour 24)</li> </ul> |
| Blinatumomab | Bone marrow: |
| Pharmacodynamics (PD) | • End Block 1 (All patients) |
| ( <u>Section 13.5</u> ) | • End Block 2 (LR patients on Arm D only) |

<sup>\*\*</sup> See lab manual on protocol webpage for sample collection and shipping details

In cases where blinatumomab treatment will not continue to Cycle 2, collect sample at end of Cycle 1.



| Peripheral blood: |
|--------------------------------------------------------------------|
| <ul> <li>Prior to (Hour 0) start of first blinatumomab</li> </ul> |
| infusion |
| <ul> <li>During (Hour 6, Hour 12, Day 2, Day 7, Day 14,</li> </ul> |
| Day 21) first blinatumomab infusion** |

<sup>\*</sup> For cases with a limited amount of tissue available for analysis, please prioritize specimen for tissue banking.

## 7.3 **At Relapse**

Patients who relapse and have consented to cell banking <u>at time of enrollment</u> should have samples of bone marrow sent to the Molecular Reference Laboratory for cell banking (see <u>Section 13.1</u>.)

# 7.4 Follow-up

See COG Late Effects Guidelines for recommended post treatment follow-up: <a href="http://www.survivorshipguidelines.org/">http://www.survivorshipguidelines.org/</a>

**Note:** Follow-up data are expected to be submitted per the Case Report Forms (CRFs) schedule.

# 8.0 CRITERIA FOR REMOVAL FROM PROTOCOL THERAPY AND OFF STUDY CRITERIA

## 8.1 Criteria for Removal from Protocol Therapy

- a) Treatment failure but not eligible to receive blinatumomab salvage
- b) Treatment failure that receives blinatumomab salvage but does not achieve CR after 2 cycles of blinatumomab
- c) Adverse events requiring removal from protocol therapy
- d) Refusal of further protocol therapy by patient/parent/guardian.
- e) Completion of planned therapy.
- f) Physician determines it is in patient's best interest.
- g) Development of a second malignancy.
- h) Second relapse at any site.
- i) Repeat eligibility studies are outside the parameters required for eligibility (if applicable, see Section 3.2).
- j) Inevaluable
- k) Found to be ineligible for HSCT (See Section 4.9.1)
- l) **Pre-Randomization (HR/IR or LR):** Interval development of significant central nervous system pathology that would preclude treatment with blinatumomab (see Section 3.2.6.12 for definition).
- m) Amendment #10: Patient found to be HR/IR at the completion of Block 1.

Patients who are off protocol therapy are to be followed until they meet the criteria for Off Study (see below). Follow-up data will be required unless consent was withdrawn.

<sup>\*\*</sup>In the event that the infusion is interrupted, the peripheral blood collection should likewise be delayed to account for the interruption. i.e. collect the timed sample after X days of infusion rather than X days from start of infusion.



#### 8.2 Off Study Criteria

- a) Death.
- b) Lost to follow-up.
- c) Patient enrollment onto another COG study with tumor therapeutic intent (e.g., at recurrence).
- d) Withdrawal of consent for any further data submission.
- e) Tenth anniversary of the date the patient was enrolled on this study.

#### 9.0 STATISTICAL CONSIDERATIONS

# 9.1 Statistical Design

# 9.1.1 Primary Endpoint

A primary objective (HR/IR Randomization) of AALL1331 is to compare disease-free survival (DFS) of HR and IR relapse patients randomized to Block 2 and 3 chemotherapy (Control) vs. two blocks of blinatumomab (Experimental), followed by allogeneic HSCT. DFS is defined as time from start of randomization to event (treatment failure, relapse, second malignancy, death) or last follow-up for those who are event-free. DFS event date will be set at Day 1 if patients are deemed as TF after randomization.

Another primary objective (LR Randomization) of AALL1331 is to compare DFS of LR relapse patients randomized to chemotherapy alone (Control: Block 3, Continuation 1, Continuation 2 and Maintenance) vs. blinatumomab/chemotherapy (Experimental: blinatumomab, Continuation 1, blinatumomab, Continuation 2, blinatumomab, Maintenance). DFS is defined as time from start of randomization to first event (relapse, second malignant neoplasm, remission death) or last follow up for those who are event-free.

The primary analyses of DFS will include all randomized patients provided that randomization is performed per protocol. The analyses will be based on the intent-to-treat principle.

# 9.1.2 <u>Secondary Endpoints</u>

A secondary objective (HR/IR Randomization) of AALL1331 is to compare overall survival (OS) of HR and IR relapse patients randomized to Block 2 and 3 chemotherapy (Control) vs. two blocks of blinatumomab (Experimental), followed by allogeneic HSCT. OS is defined as time from start of randomization to death or last date of contact.

Another secondary objective (LR Randomization) of AALL1331 is to compare OS of LR relapse patients randomized to chemotherapy alone (Control: Block 3, Continuation 1, Continuation 2 and Maintenance) vs. blinatumomab/chemotherapy (Experimental: blinatumomab, Continuation 1, blinatumomab, Continuation 2, blinatumomab, Maintenance). OS is defined as time from start of randomization to death or last date of contact.



#### 9.1.3 Exploratory Endpoints

The exploratory endpoints associated with HR/IR Randomization are to compare the rates of MRD positivity (>0.01%) at the end of Block 2 and 3 between randomized arms for HR and IR relapse patients.

Other exploratory endpoints include estimating the CR rate, MRD negativity (< 0.01%) rate and proportion that proceed to HSCT after treatment with blinatumomab for treatment failure patients not previously receiving blinatumomab, assessing the feasibility and safety of rapid taper of immune suppression for subset of HSCT patients with MRD  $\geq$  0.01% pre- and/or post-HSCT with no aGVHD, and collecting biologic samples for the prospective correlative biology studies described in Section 7.0.

Blinatumomab PK will be evaluated by summarizing blinatumomab steady state concentrations and systemic clearance obtained from non-compartmental analysis. In addition, a population PK approach using a non-linear mixed effect model will also be used to assess blinatumomab PK. Exposure-response analyses will be performed to explore associations among blinatumomab exposure, relevant clinical covariates and clinical measures of saftery and efficacy.

# 9.2 Patient Accrual and Expected Duration of Trial

#### 9.2.1 Stratification to be used in the randomization

All patients are assigned to Stratum 1 at enrollment. All HR/IR relapse patients who do not meet the treatment failure criteria at the end of Block 1 will be eligible for HR/IR randomization and randomized equally between experimental (blinatumomab) and control (chemotherapy) arms. The randomization will occur upon recovery from Block 1 of therapy, and will be stratified by: 1) Risk Group (HR vs. IR); 2) For HR patients, site of relapse (marrow vs. IEM); 3) For HR – marrow patients, duration of first remission (< 18 months vs. 18-36 months from diagnosis); 3) For HR-marrow patients, MRD level end Block 1 (< 0.1% vs.  $\geq$  0.1%) to ensure balanced randomization within these subsets (see table below).

| Stratum # | Risk-Site | CR1 mos | MRD status |
|-----------|-----------|---------|------------|
| 2 | HR-Marrow | < 18 | MRD < 0.1% |
| 3 | HR-Marrow | < 18 | MRD ≥ 0.1% |
| 4 | HR-Marrow | 18-36 | MRD < 0.1% |
| 5 | HR-Marrow | 18-36 | MRD ≥ 0.1% |
| 6 | HR-IEM | <18 | - |
| 7 | IR | - | - |

All late B-ALL marrow and late B-ALL IEM relapse patients with end Block 1 MRD < 0.1% will eligible for LR randomization and randomized equally between experimental (blinatumomab) and control (chemotherapy) arms. The randomization will occur upon recovery from Block 1 of therapy, and will be stratified by: 1) site of relapse (marrow vs. IEM); and 2) MRD level at time of randomization (< 0.01% vs.  $\geq$  0.01%) to ensure balanced randomization within these subsets.



| Stratum # | Site | CR1 mos | MRD status |
|-----------|-----------|---------|-----------------------------------|
| 8 | LR-Marrow | ≥ 36 | MRD < 0.01% |
| 9 | LR-Marrow | ≥ 36 | $MRD \ge 0.01\%$ or $MRD < 0.1\%$ |
| | | | with sensitivity 1/1000 |
| 10 | LR-IEM | ≥ 18 | MRD < 0.01% |
| 11 | LR-IEM | ≥ 18 | $MRD \ge 0.01\%$ or $MRD < 0.1\%$ |
| | | | with sensitivity 1/1000 |

#### 9.2.2 Sample size with power calculation (Activation Protocol)

Sample size calculations driving this study are based on the two randomized questions HR/IR Randomization and LR Randomization.

For HR/IR Randomization, approximately 170 evaluable HR/IR B-ALL patients are to be randomized between experimental (blinatumomab) and control (chemotherapy) arms after recovery from Block 1. As described in Section 9.3.1, the test of the randomization question has a power of 80.0% at a one-sided significance level of 2.5% to detect the desired improvement in 2-year DFS rate. The 170 evaluable HR/IR B-ALL patients are expected to take 3 years to be enrolled with the total rate of accrual to HR/IR Randomization to be 56 per year after adjusting for approximate 10% refusal rate to randomization. This estimate is based on the following estimates of annual accrual and dropout rate from past studies AALL01P2, AALL02P2, AALL0433 and ADVL04P2:

| | Early<br>marrow | Early<br>IEM | Late<br>marrow | Late<br>IEM |
|---|---|---|---|---|
| # entering study | 60 | 5 | 44 | 28 |
| Rate of MRD $\geq 0.1\%$ | - | - | 38% | 12% |
| Rate of not dropping out prior to block 2 (due to toxicity and/or treatment failure) | 70% | 70% | 90% | 90% |
| # eligible for randomization | 42 | 3 | 15 | 3 |

For LR randomization, approximately 206 evaluable LR B-ALL patients are to be randomized between experimental (blinatumomab) and control (chemotherapy) arms after recovery from Block 1. As described in Section 9.3.2, the test of the randomization question has a power of 80.4% at a one-sided significance level of 5% to detect the desired improvement in 3-year DFS rate. The 206 evaluable LR B-ALL patients are expected to accrue over 5.6 years with total rate of accrual to LR Randomization to be 37 per year after adjusting for approximate 10% refusal rate to randomization. This estimate is based on the following estimates of annual accrual and dropout rate from past studies AALL01P2, AALL02P2, AALL0433 and ADVL04P2:

| | Late marrow | Late IEM |
|--------------------|-------------|----------|
| # entering study | 44 | 28 |
| Rate of MRD < 0.1% | 62% | 88% |



| Rate of not dropping out prior to block 2 (due to toxicity and/or treatment failure) | 80% | 80% |
|---|---|---|
| # eligible for randomization | 22 | 20 |

Therefore, in order to enroll 170 and 206 evaluable patients for HR/IR and LR Randomization respectively, a total of 195 early marrow/IEM and 403 late marrow/IEM patients are expected be accrued at the beginning of the study.

# 9.2.3 Extension of accrual duration for both the LR cohort and the HR/IR cohort (Amendment #8)

With Amendment #8, for both the LR cohort and the HR/IR cohort, the accrual duration will be extended until 10/31/2019, provided that there is no prolonged interruption of study enrollment.

The AALL1331 study has demonstrated a steady accrual rate for both the LR cohort and the HR/IR cohort. The observed accrual rate is approximately 53 patients/year in the LR cohort, much faster than the anticipated 37/year, and is 50 patients/year in the HR/IR cohort, slightly smaller than but very close to the anticipated 56/year. With the faster accrual rate in the LR cohort and steady observed accrual rate in HR/IR, we amend the accrual duration for both cohorts to be until 10/31/2019 to ensure that the primary analyses maintain sufficient statistical power for the LR cohort and that the timing of completion of accrual be the same between the two cohorts. This amendment in accrual target will increase the power of statistical analyses and the sensitivity of the study, help us to gather more accurate information regarding the treatment regimens, and will not cause delay in addressing the primary objectives of the study or delay in opening the planned successor trial to AALL1331 (AALL1821). AALL1331 is the first pediatric ALL study to substitute blocks of immunotherapy for conventional chemotherapy and the increased power of the analyses may be very beneficial in moving this general approach forward in future studies.

#### 9.2.3.1 The LR Cohort

For the LR cohort, the study was originally designed to have approximately power of 0.80 to detect a hazard ratio of 0.55 with a one-sided logrank test and Type I error of 0.05, which corresponds to an increase in 3-year DFS rate from 73% in the control arm to 84% in the experimental arm. This cohort was planned to enroll a total of 206 randomized, evaluable patients. It was expected to accrue for 5.6 years, with 3 years of additional follow-up after completion of enrollment. With the observed accrual rate of 53 patients/year, the anticipated accrual completion date (ACD) with the original sample size of 206 is approximately 03/2019, and the anticipated analysis date (AAD) is 3 years after that, i.e., 03/2022.

Given the faster-than-expected observed accrual rate, if this cohort follows the original plan to enroll 206 evaluable patients and have 3 years of additional follow-up, the power of the study will be smaller than planned due to the shorter average follow-up time among the patients. This is


demonstrated by the comparison of the dotted black line to the solid red line in the figure below. As shown by the dotted black line, with the observed accrual rate of 53/year, the study will only have power of 0.77 to detect a hazard ratio of 0.55, smaller than the planned power of 0.80.



The faster observed accrual rate in the LR cohort gives us the opportunity to address this issue by enrolling more patients, resulting in an increase in the power of the analysis, an increase in the sensitivity of the study, and the ability to gather more accurate information regarding the treatment regimens. With Amendment #8, we extend the accrual duration for the LR cohort to be until 10/31/2019. This will increase the number of evaluable patients from 206 to approximately 236. With this extended accrual duration, the ACD and AAD will be 10/2019 and 10/2022, respectively (please see Section 9.3.2.1 for more details on the primary analysis with Amendment #8). (Note that the AAD of 10/2022 is still earlier than the AAD had the accrual rate been the assumed 37 patients/year.) With 236 evaluable patients, the study will have approximately power of 0.83 to detect a hazard ratio of 0.55, and power of 0.75 to detect a hazard ratio of 0.59.

The following table presents a comparison in characteristics of the trial for the LR cohort under the scenarios of (1) the original accrual target with the expected accrual rate, (2) the original accrual target with the observed accrual rate, and (3) the extended accrual duration with Amendment #8.

| | Characteristics | Original Accrual Target (assuming expected accrual rate) | Original Accrual Target (with observed accrual rate) | Extended Accrual Duration (Amendment #8) |
|---|---|---|---|---|
| 1 | Accrual rate | 37 pts/year | 53 pts/year | 53 pts/year |
| 2 | Sample size | 206 | 206 | 236 |
| 3 | Accrual completion date (ACD) | 06/2020 | 03/2019 | 10/2019 |
| 4 | Anticipated analysis date (AAD) | 06/2023 | 03/2022 | 10/2022 |



| 5 | Power of detecting a hazard ratio of 0.55 (corresponding to 3-year DFS of 84% vs. 73%) | 0.80 | 0.77 | 0.83 |
|---|---|---|---|---|
| 6 | Power of detecting a hazard ratio of 0.59 (corresponding to 3-year DFS of 83% vs. 73%) | 0.72 | 0.69 | 0.75 |
| 7 | Sample size for evaluation of toxicities and biologic aims | | | Increased by 14% |
| 8 | Delay in addressing primary<br>aim, compared to the original<br>accrual target | | | No delay |
| 9 | Timing of completion of accrual compared to the HR/IR cohort | | 5~6 more months<br>of accrual if<br>without<br>amendment of<br>accrual target of<br>the two cohorts. | The same as<br>the HR/IR<br>cohort with<br>Amendment<br>#8. |

#### 9.2.3.2 The HR/IR Cohort

For the HR/IR cohort, the study was originally designed to have approximately power of 0.80 to detect a hazard ratio of 0.58 with a one-sided logrank test and Type I error of 0.025, which corresponds to an increase in 2-year DFS rate from 45% in the control arm to 63% in the experimental arm. This cohort was planned to enroll a total of 170 randomized, evaluable patients. It was expected to accrual for approximately 3 years, with 2 years of additional follow-up after completion of enrollment. With the original sample size of 170 patients, the ACD is approximately 10/2018, and the AAD is 2 years after that, i.e., 10/2020.

If staying with the originally planned accrual target, the HR/IR randomization would be closed approximately 5-6 months earlier than the LR cohort. After closure of the HR/IR randomization, we would need to continue to enroll patients with late relapses to fulfill the accrual target for the LR cohort. A subset of patients with late relapses would be assigned the IR group at the completion of the induction therapy, and would subsequently need to be taken off therapy due to the closure of the HR/IR randomization.

To avoid having to reject patients from further protocol therapy, with Amendment #8, we extend the accrual duration for HR/IR so that this cohort will complete accrual at the same time as the LR cohort. That is, we extend accrual duration of HR/IR to be until 10/31/2019, the same as the LR cohort. We plan that the primary analysis for the HR/IR cohort be conducted approximately 1 year later (please see Section 9.3.1.1 for more details on the primary analysis with Amendment #8). Hence the AAD will be approximately 10/2020. Given that the protocol therapy duration for HR/IR patients is typically 7 months, by 10/2020 all patients in the HR/IR cohort should have completed protocol therapy. This AAD is the same as the AAD for HR/IR if we did not amend the accrual target.



In summary, the increased accrual target of the HR/IR cohort will give us the same timing of completion of accrual between the HR/IR cohort and the LR cohort, without causing any delay in addressing the primary objectives. The increased accrual target will also improve the sensitivity of this cohort and increase the power to detect a smaller difference in treatment effect between the experimental arm vs. the control arm. As shown in the figure below, the sample size of 220 evaluable patients will increase the power to detect a hazard ratio of 0.58 from 0.80 to 0.85.



The following table presents a comparison in characteristics of the trial for the HR/IR cohort under the scenarios of (1) the original accrual target, and (2) the extended accrual duration with Amendment #8.

| | Characteristics | Original<br>Accrual Target | Extended Accrual Duration (Amendment #8) |
|---|---|---|---|
| 1 | Sample size | 170 | 220 |
| 2 | Accrual completion date (ACD) | 10/2018 | 10/2019 |
| 3 | Anticipated analysis date (AAD) | 10/2020 | 10/2020 |
| 4 | Power of detecting a hazard ratio of 0.58 (corresponding to 2-year DFS of 63% vs. 45%) | 0.80 | 0.85 |
| 5 | Sample size for evaluation of toxicities and biologic aims | | Increased by 29% |
| 6 | Delay in addressing primary<br>aim, compared to the original<br>accrual target | | No delay |
| 7 | Timing of completion of accrual compared to the LR cohort | 5~6 months ahead if without amendment of accrual target of the two cohorts. | The same as the LR cohort with Amendment #8. |



## 9.2.3.3 Accrual target (Amendment #8)

With Amendment #8, both the LR cohort and the HR/IR cohort will enroll until 10/31/2019, provided that there is no prolonged interruption of study enrollment. Based on the observed accrual rates, it is anticipated, but not required, that we will enroll approximately a total of 220 randomized HR/IR patients and a total of 236 randomized LR patients. By 10/31/2019, it is expected that the total accrual on this study will not surpass 700 patients, including patients who are not eligible for or refuse randomization.

#### 9.3 Statistical Analysis Methods

#### 9.3.1 HR/IR Randomization for HR and IR relapse patients

# 9.3.1.1 Primary endpoint: intent-to-treat DFS

# The original design (Activation Protocol)

The primary efficacy analysis for HR/IR Randomization will be an intentto-treat comparison of the DFS curves between the randomized arms based on the Log-rank test. All HR/IR relapse patients who are not deemed as treatment failures at the end of Block 1 will be eligible for HR/IR Randomization. The randomization will occur upon recovery from Block 1 of therapy, and will be stratified as described in Section 9.2. From the past studies of AALL01P2, AALL02P2 and ADVL04P2, the overall 2-year DFS rate for HR/IR patients was approximately 45%. Although most events are projected to occur within 2 years, events continue to occur in subsequent years, and hence an exponential distribution is considered more appropriate than a cure-rate model for comparing survival curves for this cohort of patients at the time of final analysis. Assuming a minimum of 2 years of follow up, an estimate of 170 evaluable patients will need to be randomized to achieve the goal of 18% improvement in 2-year DFS rate with blinatumomab over the expected 2-year DFS rate of 45% with chemotherapy backbone alone, with 80.0% power at a one-sided significance level of 2.5%, which represents a 42.1% reduction in hazard rate. The power calculations are based on the assumption of proportional hazards and using the log rank test.

Interim analysis will be conducted to monitor for efficacy and futility. The efficacy stopping boundaries to be used will be based on the O' Brien-Fleming spending function. The futility boundaries are based on testing the alternative hypothesis at the 0.024 level. E This monitoring rule can be applied to any interim analysis schedule and maintains the overall significance level of 0.025. Assuming exponential distribution and the final analysis is performed at the 2 years after the completion of enrollment, the expected maximum number of events to be observed is estimated to be 109. The first interim analysis will be performed after 36 events have been observed. The cumulative power to detect the desired improvement is approximately 78%. The sample of monitoring boundaries for efficacy and futility with 3 interim analyses are given in the table below.



| Looks | # of events | # of events Information Effica | | Futility<br>Boundary |
|---|---|---|---|---|
| 1 | 36 | 33% | 3.731 | -0.392 |
| 2 | 73 | 67% | 2.504 | 0.280 |
| 3 | 109 | 100% | 1.994 | 1.994 |

## Re-design for the HR/IR cohort (Amendment #8)

## Summary of the original design

For the HR/IR cohort, the study was originally designed to have approximately power of 0.80 to detect a hazard ratio of 0.58 using a one-sided logrank test with Type I error of 0.025, which corresponds to an increase in 2-year DFS rate from 45% in the control arm to 63% in the experimental arm. This cohort was originally planned to enroll a total of 170 randomized, evaluable patients. It was expected to accrual for approximately 3 years, with 2 years of additional follow-up after completion of enrollment.

#### Extended accrual duration and increased sample size

With the extended accrual duration, the HR/IR cohort will continue to enroll until 10/31/2019. Based on the observed accrual rate of 50 patients/year, this extended accrual duration will lead to a sample size of approximately 220 randomized patients in the HR/IR cohort. As initially planned, the primary analysis on efficacy will be based on a one-sided logrank test, with one-sided Type I error of 0.025. The primary analysis is planned to be conducted 1 year after completion of accrual provided that the expected total number of events is observed by then. Otherwise the primary analysis will be conducted when the expected total number of events is observed, or at 1.5 years after completion of accrual, whichever comes first. Assuming exponential distribution for the survival function, with 4.4 years of enrollment and 1 year of additional follow-up, the expected total number of events is 131. With the sample size of 220, the study will have approximately power of 0.85 to detect a hazard ratio of 0.58.

#### Interim analysis performed to date

One interim analysis of DFS has been conducted for the HR/IR cohort using data freeze as of 12/31/2017. At the time of this first interim analysis, the observed number of events was 39 (35.8% of the information based on the original full information of 109 events), and the alpha (Type I error) that was spent was 0.00018. The first interim analysis did not cross either the efficacy or futility boundaries.

#### Amended statistical monitoring plan for DFS

With the extension of the accrual duration, the full information now



increases from the original 109 events to 131 events. With the increased expected number of events, the first interim analysis was actually conducted when we had 29.8% of information (rather than 35.8%), and the alpha that would have been spent would be 0.00004 instead of 0.00018. That is, more alpha was spent in the first interim analysis.

A new interim monitoring plan for the future looks for the HR/IR cohort was developed by an independent statistician.

The new monitoring plan for the HR/IR cohort accounts for the alphaspending that has already occurred. Specifically, with the new monitoring plan, the overall alpha to be expended is the original significance level minus the alpha expended with the initial interim monitoring that has been conducted. In the case of the HR/IR cohort, given that for the first look the alpha expended was 0.00018, the remaining alpha of 0.02482 can be used for the new monitoring plan. A monitoring plan that includes two more looks (the second look and the final look) was developed using the O'Brien-Fleming boundaries, with an overall significance level of 0.02482, scheduled at 66.4% and 100% of the total expected information. This way the cohort-wide significance level of 0.025 is maintained. The futility boundaries are based on testing the alternative hypothesis at the 0.024 level. The boundaries are shown in the following table.

| | | Original Efficacy Boundaries | | | | | New Efficacy Boundaries | | | | Futility |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Looks | # of<br>Events | Inf.<br>Time | Upper<br>Boundary<br>of Z value | Nominal<br>Alpha | Cumu.<br>Alpha | Inf. Time<br>Revised | Roundary | | Overall alpha | Futility<br>Boundary<br>of Z value | |
| 1 (done) | 39 | 35.8% | 3.568 | 0.00018 | 0.00018 | 29.8% | | | | 0.00018 | -0.327 |
| 2 | 87 | | | | | 66.4% | 2.519 | 0.00588 | 0.00588 | 0.00606 | 0.363 |
| 3 | 131 | | | | | 100% | 1.995 | 0.02301 | 0.02482 | 0.025 | 1.995 |

# Confirmatory follow-up analysis of DFS of the HR/IR randomized cohort (Amendment #10)

On 09/18/2019, the COG DSMC has recommended closing accrual to the HR/IR arms of AALL1331 and releasing the results of the HR/IR cohort to the study committee. This recommendation is primarily based on the significantly more favorable tolerability profile of the experimental (blinatumomab) arm, coupled with trending or superior DFS and OS of the blinatumomab arm (per interim analyses performed using data as of 06/30/2019). DSMC has recommended that HR/IR patients assigned to the control arm (Arm A) who are at an appropriate point in their treatment program (prior to receiving Block 3) be offered the opportunity to cross over to the experimental arm (Arm B) to receive blinatumomab.



The following table summarizes the analysis of DFS (the second look) using data as of 06/30/2019.

| | | | Ori | ginal Effica | cy Bound | aries | | New Efficacy Boundaries | | | | Futility | Observed |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Looks | Data Cutoff | # of<br>Events | Inf.<br>Time | Roundary | Nominal<br>Alpha | Cumu.<br>Alpha | Inf. Time<br>Revised | Upper<br>Boundary<br>of Z value | Nominal<br>Alpha | Cumu.<br>Alpha | Overall<br>alpha | Futility<br>Boundary<br>of Z value | Z Statistic |
| 1 | 12/31/2017 | 39 | 35.8% | 3.568 | 0.00018 | 0.00018 | 29.8% | | | | 0.00018 | -0.327 | 1.233 |
| 2 | 06/30/2019 | 80 | | | | | 61.1% | 2.644 | 0.00409 | 0.00409 | 0.00427 | 0.267 | 1.649 |

A confirmatory follow-up analysis comparing DFS of the control arm vs. the experimental arm will be conducted using the 12/31/2020 data freeze or when 131 events are observed, whichever occurs earlier. This confirmatory analysis will use the HR/IR patients randomized on or prior to 06/30/2019 (103 in the control arm and 105 in the experimental arm).

#### 9.3.1.2 Secondary Endpoint: Intent-to-treat OS

From the past studies of AALL01P2, AALL02P2 and ADVL04P2, the 3-year OS rate for HR/IR patients was approximately 48%, and most deaths occurred within the first 3 years. Therefore, a cure-rate model with exponential distribution assumed during the first 3 years followed by a flat curve is considered for OS analysis. An interim OS analysis will be conducted at the time of the final DFS analysis, i.e. when all the 170 randomized patients are followed up for 2 years. Assuming 17% improvement in 3-year OS rate with blinatumomab over the expected 3-year OS rate of 48% with chemotherapy backbone alone, approximate 70 deaths are to be observed by the time of the interim OS analysis. The power to detect such improvement at a one-sided significance level of 2.5% is approximate 61% based on the log-rank test.

If DFS analysis meets its target level of improvement (i.e. one-sided p-value < 0.025), the formal OS analysis will be performed at at 1 year after the interim OS analysis, by which time approximate 74 deaths are to be observed. The power to detect the above desired improvement is approximately 63%.

# Power of the analysis of OS with the extended accrual duration (Amendment #8)

With the accrual duration extended to 10/31/2019, the power of the analysis of OS for the HR/IR cohort will be approximately 0.67 if conducted at 1 year after completion of accrual, and will be approximately 0.72 if conducted at 2 years after completion of accrual.

# Confirmatory follow-up analysis of OS of the HR/IR randomized cohort (Amendment #10)

A confirmatory follow-up analysis comparing OS of the control arm vs. the experimental arm will be conducted at the time of the confirmatory analysis of DFS, as well as one year following it. Same as for DFS, this



analysis will also be utilizing the HR/IR patients randomized on or prior to 06/30/2019 (103 in the control arm and 105 in the experimental arm).

#### 9.3.1.3 Secondary endpoint: MRD+ rates

MRD comparisons (using an MRD+ threshold of 0.01%) will be performed at the end of Blocks 2 and 3 for marrow relapse patients participating in HR/IR Randomization. From past experience with studies AALL01P2, ADVL04P2, AALL07P1 and AALL0433, we anticipate that over the 3 years of the study, there will be 56 patients per arm evaluable for the MRD comparison at the end of Block 2 and 50 patients per arm evaluable for the MRD comparison at the end of Block 3 (see table below for derivation).

| | Early<br>marrow | Late marrow with MRD≥ 0.1% | Total |
|---|---|---|---|
| # randomized on HR/IR<br>Randomization (per arm) | 61 | 24 | 85 |
| Rate of not dropping out prior to end Block 2 | 63% | 75% | |
| # evaluable for end Block 2<br>MRD testing | 38 | 18 | 56 |
| Rate of not dropping out prior to end Block 3 | 89% | 88% | |
| # evaluable for end Block 3<br>MRD testing | 34 | 16 | 50 |

Further, we anticipate that the rates of MRD  $\geq$  0.01% in the control arm will be 67% (67% for early and 68% for late) at the end of Block 2 and 47% (43% for early and 55% for late) at the end of Block 3. A two-sample Fisher's exact test of proportions (one-sided, alpha = 5%) will be used to test the hypothesis that the proportion of patients who are MRD+ on each experimental arm (with blinatumomab) is smaller than the control arm (without blinatumomab) at the end of Block 2 and 3. The corresponding power to detect various degrees of reduction in MRD+ rates is shown in the table below:

| | Expected # per arm with | % MRD+<br>(control | | | MRD+ rational arm | |
|---|---|---|---|---|---|---|
| | successful MRD determination | arm) | 10% | 15% | 20% | 25% |
| End Block 2 | 56 | 67% | 22.6% | 41.8% | 63.2% | 81.2% |
| End Block 3 | 50 | 47% | 19.2% | 37.1% | 59.5% | 79.8% |

With the accrual duration extended to 10/31/2019, the analysis on MRD+ rates should have more statistical power.



# 9.3.1.4 Safety monitoring (Activation Protocol)

According to the past study ALLR3, the cumulative toxic death rate of Blocks 2 and 3 of chemotherapy was estimated to be 4% (1.6% for Block 2 and 2.7% for Block 3). The toxic death rate is expected to be lower in the experimental arm than the control arm because the myelosuppressive cytotoxic chemotherapy blocks are replaced with targeted immunotherapy. Therefore, toxic deaths will be closely monitored on all patients enrolled to each arm of HR/IR Randomization separately through blocks 2 and 3 of therapy. HR/IR Randomization will be temporarily closed for detailed review and possible therapy modifications if the number of toxic deaths in either arm is greater than or equal to that specified in the table. The boundary of toxic death was computed based on Pocock-type spending function at one-sided 20% significant level.

| Looks | # evaluable<br>patients | Information | Pocock boundary of excessive toxic death | Excessive toxic death rate |
|---|---|---|---|---|
| 1 | 28 | 33% | 4 | 14.29% |
| 2 | 57 | 67% | 5 | 8.77% |
| 3 | 85 | 100% | 7 | 8.24% |

Either arm of HR/IR Randomization will be rejected for excessive toxicity if the number of observed toxic deaths is greater than or equal to the corresponding boundary at any interim analysis. The actual power (based on exact binomial test) of declaring an arm too toxic are approximately 95.2%, 80.8%, 47.2% and 10.1% when the true toxic death rate is 13%, 10%, 7% and 4%, respectively.

In addition, occurred during Block 2 and 3 of chemotherapy the toxic deaths and all toxicities of all grades between the two arms will be monitored/compared during the study. If the toxic death rate or the rate for any specific toxicity is significantly higher on the blinatumomab arm compared to the control arm (ALLR3 backbone), the data will be reviewed for possible suspension of the randomization and modification of therapy.

## 9.3.1.5 <u>Amended Safety Monitoring (Amendment 6)</u>

As of April 2017, there have been 4 deaths during blocks 2 and 3, among 47 randomized patients on Arm A. Of these, three deaths occurred in 14 AYA patients (ages 17, 23, and 26 years), with a death rate of 21.4%. The death rate among the younger patients is 1/33 (3%). The published UKALLR3 clinical trial only enrolled patients up to 18 years of age at the time of first relapse. Hence the toxic death rate from that study (used as the baseline rate on this study), was based on a younger population than those enrolling on AALL1331. About 15% of enrollments on this study are currently greater than 18 years old. Based on prior studies in COG and other groups, it is known that the risk of toxic deaths may be higher in older patients relative to younger ones.



Based on this, the monitoring for toxic deaths during Blocks 2 and 3, among HR/IR patients randomized to Arm A, has been modified to apply only to patients  $\leq 18$  years of age at enrollment. The modified rule is given in the table below.

| Monitoring (HR/IR | #Evaluable patients | Pocock Boundary<br>of Excessive Toxic<br>deaths |
|---|---|---|
| patients ≤18 years | 4-40 | 4 |
| of age on Arm A) | 41-57 | 5 |
| | 58-72 | 6 |

With this rule, the probability of stopping due to excessive toxic deaths is 12% if the true toxic death rate is 4%, 48% if the true rate is 7%, and 79.2% if the true rate is 10%.

Since it is estimated that only about 13 patients on each arm will be >18 years of age at enrollment, separate stopping rules for this subset would not have much power (~74% at a true rate of 30%, or 13% power at a true rate of 10%). Instead of a formal monitoring rule for AYA patients, continuous monitoring will be done, such that any death occurring among the older patients, after the proposed supportive care changes are initiated, will trigger a study committee review and communication to the COG Data Safety Monitoring Committee.

With Amendment #8, more patients will be enrolled in the HR/IR cohort. The above safety monitoring rule on toxic deaths will be implemented until the originally planned sample size of 170 evaluable patients are enrolled and completed protocol treatment. If the toxic death rates are not concerning with the 170 patients, then no formal statistical monitoring rule on toxic deaths will be implemented for the remaining patients who will be enrolled in this cohort. However, informal continuous monitoring of occurrences of toxic deaths will continue to be conducted.

# 9.3.2 LR Randomization for LR relapse patients

## 9.3.2.1 Primary endpoint: intent-to-treat DFS from randomization

# The original design (Activation Protocol)

The primary efficacy analysis for LR Randomization will be an intent-to-treat comparison of the DFS curves between the randomized arms based on the Log-rank test. All late B-ALL marrow and IEM relapse patients with end Block 1 MRD < 0.1% who are not deemed to be treatment failures at the end of Block 1 or Block 2 will be eligible for LR Randomization. For IEM patients, uninterpretable MRD (due to lack of diagnostic marker) will be considered to be MRD negative. The randomization will occur upon recovery from Block 2 of therapy, and will be stratified as described in Section 9.2. Data from past studies suggest that most events are to occur within 3 years, but events continue to occur in subsequent years, and hence an exponential distribution is considered



more appropriate than a cure-rate model for comparing survival curves for this cohort of patients at the time of final analysis. An estimate of 206 evaluable patients will be randomized 1:1 (103 evaluable patients per arm) between randomized experimental (blinatumomab) and control (chemotherapy) arms. Assuming a minimum of 3-years of follow up, this sample size estimate is based on a goal of achieving a 11% improvement in 3-year DFS rate with blinatumomab over the expected 3-year DFS rate of 73% with chemotherapy backbone alone, with 80.4% power at a one-sided significance level of 5%, which represents a 44.6% reduction in the hazard rate. The power calculations are based on the assumption of proportional hazards and using the log rank test.

Interim analysis will be conducted to monitor for efficacy and futility. The efficacy stopping boundaries to be used will be based on the O' Brien-Fleming spending function. The futility boundaries are based on testing the alternative hypothesis at the 0.039 level. This monitoring rule can be applied to any interim analysis schedule and maintains the overall significance level of 0.05. Assuming exponential distribution and the final analysis is performed at the 3 years after the completion of enrollment, the expected maximum number of events to be observed is estimated to be 75. The first interim analysis will be performed after 25 events have been observed. The cumulative power to detect a difference is approximately 80%. The sample of monitoring boundaries for efficacy and futility with 3 interim analyses are given in the table below.

| Looks | # of events | Information | Efficacy Boundary | Futility<br>Boundary |
|-------|-------------|-------------|-------------------|----------------------|
| 1 | 25 | 33% | 3.202 | -0.312 |
| 2 | 50 | 67% | 2.140 | 0.288 |
| 3 | 75 | 100% | 1.695 | 1.695 |

#### Re-design for the LR cohort (Amendment #8)

#### **Summary of the original design**

For the LR cohort, the study was originally designed to have approximately power of 0.80 to detect a hazard ratio of 0.55 using a one-sided logrank test with Type I error of 0.05. The hazard ratio of 0.55 corresponds to an increase in 3-year DFS rate from 73% in the control arm to 84% in the experimental arm, assuming exponential distribution in survival function. This cohort was originally planned to enroll a total of 206 randomized, evaluable patients. It was expected to accrue for 5.6 years, with 3 years of additional follow-up after completion of enrollment.

# Extended accrual duration and increased sample size

With the extended accrual duration, the LR cohort will continue to enroll until 10/31/2019. Based on the observed accrual rate of 53 patients/year, this extended accrual duration will lead to a sample size of approximately



236 randomized patients in the LR cohort. As initially planned, the primary analysis on efficacy will be based on a one-sided logrank test, with one-sided Type I error of 0.05. The primary analysis will be conducted 3 years after completion of enrollment or when the expected total number of events is observed, whichever comes first. Assuming exponential distribution for the survival function, with 4.4 years of enrollment and 3 years of additional follow-up, the expected total number of events is 80. With the sample size of 236, the study will have approximately power of 0.83 to detect a HR of 0.55.

#### Amended statistical monitoring plan for DFS

With the extended accrual duration, the full information increases from the original 75 events to 80 events. The new interim monitoring plan, developed by an independent statistician, accounts for the alpha-spending that has already occurred. Specifically, with the new monitoring plan, the overall alpha to be expended is the original significance level (0.05) minus the alpha expended with the first interim monitoring that has been conducted (0.00068). That is, the remaining alpha of 0.04932 can be used for the new monitoring plan. A monitoring plan that includes two more looks (the second look and the final look) was developed using the O'Brien-Fleming monitoring boundaries, with an overall significance level of 0.04932, scheduled at 66.25% and 100% of the total expected information. This way the cohort-wide significance level of 0.05 is maintained. The futility boundaries are based on testing the alternative hypothesis at the 0.039 level. The boundaries are shown in the following table.

| | | | New Efficacy Boundaries | | | | |
|---|---|---|---|---|---|---|---|
| Looks | # of<br>Events | Inf. Time<br>Revised | Roundary | | | | |
| 2 | 53 | 66.25% | 2.151 | 0.01573 | 0.01573 | 0.01641 | 0.361 |
| 3 | 80 | 100% | 1.702 | 0.04462 | 0.04932 | 0.05 | 1.702 |

### 9.3.2.2 Secondary Endpoint: Intent-to-treat OS

From past studies suggest that most events for LR patients are to occur within 4 years after randomization and the 4-year OS rate is estimated to be 77%. Therefore, a cure-rate model with exponential distribution assumed during the first 4 years followed by a flat curve is considered for OS analysis for LR randomized patients. An interim OS analysis will be conducted at the time of the final DFS analysis, i.e. when all the 206 randomized patients are followed up for 3 years. Assuming 10% improvement in 4-year OS rate with blinatumomab over the expected 4-year OS rate of 77% with chemotherapy backbone alone, approximate 36 deaths are to be observed by the time of the interim OS analysis. The



power to detect such improvement at a one-sided significance level of 5% is approximate 60% based on the log-rank test.

If DFS analysis meets its target level of improvement (i.e. one-sided p-value < 0.05), the formal OS analysis will be performed at 1 year after the interim OS analysis, by which time approximate 37 deaths are to be observed. The power to detect the above desired improvement is approximately 61%.

# Power of the analysis of OS with the extended accrual duration (Amendment #8)

With the accrual duration extended to 10/31/2019, the power of the analysis of OS for the LR cohrt will be approximately 0.63 if conducted at 3 years after completion of accrual, and will be approximately 0.64 if conducted at 4 years after completion of accrual.

# 9.3.2.3 Monitoring for severe toxicities and toxic deaths

According to the past study of ALLR3, the cumulative toxic death rate of Block 3, Continuation and Maintenance chemotherapy was estimated to be 4% (2.7% for Block 3 and 1.5% for Continuation and Maintenance). The toxic death rate is expected to be lower in the experimental arm than the control arm because the myelosuppressive Block 3 is replaced with targeted immunotherapy. Therefore, toxic deaths will be closely monitored on all patients enrolled on to each arm of LR Randomization separately from the start of Block 3 of therapy to the completion of protocol therapy. LR Randomization will be temporarily closed for detailed review and possible therapy modifications if the number of toxic deaths in either arm is greater than or equal to that specified in the table below. The boundary of toxic death was computed based on Pocock-type spending function at one-sided 20% significant level.

| Looks | # evaluable patients | Information | Pocock boundary of excessive toxic death | Excessive toxic death rate |
|---|---|---|---|---|
| 1 | 34 | 33% | 4 | 11.76% |
| 2 | 69 | 67% | 6 | 8.70% |
| 3 | 103 | 100% | 7 | 6.80% |

Either arm of LR <u>Randomization</u> will be rejected for excessive toxicity if the number of observed toxic deaths is greater than or equal to the corresponding boundary at any interim analysis. The actual power (based on exact binomial test) of declaring an arm too toxic are approximately 98.7%, 90.9%, 61.5% and 14.4% when the true toxic death rate is 13%, 10%, 7% and 4%, respectively.

In addition, during Block 3, Continuation 2 (Week 1 - 5) and Maintenance (Week 6 - 10) the toxic deaths and all toxicities of all grades between the two arms will also be monitored/compared. If the toxic death rate or the rate for any specific toxicity is significantly higher on the blinatumomab



arm compared to the control arm, the data will be reviewed for possible suspension of the randomization and modification of therapy.

The potential for late adverse effects due to long term depletion of CD19<sup>+</sup> normal lymphocytes following blinatumomab treatment is unknown. We will monitor for lymphocyte recovery and late events related to delayed recovery. Since HR/IR/TF patients go to HSCT soon after blinatumomab, it would be difficult to make sense of lymphocyte recovery/late events after blinatumomab for them. However, the LR patients that are randomized to +/- blinatumomab and do not proceed to HSCT serve as an excellent population to monitor for these delayed adverse effects. For all patients, we will collect absolute lymphocyte (ALC)/lymphocyte subset counts (total T and B cells) and data regarding late infections and progressive multifocal leukoencephalopathy (PML) after each 12-week maintenance cycle and every 3 months after completion of therapy for 1 year. The peripheral B-cell recovery rates and rates of late events by randomized arms will be monitored and compared descriptively between the two randomized arms every 6 months in the biannual study progress report and DSMC report.

With Amendment #8, more patients will be enrolled in the LR cohort. The above safety monitoring rules on severe toxicities and toxic deaths will be implemented until the originally planned sample size of 206 evaluable patients are enrolled and completed protocol treatment. If the toxic death rates are not concerning with the 206 patients, then no formal statistical monitoring rule on severe toxicities and toxic deaths will be implemented for the remaining patients who will be enrolled in this cohort. However, informal continuous monitoring of occurrences of toxic deaths will continue to be conducted.

# 9.3.3 Pilot intervention for very high risk subset of HSCT recipients based on MRD and aGVHD

## 9.3.3.1 Primary endpoint

The primary endpoint of this non-randomized exploratory pilot intervention (accelerated taper of immune suppression) is feasibility and safety, with "success" defined as < 25% rate of Grade III-IV aGVHD and < 5% rate of treatment-related mortality (TRM) associated with the accelerated taper. We anticipate that 36 patients will meet the criteria to receive the intervention. We will calculate the observed rates of Grade III – IV aGVHD and TRM among this subset with 95% confidence intervals and compare descriptively to our target rates.

# 9.3.3.2 Exploratory endpoint

As secondary endpoints, we will calculate the percent of patients able to wean off immunosuppression without significant aGVHD (future intervention group), DFS of intervention group (vs. similar pts in ASCT0431 historical controls), rate of conversion from MRD+ to MRD-among preMRD-/postMRD+ subset (correlated with DFS), aGVHD rates



post-intervention (correlated with DFS). These data will be analyzed descriptively.

## 9.3.3.3 Safety monitoring

The toxic death and Grade 3+ GVHD rates will be closely monitored for the subset of HSCT patients with MRD  $\geq$  0.01% pre- and/or post-HSCT with no acute graft versus host disease (aGVHD) who undergo accelerated taper of immune suppression during the study. According to past studies, the cumulative toxic death rate was estimated to be 5% and the cumulative incidence rate of Grade 3+ GVDH was approximately 25%.

The safety stopping boundaries to be used for toxic death and Grade 3+ GVHD, respectively, will be based on the Pocock-type spending function at one-sided 20% significance level. Assuming 85% of evaluable HR/IR patients will proceed to HSCT study and approximately 25% of them will have MRD  $\geq$  0.01% pre- and/or post-HSCT with no evidence of aGVHD, an estimate of 36 patients will be monitored in this subset. The intervention (accelerated taper of immune suppression) will be temporarily closed for detailed review and possible therapy modifications if the number of toxic deaths or the number of Grade 3+ GVHD is greater than or equal to that specified in the corresponding table below.

Table for toxic death monitoring boundary:

| Looks | # evaluable<br>patients | Information | Pocock boundary of excessive toxic deaths | Excessive toxic death rate |
|---|---|---|---|---|
| 1 | 12 | 33% | 3 | 25.00% |
| 2 | 24 | 67% | 4 | 16.67% |
| 3 | 36 | 100% | 4 | 11.110% |

The intervention will be rejected for excessive toxicity death if the number of observed toxic deaths is greater than or equal to the corresponding boundary at any interim analysis. The actual power (based on exact binomial test) of declaring the intervention too toxic are approximately 88.5%, 71.1%, 41.6% and 10.9% when the true toxic death rate is 17%, 13%, 9% and 5%, respectively.

<u>Table for Grade 3+ GVHD monitoring boundary:</u>

| Looks | # evaluable<br>patients | Information | Pocock boundary of excessive toxicity | Excessive toxicity rate |
|---|---|---|---|---|
| 1 | 12 | 33% | 6 | 50.00% |
| 2 | 24 | 67% | 10 | 41.67% |
| 3 | 36 | 100% | 13 | 36.11% |

The intervention will be rejected for excessive Grade 3+ GVHD if the number of observed Grade 3+ GVHD is greater than or equal to the corresponding boundary at any interim analysis. The actual power (based on exact binomial test) of declaring the intervention too toxic are approximately 96.4%, 80.5%, 45.9% and 13.2% when the true rate of Grade 3+ GVHD is 49%, 41%, 33% and 25%, respectively.



See <u>Appendix XII</u> for guidelines for establishing organ stage and overall grade of acute GVHD.

With Amendment #8, the above monitoring of toxic deaths and Grade 3+ GVHD in the subset of HSCT patients with MRD  $\geq$  0.01% pre- and/or post-HSCT with no aGVHD who undergo accelerated taper of immune suppression during the study will continue to be conducted until the HR/IR cohort meet the original planned accrual target of 170 evaluable patients. After that, no formal monitoring of toxic deaths or Grade 3+ GVHD will be conducted in this subset of patients. However, informal continuous monitoring of occurrences of toxic deaths will continue to be conducted.

9.3.4 <u>Treatment Failure (TF) patients who are non-randomly assigned to blinatumomab</u> Point estimate and the corresponding exact 95% confidence interval based on Clopper-Pearson's method will be provided to estimate the hematologic CR, the rate of MRD < 0.01%, and the proportion treatment failure patients able to proceed to hematopoietic stem cell transplant (HSCT).

The toxic death will be closely monitored for TF patients who are non-randomly assigned to blinatumomab. According to past studies, an approximate 60 (10%) of enrolled patients will be deemed as TF, and the cumulative toxic death rate is estimated to be 6%. The safety stopping boundaries to be used for toxic death will be based on the Pocock-type spending function at one-sided 20% significance level. The intervention for TF patients will be temporarily closed for detailed review and possible therapy modifications if the number of toxic deaths is greater than or equal to that specified in the corresponding table below.

Table for toxic death monitoring boundary:

| Looks | # evaluable patients | Information | Pocock boundary of excessive toxicities | Excessive toxic death rate |
|---|---|---|---|---|
| 1 | 12 | 20% | 3 | 25.00% |
| 2 | 24 | 40% | 4 | 16.67% |
| 3 | 36 | 60% | 5 | 13.89% |
| 4 | 48 | 80% | 6 | 12.50% |
| 5 | 60 | 100% | 7 | 11.67% |

The intervention will be rejected for excessive toxicity death if the number of observed toxic deaths is greater than or equal to the corresponding boundary at any interim analysis. The actual power (based on exact binomial test) of declaring the intervention too toxic are approximately 85.9%, 67.1%, 39.1% and 12.9% when the true toxic death rate is 15%, 12%, 9% and 6%, respectively.

With Amendment #8, after monitoring toxic death rates in 60 evaluable TF patients, no further formal monitoring of toxic deaths among TF patients will be conducted. However, informal continuous monitoring of occurrences of toxic deaths will continue to be conducted.



## 9.3.5 <u>Blinatumomab related reportable adverse event (RAE)</u>

A reportable adverse event (RAE) with respect to blinatumomab is defined in Section 5.2. The reporting period case report form (CRF) for each blinatumomab course will specifically collect data regarding blinatumomab RAEs. Due to limited experience with blinatumomab, very little information is available estimate the expected incidence of blinatumomab RAEs. We will prospectively monitor the blinatumomab RAE rate on monthly study committee calls, and will report the blinatumomab RAE rate every 6 months in the biannual study progress report and DSMC report. RAE rates  $\geq 10\%$  will be of particular concern and will prompt discussion with the DSMC.

# 9.3.6 <u>Monitoring for infection rate of 96-hour bag changes in Blinatumomab</u> administration (Amendment #2)

The rate of Grade 3 or higher relevant infections (defined as sepsis, bacteremia, device or catheter-related infection) will be monitored among patients who received blinatumomab with the infusion bag changed up to 96 hours. We will consider 96 hour bag change acceptable if the infection rate is 5% or less. All Grade 3 or higher relevant infections will be evaluated every six months and the infection rate will be tested to determine whether the true rate is greater than 5% using exact one-sided one-sample binomial test, and the results will be presented to DSMC. If at one of scheduled analyses, the one-sided p-value of the test is less than 0.05, the 96 hour bag change would be considered unacceptable and the DSMC will be consulted regarding whether the bag change frequency should be changed back to 48 hours. The two-sided 90% confidence interval for the infection rate will also be provided.

# 9.3.7 <u>Monitoring for infection rate of 7-day bag changes in Blinatumomab</u> administration (Amendment #8)

Amendment #8 incorporates the allowance of a 7-day (168 hours) bag change schedule for Blinatumomab. This infusion schedule is added as an additional option to the existent 24-hour, 48-hour, and 96-hour infusion schedules.

To ensure safety of using the 7-day bag change schedule, after the activation of this amended protocol, the rate of grade 3 or higher relevant infections (defined as sepsis, bacteremia, device or catheter-related infection) will be monitored among patients weighing  $\geq 22$  Kg who are enrolled after activation of the amended protocol and randomized to receive blinatumomab.

We will conduct monthly monitoring of rate of relevant infections of grade 3+ using a Bayesian safety monitoring approach. Based on the observed accrual rate, we expect that every month we will have approximately 4 to 5 patients randomized to the blinatumomab arms (LR and HR/IR cohorts combined), and that the majority of them will be using 7-day bag change schedule. For this monitoring we will assume that from the date of the activation of this amended protocol, every patient weighing  $\geq$  22 Kg who are enrolled and randomized to receive blinatumomab will be using 7-day bag change schedule. We expect that the rate of grade 3+ infections related to the use of 7-day bag change schedule is 5% or less.



We assume that the number of patients experiencing relevant grade 3+ infections among those who use 7-day bag change schedule follows a binomial distribution, and that the probability for a patient to have relevant infections has a prior distribution of Beta(0.05,0.95). The first interim monitoring of infections for 7-day bag change will be undertaken after an initial 6 patients have received at least 1 cycle of blinatumomab using 7-day bag change schedule and have AE data reported in Medidata RAVE, which is expected to occur 3 to 4 months after the activation of the amended protocol. After that, we will conduct monthly interim monitoring of the infection rate.

At each interim monitoring, the posterior distribution of the probability for a patient to experience relevant grade 3+ infection ( $p_{infection}$ ) will be calculated. If it is >95% likely that  $p_{infection} > 5\%$ , the study committee will conduct toxicity review related to 7-day bag change, consider the necessity of changing the bag change frequency back to 96 hours, and report the analysis results to DSMC. A simulation study showed that the probability for the rule to be triggered is approximately 0.97, 0.84, 0.50 and 0.10 when the true rate of relevant grade 3+ infection is 20%, 15%, 10% and 5%, respectively.

# 9.4 Gender and Minority Accrual Estimates

The gender and minority distribution of the study population is expected to be (Activation Protocol):

| Accrual Targets | | | |
|--------------------------------------------|------------|-------|-------|
| Ethnic Category | Sex/Gender | | |
| Dennie Category | Females | Males | Total |
| Hispanic or Latino | 85 | 79 | 164 |
| Not Hispanic or Latino | 225 | 209 | 434 |
| Ethnic Category: Total of All Participants | 310 | 288 | 598 |
| Racial Category | | | |
| American Indian/Alaska Native | 5 | 3 | 8 |
| Asian | 12 | 14 | 26 |
| Black or African American | 35 | 22 | 57 |
| Native Hawaiian or Other Pacific Island | 2 | 1 | 3 |
| White | 256 | 248 | 504 |
| Racial Categories: Total of All Subjects | 310 | 288 | 598 |

<sup>\*</sup> These totals must agree

This distribution was derived from past studies on AALL01P2, AALL02P2, ADVL04P2 and AALL0433.

The gender and minority distribution of the study population is expected to be (Amendment #8):

| Accrual Targets | |
|-----------------|------------|
| | Sex/Gender |



| Ethnic Category | Females | Males | Total |
|--------------------------------------------|---------|-------|-------|
| Hispanic or Latino | 99 | 93 | 192 |
| Not Hispanic or Latino | 263 | 245 | 508 |
| Ethnic Category: Total of All Participants | 363 | 337 | 700 |
| Racial Category | • | | |
| American Indian/Alaska Native | 5 | 4 | 9 |
| Asian | 14 | 16 | 30 |
| Black or African American | 41 | 26 | 67 |
| Native Hawaiian or Other Pacific Island | 3 | 1 | 4 |
| White | 300 | 290 | 590 |
| Racial Categories: Total of All Subjects | 363 | 337 | 700 |

This distribution was derived from past studies on AALL01P2, AALL02P2, ADVL04P2 and AALL0433.

#### 10.0 EVALUATION CRITERIA

# 10.1 Common Terminology Criteria for Adverse Events (CTCAE)

This study will utilize version 4.0 of the CTCAE of the National Cancer Institute (NCI) for toxicity and performance reporting. A copy of the CTCAE version 4.0 can be downloaded from the CTEP website

(<a href="http://ctep.cancer.gov/protocolDevelopment/electronic\_applications/ctc.htm">http://ctep.cancer.gov/protocolDevelopment/electronic\_applications/ctc.htm</a>). Additionally, toxicities are to be reported on the appropriate case report forms.

<u>Please note:</u> 'CTCAE v4.0' is understood to represent the most current version of CTCAE v4.0 as referenced on the CTEP website (i.e., v4.02 and all subsequent iterations prior to version 5.0).

# 10.2 Response Criteria

See definitions in <u>Section 3.3</u>.



## 11.0 ADVERSE EVENT REPORTING REQUIREMENTS

# 11.1 Purpose

Adverse event (AE) data collection and reporting, which are required as part of every clinical trial, are done to ensure the safety of patients enrolled in the studies as well as those who will enroll in future studies using similar agents. Certain adverse events must be reported in an expedited manner to allow for timelier monitoring of patient safety and care. The following sections provide information about expedited reporting.

## 11.2 **Determination of reporting requirements**

Reporting requirements may include the following considerations: 1) whether the patient has received an investigational or commercial agent; 2) the characteristics of the adverse event including the *grade* (severity), the *relationship to the study therapy* (attribution), and the *prior experience* (expectedness) of the adverse event; 3) the Phase (1, 2, or 3) of the trial; and 4) whether or not hospitalization or prolongation of hospitalization was associated with the event.

An <u>investigational agent</u> is a protocol drug administered under an Investigational New Drug Application (IND). In some instances, the investigational agent may be available commercially, but is actually being tested for indications not included in the approved package label.

<u>Commercial agents</u> are those agents not provided under an IND but obtained instead from a commercial source. The NCI, rather than a commercial distributor, may on some occasions distribute commercial agents for a trial.

When a study includes both investigational and commercial agents, the following rules apply

- Concurrent administration: When an investigational agent is used in combination with a commercial agent, the combination is considered to be investigational and expedited reporting of adverse events would follow the guidelines for investigational agents.
- Sequential administration: When a study includes an investigational agent and a commercial agent on the same study arm, but the commercial agent is given for a period of time prior to starting the investigational agent, expedited reporting of adverse events that occur prior to starting the investigational agent would follow the guidelines for commercial agents. Once therapy with the investigational agent is initiated, all expedited reporting of adverse events follow the investigational agent reporting guidelines.

# 11.3 Expedited Reporting Requirements – Serious Adverse Events (SAEs)

To ensure compliance with these regulations/this guidance, as IND/IDE sponsor, NCI requires that AEs be submitted according to the timeframes in the AE reporting tables assigned to the protocol, using the CTEP Adverse Event Reporting System (CTEP-AERS).

Any AE that is serious qualifies for expedited reporting. An AE is defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not



considered drug related. A Serious Adverse Event (SAE) is any adverse drug event (experience) occurring at any dose that results in ANY of the following outcomes:

- 1) Death
- 2) A life-threatening adverse drug experience.
- 3) An adverse event resulting in inpatient hospitalization or prolongation of existing hospitalization (for  $\geq$  24 hours). This does not include hospitalizations that are part of routine medical practice.
- 4) A persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions.
- 5) A congenital anomaly/birth defect.
- 6) Important Medical Events (IME) that may not result in death, be life threatening, or require hospitalization may be considered a serious adverse drug experience when, based upon medical judgment, they may jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the outcomes listed in this definition.

## 11.4 Special Situations for Expedited Reporting

# 11.4.1 SAEs Occurring More than 30 Days After Last Dose of Study Drug

Any Serious Adverse Event that occurs more than 30 days after the last administration of the investigational agent/intervention <u>and</u> has an attribution of a possible, probable, or definite relationship to the study therapy must be reported according to the CTEP-AERS reporting tables in this protocol.

#### 11.4.2 Persistent or Significant Disabilities/Incapacities

Any AE that results in persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions (formerly referred to as disabilities), congenital anomalies or birth defects, must be reported via CTEP-AERS if it occurs at any time following treatment with an agent under a NCI IND/IDE since these are considered to be serious AEs.

## 11.4.3 <u>Death</u>

Reportable Categories of Death

- Death attributable to a CTCAE term.
- Death Neonatal: Newborn death occurring during the first 28 days after birth.
- Sudden Death NOS: A sudden (defined as instant or within one hour of the onset of symptoms) or an unobserved cessation of life that cannot be attributed to a CTCAE term associated with Grade 5.
- Death NOS: A cessation of life that cannot be attributed to a CTCAE term associated with Grade 5.
- Death due to progressive disease should be reported as *Grade 5 "Disease progression: in the system organ class (SOC) "General disorders and administration site conditions."* Evidence that the death was a manifestation of underlying disease (*e.g.*, radiological changes suggesting tumor growth or progression: clinical deterioration associated with a disease process) should be submitted.



Any death occurring *within 30 days* of the last dose, regardless of attribution to the investigational agent/intervention requires expedited reporting within 24 hours.

Any death occurring *greater than 30 days* after the last dose of the investigational agent/intervention requires expedited reporting within 24 hours **only if** it is possibly, probably, or definitely related to the investigational agent/intervention.

# 11.4.4 Secondary Malignancy

A **secondary malignancy** is a cancer caused by treatment for a previous malignancy (e.g., treatment with investigational agent/intervention, radiation or chemotherapy). A metastasis of the initial neoplasm is not considered a secondary malignancy.

The NCI requires all secondary malignancies that occur following treatment with an agent under an NCI IND/IDE be reported via CTEP-AERS. Three options are available to describe the event:

- Leukemia secondary to oncology chemotherapy
- Myelodysplastic syndrome
- Treatment related secondary malignancy

Any malignancy possibly related to cancer treatment (including AML/MDS) must also be reported via the routine reporting mechanisms outlined in this protocol.

## 11.4.5 Second Malignancy

A second malignancy is one unrelated to the treatment of a prior malignancy (and is **NOT** a metastasis from the initial malignancy). Second malignancies require **ONLY** routine reporting via CDUS unless otherwise specified.

# 11.4.6 Pregnancy, Pregnancy Loss, and Death Neonatal

NOTE: When submitting CTEP-AERS reports for "Pregnancy", "Pregnancy loss", or "Neonatal loss", the Pregnancy Information Form, available at <a href="http://ctep.cancer.gov/protocolDevelopment/electronic\_applications/docs/PregnancyReportForm.pdf">http://ctep.cancer.gov/protocolDevelopment/electronic\_applications/docs/PregnancyReportForm.pdf</a>, needs to be completed and faxed along with any additional medical information to (301) 897-7404. The potential risk of exposure of the fetus to the investigational agent(s) or chemotherapy agent(s) should be documented in the "Description of Event" section of the CTEP-AERS report.

#### 11.4.6.1 Pregnancy

Patients who become pregnant on study risk intrauterine exposure of the fetus to agents that may be teratogenic. For this reason, pregnancy needs to be reported in an expedited manner via CTEP-AERS as **Grade 3** "Pregnancy, puerperium and perinatal conditions - Other (pregnancy)" under the Pregnancy, puerperium and perinatal conditions SOC.

There is a possibility that the sperm of male patients treated on studies involving possible teratogenic agents may have been damaged. For this



reason, pregnancy in partners of men on study needs be reported and followed in the same manner as a patient pregnancy.

Pregnancy needs to be followed **until the outcome is known**. If the baby is born with a birth defect or anomaly, then a second CTEP-AERS report is required.

### 11.4.6.2 **Pregnancy Loss (Fetal Death)**

Pregnancy loss is defined in CTCAE as "Death in utero." Any Pregnancy loss should be reported expeditiously, as **Grade 4** "Pregnancy loss" under the "Pregnancy, puerperium and perinatal conditions" **SOC.** Do NOT report a pregnancy loss as a Grade 5 event since CTEP-AERS recognizes any Grade 5 event as a patient death.

#### 11.4.6.3 **Death Neonatal**

Neonatal death, defined in CTCAE as "Newborn death occurring during the first 28 days after birth", should be reported expeditiously as Grade 4 "Death neonatal" under the "General disorders and administration" SOC, when the death is the result of a patient pregnancy or pregnancy in partners of men on study. Do NOT report a neonatal death resulting from a patient pregnancy or pregnancy in partners of men on study as a Grade 5 event since CTEP-AERS recognizes any Grade 5 event as a patient death.

# 11.5 Reporting Requirements for Specialized AEs

#### 11.5.1 Baseline AEs

Although a pertinent positive finding identified on baseline assessment is not an AE, when possible it is to be documented as "Course Zero" using CTCAE terminology and grade. An expedited AE report is not required if a patient is entered on a protocol with a pre-existing condition (e.g., elevated laboratory value, diarrhea). The baseline AE must be re-assessed throughout the study and reported if it fulfills expedited AE reporting guidelines.

- a. If the pre-existing condition worsens in severity, the investigator must reassess the event to determine if an expedited report is required.
- b. If the AE resolves and then recurs, the investigator must re-assess the event to determine if an expedited report is required.
- c. No modification in grading is to be made to account for abnormalities existing at baseline.

## 11.5.2 Persistent AEs

A persistent AE is one that extends continuously, without resolution between treatment cycles/courses.

ROUTINE reporting: The AE must be reported only once unless the grade becomes more severe in a subsequent course. If the grade becomes more severe the AE must be reported again with the new grade.



EXPEDITED reporting: The AE must be reported only once unless the grade becomes more severe in the same or a subsequent course.

### 11.5.3 Recurrent AEs

A recurrent AE is one that occurs and resolves during a cycle/course of therapy and then reoccurs in a later cycle/course.

ROUTINE reporting: An AE that resolves and then recurs during a subsequent cycle/course must be reported by the routine procedures.

EXPEDITED reporting: An AE that resolves and then recurs during a subsequent cycle/course does not require CTEP-AERS reporting unless:

- 1) The grade increases OR
- 2) Hospitalization is associated with the recurring AE.

## 11.6 Exceptions to Expedited Reporting

## 11.6.1 Specific Protocol Exceptions to Expedited Reporting (SPEER)

SPEER: Is a subset of AEs within the Comprehensive Adverse Events and Potential Risks (CAEPR) that contains a list of events that are considered expected for CTEP-AERS reporting purposes. (Formerly referred to as the Agent Specific Adverse Event List (ASAEL).)

AEs listed on the SPEER should be reported expeditiously by investigators to the NCI via CTEP-AERS <u>ONLY</u> if they exceed the grade of the event listed in parentheses after the event. If the CAEPR is part of a combination IND using multiple investigational agents and has an SAE listed on different SPEERs, use the lower of the grades to determine if expedited reporting is required.

### 11.6.2 Special Situations as Exceptions to Expedited Reporting

An expedited report may not be required for a specific protocol where an AE is listed as expected. The exception or acceptable reporting procedures will be specified in the protocol. The protocol specific guidelines supersede the NCI Adverse Event Reporting Guidelines. These special situations are listed under the CTEP-AERS reporting <u>Table A</u> for this protocol.

## 11.7 Reporting Requirements - Investigator Responsibility

Clinical investigators in the treating institutions and ultimately the Study Chair have the primary responsibility for AE identification, documentation, grading, and assignment of attribution to the investigational agent/intervention. It is the responsibility of the treating physician to supply the medical documentation needed to support the expedited AE reports in a timely manner.

Note: All expedited AEs (reported via CTEP-AERS) must also be reported via routine reporting. Routine reporting is accomplished via the Adverse Event (AE) Case Report Form (CRF) within the study database.

## 11.8 General Instructions for Expedited Reporting via CTEP-AERS

The descriptions and grading scales found in the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 will be utilized for AE reporting. All appropriate



treatment areas should have access to a copy of the CTCAE version 5.0. A copy of the CTCAE version 5.0 can be downloaded from the CTEP web site <a href="http://ctep.cancer.gov/protocolDevelopment/electronic\_applications/ctc.htm">http://ctep.cancer.gov/protocolDevelopment/electronic\_applications/ctc.htm</a>.

An expedited AE report for all studies utilizing agents under an NCI IND/IDE must be submitted electronically to NCI via CTEP-AERS at: <a href="https://eapps-ctep.nci.nih.gov/ctepaers">https://eapps-ctep.nci.nih.gov/ctepaers</a>.

In the rare situation where Internet connectivity is disrupted, the 24-hour notification is to be made to the NCI for agents supplied under a CTEP IND by telephone call to (301) 897–7497.

In addition, once Internet connectivity is restored, a 24-hour notification that was phoned in must be entered into the electronic CTEP-AERS system by the original submitter of the report at the site.

- Expedited AE reporting timelines are defined as:
  - 24-Hour; 5 Calendar Days The AE must initially be reported via CTEP-AERS within 24 hours of learning of the event, followed by a complete expedited report within 5 calendar days of the initial 24-hour report.
  - o **7 Calendar Days** A complete expedited report on the AE must be submitted within 7 calendar days of the investigator learning of the event.
- Any event that results in a persistent or significant incapacity/substantial disruption of
  the ability to conduct normal life functions, or a congenital anomaly/birth defect, or is
  an IME, which based upon the medical judgment of the investigator may jeopardize
  the patient and require intervention to prevent a serious AE, must be reported via
  CTEP-AERS if the event occurs following investigational agent administration.
- Any death occurring within 30 days of the last dose, regardless of attribution to an agent/intervention under an NCI IND/IDE requires expedited reporting within 24 hours.
- Any death occurring greater than 30 days of the last dose with an attribution of possible, probable, or definite to an agent/intervention under an NCI IND/IDE requires expedited reporting within 24 hours.

CTEP-AERS Medical Reporting includes the following requirements as part of the report: 1) whether the patient has received at least one dose of an investigational agent on this study; 2) the characteristics of the adverse event including the *grade* (severity), the *relationship to the study therapy* (attribution), and the *prior experience* (expectedness) of the adverse event; 3) the Phase (1, 2, or 3) of the trial; and 4) whether or not hospitalization or prolongation of hospitalization was associated with the event.

Any medical documentation supporting an expedited report (e.g., H & P, admission and/or notes, consultations, ECG results, etc.) MUST be faxed within 48-72 hours to the NCI. NOTE: English is required for supporting documentation submitted to the numbers listed below in order for the NCI to meet the regulatory reporting timelines.



Fax supporting documentation for AEs related to investigational agents supplied under a CTEP IND to: (301) 897-7404.

Also: Fax or email supporting documentation to COG for **all** IND studies (fax # (310) 640-9193; email: <u>COGAERS@childrensoncologygroup.org</u>; Attention: COG CTEP-AERS Coordinator).

- ALWAYS include the ticket number on all faxed documents.
- Use the NCI protocol number and the protocol-specific patient ID provided during trial registration on all reports.
- 11.9 Reporting Table for Late Phase 2 and Phase 3 Studies Table A

  Expedited Reporting Requirements for Adverse Events that Occur on Studies under an IND/IDE within 30 Days of the Last Administration of the Investigational Agent/Intervention<sup>1</sup>

## FDA REPORTING REQUIREMENTS FOR SERIOUS ADVERSE EVENTS (21 CFR Part 312)

**NOTE:** Investigators **MUST** immediately report to the sponsor (NCI) **ANY** Serious Adverse Events, whether or not they are considered related to the investigational agent(s)/intervention (21 CFR 312.64) An adverse event is considered serious if it results in **ANY** of the following outcomes:

- 1) Death.
- 2) A life-threatening adverse event.
- 3) Any AE that results in inpatient hospitalization or prolongation of existing hospitalization for ≥ 24 hours. This does not include hospitalizations that are part of routine medical practice.
- 4) A persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions.
- 5) A congenital anomaly/birth defect.
- 6) Important Medical Events (IME) that may not result in death, be life threatening, or require hospitalization may be considered serious when, based upon medical judgment, they may jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the outcomes listed in this definition. (FDA, 21 CFR 312.32; ICH E2A and ICH E6.)

**ALL SERIOUS** adverse events that meet the above criteria **MUST** be immediately reported to the NCI via CTEP-AERS within the timeframes detailed in the table below.

| Hospitalization | Grade 1 | Grade 2 | Grade 3 | Grade 4 & 5 |
|---|---|---|---|---|
| | Timeframes | Timeframes | Timeframes | Timeframes |
| Resulting in<br>Hospitalization<br>≥ 24 hrs | 7 Calendar Days | | 24-Hour Notification | |
| Not resulting in<br>Hospitalization<br>≥ 24 hrs | Not Required | | 7 Calendar Days | 5 Calendar Days |

**NOTE:** Protocol specific exceptions to expedited reporting of serious adverse events are found in the Specific Protocol Exceptions to Expedited Reporting (SPEER) portion of the CAEPR. Additional Special Situations as Exceptions to Expedited Reporting are listed below.

### Expedited AE reporting timelines are defined as:

"24-Hour; 5 Calendar Days" - The AE must initially be reported via CTEP-AERS within 24 hours of learning of the AE, followed by a complete expedited report within 5 calendar days of the initial 24-hour notification. "7 Calendar Days" - A complete expedited report on the AE must be submitted within 7 calendar days of learning of the AE.



<sup>1</sup>SAEs that occur more than 30 days after the last administration of investigational agent/intervention and have an attribution of possible, probable, or definite require reporting as follows:

# Expedited 24-hour notification followed by complete report within 5 calendar days for:

• All Grade 4, and Grade 5 AEs

## **Expedited 7 calendar day reports for:**

- Grade 2 adverse events resulting in hospitalization or prolongation of hospitalization
- Grade 3 adverse events

### 11.10 Protocol Specific Additional Instructions and Reporting Exceptions

- Grades 1 4 myelosuppression (anemia, neutropenia, thrombocytopenia) do not require expedited reporting.
- Any blinatumomab-related AE that results in interruption of dosing as described in <u>Section 5.2</u> requires expedited reporting.
- Any Grade 3 or higher infection (defined as sepsis, bacteremia, device or catheterrelated infection) that occurs more than 30 days after the last administration of blinatumomab and has an attribution of possible, probable, or definite must also be reported via CTEP-AERS.

# 11.11 Reporting of Adverse Events for <u>commercial</u> agents – CTEP-AERS abbreviated pathway

The following are expedited reporting requirements for adverse events experienced by patients on study who have <u>not</u> received any doses of an investigational agent on this study.

Commercial reporting requirements are provided in Table B.

COG requires the CTEP-AERS report to be submitted within 7 calendar days of learning of the event.

#### Table B

Reporting requirements for adverse events experienced by patients on study who have NOT received any doses of an investigational agent on this study.

# CTEP-AERS Reporting Requirements for Adverse Events That Occur During Therapy With a Commercial Agent or Within 30 Days<sup>1</sup>

| Attribution | Grade 4 | | Grade 5 |
|------------------------------|------------|----------|-----------|
| | Unexpected | Expected | |
| Unrelated or Unlikely | | | CTEP-AERS |
| Possible, Probable, Definite | CTEP-AERS | | CTEP-AERS |

<sup>1</sup>This includes all deaths within 30 days of the last dose of treatment with a commercial agent, regardless of attribution. Any death that occurs more than 30 days after the last dose of treatment with a commercial agent that can be attributed (possibly, probably, or definitely) to the agent and is <u>not</u> due to cancer recurrence must be reported via CTEP-AERS.



## 11.12 Routine Adverse Event Reporting

**Note:** The guidelines below are for routine reporting of study specific adverse events on the COG case report forms and do not affect the requirements for CTEP-AERS reporting.

Routine reporting is accomplished via the Adverse Event (AE) Case Report Form (CRF) within the study database. For this study, routine reporting is split into three categories:

- 1. During all blinatumomab cycles as well as parallel control arm cycles, routine reporting will include all toxicities of all grades (see table).
- 2. HSCT routine reporting will include All toxicities reported via CTEP-AERS and all Grade 4 and higher non-hematological Adverse Events
- 3. During all other blocks of therapy, routine reporting will include all toxicities reported via CTEP-AERS and all Grade 3 and higher non-hematological Adverse Events (see table).

| ADV | FDSF FVFNT DFDADTI | NG BY TREATMENT PHASE |
|---|---|---|
| ALL PATIENTS | EKSE EVENT KEFOKTI | REPORTING REQUIREMENT |
| Block 1 | | Grade 3 and higher non-hematological Adverse Events and all toxicities reported via CTEP-AERS |
| HR/IR | | |
| Arm A<br>(Control) | Arm B<br>(Experimental) | |
| Block 2 | Blinatumomab: Cycle 1 | Grade 1-5 hematological and non-hematological Adverse Events |
| Block 3 | Blinatumomab: Cycle 2 | Grade 1-5 hematological and non-hematological Adverse Events |
| Bridging | Therapy | Grade 3 and higher non-hematological Adverse Events and all toxicities reported via CTEP-AERS |
| HSCT | HSCT | Grade 4 and higher non-hematological Adverse Events and all toxicities reported via CTEP-AERS |
| LR | | |
| Arm C<br>(control) | Arm D (Experimental) | |
| Block 2 | Block 2 | Grade 3 and higher non-hematological Adverse Events and all toxicities reported via CTEP-AERS |
| Block 3 | Blinatumomab cycle 1 | Grade 1-5 hematological and non-hematological Adverse Events |
| Continuation 1 | Continuation 1 | Grade 3 and higher non-hematological Adverse Events and all toxicities reported via CTEP-AERS |
| Continuation 2 (first 5 weeks – days 1-35) | Blinatumomab cycle 2 | Grade 1-5 hematological and non-hematological Adverse Events |
| Continuation 2 (last 3 weeks – days 36-53) Maintenance (first 5 weeks – days 1-35) | Continuation 2 | Grade 3 and higher non-hematological Adverse Events and all toxicities reported via CTEP-AERS |
| Maintenance<br>(second 5 weeks – days 36-<br>70) | Blinatumomab cycle 3 | Grade 1-5 hematological and non-hematological Adverse Events |



| Maintenance (remainder) | Maintenance (all) | Grade 3 and higher non-hematological Adverse Events and all toxicities reported via CTEP-AERS |
|---|---|---|
| <b>TF-Salvage Therapy</b> | | |
| Blinatumomab-S 1 | | Grade 1-5 hematological and non-hematological |
| Blinatumo | omab-S 2 | Adverse Events |



#### 12.0 RECORDS AND REPORTING

See the Case Report Forms posted on the COG web site with each protocol under "Data Collection/Specimens". A submission schedule is included.

#### 12.1 **CDUS**

This study will be monitored by the Clinical Data Update System (CDUS). Cumulative CDUS data will be submitted quarterly to CTEP by electronic means. Reports are due January 31, April 30, July 31 and October 31. This is not a responsibility of institutions participating in this trial.

### 12.2 CTA/CRADA

The agent(s) supplied by CTEP, DCTD, NCI used in this protocol is/are provided to the NCI under a Collaborative Agreement (CRADA, CTA, CSA) between the Pharmaceutical Company(ies) (hereinafter referred to as "Collaborator(s)") and the NCI Division of Cancer Treatment and Diagnosis. Therefore, the following obligations/guidelines, in addition to the provisions in the "Intellectual Property Option to Collaborator" (http://ctep.cancer.gov/industryCollaborations2/intellectual\_property.htm) contained within the terms of award, apply to the use of the Agent(s) in this study:

- 12.2.1 Agent(s) may not be used for any purpose outside the scope of this protocol, nor can Agent(s) be transferred or licensed to any party not participating in the clinical study. Collaborator(s) data for Agent(s) are confidential and proprietary to Collaborator(s) and shall be maintained as such by the investigators. The protocol documents for studies utilizing Agents contain confidential information and should not be shared or distributed without the permission of the NCI. If a copy of this protocol is requested by a patient or patient's family member participating on the study, the individual should sign a confidentiality agreement. A suitable model agreement can be downloaded from: http://ctep.cancer.gov.
- 12.2.2 For a clinical protocol where there is an investigational Agent used in combination with (an)other Agent(s), each the subject of different Collaborative Agreements, the access to and use of data by each Collaborator shall be as follows (data pertaining to such combination use shall hereinafter be referred to as "Multi-Party Data"):
  - a. NCI will provide all Collaborators with prior written notice regarding the existence and nature of any agreements governing their collaboration with NCI, the design of the proposed combination protocol, and the existence of any obligations that would tend to restrict NCI's participation in the proposed combination protocol.
  - b. Each Collaborator shall agree to permit use of the Multi-Party Data from the clinical trial by any other Collaborator solely to the extent necessary to allow said other Collaborator to develop, obtain regulatory approval or commercialize its own Agent.
  - c. Any Collaborator having the right to use the Multi-Party Data from these trials must agree in writing prior to the commencement of the trials that it will use

210



the Multi-Party Data solely for development, regulatory approval, and commercialization of its own Agent.

- 12.2.3 Clinical Trial Data and Results and Raw Data developed under a Collaborative Agreement will be made available to Collaborator(s), the NCI, and the FDA, as appropriate and unless additional disclosure is required by law or court order as described in the IP Option to Collaborator

  (<a href="http://ctep.cancer.gov/industryCollaborations2/intellectual\_property.htm">http://ctep.cancer.gov/industryCollaborations2/intellectual\_property.htm</a>).

  Additionally, all Clinical Data and Results and Raw Data will be collected, used and disclosed consistent with all applicable federal statutes and regulations for the protection of human subjects, including, if applicable, the Standards for Privacy of Individually Identifiable Health Information set forth in 45 C.F.R. Part 164.
- 12.2.4 When a Collaborator wishes to initiate a data request, the request should first be sent to the NCI, who will then notify the appropriate investigators (Group Chair for Cooperative Group studies, or PI for other studies) of Collaborator's wish to contact them.
- 12.2.5 Any data provided to Collaborator(s) for Phase 3 studies must be in accordance with the guidelines and policies of the responsible Data Monitoring Committee (DMC), if there is a DMC for this clinical trial.
- 12.2.6 Any manuscripts reporting the results of this clinical trial must be provided to CTEP by the Group office for Cooperative Group studies or by the principal investigator for non-Cooperative Group studies for immediate delivery to Collaborator(s) for advisory review and comment prior to submission for publication. Collaborator(s) will have 30 days from the date of receipt for review. Collaborator shall have the right to request that publication be delayed for up to an additional 30 days in order to ensure that Collaborator's confidential and proprietary data, in addition to Collaborator(s)'s intellectual property rights, are protected. Copies of abstracts must be provided to CTEP for forwarding to Collaborator(s) for courtesy review as soon as possible and preferably at least three (3) days prior to submission, but in any case, prior to presentation at the meeting or publication in the proceedings. Press releases and other media presentations must also be forwarded to CTEP prior to release. Copies of any manuscript, abstract and/or press release/ media presentation should be sent to:

Email: ncicteppubs@mail.nih.gov

The Regulatory Affairs Branch will then distribute them to Collaborator(s). No publication, manuscript or other form of public disclosure shall contain any of Collaborator's confidential/proprietary information.



## 13.0 SPECIAL STUDIES AND SPECIMEN REQUIREMENTS

NOTE: Enrollment APEC14B1 is ENCOURAGED, but NOT REQUIRED. APEC14B1 only require a single cell bank specimen (i.e. not separate AALL1331 and APEC14B1 specimens).

# 13.1 Banking for Future Research (optional)

For cases with a limited amount of tissue available for analysis, please prioritize specimen for tissue banking. Samples will be collected at different time points. See <u>Section 7.2</u> for time points.

This study is designed to provide material for banking for the purpose of performing retrospective studies to refine risk stratification, identify new targets for therapy, identify biomarkers to predict response, and to link host polymorphisms with various disease characteristics and toxicities. See <u>Appendix VI</u> for details.

#### Sample Collection Procedures

A Specimen Transmittal Form should accompany every shipment of specimen(s) to the COG Reference Laboratory. Please complete one form per patient per shipment.

<u>Please note:</u> The AALL1331 Specimen Transmittal Form should be used. This is a protocol specific form.

## Shipping Media (SM)

Samples for the Reference Laboratories are to be collected in shipping media (SM) in special 15 mL conical tubes. The SM contains RPMI with EDTA as the anticoagulant. These tubes will be prepared in the Molecular Reference Laboratory and shipped in batches to each participating institution, where they can be stored frozen at -20°C until use. Tubes are stable for 3 months if refrigerated and stable for 1 year if frozen. To request prepared and pre-packaged sample shipping tubes, order tubes through the Biopathology Center kit management system <a href="https://ricapps.nationwidechildrens.org/KitManagement/">https://ricapps.nationwidechildrens.org/KitManagement/</a>.

Please note: The receiving institutions are strongly encouraged to make requests for sample tubes well in advance of their first patient registration on AALL1331; it will not be possible to expedite shipping because of prohibitive costs.

#### **Bone Marrow/Peripheral Blood Collection Procedures for Reference Laboratories:**

- a. Collect BM/PB into a syringe and transfer the specimen immediately into the SM tube with RPMI/EDTA.
- b. Mix well. At least 2 mL and up to 5 mL of BM/PB can be placed in 1 SM tube. If you don't have SM tubes, you can place the BM/PB into large purple EDTA tubes that are commonly available in most hospitals. However, the viability of the cells is greatly enhanced in the SM tubes.
- c. For BM, use multiple syringes and tubes as necessary. Reposition the BM aspirate needle at least once during the diagnostic procedure to ensure the maximum quality of BM. DO NOT SHIP SYRINGES.
- d. Label each tube with COG registration number, patient name and date of birth, collection date, institution and type of specimen (bone marrow).
- e. Samples are to be shipped at room temperature except for international samples that are expected to be delayed for more than 48 hours place a cold pack (not ice pack) in shipment.



**NOTE**: For patients who are not having a BM for medical reasons at diagnosis or other time points and have an <u>absolute blast count of at least 1,000/µL</u>, PB may be submitted to the Reference Laboratories instead of BM. Submit 2 mL of PB for each 1 mL of required marrow.

#### Reference Laboratory – Shipping Address (including Saturday delivery):

COG Leukemia Biospecimen Bank Nationwide Children's Hospital 575 Children's Crossroads, Room WB2255 Columbus, OH 43215

Phone: (614) 722-2866 Fax: (614) 722-2887

Email: mglab@nationwidechildrens.org

All samples should be mailed by overnight carrier (Federal Express) PRIORITY (delivery before 10 am). Use the COG FedEx account number, which may be found at: https://members.childrensoncologygroup.org/ files/reference/FEDEXmemo.pdf.

Notify Laboratory of each Saturday delivery (email or phone) and remember to mark "For Saturday Delivery" on the FedEx paperwork.

#### 13.2 Local Bone Marrow: Central review of cytogenetics/FISH

Bone marrow aspiration to confirm relapse (and/or to detect potential marrow disease in presumed isolated extramedullary relapse patients) is required for <a href="study entry">study entry</a>. Morphologic, immunophenotypic, & cytogenetic/FISH analysis should be performed by the local institution. Cytogenetic analysis should include FISH for any cytogenetic abnormalities known from the patient's original leukemia if applicable. All FISH should be performed on uncultured, directly-harvested cells or unstimulated overnight cultured cells if the former is not possible. FISH for abnormalities shown by cytogenetics to be unique to the relapse specimen should also be done on directly harvested cells or unstimulated overnight cultured cells if the former is not possible. Cytogenetic/FISH analysis must be performed at a COG approved cytogenetics lab and cases will be reviewed retrospectively by the COG Cytogenetics Committee.

Please see the following link for a list of COG approved cytogenetics labs: <a href="https://www.cogmembers.org/site/admin/default.aspx">https://www.cogmembers.org/site/admin/default.aspx</a>

### **Required Material:**

- a) Two **original** karyotypes of different cells from each abnormal clone or of two normal cells when no abnormalities are found; full-size metaphase images of the karyotypes cells.
- b) A completed COG Cytogenetics Reporting Form and FISH Form (if done). These reporting forms are available on the AALL1331 protocol web page. Electronic submission of the karyotypes/FISH images is required.

**Shipping**: The review materials on each case should be sent to the COG ALL Cytogenetic Coordinators within 4 weeks of study entry. If the institution is west of the Mississippi River, send these materials to Dr. Andrew Carroll (University of Alabama). If the



institution is east of Mississippi River (except Minnesota and Wisconsin, which go to Dr. Carroll), send all materials to Dr. Nyla Heerema (The Ohio State University).

## Western Laboratory – Shipping Address:

Dr. Andrew Carroll, Ph.D. Ph.D. Department of Genetics University of Alabama at Birmingham 720 20th St. So. Kaul Bldg. Room 314B Birmingham, AL 35294

Phone: 205-934-0665 Fax: 205-934-1078 Email: acarroll@ uab.edu

#### **Eastern Laboratory – Shipping Address:**

Dr. Nyla Heerema, Ph.D.
Professor and Director of Cytogenetics
The Ohio State University
Division of Clinical Pathology
Hamilton Hall, Room 167
1645 Neil Ave. Columbus, OH 43210

Phone: 614-292-7815 Fax: 614-292-7072

Email: Nyla.Heerema@osumc.edu

# 13.3 Bone Marrow for Central Flow-Immunophenotyping and MRD (required)

Immunophenotyping will be done on fresh bone marrow specimens collected <u>at study entry</u> (see <u>Section 7.1</u>). Minimal residual disease will be detected using 6 color flow cytometry (Dr. Michael Borowitz, Johns Hopkins University) on fresh bone marrow specimens collected <u>during therapy at various designated time points</u> (see <u>Section 7.1</u>). Sample Collection Procedures

A Specimen Transmittal Form should accompany every shipment of specimen(s) to the COG Reference Laboratory. Please complete one form per patient per shipment.

<u>Please note:</u> The AALL1331 Specimen Transmittal Form should be used. This is a protocol specific form.

#### Shipping Media (SM)

Samples for the Reference Laboratories are to be collected in shipping media (SM) in special 15 mL conical tubes. The SM contains RPMI with EDTA as the anticoagulant. These tubes will be prepared in the Molecular Reference Laboratory and shipped in batches to each participating institution, where they can be stored frozen at -20°C until use. Tubes are stable for 3 months if refrigerated and stable for 1 year if frozen. To request prepared and pre-packaged sample shipping tubes, order tubes through the Biopathology Center kit management system <a href="https://ricapps.nationwidechildrens.org/KitManagement/">https://ricapps.nationwidechildrens.org/KitManagement/</a>.

**Please note:** The receiving institutions are strongly encouraged to make requests for sample tubes well in advance of their first patient registration on AALL1331; it will NOT be possible to expedite shipping because of prohibitive costs.

#### **Bone Marrow Collection Procedures for Reference Laboratories:**



- a. Collect BM into a syringe and transfer the specimen immediately into the SM tube with RPMI/EDTA.
- b. Mix well. At least 2 mL and up to 5 mL of BM can be placed in 1 SM tube. If you don't have SM tubes, you can place the BM into large purple EDTA tubes that are commonly available in most hospitals. However, the viability of the cells is greatly enhanced in the SM tubes.
- c. Use multiple syringes and tubes as necessary. Reposition the BM aspirate needle at least once during the diagnostic procedure to ensure the maximum quality of BM. DO NOT SHIP SYRINGES.
- d. Label each tube with COG registration number/Biopathology number, patient name and date of birth, date, institution and type of specimen (bone marrow).
- e. Samples are to be shipped at room temperature except for international samples that are expected to be delayed for more than 48 hours place a cold pack (not ice pack) in shipment.

**NOTE**: For patients who are not having a BM for medical reasons at diagnosis or other time points and have an <u>absolute blast count of at least  $1,000/\mu L$ </u>, PB maybe submitted to the Reference Laboratories instead of BM. Submit 2 mL of PB for each 1 mL of BM required.

**Please note:** Specimens will be shipped to the COG Reference Laboratory at Johns Hopkins (Eastern) ONLY.

# **Reference Laboratory – Shipping Address (including Saturday delivery):**

Michael Borowitz, MD, PhD

Flow Cytometry Laboratory, Johns Hopkins Medical Institutions

Weinberg Building – Room 2300

401 N. Broadway

Baltimore, MD 21287 Phone: 410-614-2968 Fax: 410-502-1493

Email: mborowit@jhmi.edu

All samples should be mailed by overnight carrier (Federal Express) PRIORITY (delivery before 10 am). Use the COG FedEx account number, which may be found at: <a href="https://members.childrensoncologygroup.org/files/reference/FEDEXmemo.pdf">https://members.childrensoncologygroup.org/files/reference/FEDEXmemo.pdf</a>.

Notify Laboratory of each Saturday delivery at 410-614-2968 or via email at kbowles3@jhmi.edu

#### 13.4 Bone Marrow for CRLF2 expression (optional)

We will quantify surface CRLF2 expression by flow cytometry and correlate with outcome. This assay will be done in conjunction with the immunophenotyping performed at study entry in Dr. Mike Borowitz's lab at Johns Hopkins University (see <u>Section 13.3</u>). For details, refer to Appendix IX.

## Sample Collection Procedures

**NOTE:** A separate specimen is NOT REQUIRED. Please note on the specimen transmittal forms that accompany the required immunophenotyping specimen whether the patient has consented for the optional CRLF2 expression assay.



## 13.5 Blinatumomab Pharmacodynamics (PD) (optional)

Immunopharmacologic testing will be performed using blood and bone marrow specimens in consenting patients treated with blinatumomab during the first exposure to blinatumomab in an effort to identify biomarkers of blinatumomab response. For details, refer to Appendix X.

NOTE: All patients will be offered participation in this study at Block 1, prior to treatment assignment/randomization. Bone marrow samples will be drawn on all consenting patients at end Block 1. If the patient is subsequently randomized or assigned to treatment with blinatumomab (Arm B, Arm D, or Salvage Therapy), the Block 1 bone marrow sample will be analyzed and subsequent blood samples should be obtained. If the patient is randomized to treatment on the control arm (Arm A or Arm C), the Block 1 bone marrow sample will be destroyed and no further samples will be collected.

## Sample Collection Procedures

A Specimen Transmittal Form should accompany every shipment of specimen(s) to the Brown Laboratory. Please complete one form per patient per shipment.

In the event that the infusion is interrupted, the peripheral blood collection should likewise be delayed to account for the interruption. i.e. collect the timed sample after X days of infusion rather than X days from start of infusion.

<u>Please note:</u> The AALL1331 Specimen Transmittal Form should be used. This is a protocol specific form.

#### Blood and marrow collection schedule (see Section 7.2)

- Bone Marrow (1 sample, 5-10mL in sodium heparin tube)
  - o End Block 1 (All patients)
  - o End Block 2 (LR patients on Arm D only)
- Blood during first blinatumomab cycle (7 samples, 3mL each in sodium heparin tubes)
  - o Day 1
    - 0 hr (just prior to start of blinatumomab infusion)
    - 6 hr
    - 12 hr
  - o Day 2
  - o Day 7
  - o Day 14
  - o Day 21

Samples should be shipped at room temperature.

### **Brown Laboratory – Shipping Address (including Saturday delivery):**

Dr. Patrick Brown Johns Hopkins Oncology Cancer Research Building I, Room 262 1650 Orleans Street Baltimore, MD 21231


Laboratory phone: 410-955-8688

Pager no: 410-434-0732 E-mail: pbrown2@jhmi.edu

All samples should be mailed by overnight carrier (Federal Express) PRIORITY (delivery before 10 am). Use the COG FedEx account number, which may be found at: <a href="https://members.childrensoncologygroup.org/files/reference/FEDEXmemo.pdf">https://members.childrensoncologygroup.org/files/reference/FEDEXmemo.pdf</a>.

Saturday deliveries are permissible. If a Saturday delivery is required, please notify Dr. Brown of the planned shipment via email (pbrown2@jhmi.edu) PRIOR to the time of shipment and clearly mark the package "For Saturday Delivery".

#### 13.6 Protein Cell Stress Pathways (optional)

Note: Isolated extramedullary relapse patients are not eligible for this sub-study.

This study is designed to analyze two specific aims: 1) To determine if specific protein expression profiles, as determined by reverse-phase protein lysate array (RPPA) analysis and phospho-flow analysis, correlate with therapy response and 2) To determine if alterations in specific cell stress proteins (such as the UPR) during chemotherapy can identify low risk patients with "high risk" protein signatures. For details, refer to Appendix XI.

Consenting patients will have peripheral blood samples (5mL for those  $\geq$  10kg, 3 mL for those < 10 kg) collected at 0 hours (prior to start of Block 1 systemic chemotherapy), and at 2 time points after the initiation of therapy (6 hours and 24 hours after the first dose of Block 1 systemic chemotherapy) to examine for changes in protein expression patterns. Blood samples for RPPA using sucrose centrifugation and (if necessary) the lymphoblast population will be isolated by either bead technology or flow cytometry. Sample collected for phospho-flow will be analyzed directly from whole blood. Sorted lymphoblasts will be made into lysates for RPPA analysis prior to freezing. Remaining samples will be frozen as pellets for protein analysis.

## **Eligible samples:**

Sample should be sent to the Horton lab only if the patient has an initial absolute blast count of at least 1,000 lymphoblasts/ $\mu L$ . To calculate the absolute blast percentage, multiply the total WBC by the % peripheral blasts:

 $(WBC)(\% blast)(1000) = absolute blast count/\mu L$ 

Example: If the patient has a WBC of 10 and 50% blasts, the absolute blast count is:  $(10)(.5)(1000) = 5000/\mu L$ 

If the initial % blasts is unknown, send samples only if the total WBC is more than 10,000 and notify the Horton lab of the % blast as soon as available (contact info provided below).

# Sample Collection Procedures

A Specimen Transmittal Form should accompany every shipment of specimen(s) to the Horton Laboratory. Please complete one form per patient per shipment. **Please note:** The AALL1331 Specimen Transmittal Form should be used. This is a protocol specific form.



**Sample collection time points:** 

| | Day 1, Hour 0 | Day 1, Hour 6-8 | Day 1, Hour 24 |
|---|---|---|---|
| | (before start of systemic | | |
| | chemotherapy) | | |
| Peripheral | • 3 – 5 mL <sup>#</sup> in CellSave | • 3mL in CellSave | • 3mL in CellSave |
| Blood | Preservative Tube* | Preservative | Preservative |
| (Block 1 | • 3mL in heparin tube | Tube* | Tube* |
| only) | • | • 3mL in heparin | • 3mL in heparin |
| | | tube | tube |

<sup># 5</sup> mL for those  $\geq$  10kg, 3 mL for those  $\leq$  10kg

Store samples in refrigerator until shipment, and use Thermosafe with ice pack (or similar Styrofoam shipping containers with sufficient ice packs if these are not available at your site.) These containers maintain biology samples at a constant temperature and are strongly recommended for biology sample shipment, particularly in warm weather months.

## **Horton Laboratory – Shipping Address (including Saturday delivery):**

Dr. Terzah Horton c/o Gaye Jenkins Feigin Center, Room 760.01 1102 Bates St. Baylor College of Medicine Houston, TX 77030

Phone: (832) 824-4676 or (832) 824-4269

Email tmhorton@txccc.org

All samples should be mailed by overnight carrier (Federal Express) PRIORITY (delivery before 10 am). Use the COG FedEx account number, which may be found at: https://members.childrensoncologygroup.org/ files/reference/FEDEXmemo.pdf.

The Horton lab can accept Saturday shipments if we are contacted ahead of time. Please contact Gaye Jenkins or Dr. Horton (832-824-4676 or 832-824-4269) for alternative address and shipping information for Saturday delivery.

13.7 Blinatumomab Immunogenicity Assessment (Required)
(See lab manual on protocol webpage for sample collection and shipping details)

Blinatumomab is a novel protein therapeutic under clinical development. As outlined in the Draft Guidance: Immunogenicity Assessment for Therapeutic Protein Products (Feb 2013) pre-specified immunogenicity sampling will be performed to evaluate and mitigate risk (<a href="http://www.fda.gov/downloads/Drugs/GuidanceComplianceRegulatoryInformation/Guidances/UCM338856.pdf">http://www.fda.gov/downloads/Drugs/GuidanceComplianceRegulatoryInformation/Guidances/UCM338856.pdf</a>).

Blood samples for the assessment of blinatumomab immunogenicity will be collected to determine whether anti-idiotype antibodies directed against blinatumomab have been

<sup>\*</sup> CellSave tubes will be provided by the Horton lab to each institution upon IRB approval. To obtain more CellSave tubes, contact the Horton lab at the numbers provided below. If the CellSave tubes are not available, submit entire 6 mL sample in 2 heparin tubes. Note that the sample integrity is greatly enhanced by the use of CellSave tubes.



developed. Screening for these antibodies will be done by ELISA assay on ECL Basis (electrochemiluminescence), and binding will be confirmed with a Biacore assay to measure protein-protein interaction and binding affinity.

In a tiered approach patient samples are initially tested in a screening assay. Samples that produce signals above a certain screening cut point (classified as "positive") may be subjected to a confirmatory assay. The screening assay is designed to minimize false negatives, so positive screening assays need to be confirmed as positive. These are performed using the same format as the screening assay. A comparison of patient serum in the presence and absence of excess blinatumomab is used to confirm or deny the existence of anti blinatumomab antibodies. The screening and confirmation assay in the context of blinatumomab clinical studies will be performed according to an internal standardized protocol using a validated assay.

Immunoassay-positive samples will be analyzed in a third step using a cell based blinatumomab-mediated cytotoxicity assay to determine if the detected antibodies have neutralizing properties. Detection of neutralizing anti-blinatumomab antibodies relies on a validated bioassay measuring changes in the biologic activity of blinatumomab triggered by the presence of the antibody.

Blood Serum samples for antibody testing are being collected on all patients randomized to receiving blinatumomab for the measurement screening of anti-blinatumomab binding antibodies. Samples testing positive for binding antibodies will also be tested for neutralizing antibodies and may be further characterized for quantity/titer, isotype, affinity and presence of immune complexes. The 'cell-based assay' for neutralizing antibody detection tests patient sera in a model cell based system. This does not require patient cells or additional serum to be collected. Both the screening and the neutralizing assays are well-established at the Amgen Research Munich laboratory.

COG will be notified of any positive neutralizing antibody results to blinatumomab. If results are not provided, no neutralizing antibodies to blinatumomab have been detected. Patients who test positive for neutralizing antibodies to blinatumomab at the final scheduled study visit will be asked to return for additional follow-up testing. This testing is to occur approximately every three months starting from when the site has been notified of the positive result, until: (1) neutralizing antibodies are no longer detectable or (2) the subject has been followed for a period of at least one year ( $\pm$  4 weeks) post administration of blinatumomab. All follow-up results, both positive and negative will be communicated to COG. More frequent testing (e.g. every month) or testing for a longer period of time may be requested in the event of safety-related concerns. Follow-up testing is not required where it is established that the subject did not receive blinatumomab. Patients who test positive for binding, non-neutralizing antibodies and have clinical sequelae that are considered potentially related to an anti-blinatumomab antibody response may also be asked to return for additional follow-up testing.

# 13.8 Blinatumomab PK (required)

Please see the Lab Manual posted on the protocol web page for sample collection and shipping details.

219



#### 14.0 RADIATION THERAPY GUIDELINES FOR ALL PATIENTS

Radiation therapy (RT) for patients on COG protocols can only be delivered at approved COG RT facilities (per COG administrative policy: Other Membership: Radiation Oncology Paritipcation Requirements).

Timing of protocol therapy administration, response assessment studies, and surgical interventions are based on schedules derived from the experimental design or on established standards of care. Minor unavoidable departures (up to 72 hours) from protocol directed therapy and/or disease evaluations (and up to 1 week for surgery) for valid clinical, patient and family logistical, or facility, procedure and/or anesthesia scheduling issues are acceptable per COG administrative Policy 5.14 (except where explicitly prohibited within the protocol).

#### 14.1 General Guidelines

The objective of this protocol is to compare the benefits and risks of Blinatumomab in the treatment of first relapse B-ALL. Patients eligible for this study will undergo risk classification after an initial block of chemotherapy (Block 1). Risk classification and the indications for irradiation will be based on site of first relapse, time to first relapse, MRD status following Block1 chemotherapy and clinical response to chemotherapy (when testicular leukemia is present at protocol entry).

Patients determined to be low risk (LR) after Block 1, will receive additional chemotherapy (Block 2) post randomization to a control arm or an experimental arm. The experimental arm includes blinatumomab. Both the control and experimental arms include maintenance chemotherapy to complete the respective regimens. LR patients with testicular leukemia at protocol entry will receive testicular irradiation (2400cGy) during Block2 if they do not have a clinical complete response after Block1. LR patients with CNS leukemia at protocol entry will receive cranial irradiation (1800cGy) during maintenance chemotherapy.

Intermediate Risk (IR) and High Risk (HR) patients will proceed to protocol-specified hematopoietic stem cell transplant (HSCT). Selected patients that do not respond to Block1 and HR and IR patients that do not respond to the control arm will receive blinatumomab in a separate treatment arm and may proceed to HSCT depending on their response to Blinatumomab provided they do not have a history of CNS leukemia (CNS3) at or after protocol entry. IR/HR patients with testicular leukemia at protocol entry will receive testicular irradiation (2400cGy) during the first cycle of Blinatumomab (experimental arm) if they do not have a complete response after Block1. IR/HR patients with testicular leukemia who have a complete clinical response to Block 1 will receive *supplemental* testicular irradiation (600cGy) sequentially with total body irradiation (TBI). IR/HR patients with CNS leukemia at protocol entry will receive *supplemental* cranial irradiation (600cGy) sequentially with TBI. *Supplemental* irradiation refers to irradiation of any site performed sequentially with TBI.

Treatment failure (TF) patients are select patients that do not respond to Block1 and HR and IR patients that do not respond to the control arm. They will receive Blinatumomab in a separate treatment arm and may proceed to HSCT depending on their response to Blinatumomab provided they do not have a history of CNS leukemia (CNS3) at or after protocol entry. They may also receive testicular or cranial irradiation therapy when indicated. TF patients after block1 will receive testicular irradiation (2400cGy) during their first course of Blinatumomab. TF patients with testicular leukemia who have a complete clinical response to Block1 will receive supplemental testicular irradiation (600cGy)



sequentially with total body irradiation (TBI). TF patients after block2 with CNS leukemia at protocol entry will receive supplemental cranial irradiation (600cGy) sequentially with TBI.

Because there is no consensus on fractionated TBI or supplemental irradiation regimens, the radiation therapy guidelines for this study were designed to promote protocol participation and match guidelines used at the majority of approved transplant institutions and evolved from guidelines developed for other COG protocols. Questions about these guidelines should be directed to the radiation therapy coordinator or principal investigator. *Complete clinical response* refers only to the testes. *Supplemental irradiation* refers to irradiation of any site performed sequentially with TBI.

## 14.1.1 Required Benchmark and Questionnaires

Radiation therapy will be administered using photons or electrons according to treatment site. All centers administering TBI must have completed the TBI benchmark for the specific TBI technique to be used for patients treated on this study. Benchmark instructions are available at the IROC Rhode Island website: <a href="https://www.qarc.org/">https://www.qarc.org/</a>.

The calibration of therapy units used in this protocol must be verified by IROC Houston (RPC) (http://irochouston.mdanderson.org).

# 14.2 Indications for Radiation Therapy

# 14.2.1 Total Body Irradiation

TBI is indicated as part of the preparative regimen for IR/HR patients undergoing HSCT.

- 14.2.1.1 Supplemental cranial irradiation is indicated for HSCT patients with a history of CNS leukemia at protocol entry and shall be given sequentially.
- 14.2.1.2 Supplemental testicular irradiation is indicated for HSCT patients with the diagnosis of testicular leukemia and complete response after Block1 and shall be given sequentially. Those with testicular leukemia and without complete response after Block1 will not require supplemental testicular irradiation because they will have already received 2400cGy earlier in the regimen.
- 14.2.1.3 Patients who require irradiation to extra-medullary sites other than brain and testes should contact the Study Chair.

# 14.2.2 Cranial Irradiation

LR patients with a history of CNS leukemia at protocol entry should receive cranial irradiation. Cranial irradiation will be given between the first and second 12 week blocks of Maintenance chemotherapy. This corresponds to Week 40 for LR patients treated on the control arm and Week 54 for LR patients treated on the experimental arm. IR/HR patients will receive supplemental cranial irradiation sequentially with TBI prior to HSCT. Exceptions to the use of cranial irradiation include concerns about additional effects due to patient age, history of prior cranial



irradiation and history or imaging evidence of CNS toxicity including leukoencephalopathy, stroke and necrosis.

# 14.2.3 Testicular Irradiation

Patients with persistent testicular leukemia at the end of Block 1 will receive 2400 cGy of testicular radiation during either Block 2 chemotherapy (for LR patients and HR/IR patients randomized to the control arm) or during blinatumomab (for HR/IR patients randomized to the experimental arm and TF patients after Block 1). Prior testicular irradiation will not be a contraindication to supplemental testicular irradiation on this protocol.

## **14.3 Timing**

- 14.3.1 All patients who might require irradiation should be seen in consultation by a radiation oncologist in advance of treatment. The purpose of the consultation is to participate in planning the sequence of treatment and to determine the need for extra medullary (cranial, testicular and other) and supplemental irradiation in conjunction with HSCT.
- 14.3.2 The timing of TBI and supplemental irradiation will be determined in part by the TBI fractionation regimen. Supplemental irradiation should precede TBI and be performed during weekdays.

# 14.4 Emergency Irradiation

There may be instances when radiation therapy has been administered prior to enrollment on this protocol because of potentially life-threatening or function-threatening extramedullary involvement. Although it is not expected that prior treatment would make total body irradiation contraindicated, it should be considered when describing to the patient or parent the potential complications of treatment on this protocol.

## 14.5 Equipment and Methods of Delivery

| <u> </u> | • | |
|------------------------|------------|------------|
| Treatment Site | Photons | Electrons |
| TBI | Any Energy | |
| Cranial Irradiation | 4 or 6MV | |
| Testicular Irradiation | Any Energy | Any Energy |

Any energy for photons or electrons can be used as long as the skin and target dose requirements are met.

## 14.6 Treatment Volumes

#### 14.6.1 Total Body Irradiation

The entire body will be treated including the head and feet in one field. Care should be taken to insure that the patient is entirely within the 90% isodose line of the beam and not in the penumbra region.



#### 14.6.2 Cranial Irradiation

The treatment site consists of the entire brain and intracranial subarachnoid volume as well as the optic nerves and the posterior halves of the optic globes. The caudal border shall be the C2/3 vertebral interspace.

#### 14.6.3 Testicular Irradiation

The treatment site consists of the testes in the scrotal sac.

## 14.7 Target Dose

#### 14.7.1 Dose Definition

Photon and electron dose is to be specified in centigray (cGy)-to-muscle.

#### 14.7.2 Prescribed Dose, Fractionation and Dose Rate for TBI

TBI may be administered with either of the following two regimens:

- 1200 cGy administered over 3 consecutive treatment days (Days -7, -6, -5) at 200cGy BID
- 1200 cGy administered over 4 consecutive treatment days (Days -8, -7, -6, -5) at 150cGy BID

#### Allowable but not preferred TBI regimen:

• 1320 cGy given over 4 consecutive treatment days (Days -8, -7, -6, -5) at 165 cGy BID

Important considerations for TBI:

- Effort should be made to avoid interruptions in TBI administration
- The inter-fraction interval shall be no less than 5 hours between treatments (start to start)
- A mid-plane dose rate of between 6 and 15 cGy per minute is required

## 14.7.3 Prescribed Dose and Fractionation for Cranial Irradiation

- 14.7.3.1 LR patients will receive 1,800 cGy administered in 10 daily fractions of 180 cGy during Maintenance chemotherapy.
- 14.7.3.2 IR/HR patients will receive 600 cGy administered in 3 daily fractions of 200 cGy immediately before TBI
- 14.7.4 <u>Prescribed Dose and Fractionation for Testicular Irradiation (testicular leukemia at</u> protocol entry)
  - 14.7.4.1 LR patients will not receive testicular irradiation if a complete clinical response is observed after Block1.



- 14.7.4.2 LR patients will receive 2400 cGy testicular irradiation administered in 12 daily fractions of 200 cGy during Block 2 if a complete clinical response is not observed after Block 1.
- 14.7.4.3 IR/HR patients will receive 600 cGy administered in 3 daily fractions of 200 cGy immediately before TBI if complete clinical response is observed after Block 1.
- 14.7.4.4 IR/HR patients will receive 2400 cGy testicular irradiation administered in 12 daily fractions of 200 cGy During Block 2 if a complete clinical response is not observed after Block 1.
- 14.7.5 <u>Prescribed dose and fractionation for testicular irradiation (testicular leukemia not present at protocol entry)</u>
  - 14.7.5.1 Supplemental testicular irradiation of 400 cGy in 1 or 2 daily fractions prior to or during TBI may be administered according to institutional preference but is not required.

#### 14.8 **Treatment Technique**

#### 14.8.1 TBI

Supine and prone, lateral decubitus, upright seated and standing positions are allowed. Treatment will be delivered with equally weighted parallel opposed portals. Each treatment will include both fields. All treatment techniques and patient positions should meet the criteria on dose, dose rate, and dose uniformity. Beam spoilers or other equally effective devices may be used to increase skin dose to meet the dose uniformity requirements. Changes in patient positioning after the patient has started TBI must be documented. Changes in lung blocking and dose recalculation should be reported.

#### 14.8.2 TBI - Lung Shielding

Lung shielding is mandated to restrict the lung dose (see <u>Section 14.9.1</u>). Lung shielding to achieve dose reduction should conform to the following guidelines:

- The lateral edges will be 1.0 1.5 cm inside the inner border of the ribs;
- The inferior edges will be 1.0 1.5 cm superior from the dome of the apex of the diaphragm;
- The superior borders will be 1.0 1.5 cm below the clavicles;
- The medial border 2.0 2.5 cm lateral to edges of the thoracic vertebral bodies.
- No contouring of the lung shields will be done around the hilum unless there is residual hilar adenopathy in which case the margins around the hilar abnormality will be 1.0-1.5 cm. When utilized, lung blocks should be employed for sequential treatments starting with the first treatment.
- Compensatory electron boost of the portion of the chest wall shielded by the lung blocks is not required.



#### 14.8.3 <u>Cranial Irradiation</u>

Supine treatment is recommended with immobilization appropriate for the age of the child. Two opposed lateral equally weighted photon beams are preferred. The fields shall extend at least 1 cm beyond the periphery of the scalp. Customized field-shaping is required with blocks that are at least 5 HVL thick. Alternatively, a multi-leaf collimator may be used provided the leaf width is less than or equal to 5 mm.

Lens sparing techniques are encouraged with 1 of 2 techniques:

- Angling of the 2 lateral fields in the anterior direction (RAO/LAO) using the lateral canthus markers to "flatten" the beam edge. Shielding blocks are used to block the anterior halves of the eyes, the nose, and mouth.
- Set the central axes of the horizontal cranial beams so that they are aligned to the lateral canthi (half-beam blocking technique). The anterior edges of the beams are defined by an external block or by an independently controlled collimator and meet at a point 1 cm anterior to the frontal lobe meninges. Shielding blocks cover the anterior halves of the eyes and protect the nose and mouth.

#### 14.8.4 Testicular Irradiation

The patient shall be treated in the supine position. Field shaping for photons and electrons will be done with either customized cerrobend blocking or multi-leaf collimation. The testes may be supported posteriorly and, if possible, extended caudally in order to minimize perineal irradiation. The penis should be excluded from the field.

## 14.9 **Organs at Risk**

#### 14.9.1 Normal tissue sparing for TBI

Restricting the lung dose to  $\leq 800$  cGy is required on this protocol. This requirement applies to both AP/PA and lateral treatments. Institutions are allowed to use their preferred method of beam attenuation to achieve the dose reduction to lungs. The lung dose shall be reported as reference point C for lateral treatments and reference point D for AP/PA treatments (see Section 14.10.1.2). It should be reported on the TBI Summary form.

# 14.9.2 Normal tissue sparing for cranial irradiation

• Lens sparing techniques, as outlined in <u>Section 14.8.3</u>, are encouraged.

# 14.9.3 Normal tissue sparing for testicular irradiation

• Techniques for sparing perineum and penis are outlined in <u>Section 14.8.4</u>.

## 14.10 Dose Calculation and Reporting

## 14.10.1 Dose calculations for TBI

14.10.1.1 Suggested Methods for Dose Calculations for TBI



The TBI percent depth dose (PDD) or Tissue Maximum Ratio (TMR) and output factors may be measured under TBI treatment conditions for a range of phantom sizes to establish the database for TBI beam-on time calculations and to validate the calculation method. Measurements of entrance and exit dose at the center of a phantom equivalent to the size of the typical patient are performed and compared to the calculated dose. If differences are found, additional correction factors should be introduced to the calculation method. The prescription point is defined as the point along the longitudinal axis of the patient at the mid-plane at the level of the umbilicus (Point E below). Tissue inhomogeneity correction is not required in the calculation of dose to the prescription point.

14.10.1.2 Dose Calculations and Measurements to Selected Anatomical Reference Points for TBI

**Prescription Point:** 

The following reference points will be determined:

The calculated and measured doses to selected anatomical points must be submitted to IROC RI as part of the quality assurance documentation:

(Point A - Head) This reference point is defined along the longitudinal axis of the skull at the greatest mid-separation (immediately superior to the nasal bridge). The depth should be taken as midway between the entrance and exit points of the opposed radiation beams.

(Point B – Neck) This reference point is defined along the patient's longitudinal axis at the level of C3/C4 (approximate mid-neck, but chosen for the thinnest mid-separation of the neck). The point is taken to be midway between the entrance and exit point of the beam.

(Point C - Mid-mediastinum) For APPA: The point is in the center of the chest along the sagittal plane midway between the anterior and posterior surfaces (Usually at the level of the carina). For opposed laterals: this point is located midway between the entrance and exit points of the beams at the level of the carina. Calculations at this reference point should include lung shielding if present.

(Point D – Mid-Lung) APPA only: This reference point is centered in the middle of the right or left lung (both medial/lateral and cephalocaudad directions). The depth should be taken as midway between the entrance and exit points of the opposed radiation beams. Calculations at this reference point should include lung shielding if present.

(Point E – Umbilicus) This is the PRESCRIPTION POINT. This point is located along the patient's longitudinal axis at the level of the umbilicus and midway between the entrance and exit points of the opposed beams.



(Point F – Hip or Pelvis) This reference point is defined at the level approximately 1 cm superior to pubic symphysis midway between the entrance and exit points of the beam.

(Point G - Knee) This reference point is defined along the midline in the mid-plane of the knee at the level of the patella.

(Point H -Ankle) This reference point is defined along the midline at the mid-plane of the ankle at the level of the lateral malleolus.

#### 14.10.1.3 Lung Dose Calculation

Tissue heterogeneity must be accounted for in the calculation of dose to lung. The preferred method is use of CT to enable use of CT numbers in the calculation. Alternatively, other methods as developed by the participating institution may be used. Lung density value estimates, based on methods adopted by treating institutions, may be incorporated into the dose calculation. The methodology used by each participating institution for lung dose determination will be evaluated as part of the benchmark approval process.

## 14.10.2 <u>Dose Uniformity and Treatment Site Coverage</u>

14.10.2.1 TBI Dose Uniformity and Treatment Site Coverage

The TBI fields should be set up to cover the patient's entire body without any part of the patient extending into the penumbra region. The dose difference between the prescription point and each reference point (see separate guidance for lung dose in Section 14.9.1) shall be within  $\pm$  10% of the prescribed dose. The calculated dose to the lung shall be in accordance with the lung dose requirements specified in Section 14.9. To limit overall total lung dose to  $\leq$  800 cGy, partial transmission lung blocks can be used. For AP/PA treatments the lung blocks may be placed in both AP and PA fields or alternatively in just the AP or PA field alone.

- 14.10.2.2 Cranial Irradiation Dose Uniformity and Treatment Site Coverage

  The prescription point for the cranial treatment is at or near the center of
  the field. Regardless of the location of the central axis, the dose should
  be prescribed at the center of the cranial volume –midway between the
  points of maximum separation. The variations of dose within the
  treatment site shall be within +7%, -5% of the dose to the prescription
  point.
- 14.10.2.3 Testicular Irradiation Dose Uniformity and Treatment Site Coverage
  The scrotum should be treated with en face electrons with the
  prescription depth covered by the 90% isodose. If electron beam is used
  for testicular irradiation, the prescription should include the beam
  energy and the dose coverage. Photon irradiation is allowed.



#### 14.10.3 <u>Tissue heterogeneity</u>

There shall be no required correction for tissue heterogeneity for the cranial and testicular treatment.

#### 14.10.4 Interruption of therapy

Excluding weekends and holidays, supplemental cranial irradiation, testicular irradiation and fractionated TBI should be continuous. All efforts should be made not to have treatment delay or interruption. Once patients have begun testicular treatment, they should immediately proceed to TBI for transplantation. If interruptions occur, the radiation therapy coordinator should be notified.

# 14.11 Quality Assurance Documentation and Review

There are no on-treatment review or image submission requirements for this study. A post-treatment review will be conducted by IROC RI.

Within 1 week of the completion of radiotherapy, the following data shall be submitted for TBI and/or cranial and testicular irradiation:

- TBI Summary Form for Total Body Irradiation.
- Measured and/or calculated doses for the TBI reference points.
- A copy of the radiotherapy record including the prescription, and daily and cumulative doses for all treated sites including TBI and supplemental sites (cranial, testicular).
- The "RT-2 Radiotherapy Total Dose Record" forms must be completed for cranial and testicular irradiation.
- If the treatment technique differs from an approved benchmark, a new benchmark must be completed and approved (see Section 14.1.1).

Data should be sent by email to the IROC Rhode Island QA Center: <a href="mailto:datasubmission@qarc.org">datasubmission@qarc.org</a>

Questions regarding the dose calculations or documentation should be directed to the COG Protocol Dosimetrist at the IROC Rhode Island QA Center.

Email: physics@qarc.org Phone: (401) 753-7600

#### 14.12 **Definitions of Deviation in Protocol Performance**

## 14.12.1 TBI

14.12.1.1 Deviations for prescription dose Deviations for TBI Dose

Variation Acceptable:

• The dose to the prescription point and to any of the reference points (except points C and D lung dose points) differs from the protocol specified dose by >10% or <15%.



# Deviation Unacceptable:

• The dose to the prescription point and to any of the reference points (except points C and D lung dose points) differs from the protocol specified dose by >15%.

#### 14.12.1.2 Deviations for TBI Dose Rate

 A dose rate exceeding 15cGy/min will be considered as an unacceptable deviation.

# 14.12.1.3 Deviations for Lung Dose

• The dose to the lungs (reference points C and D) that is < 700 cGy or > 900 cGy will be considered an unacceptable deviation.

## 14.12.2 <u>Deviations for Cranial Irradiation Dose</u>

# Variation Acceptable:

• The dose to the prescription point differs from the protocol specified dose by > 6 but ≤ 10%.

# Deviation Unacceptable:

• The dose to the prescription point differs from the protocol specified dose by >10%.

# 14.12.3 <u>Deviations for Testicular Irradiation Dose</u>

## Variation Acceptable:

• The dose to the prescription point differs from the protocol specified dose by > 6% but ≤ 10%.

## Deviation Unacceptable:

• The dose to the prescription point differs from the protocol specified dose by > 10%.



#### APPENDIX I: SUPPORTIVE CARE

**NOTE:** For blinatumomab-specific supportive care guidelines, please refer to <u>Section 5.2</u>.

#### **General Guidelines**

Aggressive supportive care improves outcome. The following guidelines are intended to give general direction for optimal patient care and to encourage uniformity in the treatment of this study population. Notify Study Chair of any unexpected or unusually severe complications. Please also see the COG Supportive Care Guidelines at: <a href="https://childrensoncologygroup.org/index.php/cog-supportive-care-guidelines">https://childrensoncologygroup.org/index.php/cog-supportive-care-guidelines</a>.

#### **Blood Components**

Blood products should be irradiated following current FDA guidelines.

Investigators in Canadian institutions need to follow the CSA standards for Blood and Blood Components.

# Red Blood Cells (RBC)

Transfusion with RBC is indicated to correct severe or symptomatic anemia or acute blood loss. In the setting of extreme hyperleukocytosis investigators should be mindful that peripheral red blood cells (PRBC) may contribute to hyperviscosity.

#### **Platelets**

Transfusion with platelets is indicated to correct bleeding manifestations and may be indicated for severe thrombocytopenia without bleeding particularly prior to an invasive procedure.

## **Special Guidelines During Induction (Block 1)**

Patients may experience profound myelosuppression and immune suppression during this time. Since steroids may mask fever as well as other components of the inflammatory response, sepsis during Induction may be associated with very mild and subtle symptoms. Caregivers must also be made aware that patients may experience very rapid clinical deterioration. This suggests the need for a supportive care network that can recognize and respond to sudden changes in a patient's condition. In addition it should be noted that serious toxic events may have an intestinal component. Patients with subtle GI symptoms should be monitored very closely. Taken together, the risks of significant morbidity and mortality, including sudden death in patients with relapsed leukemia, are sufficient to strongly recommend hospitalization during remission Induction, until patients show consistent neutrophil recovery and transfusion needs that are deemed to be manageable in the outpatient setting.

# Tumor Lysis Syndrome

In this population with ALL, rapidly assess patients clinically and by appropriate laboratory parameters for evidence of symptomatic hyperleukocytosis, tumor lysis syndrome, and coagulopathy. Suggested studies to be obtained prior to initiating antileukemia therapy include complete blood count (CBC), prothrombin and activated partial thromboplastin times, fibrinogen, D-dimer, and serum electrolytes, including creatinine, BUN, uric acid, phosphorous, and calcium. Continued monitoring of these studies should be carried out at suitable intervals until abnormalities have resolved or the risk has abated. Begin allopurinol at a dose of 300 mg/m²/day or 10 mg/kg/day (maximum 800 mg/day) in 2-3 divided doses and continue until peripheral blasts and extramedullary disease are reduced. In some situations it may be appropriate to use rasburicase. Hydrate at 2,400 – 3,000 mL/m²/day (potassium should not be added to hydration fluids) to maintain urine output > 100 mL/m²/hour until peripheral blasts and extramedullary disease are reduced.



## **Infection Prophylaxis**

Patients undergoing transplantation for ALL on this protocol are at high risk for infection. This risk may be increased due to infections that occur during the intensive chemotherapy most patients will receive prior to stem cell transplant on this protocol. Centers should be especially mindful of this as they choose anti-bacterial, anti-fungal, anti-viral, and PCP prophylactic regimens. Aside from well established screening approaches for CMV, centers may wish to consider routine screening for other viral pathogens such as Adenovirus or HHV-6. Any prophylaxis regimen chosen must be the same for patients on both arms of the protocol. Special considerations should be given for antifungal prophylaxis (see below).

# Supportive Care for Patients Age 15 Years and Older

It is recommended that adolescent and young adult (AYA) patients enrolled on this protocol (defined as patients between the ages of 15 and 31 years) be monitored in the hospital during Block 1, Block 2 and Block 3 of chemotherapy until they show signs of bone marrow recovery (specifically evidence that the absolute neutrophil count (ANC) is rising for 2 successive days) and the patient is afebrile and clinically stable. If a patient should experience profound myelosuppression at any other time, there should also be a very low threshold to hospitalize AYA patients with inpatient management continued until there is evidence of bone marrow recovery. Antibiotic prophylaxis against Gram-positive and Gram-negative organisms (e.g. levofloxacin) may be considered during these hospitalizations until patients meet the criteria for discharge. If the patient should develop febrile neutropenia while on antibiotic prophylaxis, the patient should be started on broad-spectrum intravenous antibiotics per institutional guidelines. Antifungal prophylaxis may also be considered during periods of myelosuppression. Options include an echinocandin such as caspofungin or micafungin, or an azole. Azole antifungal agents (i.e., fluconazole, itraconazole, posaconazole, voriconazole) given concurrently with vincristine may increase the risk of neurotoxicity. Investigator caution is advised if azole antifungals are used. If antibiotic and/or antifungal prophylaxis is utilized, consultation with Infectious Disease may be considered.

#### Pneumocystis iiroveci

All patients should receive trimethoprim/sulfamethoxazole (TMP/SMX) at a dose of TMP 2.5 mg/kg/dose (maximum dose 160 mg/dose) by mouth twice daily on 2 or 3 sequential days per week. For patients allergic to or experiencing excessive myelosuppression with TMP/SMX, alternative prophylaxis with dapsone (2 mg/kg/day by mouth, maximum dose 100 mg/day), aerosolized pentamidine (300 mg/q month ≥ 5 years of age), or atovaquone (4 - 24 month: 45 mg/kg/day; > 24 months: 30 mg/kg/day) by mouth may be considered. For children in whom TMP/SMX, dapsone, atovaquone, and inhaled pentamidine cannot be administered, IV pentamidine (4 mg/kg/dose IV every 2 to 4 weeks) should be given. (REF: Centers for Disease Control and Prevention. Guidelines for preventing infectious complications among hematopoietic stem cell transplant recipients: a global perspective. (https://www.cdc.gov/mmwr/preview/mmwrhtml/rr6002a1.htm)

## Varicella Vaccine

May be given to the siblings of patients in remission and stable at the physician's discretion. Varicella vaccination is not recommended for ALL patients during therapy.

#### Gamma globulin

If clinically indicated, IgG levels may be monitored throughout treatment. If the IgG level falls below age-determined normal levels, IVIG at 400 mg/kg may be administered at the discretion of the investigator. Note of IVIG administration should be recorded on data form.

#### Antifungals

Azole antifungal agents (i.e. fluconazole, itraconazole, voriconazole) given concurrently with vincristine may increase the risk of neurotoxicity. Investigator caution is advised if azole antifungals are used.



Fluconazole and other azoles are expected to increase serum tacrolimus and sirolimus levels. Therefore, dosages of sirolimus and tacrolimus should be adjusted accordingly. Due to extreme interactions with sirolimus, voriconazole is contraindicated during sirolimus. Patients on voriconazole prior to transplant should have another drug substituted for voriconazole prior to starting sirolimus therapy.

# Hospitalization after High-Dose Cytarabine

Empiric hospitalization after Day 8 of Induction 3 (intensively-timed Capizzi-II) until there is evidence of marrow recovery should be considered due to the risk of neutropenic sepsis; patients not hospitalized should be monitored very closely.

#### **Treatment of Established or Presumed Infections**

# Fever with Neutropenia

For patients with ANC  $< 500/\mu L$  or expected to fall to this level within the next 48 hours and an oral-equivalent temperature  $\ge 38.3$  °C once or between 38.0 °C and 38.3 °C twice within 12 hours, empiric broad spectrum antibiotics should be instituted after obtaining appropriate cultures. Patients who present with severe sepsis should have empiric antibiotic coverage widened to include resistant Gram-negative, Gram-positive, and anaerobic bacteria.

The risk of bacteremia and infectious mortality is higher during Induction and during profound neutropenia. For prolonged fever and neutropenia (≥ 96 hours), empiric antifungal therapy with either caspofungin or liposomal amphotericin B should be given during periods of anticipated prolonged neutropenia including induction.

Also, please see the COG Fever and Neutropenia Guidelines at:

https://childrensoncologygroup.org/downloads/COG SC FN Guideline Document Dec 2017.pdf

#### Use of filgrastim (G-CSF)

Filgrastim may be used for severe infections with neutropenia, but routine use is discouraged.

Filgrastim at a dose of 5 micrograms/kg/day given IV or subcutaneously is required for recipients of cord blood starting at Day +1 and continuing until patients are fully engrafted. Filgrastim is generally not necessary for BM/PBSC recipients and is not recommended, unless engraftment is delayed.

## Primary Varicella Infection (Chickenpox)

Patients should be treated promptly with acyclovir 1500 mg/m²/day intravenously divided q8 hours, and monitored closely for the development of invasive systemic disease.

# **Empiric Management of Pulmonary Infiltrates**

Pulmonary infiltrates should be evaluated with bronchoscopy and biopsy, lavage or open lung biopsy. If a procedure cannot be tolerated, begin empiric antifungal therapy given the high likelihood of fungal disease during Induction, Re-induction and periods of intensive chemotherapy (HDAraC). Empiric coverage should include treatment for gram-negative and positive bacteria, Legionella (erythromycin), Pneumocystis (TMP/SMX), and fungi (amphotericin) pending culture results. If fungal pulmonary disease is documented, surveillance radiographic imaging studies of the sinuses, abdomen/pelvis and brain are indicated. Surgical excision of pulmonary lesions should be considered at the discretion of the treating physician. Treatment of fungal infections with amphotericin B and/or other antifungal agents will be at the discretion of the treating physician. Azole antifungal agents (i.e. fluconazole, itraconazole, voriconazole) given concurrently with vincristine may increase the risk of neurotoxicity. Investigator caution is advised if azole antifungals are used.



# Management of Mucositis/Perirectal Cellulitis

Mucositis should be managed with IV hydration and hyperalimentation if indicated, effective analgesia, broad-spectrum gram-positive and gram-negative antibiotic therapy and empiric antiviral and antifungal therapy as indicated. Management of perirectal cellulitis should include broad-spectrum antibiotic therapy with dual gram-negative coverage as well as anaerobic coverage (i.e. ceftazidime + aminoglycoside + metronidazole; or piperacillin-tazobactam + aminoglycoside), Sitz baths, a strong barrier technique and effective analgesia.

# Prevention and Management of Chemotherapy-induced Nausea and Vomiting (CINV)

Please refer to the COG Endorsed guidelines on prevention and management of CINV at: https://childrensoncologygroup.org/downloads/COG SC CINV Guidelines Document Feb 2018.pdf

The routine use of steroids including dexamethasone, as an antiemetic is discouraged but may be appropriate in select patients with demonstrated intolerance to higher-dose chemotherapeutic agents.

#### Gastrointestinal (GI) Protection

While patients are on steroid therapy, consider using an H2 receptor antagonist (e.g., ranitidine, famotidine).

# Constipation

As vincristine may cause severe constipation, prophylactic stool softeners/laxatives (per investigator's discretion) are recommended during all phases in which VCR is given.



#### APPENDIX II: THERAPY DELIVERY MAPS

| APPENDIX II-A Block 1 (All patients) | | |
|---|---|---|
| Block 1 therapy is common to all patients on study | Patient COG ID number | DOB |

Block 1 lasts 4 weeks (28 days). Please see Section 4.2 for treatment details. This therapy delivery map is on two (2) pages. ROUTE DAYS DRUG DOSAGE **IMPORTANT NOTES OBSERVATIONS** Age (yrs) Dose ALL PATIENTS a. Hx, PE [VS/Wt (BSA)] Intrathecal Methotrexate (IT MTX) IT 1-1.99 8 mg b. CBC/diff/platelets 2-2.99 10 mg c. Local BM evaluation % 3-8.99 12 mg Note age-based dosing d. BM for Immunophenotyping >9 15 mg e. CSF cell count, cytospin<sup>1</sup> CNS1/2 ONLY IT Age (yrs) Dose Intrathecal Methotrexate (IT MTX) 1-1.99 8 mg f. Bilirubin, ALT & creatinine. \*For CNS2: Continue weekly until 2 clear csf 2-2.99 10 mg BUN samples are obtained i.e. CNS1 3-8.99 12 mg g. Echocardiogram Note age-based dosing >9 15 mg h. Pregnancy test CNS3 ONLY Intrathecal Triple Therapy (ITT): 8, 15, 22 Age (yrs) Dose i. Testicular Exam & Testicular Methotrexate (MTX)/ 1-1.99 MTX:8mg, biopsy, if indicated® Hydrocortisone (HC)/Cytarabine HC: 8mg, ARAC: 16mg (ARAC) Note age-based dosing 2-2.99 MTX: 10mg Obtain with each IT/ITT HC: 10 mg ARAC: 20 mg See Section 7.0 for details. 3-8.99 MTX: 12 mg HC: 12 mg **Optional studies** ARAC: 24 mg Banking for future research ≥9 MTX: 15 mg k Protein cell stress pathways HC: 15 mg CRLF2 expression ARAC: 30 mg m. BM sample for Administer through the tubing of a freely MitoXANTRONE (MITOX) IV over 15-30 10 mg/m<sup>2</sup>/dose 1, 2 Blinatumomab PD minutes infusing solution of D<sub>5</sub>W or 0.9% NaCl 10 mg/m<sup>2</sup>/dose BID Total Daily Dose 20 mg/m<sup>2</sup>/day divided BID Dexamethasone (DEX) PO 1-5, 15-19 Cap dose at 40 mg per day. +Or infusion via minibag as per institutional See Section 7.2 for details. VinCRIStine (VCR) IV push over 1.5 mg/m<sup>2</sup> 1, 8, 15, 22 1 minute+ policy. Maximum dose: 2mg 2500 International 3, 17 Administer through the tubing of a freely Pegaspargase (PEG-ASP) IV over 1-2 **OBTAIN OTHER STUDIES AS** hours units/m2/dose infusing solution of D<sub>5</sub>W or 0.9% NaCl REQUIRED FOR GOOD PATIENT CARE



APPENDIX II-A Block 1 (All patients)
Block 1 therapy is common to all patients on study

Patient COG ID number

DOB

| Ht | cm | | Wtkg | BSA | m² | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Date | Date | Day | IT MTX | IT MTX | ITT | MITOX | DEX | VCR | PEG-ASP | Studies | Comments (Include |
| Due | Given | | ALL PATIENTS | CNS1/2 ONLY* | CNS3 ONLY | | | | | | any held doses, or |
| | | | mg | mg | mg | mg | mg | mg | IU | | dose modifications) |
| | | | | Enter calculated | d dose above and ac | tual dose adı | ministered b | elow | | a, b, c% d-i, 1\$,j+ | |
| | | 1 | mg | | | mg | mg | mg | | k <sup>¥</sup> | |
| | | 2 | | | | mg | | | | | |
| | | 3 | | | | | | | IU | | |
| | | 4 | | | | | | | | | |
| | | 5 | | | | | • | | | | |
| | | 8 | | mg | mg | | | mg | | b, e, f | |
| | | 15 | | mg* | mg | | mg | mg | | b, e*, f | |
| | | | | nig | mg | | n | mg | | 0, 0 , 1 | |
| | | 17 | | | | | | | IU | | |
| | | 19 | | | | | ▼ | | | | |
| | | 22 | | mg* | mg | | | mg | | b, e*, f | |
| | | 29 | | | | | | | | b, c, e^, f, i <sup>®</sup> , j <sup>+</sup> , m | |
| | | | | and will be removed f<br>(experimental arm). A<br>Block 1 with M3 marr<br>(Blinatumomab-S) (See | gin next course based on Day 29 risk assignment and treatment randomization. IR/HR patients are not eligible for post-Induction treatment divill be removed from protocol therapy at the end of Induction. LR patients will be randomized to Arm C (control arm) or Arm D reperimental arm). All LR patients (Arm C and Arm D) receive Block 2 therapy (Section 4.3, APPENDIX II-B). Treatment failures post-ock 1 with M3 marrow without residual CNS disease (CNS1) are eligible for treatment with at least 2 blocks of Salvage Therapy linatumomab-S) (Section 4.7, APPENDIX II-F); treatment failures with residual CNS disease (CNS2/3), irrespective of marrow status will off protocol therapy. See Section 4.3 for further details on time frame for end-Block 1 evaluations and criteria to fulfill prior to subsequent | | | | | | |

\*For CNS2 patients, continue weekly until 2 clear CSF (CNS1) samples are obtained; can be a max of 4 (Days 1, 8, 15 and 22). If still unclear, patients are treatment failures and will be off protocol therapy regardless of marrow status.

- ^ A diagnostic LP should be performed on Day 29 for CNS2 or CNS3 patients for whom clearance of CSF blasts has not yet been documented.
- <sup>®</sup> Testicular biopsy is only done in the setting of persistent testicular enlargement. Patients with persistent testicular leukemia at the end of Block 1 who are deemed treatment failure (TF) will receive 2400 cGy of testicular radiation during Blinatumomab.
- No separate specimen needed-cell pellet from required central flow MRD assays will be used (see Section 13.4 for complete details).
- <sup>¥</sup> PB before and after chemotherapy on Day 1 of Block 1 (see <u>Section 13.6</u>) for complete details).
- <sup>%</sup> BM evaluation to confirm relapse and/or detect marrow disease in presumed isolated extramedullary relapse patients should include morphology, immunophenotyping & cytogenetics/FISH. Cytogenetic/FISH analysis must be performed at a COG approved cytogenetics lab and cases will be reviewed retrospectively
- + Bone marrow: at Baseline and End Block 1. Peripheral blood: At Baseline and End Block 1. (See Section 13.1 for complete details)

  See Section 5.0 for Dose Modifications for Toxicities and Appendix I for Supportive Care Guidelines.

DOB



## APPENDIX II-B Block 2

Block 2 therapy is for all LR patients post Block-1 (Arm C and Arm D)

Patient COG ID number

Block 2 lasts 4 weeks (28 days). Block 2 should begin after receipt of risk assignment according to timing outlined in Section 4.2.7. All patients can proceed with Day 1 of Block 2 without awaiting count recovery (must be no later than 5 calendar days after callback). Patients with M1 marrow after Block 1 should await count recovery to ANC  $\geq 500/\mu$ L and platelets  $\geq 50,000/\mu$ L prior to beginning Day 8 ID MTX; Patients with M2 marrow after Block 1 should not await recovery prior to beginning Day 8 ID MTX. All patients should await count recovery to ANC  $\geq 500/\mu$ L and platelets  $\geq 50,000/\mu$ L prior to beginning Day 15 cyclophosphamide and etoposide. Please see Section 4.3 for treatment details. This Therapy Delivery Map is on two (2) pages.

| DRUG | ROUTE | DOSAGE | | DAYS | IMPORTANT NOTES | OBSERVATIONS |
|---|---|---|---|---|---|---|
| Dexamethasone (DEX) | РО | 3 mg/m²/dose BID | | 1-5 | Total Daily Dose: 6 mg/m²/day, divided BID. | a Hx, PE [VS/Wt (BSA)] b CBC/diff/platelets c Local BM evaluation |
| VinCRIStine (VCR) | IV push over 1<br>minute+ | 1.5 mg/m²/dose | | 1 | + Or infusion via minibag as per institutional policy Maximum dose: 2 mg | d BM for MRD evaluation<br>e CSF cell count, cytospin <sup>1</sup> |
| Intrathecal Methotrexate (IT MTX) | IT | 1-1.99<br>2-2.99<br>3-8.99 | Dose<br>8 mg<br>10 mg<br>12 mg<br>15 mg | 8 | CNS 1/2 ONLY Note age-based dosing When IT therapy and ID MTX are scheduled for the same day, deliver the IT therapy within 6 hours of the beginning of the IV MTX infusion (hour -6 to +6, with 0 being the start of the MTX bolus). | f Bilirubin, ALT & creatinine, BUN g Testicular Exam Optional studies h Banking for future research i Bone Marrow for Blinatumomab PD (Arm D ONLY) |
| Intrathecal Triple Therapy<br>(ITT):<br>Methotrexate (MTX)<br>Hydrocortisone (HC)<br>Cytarabine (ARAC) | IT | 1-1.99<br>2-2.99<br>3-8.99<br>≥9 | Dose MTX:8mg, HC: 8mg, ARAC: 16mg MTX: 10mg HC: 10 mg ARAC: 20 mg MTX: 12 mg HC: 12 mg HC: 12 mg MTX: 15 mg HC: 15 mg ARAC: 24 mg MTX: 15 mg ARAC: 30 mg | 8, 22 | CNS3 ONLY. Note age-based dosing. | ¹ Obtain with each IT/ITT See Section 7.0 for details. See Section 7.2 for details. OBTAIN OTHER STUDIES AS REQUIRED FOR GOOD PATIENT CARE |
| Intermediate Dose<br>Methotrexate (ID MTX) | IV over 36 hours | 1000 mg/m²/dose | <u> </u> | 8 | See Section 5.8 for admin guidelines. | |
| Leucovorin (LCV) | PO/IV | 15 mg/m²/dose Q6H | | 10, 11 | 48 hours after the start of ID MTX infusion. See Section 5.8 for admin guidelines | |
| Pegaspargase (PEG-ASP) | IV over 1-2 hours | 2500 International unit | ts/m²/dose | 9 or 10* | *Administer 4 hours after completion of Day 8 IV MTX. | |
| Cyclophosphamide (CPM) | IV over 15-30 mins. | 440 mg/m²/dose | | 15-19 | | |
| Etoposide (ETOP) | IV over 60-120 mins. | 100 mg/m <sup>2</sup> /dose | | 15-19 | | |
| Testicular Radiotherapy: Pat | ients with persistent testic | ular disease will receive t | testicular radiation | during Block | k 2 therapy. See Section 14.2 for details of TRT. | |



| APPENDIX II-B Block 2 | | |
|---|---|---|
| Block 2 therapy is for all LR patients post Block-1 (Arm C and Arm D) | Patient COG ID number | DOB |

| | Ht | cm | | , | Wtkg | | BSA | m² | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Date<br>Due | Date<br>Given | Day | DEX. | VCR | IT MTX<br>CNS1/2 ONLY | ITT<br>CNS3 ONLY | ID MTX | LCV | PEG-ASP | CPM | ETOP | Studies | Comments (Include any held doses, or dose |
| Due | Given | | mg | mg | mg | mg | mg | mg | IU | mg | mg | | modifications) |
| | | | | | dose above and actua | | | 8 | | 8 | 8 | | / |
| | | 1 | mg | mg | | | | | | | | a, b, f | |
| | | 5 | | | | | | | | | | | |
| | | | • | | | | | | | | | | |
| | | 8 | | | mg | mg | mg^ | | | | | b, e, f | |
| | | 9 | | | | | | | IU* | | | | |
| | | 10 | | | | | | mg | | | | | |
| | | 11 | | | | | | mg | | | | | |
| *** | | 15 | | | | | | | | mg& | mg& | b, f | |
| | | 19 | | | | | | | | <b>\</b> | $\forall$ | | |
| | | 22 | | | | mg | | | | | | b, e <sup>#</sup> , f | |
| | | 29 | | | | | | | | | | b,c,d,f,g,h <sup>+</sup> ,i | |
| | | | | ollowing count recovery, <b>LR patients randomized to Arm C</b> receive Block 3 therapy (Section 4.4, APPENDIX II-C), and <b>LR patients randomized to Arm D</b> receinatumomab Block 1: Cycle 1 therapy (Section 4.15, APPENDIX II-M. | | | | | | | | | |

<sup>^</sup> All patients with M1 marrow are recommended to await count recovery to ANC ≥ 500/µL and platelets ≥ 50,000/µL prior to beginning Day 8 ID MTX. Day 8 treatment must begin no later than 14 calendar days after giving the Day 1 vincristine and dexamethasone to continue to receive protocol therapy.

See Section 5.0 for Dose Modifications for Toxicities and Appendix I for Supportive Care Guidelines.

<sup>&</sup>amp; Await count recovery to ANC  $\geq 500/\mu$ L and platelets  $\geq 50,000/\mu$ L prior to beginning Day 15 cyclophosphamide and etoposide.

<sup>+</sup> **Peripheral blood:** End Block 2 (See Section 13.1 for complete details)

<sup>\*</sup>Administer 4 hours after completion of Day 8 IV MTX. (Day 9 or 10)

<sup>#</sup> CNS3 ONLY



APPENDIX II-C Block 3
Block 3 therapy is for all LR patients randomized to the control arm (Arm C).

Patient COG ID number DOB

Block 3 lasts 4 weeks (28 days) and starts when ANC  $\geq$  500/ $\mu$ L and platelets  $\geq$  50,000/ $\mu$ L. Await count recovery to ANC  $\geq$  500/ $\mu$ L and platelets  $\geq$  50,000/ $\mu$ L prior to beginning Day 22 ID MTX. See Section 4.4 for treatment details. This Therapy Delivery Map is on two (2) pages.

| DRUG ROUTE | | DOSAGE | | DAYS | IMPORTANT NOTES | OBSERVATIONS |
|---|---|---|---|---|---|---|
| Dexamethasone (DEX) | PO (May be given IV) | 3 mg/m²/dose BID | | 1-5 | Total Daily Dose: 6 mg/m²/day, divided BID. | a Hx, PE [VS/Wt (BSA)] b CBC/diff/platelets c Local BM evaluation |
| VinCRIStine (VCR) | IV push over 1 minute <sup>+</sup> | 1.5 mg/m²/dose | | 1 | <sup>†</sup> Or infusion via minibag as per institutional policy<br>Maximum dose: 2 mg | d BM for MRD evaluation e CSF cell count, cytospin <sup>1</sup> |
| Cytarabine (ARAC) | IV over 3 hours | 3000 mg/m²/dose | Q12H | 1, 2, 8, 9 | | f Bilirubin, ALT & creatinine, BUN |
| Asparaginase (Erwinia) | IM or IV over 1 hour | 25, 000 Internation | nal units/m²/dose | 2, 4, 9, 11, 23 | See Section 4.4 for administration guidelines. On Days 2 and 9, Erwinia should be given 4 hours after last cytarabine infusions. On Day 23, Erwinia is to be given 4 hours after the completion of the Day 22 MTX infusion. | <sup>1</sup> Obtain with each IT/ITT See Section 7.0 for further details. |
| Intermediate Dose<br>Methotrexate (ID MTX) | IV over 36 hours | 1000 mg/m²/dose | | 22 | See Section 5.8 for admin guidelines. | |
| Leucovorin (LCV) | PO/IV | 15 mg/m²/dose | | 24, 25 | 48 hours after the start of ID MTX infusion. See<br>Section 5.8 for admin guidelines | OBTAIN OTHER STUDIES AS REQUIRED FOR GOOD |
| Intrathecal Methotrexate<br>(IT MTX) | IT | Age (yrs)<br>1-1.99<br>2-2.99<br>3-8.99<br>≥9 | Dose<br>8 mg<br>10 mg<br>12 mg<br>15 mg | 1 All Patients 22 CNS 1/2 ONLY | When IT therapy and ID MTX are scheduled for the same day, deliver the IT therapy within 6 hours of the beginning of the IV MTX infusion (hour -6 to +6, with 0 being the start of the MTX bolus). Note age-based dosing | PATIENT CARE |
| Intrathecal Triple Therapy<br>(ITT):<br>Methotrexate (MTX)<br>Hydrocortisone (HC)<br>Cytarabine (ARAC) | IT | Age (yrs) 1-1.99 2-2.99 3-8.99 ≥9 | Dose MTX:8mg, HC: 8mg, ARAC: 16mg MTX: 10mg HC: 10 mg ARAC: 20 mg MTX: 12 mg HC: 12 mg ARAC: 24 mg MTX: 15 mg HC: 15 mg ARAC: 30 mg | 22 | CNS3 ONLY When ITT therapy and ID MTX are scheduled for the same day, deliver the ITT therapy within 6 hours of the beginning of the IV MTX infusion (hour -6 to +6, with 0 being the start of the MTX bolus). Note age-based dosing | |



| APPENDIX II-C | Block 3 | | |
|---|---|---|---|
| Block 3 therapy is for | all LR patients randomized to the control arm (Arm C). | Patient COG ID number | DOB |

| | | | Ht | cı | n V | Vt | kg | BSA | | $m^2$ | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Date Due | Date<br>Given | Day | DEX. | VCR | ASP<br>ERWINIA | ID MTX | LCV | ARAC | | IT MTX All Patients | IT MTX<br>CNS1/2 ONLY | ITT<br>CNS3 ONLY | Studies | Comments (Include any held |
| | | | mg | mg | IU | mg | mg | mg | mg | mg | mg | mg | | doses, or dose<br>modifications) |
| | | | Enter calc | ulated dose | above and actua | ıl dose admin | istered belov | V | | | | | | |
| | | 1 | mg | mg | | | | mg | _mg | mg | | | a, b, e, f | |
| | | 2 | 1 1 | | IU | | | mg | _mg | | | | | |
| | | 3 | | | | | | | | | | | | |
| | | 4 | | | IU | | | | | | | | | |
| | | 5 | \ \ | | | | | | | | | | | |
| | | 8 | | | | | | mg | _mg | | | | b, f | |
| | | 9 | | | IU | | | mg | _mg | | | | | |
| | | | | | *** | | | | | | | | | |
| | | 11 | | | IU | | | | | | | | | |
| | | 1.5 | | | | | | | | | | | 1 6 | |
| | | 15 | | | | | | | _ | | | | b, f | |
| | | 22 | | | | ma^ | | | | | ma | ma | b, e, f | |
| | | 23 | | | IU | mg^ | | | | | mg | mg | 0, 6, 1 | |
| | | 24 | | | 10 | | mg | | | | | | | |
| | | 25 | | | | | mg | | | | | | | |
| | | 29 | | | | | | | | | | | b, (c, d)* f | |
| | | | ing count r | ecovery AN | L<br>NC > 500/uL. aı | nd platelets: | > 50,000/uI | HR/IR Tre | atmen | t Failures post-Blo | ock 3 have the opti | on of receiving | | I<br>Salvage Therapy – |
| | | | 3 | | | r | _ : = , = = = , pez | | | t and to post Bi | | | | |

Blinatumomab-S (Sections 4.7, 4.8, APPENDIX II-F, II-G). LR patients randomized to Arm C receive Continuation 1 therapy (Section 4.11, Appendix II-I).

See Section 5.0 for Dose Modifications for Toxicities and Appendix I for Supportive Care Guidelines.

<sup>^</sup> Await count recovery until ANC  $\geq$  500/ $\mu$ L and platelets  $\geq$  50,000/ $\mu$ L prior to beginning Day 22 ID MTX.

<sup>\*</sup>HR/IR Patients ONLY.



# APPENDIX II-D Blinatumomab Block - Cycle 1 (HR/IR Patients in Arm B)

This therapy is the 1st cycle of therapy with blinatumomab for the HR/IR patients assigned to the experimental arm (Arm B)

Patient COG ID number DOB

Blinatumomab Block-Cycle 1 lasts 5 weeks (35 Days). For patients with M1 marrow, treatment begins when ANC  $\geq 500/\mu$ L and platelets  $\geq 50,000/\mu$ L and must begin no later than 14 calendar days after risk assignment for patient to continue to receive protocol therapy. For patients with M2 marrow, treatment begins without awaiting count recovery, and must be no later than 5 calendar days after callback. See Section 4.5 for treatment details. This Therapy Delivery Map is on two (2) pages.

| DRUG | ROUTE | DOSAGE | DOSAGE | | IMPORTANT NOTES | OBSERVATIONS |
|---|---|---|---|---|---|---|
| Blinatumomab (BLIN) Do not use commercial supply | IV | 15 micrograms/1 | n²/day | 1-28 | | a Hx, PE [VS/Wt (BSA)] b CBC/diff/platelets c BM (Local evaluation & MRD) |
| Dexamethasone (DEX) | PO or IV | | 20 mg) 30 to 60 minutes of the Blinatumomab | 1 | Start prior to blinatumomab therapy | d CSF cell count, cytospin <sup>1</sup> e Bilirubin, ALT & creatinine, BUN |
| Intrathecal<br>Methotrexate (IT<br>MTX) | IT | Age (yrs) Dose<br>1-1.99<br>2-2.99<br>3-8.99<br>>9 | 8 mg<br>10 mg<br>12 mg<br>15 mg | 15, 29 | CNS1/2 ONLY Note age-based dosing | f Peripheral blood for PK g Peripheral blood for Immunogenicity Optional studies |
| Intrathecal Triple Therapy (ITT): Methotrexate (MTX) Hydrocortisone (HC) Cytarabine (ARAC) | IT | Age (yrs) 1-1.99 2-2.99 3-8.99 ≥9 | Dose MTX:8mg, HC: 8mg, ARAC: 16mg MTX: 10mg HC: 10 mg ARAC: 20 mg MTX: 12 mg HC: 12 mg ARAC: 24 mg MTX: 15 mg HC: 15 mg ARAC: 30 mg | 15, 29 | CNS3 ONLY Note age-based dosing | h Blinatumomab PD 1 Obtain with each IT/ITT See Section 7.0 for further details. OBTAIN OTHER STUDIES AS REQUIRED FOR GOOD PATIENT CARE |
| Testicular Radiother<br>Section 14.2 for detail | | persistent testicular di | sease will receive testi | cular radia | tion during Blinatumomab Block – Cycle 1. See | |



| APPENDIX II-D Blinatumomab Block - Cycle 1 (HR/IR Patients in Arm B) | | |
|---|---|---|
| This therapy is the 1st cycle of therapy with blinatumomab for the HR/IR patients assigned to the experimental arm (Arm B) | Patient COG ID number | DOB |

| Ht | | cm | Wt | kg | BSA | $m^2$ | | | |
|---|---|---|---|---|---|---|---|---|---|
| Date Due | Date<br>Given | Day | BLIN | DEX | | IT MTX<br>CNS1/2 ONLY | ITT<br>CNS3 ONLY | Studies | Comments (Include any held doses, or dose modifications) |
| | | | mcg | mg | | mg | mg | | |
| | | | Enter calculated d | ose above and actu | al dose ad | lministered below | | • | |
| | | 1 | mcg | mg | | | | a*, b, e, h+,g\$ | |
| | | 2 | | | | | | f&,h+ | |
| | | 7 | | | | | | h+ | |
| | | 8 | | | | | | b, e, | |
| | | 14 | | | | | | f&, h+ | |
| | | 15 | | | | mg | mg | b, d, e | |
| | | 21 | | | | | | h+ | |
| | | 22 | . ↓ | | | | | b, e, | |
| | | 20 | , | | | | | | |
| | | 28 | | | | | | | |
| | | 29 | | | | mg | mg | b, c, d, e | |
| | | 30-35 | Rest Period | | | | | | |
| | | | Following cou<br>protocol therap | Following count recovery, start next cycle, Blinatumomab Block Cycle 2 (Section 4.6, APPENDIX II-E). Treatment failures will be taken off | | | | | |
| 1 Dania kas | al blaad | . D: 4- | | | II 12 | D 2 D 7 D | 14 D 21) £41 | -1:t1-:C | usion (saa Saation 12.5 for aamplata |

<sup>+</sup>**Peripheral blood:** Prior to (Hour 0) and during (Hour 6, Hour 12, Day 2, Day 7, Day 14, Day 21) first blinatumomab infusion (see Section 13.5 for complete details).

See Section 5.0 for Dose Modifications for Toxicities and Appendix I for Supportive Care Guidelines.

<sup>\$</sup> Prior to (Hour 0) first blinatumomab infusion (see Section 13.7 & lab manual for details)

<sup>&</sup>amp; See lab manual for collection and shipping details

<sup>\*</sup>See recommended vital sign monitoring for Blinatumomab blocks in Section 7.1e



# APPENDIX II-E Blinatumomab Block - Cycle 2 (HR/IR Patients in Arm B)

This therapy is the 2<sup>nd</sup> cycle of therapy with blinatumomab for the HR/IR patients assigned to the experimental arm (Arm B)

Patient COG ID number DOB

Blinatumomab Block-Cycle 2 lasts 5 weeks (35 Days) and begins when ANC ≥ 500/µL and platelets ≥ 50,000/µL. See Section 4.6 for treatment details. This Therapy Delivery Map is on one (1) page.

| DRUG | ROUTE | DOSAGE | DAYS | IMPORTANT NOTES | OBSERVATIONS |
|---|---|---|---|---|---|
| Blinatumomab (BLIN) Do not use commercial supply | IV | 15 micrograms/m²/day | 1-28 | | a Hx, PE [VS/Wt (BSA)] b CBC/diff/platelets c BM (Local evaluation & MRD) |
| Intrathecal Methotrexate (IT MTX) | IT | Age (yrs) Dose 1-1.99 8 mg 2-2.99 10 mg 3-8.99 12 mg ≥9 15 mg | 8, 29 | CNS1/2 ONLY Note age-based dosing | d CSF cell count, cytospin¹ e Bilirubin, ALT & creatinine, BUN f Peripheral blood for Immunogenicity |
| Intrathecal Triple Therapy (ITT): Methotrexate (MTX) Hydrocortisone (HC) Cytarabine (ARAC) | IT | Age (yrs) 1-1.99 Dose MTX:8mg, HC: 8mg, ARAC: 16mg 2-2.99 MTX: 10mg HC: 10 mg ARAC: 20 mg 3-8.99 MTX: 12 mg HC: 12 mg ARAC: 24 mg → MTX: 15 mg HC: 15 mg ARAC: 30 mg | 8, 29 | CNS3 ONLY Note age-based dosing | Obtain with each IT/ITT See Section 7.0 for further details. OBTAIN OTHER STUDIES AS REQUIRED FOR GOOD PATIENT CARE |

| Ht | cm | Wt | kg | BSA | m² |
|----|----|----|----|-----|----|
|----|----|----|----|-----|----|

| Date Due | Date | Day | BLIN | IT MTX | ITT | Studies | Comments (Include any held doses, or dose modifications) |
|---|---|---|---|---|---|---|---|
| | Given | | | CNS1/2 ONLY | CNS3 ONLY | | |
| | | | mcg | mg | mg | | |
| | | | Enter calculated | dose above and actu | al dose administered | below | |
| | | 1 | mcg | | | a*, b, e | |
| | | 8 | | mg | mg | b, d, e | |
| | | 15 | | | | | |
| | | 22 | | | | b, e | |
| | | 28 | <b>†</b> | | | | |
| | | 29 | | mg | mg | b, c, d, e,f <sup>\$</sup> | |
| | | 30-35 | Rest Period | | | | |
| | | | | Following count recovery, patients will proceed to HSCT (Section 4.9). See Section 4.10, Appendix II-H for suggested bridging therapy in the event that HSCT is delayed. Treatment failures will be taken off protocol therapy. | | | |

<sup>§</sup> In cases where blinatumomab treatment will not continue to Cycle 2, collect sample at end of Cycle 1. See Section 13.7 and lab manual for details

See Section 5.0 for Dose Modifications for Toxicities and Appendix I for Supportive Care Guidelines.



# APPENDIX II-F Blinatumomab-S: Cycle 1 (Treatment Failure)

This therapy is the 1<sup>st</sup> cycle of therapy with Salvage Therapy (Blinatumomab-S) for the HR/IR patients classified as treatment failures who have not previously had blinatumomab on study.

| - | |
|-----------------------|-----|
| Patient COG ID number | DOB |

Blinatumomab-S: Cycle 1 lasts 5 weeks (35 Days). See Section 4.7 for treatment details. This Therapy Delivery Map is on two (2) pages.

| DRUG | ROUTE | DOSAGE | DAYS | IMPORTANT NOTES | OBSERVATIONS |
|---|---|---|---|---|---|
| Blinatumomab (BLIN) Do not use commercial supply | IV | 5 micrograms/m²/day 15 micrograms/m²/day | 1-7<br>8-28 | | a Hx, PE [VS/Wt (BSA)] b CBC/diff/platelets c CSF cell count, cytospin <sup>1</sup> |
| Dexamethasone (DEX) | PO or IV | 5 mg/m <sup>2</sup> (max 20 mg) 30 to 60 minutes prior to the start of the Blinatumomab infusion | 1, 8 | Start prior to blinatumomab<br>therapy on Day 1 and prior to<br>step dose on Day 8. | d Bilirubin, ALT & creatinine, BUN e Local BM evaluation f BM for MRD- pre |
| Intrathecal<br>Methotrexate (IT<br>MTX) | IT | Age (yrs) Dose 1-1.99 8 mg 2-2.99 10 mg 3-8.99 12 mg ≥9 15 mg | 15 | Note age-based dosing | HSCT g Peripheral blood for PK h Peripheral blood for Immunogenicity Optional studies i Blinatumomab PD |
| | | | | | <sup>1</sup> Obtain with each IT/ITT |
| | | | | | See <u>Section 7.0</u> for further details. |
| | | | | | OBTAIN OTHER<br>STUDIES AS<br>REQUIRED FOR GOOD<br>PATIENT CARE |

**Testicular Radiotherapy:** Patients with persistent testicular disease will receive testicular radiation during the 1<sup>st</sup> cycle of Blinatumomab-S therapy. See Section 14.2 for details of TRT.



# APPENDIX II-F Blinatumomab-S: Cycle 1 (Treatment Failure)

This therapy is the 1<sup>st</sup> cycle of therapy with Salvage Therapy (Blinatumomab-S) for the HR/IR patients classified as treatment failures who have not previously had blinatumomab on study.

| Patient COG ID number | DOB |
|-----------------------|-----|

| Н | [t | _cm | Wt | kg | BSAr | $m^2$ | |
|---|---|---|---|---|---|---|---|
| Date<br>Due | Date<br>Given | Day | BLINmcg days 1-7 mcg days 8-28 | DEX<br>mg | IT MTXmg | Studies | Comments (Include any held doses, or dose modifications) |
| | | | | e and actual dose administered | below | | |
| | | 1 | mcg days 1-7 | mg | | a*, b, d, i+,h\$ | |
| | | 2 | | | | g& | |
| | | 3 | | | | | |
| | | 4 | | | | | |
| | | 5 | <u> </u> | | | | |
| | | 6 | <u> </u> | | | • | |
| | | / | 1 0.20 | | | 1 1 | |
| | | 8 | mcg days 8-28 | mg | | b, d | |
| | | 10 | <u> </u> | | | | |
| | | 14 | | | | b, c, d, g&, i <sup>+</sup> | |
| | | 15 | | | mg | 3, 3, 4, 8, 1 | |
| | | 16 | | | | | |
| | | 21 | | | | b, d, i <sup>+</sup> | |
| | | 22 | _ | | | | |
| | | 28 | + | | | | |
| | | 29 | D (D ) | | | b, d, e, f <sup>+++</sup> | |
| - | 1 | 30-35 | Rest Period | '. C | 0 4' 40) 4 Dl' 4 | 1 G. C1 2 (G | 4.0. ADDENDIV II. C) |
| + D . 1 | 111 | l D : | | eria for proceeding to HSCT ( | | | |

<sup>&</sup>lt;sup>+</sup> **Peripheral blood:** Prior to (Hour 0) and during (Hour 6, Hour 12, Day 2, Day 7, Day 14, Day 21) first blinatumomab infusion (see Section 13.5 for complete details).

See Section 5.0 for Dose Modifications for Toxicities and Appendix I for Supportive Care Guidelines.

<sup>\$</sup> Prior to (Hour 0) first blinatumomab infusion. In cases where blinatumomab treatment will not continue to Cycle 2, collect additional sample at end of Cycle 1. (see Section 13.7 and lab manual for details)

<sup>&</sup>amp; See lab manual for collection and shipping details

<sup>\*</sup>See recommended vital sign monitoring for Blinatumomab blocks in Section 7.1e

<sup>+++</sup> Pre-HSCT evaluation



# APPENDIX II-G Blinatumomab-S: Cycle 2 (Treatment failure)

This therapy is the 2<sup>nd</sup> cycle of therapy with Salvage Therapy (Blinatumomab-S) for the HR/IR patients classified as treatment failures who have not previously had blinatumomab on study.

| Patient COG ID number | DOB |
|-----------------------|-----|

Blinatumomab-S: Cycle 2 lasts 5 weeks (35 Days) and starts no earlier than Day 36 after the beginning of Blinatumomab-S: Cycle 1.. See Section 4.8 for treatment details. This Therapy Delivery Map is on two (2) pages.

| DRUG | ROUTE | DOSAGE | DAYS | IMPORTANT NOTES | OBSERVATIONS |
|---|---|---|---|---|---|
| Blinatumomab (BLIN) Do not use commercial supply Intrathecal | IV<br>IT | 15 micrograms/m²/day Age (vrs) Dose | 1-28<br>8, 29 | | a Hx, PE [VS/Wt (BSA)] b CBC/diff/platelets c Local BM evaluation d CSF cell count, cytospin <sup>1</sup> e Bilirubin, ALT & creatinine, BUN |
| Intrathecal Methotrexate (IT MTX) | | Age (yrs) Dose 1-1.99 8 mg 2-2.99 10 mg 3-8.99 12 mg ≥9 15 mg | 8, 29 | Note age-based dosing | f BM for MRD- pre HSCT g Peripheral blood for Immunogenicity 1 Obtain with each IT/ITT See Section 7.0 for further details. OBTAIN OTHER STUDIES AS REQUIRED FOR GOOD PATIENT CARE |



APPENDIX II-G Blinatumomab-S: Cycle 2 (Treatment failure)

This therapy is the  $2^{nd}$  cycle of therapy with Salvage Therapy (Blinatumomab-S) for the HR/IR patients classified as treatment failures who have not previously had blinatumomab on study.

| Patient COG ID number | DOB |
|-----------------------|-----|

| Ht | c | m | | Wt | kg | | BSA | $\mathbf{m}^2$ |
|---|---|---|---|---|---|---|---|---|
| | Date Due | Date | Day | BLIN | | IT MTX | Studies | Comments (Include any held doses, or dose modifications) |
| - 1 | | Given | | | | mg | | |
| | | | | mcg | | | | |
| | | | | Enter calculated | dose abo | ve and actual dose a | dministered belov | V |
| L | 1 | | mcg | | | a*, b, e | | |
| - [ | | | 8 | | | mg | b, d, e | |
| | | | 15 | | | | b, e | |
| Į | | | 22 | | | | b, e | |
| Ī | | | 29 | <b>V</b> | | mg | b, c, d, e,g\$,<br>f*** | |
| | | | 30-35 | Rest Period | | | | |
| | | | | See Section 4.8 | See Section 4.8.5 for criteria for proceeding to HSCT (Section 4.9) or to Bridging Maintenance Therapy Section 4.10, Appendix I | | | |
| | | | | Patients with M | 2/M3 ma | rrow after Blinatur | nomab-S: Cycle 2 | 2 will be taken off protocol therapy. |

In cases where blinatumomab treatment will not continue to Cycle 2, collect sample at end of Cycle 1. See Section 13.7 and lab manual for details \*See recommended vital sign monitoring for Blinatumomab blocks in Section 7.1e

See Section 5.0 for Dose Modifications for Toxicities and Appendix I for Supportive Care Guidelines.

<sup>+++</sup> Pre-HSCT evaluation



| Appendix II-H | Bridging Maintenance Therapy: Optional (HR/IR patients |
|----------------|--------------------------------------------------------|
| and TF patient | ts that are eligible for HSCT) |

Patient COG ID number DOB

This therapy is only for HR/IR patients awaiting stem cell transplant therapy due to stem cell source or facility scheduling issues causing a lag time > 2 weeks after count recovery. Bridging therapy can be given for a maximum of 6 weeks, but does not need to be given the full 6 weeks if patient is ready for HSCT earlier.

This therapy lasts for a maximum of 6 weeks (42 days) and starts when peripheral counts recover to ANC  $\geq 500/\mu$ L and platelets  $\geq 50~000/\mu$ L. See Section 4.10 for treatment details. This therapy delivery map is on one (1) page.

| DRUG | ROUTE | DOSAGE | DAYS | IMPORTANT NOTES | OBSERVATIONS |
|---|---|---|---|---|---|
| VinCRIStine (VCR) | IV push over 1 minute <sup>+</sup> | 1.5 mg/m²/dose | 1, 22 | + Or infusion via minibag as per institutional policy. Maximum dose: 2 mg | a Hx, PE [VS/Wt (BSA)] b CBC/diff/platelets c BM for MRD evaluation d BUN/creatinine e LFTs |
| Mercaptopurine (MP) | PO | 75 mg/m²/dose | 1-42 | | C LI 13 |
| Methotrexate (MTX) | PO | 20 mg/m²/dose | 1, 8, 15, 22, 29, 36 | | See <u>Section 7.1c</u> for Follow up observations. |

| Ht | :cm | | Wt | kg | BSA | m² | |
|---|---|---|---|---|---|---|---|
| Date Due | Date Given | Day | VCR<br>mg | MP<br>mg | PO MTX<br>mg | Studies | Comments (Include any held doses, or dose modifications) |
| | | | | | actual dose administe | ered below | , |
| | | 1 | mg | mg | mg | a, b, d,e | |
| | | 8 | | | mg | | |
| | | 15 | | | mg | | |
| | | 22 | mg | | mg | | |
| | | 29 | | | mg | | |
| | | 36 | | | mg | | |
| | | 42 | | <b>₩</b> | | | |
| | | 43 | | | | $c^1$ | |

Bone marrow for MRD evaluation must be repeated prior to the start of HSCT.

See Section 5.0 for Dose Modifications for Toxicities and Appendix I for Supportive Care Guidelines.

DOB



# APPENDIX II-I Continuation 1/2 (All LR patients)

This therapy is for all LR patients and is the same for Continuation 1 and Continuation 2.

Patient COG ID number

Continuation lasts 8 weeks and is given twice, for a total of 16 weeks. Begin when ANC  $\geq 500/\mu$ L and platelets  $\geq 50,000/\mu$ L. Await count recovery to ANC  $\geq 500/\mu$ L and platelets  $\geq 50,000/\mu$ L

| DRUG | ROUTE | UTE DOSAGE | | DAYS | IMPORTANT NOTES | OBSERVATIONS |
|---|---|---|---|---|---|---|
| Dexamethasone (DEX) | РО | 3 mg/m²/dose BID | | 1-5 | Total Daily Dose: 6 mg/m²/day, divided BID. | a Hx, PE [VS/Wt (BSA)] b CBC/diff/platelets c CSF cell count, cytospin <sup>1</sup> |
| VinCRIStine (VCR) | IV push over 1 minute <sup>+</sup> | 1.5 mg/m²/dose | | 1 | <sup>+</sup> Or infusion via minibag as per institutional policy Maximum dose: 2 mg | d Bilirubin, ALT & creatinine, BUN |
| Methotrexate (MTX) | PO | 20 mg/m²/dose | | 8, 15, 29, 36 | | |
| Intermediate Dose<br>Methotrexate (ID MTX) | IV over 36 hours | 1000 mg/m²/dose | | 22 | CNS3 ONLY | |
| Methotrexate (MTX) | PO | 25 mg/m²/dose Q6H | x 4 doses | 22 | CNS1/2 ONLY | Obtain with each IT/ITT |
| Mercaptopurine (MP) | PO | 75 mg/m²/dose daily | 7 | 1-42 | | See Section 7.0 for further details |
| Leucovorin (LCV) | IV/PO | 15 mg/m²/dose Q6H | | 24, 25 | CNS3 ONLY Begin 48 hrs after the START of ID MTX infusion. | details |
| Leucovorin (LCV) | PO | 10 mg/m <sup>2</sup> /dose Q6H | H x 2 | 24 | CNS1/2 ONLY Begin 48 hrs after the START of day 22 PO Methotrexate | OBTAIN OTHER STUDII |
| Cyclophosphamide (CPM) | IV over 15-30 minutes | 300 mg/m²/dose | | 43, 50 | See Section 4.11 and Appendix IV for administration | AS REQUIRED FOR GOOD<br>PATIENT CARE |
| Etoposide (ETOP) | IV over 60-120 minutes | 150 mg/m²/dose | | 43, 50 | guidelines. | |
| Thioguanine (TG) | PO | 40 mg/m²/dose | | 43-49 | | |
| Cytarabine (ARAC) | IV over 1 – 30 minutes or SQ | 50 mg/m²/dose | | 44-47, 51-54 | | |
| Intrathecal Methotrexate (IT MTX) | IT | Age (yrs) Dose<br>1-1.99<br>2-2.99<br>3-8.99<br>≥9 | 8 mg<br>10 mg<br>12 mg<br>15 mg | 1, 43 | CNS1/2 ONLY Note age-based dosing | |
| Intrathecal Triple Therapy<br>(ITT):<br>Methotrexate (MTX)<br>Hydrocortisone (HC)<br>Cytarabine (ARAC) | IT | Age (yrs)<br>1-1.99<br>2-2.99<br>3-8.99<br>≥9 | Dose<br>MTX:8mg,<br>HC: 8mg,<br>ARAC: 16mg<br>MTX: 10mg<br>HC: 10 mg<br>ARAC: 20 mg<br>MTX: 12 mg<br>HC: 12 mg<br>ARAC: 24 mg<br>MTX: 15 mg<br>HC: 15 mg<br>ARAC: 30 mg | 1, 43 | CNS3 ONLY Note age-based dosing | |



#### APPENDIX II-I Continuation 1/2 (All LR patients) This therapy is for all LR patients and is the same for Continuation 1 and Continuation 2. Patient COG ID number DOB Enter Cycle #: Ht Wt kg **BSA** $m^2$ cm DEX. MP VCR ID MTX LCV ETOP CPM TG Day PO PO MTX ARAC IT MTX ITT Studies Date Date Comments MTX CNS1/2 CNS3 CNS1/2 CNS3 \_mg (Include any held Due Given **ONLY ONLY ONLY** doses, or dose **ONLY** modifications) \_mg mg Enter calculated dose above and actual dose administered below 1 a, b, c,d mg mg mg mg mg 2 3 b,d 8 \_mg b,d 15 mg \_mg mg \_mg mg 24 mg 25 mg 29 b.d mg 36 \_mg b,d 42 43^ b, c,d mg mg mg mg mg 44 mg 47 49 50 b, d \_mg \_mg 51 \_mg 53 54 56 b,d

Following Continuation 1, upon count recovery, **LR patients randomized to Arm C** will receive Continuation 2 therapy (Section 4.11, APPENDIX II-I), **LR patients randomized to Arm D** will receive Blinatumomab Block: Cycle 2 therapy (Section 4.16, APPENDIX II-N),

Following Continuation 2, upon count recovery, LR patients randomized to Arm C will receive Maintenance Cycle 1 therapy (Section 4.12, Appendix II-J), LR patients randomized to Arm D will receive Blinatumomab Block: Cycle 3 therapy (Section 4.16, APPENDIX II-N),

<sup>^</sup> Await count recovery to ANC  $\geq 500/\mu$ L and platelets  $\geq 50,000/\mu$ L prior to beginning Day 22 and Day 43 therapy. See Section 4.11 for details See Section 5.0 for Dose Modifications for Toxicities and Appendix I for Supportive Care Guidelines.



Appendix II-J Maintenance Cycle 1 (All LR patients)
This Maintenance therapy is for all LR patients (Arm C and Arm D)

Patient COG ID number

DOB

Maintenance Cycle 1 lasts for 12 weeks (84 days) and starts when peripheral counts recover to ANC  $\geq 500/\mu$ L and platelets  $\geq 50~000/\mu$ L. See Section 4.12 for treatment details. This

therapy delivery map is for Maintenance and is on two (2) pages.

| DRUG | ROUTE | DOSAGE | | DAYS | IMPORTANT NOTES | OBSERVATIONS | | |
|---|---|---|---|---|---|---|---|---|
| Dexamethasone (DEX) | РО | 3 mg/m²/dose BID | | 3 mg/m²/dose BID | | 3 mg/m²/dose BID 1-5, 29-33, & 57-61 Total Daily Do | Total Daily Dose: 6 mg/m²/day, divided BID. | a Hx, PE [VS/Wt (BSA)] b CBC/diff/platelets c CSF cell count, cytospin <sup>1</sup> |
| VinCRIStine (VCR) | IV push over 1<br>minute <sup>+</sup> | 1.5 mg/m²/dose | | 1, 29, 57 | + Or infusion via minibag as per institutional policy. Maximum dose: 2 mg | d Bilirubin, ALT & creatinine, BUN e Absolute lymphocyte count with T and | | |
| Mercaptopurine (MP) | PO | 75 mg/m <sup>2</sup> /dose daily | | 1-84 | | B subset quantification. <sup>2</sup> | | |
| Methotrexate (MTX) | PO | 20 mg/m²/dose weekly | | 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, 78 | | f Peripheral blood for Immunogenicity | | |
| Intrathecal<br>Methotrexate (IT MTX) | IT | 2-2.99 1<br>3-8.99 1 | 3 mg<br>10 mg<br>12 mg<br>15 mg | 1 | CNS1/2 ONLY Note age-based dosing | <sup>1</sup> Obtain with each IT/ITT <sup>2</sup> To be done at the end of each 12 week maintenance cycle and every 3 months after completion of therapy for 1 year. | | |
| Intrathecal Triple Therapy (ITT): Methotrexate (MTX) | IT | 1-1.99 N | Dose<br>MTX:8mg,<br>HC: 8mg, | 1 | CNS3 ONLY | See Section 7.0 for further details. | | |
| Hydrocortisone (HC)<br>Cytarabine (ARAC) | | 2-2.99 M<br>H | ARAC: 16mg<br>MTX: 10mg<br>HC: 10 mg<br>ARAC: 20 mg | | Note age-based dosing | | | |
| | | H<br>A | MTX: 12 mg<br>HC: 12 mg<br>ARAC: 24 mg<br>MTX: 15 mg | | | | | |
| | | I | HC: 15 mg<br>ARAC: 30 mg | | | OBTAIN OTHER STUDIES AS<br>REQUIRED FOR GOOD PATIENT CAR | | |



Appendix II-J Maintenance Cycle 1 (All LR patients)
This Maintenance therapy is for all LR patients (Arm C and Arm D)

Patient COG ID number

DOB

| Ht | cm | | | Wt | kg | В | SA m <sup>2</sup> | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Date Due | Date<br>Given | Day | DEX. | VCR<br>mg | MP<br>mg | MTX<br>mg | IT MTX<br>CNS1/2 ONLY<br>mg | ITT CNS3 ONLYmg | Studies | Comments (Include any held doses, or dose modifications) |
| | | | | | above and ac | | | | | |
| | | 1 | mg | mg | mg | | mg | mg | a, b, c, d,f <sup>\$</sup> | |
| | | 2 | | | | | | | | |
| | | 3 | | | | | | | | |
| | | 5 | | | | | | | | |
| | | **** | * | | | | | | | |
| | | 8 | | | | mg | | | | |
| | | 15 | | | | mg | | | | |
| | | 22 | | | | mg | | | | |
| | | 29 | mg | mg | | mg | | | a, b, d | |
| | | 30 | | | | | | | | |
| | | 31 | | | | | | | | |
| | | 32 | | | | | | | | |
| | | 33 | * | | | | | | | |
| | | 36 | | | | mg | | | | |
| | | 43 | | | | mg | | | | |
| | | 50 | | | | mg | | | | |
| | | 57 | mg | mg | | mg | | | a, b, d | |
| | | 58 | | | | | | | | |
| | | 58 | | | | | | | | |
| | | 60 | | | | | | | | |
| | | 61 | * | | | | | | | |
| | | 64 | | | | mg | | | | |
| | | 71 | | | | mg | | | | |
| | | 78 | | | | mg | | | | |
| | | 84 | | | | | | | a, b, d, e | |
| | | 85 | Following N | I<br>Maintenance C | vcle 1 therapy. | CNS3 patients | ONLY will receive ( | L<br>CNS directed therapy with ch | | 4.13, APPENDIX II-K). All other |
| | | 00 | patients on A | Arm C and Ar | m D will contin | ue with Mainte | nance Post-Cycle 1 th | erapy (Section 4.14, APPEN | DIX II-L) | |

\$ Arm D ONLY. Prior to start of Maintenance therapy for eligible patients (see Section 13.7 and lab manual for details)

See Section 5.0 for Dose Modifications for Toxicities and Appendix I for Supportive Care Guidelines.



APPENDIX II-K Maintenance Chemoradiation-CNS Directed Therapy (LR Patients)

This therapy is for all CNS3 patients ONLY and is given between 1st and 2nd cycles of Maintenance therapy.

Patient COG ID number DOB

This CNS directed therapy lasts 3 weeks (21 days) and starts when ANC  $\geq 500/\mu$ L and platelets  $\geq 50,000/\mu$ L (whichever occurs later). See Section 4.13 for treatment details. This Therapy Delivery Map is on one (1) page

| DRUG | ROUTE | DOSAGE | DAYS | IMPORTANT NOTES | OBSERVATIONS |
|---|---|---|---|---|---|
| Dexamethasone (DEX) | PO | 5 mg/m²/dose BID | /dose BID 1-7, 15-21 Total Daily Dose: 10 mg/m²/day, divided BID. | | a Hx, PE [VS/Wt (BSA)] b CBC/diff/platelets |
| VinCRIStine (VCR) | IV push over 1 minute <sup>+</sup> | 1.5 mg/m²/dose 1, 8, 15 | | + Or infusion via minibag as per institutional policy | c Bilirubin, ALT & creatinine,<br>BUN |
| | | | | Maximum dose: 2 mg | See Section 7.0 for further details. |
| Pegaspargase (PEG-ASP) | egaspargase (PEG-ASP) IV over 1-2 hours 2500 International units/m²/dose 1 Administer through the tubing of a freely infusing solution of D5W or 0.9% NaCl | | | | |
| Cranial Radiotherapy: Pa<br>Section 14.1 for details of c | OBTAIN OTHER STUDIES AS REQUIRED FOR GOOD PATIENT CARE | | | | |

| Ente | er Cycle #: _ | | Ht_ | cm | Wtl | kg BS | Am <sup>2</sup> | |
|---|---|---|---|---|---|---|---|---|
| Date Due | Date<br>Given | Day | DEX.<br>mg | VCR<br>mg | PEG-ASP<br>IU | Studies | | Comments (Include any held doses, or dose modifications) |
| | | | | | Enter calcu | lated dose above | and actual dose admin | istered below |
| | | 1 | mg | mg | IU | a, b, c | | |
| | | 2 | 1 | | | | | |
| | | 3 | | | | | | |
| | | 4 | | | | | | |
| | | 5 | | | | | | |
| | | 6 | | | | | | |
| | | 7 | ▼ | | | | | |
| | | 8 | | mg | | | | |
| | | 15 | mg | mg | | | | |
| | | 16 | | | | | | |
| | | 17 | | | | | | |
| | | 18 | | | | | | |
| | | 19 | | | | | | |
| | | 20 | | | | | | |
| | | 21 | | | | | | |
| | | 22 | Following chem | oradiation, patients v | vill receive Maintena | nce Post-Cycle 1 | therapy (Section 4.14, A | PPENDIX II-L) when count parameters are met. |

See Section 5.0 for Dose Modifications for Toxicities and Appendix I for Supportive Care Guidelines.


| APPENDIX II-L Maintenance Post Cycle 1 (All LR patients) | | |
|---|---|---|
| THE EXPLICATION OF CYCLE I (I'M DIX patients) | Patient COG ID number | DOB |
| This therapy is for all LR patients (Arm C and Arm D) | | |

Maintenance Post Cycle 1 is given in 12 week cycles based on dose modifications for low counts and platelets. See Section 4.14 and Section 5.9 for details. This therapy delivery map is on two (2) pages.

| DRUG | ROUTE | DOSAGE | DAYS | IMPORTANT NOTES | OBSERVATIONS |
|---|---|---|---|---|---|
| Dexamethasone (DEX) | РО | 3 mg/m²/dose BID | 1-5, 29-33, & 57-61 | Total Daily Dose: 6 mg/m²/day, divided BID. | a Hx, PE [VS/Wt (BSA)] b CBC/diff/platelets c CSF cell count, cytospin <sup>1</sup> |
| VinCRIStine (VCR) | IV push over 1 minute <sup>+</sup> | 1.5 mg/m²/dose | 1, 29, 57 | + Or infusion via minibag as per institutional policy Maximum dose: 2 mg | d Bilirubin, ALT & Creatinine, BUN e Absolute lymphocyte count with T |
| Methotrexate (MTX) | PO | 20 mg/m²/dose | 1 | CNS3 ONLY | and B subset quantification <sup>2</sup> |
| Mercaptopurine (MP) | PO | 75 mg/m²/dose daily | 1-84 | | |
| Methotrexate (MTX) | PO | 20 mg/m²/dose weekly | 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, 78 | | <sup>1</sup> Obtain with each IT/ITT <sup>2</sup> To be done at the end of each 12 week |
| Intrathecal<br>Methotrexate (IT MTX) | IT | Age (yrs) Dose<br>1-1.99 8 mg | 1 | CNS1/2 ONLY | maintenance cycle and every 3 months after completion of therapy for 1 year. |
| | | 2-2.99 10 mg<br>3-8.99 12 mg<br>≥9 15 mg | | Note age-based dosing | See <u>Section 7.0</u> for further details. |
| | | | | | OBTAIN OTHER STUDIES AS |
| | | | | | REQUIRED FOR GOOD |
| | | | | | PATIENT CARE |



| APPENDIX II-L Maintenance Post Cycle 1 (All LR patients) | | |
|---|---|---|
| THE ENDING I E Maintenance 1 ost Cycle I (I'm Elk patients) | Patient COG ID number | DOB |
| This therapy is for all LR patients (Arm C and Arm D) | | |

| Cyc | cle # | | | Ht | cm | V | Vt | _kg | BSA | m² | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Date Due | Date<br>Given | Day | DEX. | VCR<br>mg | MTX (PO) CNS3 ONLY mg | MTX (PO)mg | MP<br>mg | IT MTX<br>CNS1/2 ONI<br>mg | | | Comments (Include any held doses, or dose modifications) |
| | | | | Enter o | calculated dose ab | ove and actua | l dose admin | istered below | | | |
| | | 1 | mg | mg | mg | | mg | mg | a, b, c, d | | |
| | | 3 | | | | | | | | | |
| | | 4 | | | | | | | | | |
| | | 5 | \ \ | | | | | | | | |
| | | 8 | | | | mg | | | | | |
| | | 15 | | | | mg | | | | | |
| | | 22 | | | | mg | | | | | |
| | | 29 | mg | mg | | mg | | | a, b, d | | |
| | | 30 | | | | | | | | | |
| | | 31 | | | | | | | | | |
| | | 32 | <b> </b> | | | | | | | | |
| | | 36 | • | | | mg | | | | | |
| | | 43 | | | | | | | | | |
| | | **** | | | | mg | | | | | |
| | | 50 | | | | mg | | | | | |
| | | 57<br>58 | mg | mg | | mg | | | a, b, d | | |
| | | 59 | | | | | | | | | |
| | | 60 | ] | | | | | | | | |
| | | 61 | * | | | | | | | | |
| | | 64 | | | | mg | | | | | |
| | | 71 | | | | mg | | | | | |
| | | 78 | | | | mg | | | | | |
| | | 84 | | | | | | | a, b, d, e | | |
| | | 85 | | nce cycles ar<br>female patie | | eek cycles base | d on dose mo | odifications for lov | v counts or low platel | ets until 2 yr | rs from start of Block 1 therapy for both |

See Section 5.0 for Dose Modifications for Toxicities and Appendix I for Supportive Care Guidelines.



| APPENDIX II-M Blinatumomab Block - Cycle 1 (LR Patients in Arm D) | | |
|---|---|---|
| This therapy is the 1st cycle of therapy with blinatumomab for the LR patients randomized to Arm D | Patient COG ID number | DOB |

This cycle lasts 5 weeks (35 days) and starts when peripheral counts recover to ANC  $\geq 500/\mu L$  and platelets  $\geq 50~000/\mu L$ . See Section 4.15 for treatment details. This Therapy Delivery Map is on two (2) pages.

| DRUG | ROUTE | DOSAGE | DAYS | IMPORTANT NOTES | OBSERVATIONS |
|---|---|---|---|---|---|
| Blinatumomab (BLIN) Do not use commercial supply | IV | 15 micrograms/m²/day | 1-28 | | a Hx, PE [VS/Wt (BSA)] b CBC/diff/platelets c CSF cell count, cytospin <sup>1</sup> |
| Dexamethasone (DEX) | PO or IV | 5 mg/m² (max 20 mg) 30 to 60 minutes prior to the start of the Blinatumomab infusion | 1 | Start prior to blinatumomab therapy | d Bilirubin, ALT & creatinine, BUN e Peripheral blood for PK |
| Intrathecal Methotrexate (IT MTX) | IT | Age (yrs) Dose<br>1-1.99 8 mg<br>2-2.99 10 mg<br>3-8.99 12 mg | 8, 29 | CNS1/2 ONLY Note age-based dosing | f Peripheral blood for Immunogenicity Optional studies |
| Intrathecal Triple Therapy (ITT): Methotrexate (MTX) Hydrocortisone (HC) Cytarabine (ARAC) | IT | ≥9 15 mg Age (yrs) Dose 1-1.99 MTX:8mg, HC: 8mg, ARAC: 16mg 2-2.99 MTX: 10mg HC: 10 mg ARAC: 20 mg 3-8.99 MTX: 12 mg HC: 12 mg ARAC: 24 mg MTX: 15 mg | 8, 29 | CNS3 ONLY Note age-based dosing | g Blinatumomab PD <sup>1</sup> Obtain with each IT/ITT See Section 7.0 for further details. |
| | | ≥9 MTX: 15 mg<br>HC: 15 mg<br>ARAC: 30 mg | | | OBTAIN OTHER STUDIES AS<br>REQUIRED FOR GOOD PATIENT<br>CARE |
| Testicular Radiothera | y: Patients with persis | stent testicular disease will receive testicular radia | ition.See S | Section 14.2 for details of TRT. | |



APPENDIX II-M Blinatumomab Block - Cycle 1 (LR Patients in Arm D)

This therapy is the 1st cycle of therapy with blinatumomab for the LR patients randomized to Arm D

Patient COG ID number DOB

| Ht | cr | n | Wtl | κg | BSA | m² | | | |
|---|---|---|---|---|---|---|---|---|---|
| Date Due | Date<br>Given | Day | BLIN<br>mcg | | DEX<br>mg | IT MTX CNS1/2<br>ONLY | ITT CNS3 ONLY<br>mg | Studies | Comments (Include any held doses, or dose modifications) |
| | 01,011 | | | | ms | mg | | | incumons) |
| | | | | | | Enter calculated | dose above and actua | al dose administered below | ý. |
| | | 1 | mcg | | mg | | | a*, b, d, g <sup>+</sup> ,f <sup>\$</sup> | |
| | | 2 | | | | | | e& g+ | |
| | | 7 | | | | | | $g^+$ | |
| | | 8 | | | | mg | mg | b, c, d, | |
| | | 14 | | | | | | e& g+ | |
| | | 15 | | | | | | b, d | |
| | | 21 | | | | | | g <sup>+</sup> | |
| | | 22 | | | | | | b, d | |
| | | 28 | | | | | | | |
| | | 29 | | | | mg | mg | b, c, d | |
| | | 30-35 | Rest Period | Rest Period | | | | | |
| | | 36 | Following Blina | ollowing Blinatumomab Block: Cycle 1, patients receive Continuation 1 therapy (Section 4.11, APPENDIX II-I) when count parameters are | | | | | |
| | | | met. | | | | | | |

<sup>&</sup>lt;sup>+</sup> **Peripheral blood:** Prior to (Hour 0) and during (Hour 6, Hour 12, Day 2, Day 7, Day 14, Day 21) first blinatumomab infusion (see Section 13.5 for complete details). \$ Prior to (Hour 0) first blinatumomab infusion (see Section 13.7 and lab manual for details)

<sup>&</sup>amp; See lab manual for details

<sup>\*</sup>See recommended vital sign monitoring for Blinatumomab blocks in Section 7.1e

See Section 5.0 for Dose Modifications for Toxicities and Appendix I for Supportive Care Guidelines.



# APPENDIX II-N Blinatumomab Block - Cycle 2 and 3 (LR Patients in Arm D)

This therapy is Cycles 2 and 3 of therapy with blinatumomab for the LR patients randomized to Arm D

Patient COG ID number DOB

Blinatumomab Block: Cycles 2 & 3; each last 5 weeks (35 days) and starts when peripheral counts recover to ANC  $\geq 500/\mu L$  and platelets  $\geq 50,000/\mu L$ . See Section 4.16 for treatment details.

This Therapy Delivery Map is on one (1) page.

| DRUG | ROUTE | DOSAGE | DAYS | IMPORTANT NOTES | OBSERVATIONS |
|---|---|---|---|---|---|
| Blinatumomab (BLIN) Do not use commercial supply | IV | 15 micrograms/m²/day | 1-28 | | a Hx, PE [VS/Wt (BSA)] b CBC/diff/platelets c Bilirubin, ALT & creatinine, BUN d Peripheral blood for Immunogenicity See Section 7.0 for further details. OBTAIN OTHER STUDIES AS REQUIRED FOR GOOD PATIENT CARE |

Enter Cycle #\_\_\_\_\_ kg BSA \_\_\_\_\_ m<sup>2</sup>

| Date Due | Date<br>Given | Day | BLIN | Studies | Comments (Include any held doses, or dose modifications) |
|---|---|---|---|---|---|
| | | | mcg | | |
| | | | Enter calculated d | lose above and act | ual dose administered below |
| | | 1 | mcg | a*, b, c | |
| | | 8 | | b, c | |
| | | 15 | | b, c | |
| | | 22 | | b, c | |
| | | 28 | <b>†</b> | | |
| | | 29 | | b, c,d <sup>\$</sup> | |
| | | 30-35 | Rest Period | | |
| | | 36 | Following Blinatumomab Block Cycle 2: LR B-ALL patients randomized to <b>Arm D</b> will receive Continuation 2 (Section 4.11, APPENDIX II-I) when count parameters are met. Following Blinatumomab Block Cycle 3: LR B-ALL patients randomized to <b>Arm D</b> will receive Maintenance Cycle 1 therapy-(Section 4.12, Appendix II-J) when count parameters are met. | | |

Sobtain at End Cycle 2. In cases where blinatumomab treatment will not continue to Cycle 2, collect sample at end of Cycle 1. See Section 13.7 and lab manual for details

See Section 5.0 for Dose Modifications for Toxicities and Appendix I for Supportive Care Guidelines.

<sup>\*</sup>See recommended vital sign monitoring for Blinatumomab blocks in <u>Section 7.1e</u>



# APPENDIX III: MERCAPTOPURINE DOSING GUIDELINES

# MERCAPTOPURINE 75 mg/m<sup>2</sup>

Note: The Mercaptopurine dosing nomograms in this appendix only apply to the tablet formulation.

| Body Surface Area (m²)* | Daily Dose (d) for 7 days<br>(1 tablet = 50 mg) | Cumulative Weekly Dose |
|---|---|---|
| 0.36 - 0.40 | ½ tab / d x 6; 1 tab / d x 1 | 200 mg/wk |
| 0.41 - 0.45 | ½ tab / d x 5; 1 tab / d x 2 | 225 mg/wk |
| 0.46 - 0.49 | ½ tab / d x 4; 1 tab / d x 3 | 250 mg/wk |
| 0.50 - 0.54 | 1 tab / d x 4; ½ tab / d x 3 | 275 mg/wk |
| 0.55 - 0.59 | 1 tab / d x 5; ½ tab / d x 2 | 300 mg/wk |
| 0.60 - 0.64 | 1 tab / d x 6; ½ tab / d x 1 | 325 mg/wk |
| 0.65 - 0.69 | 1 tab / day | 350 mg/wk |
| 0.70 - 0.73 | 1 tab / d x 6; 1½ tab / d x 1 | 375 mg/wk |
| 0.74 - 0.78 | 1 tab / d x 5; 1½ tab / d x 2 | 400 mg/wk |
| 0.79 - 0.83 | 1 tab / d x 4; 1½ tab / d x 3 | 425 mg/wk |
| 0.84 - 0.88 | 1½ tab / d x 4; 1 tab / d x 3 | 450 mg/wk |
| 0.89 - 0.92 | 1½ tab / d x 5; 1 tab / d x 2 | 475 mg/wk |
| 0.93 - 0.97 | 1½ tab / d x 6; 1 tab /d x 1 | 500 mg/wk |
| 0.98 - 1.02 | 1½ tab / day | 525 mg/wk |
| 1.03 - 1.07 | 1½ tab / d x 6; 2 tab / d x 1 | 550 mg/wk |
| 1.08 - 1.11 | 1½ tab / d x 5; 2 tab / d x 2 | 575 mg/wk |
| 1.12 - 1.16 | 1½ tab / d x 4; 2 tab / d x 3 | 600 mg/wk |
| 1.17 - 1.21 | 2 tab / d x 4; 1½ tab / d x 3 | 625 mg/wk |
| 1.22 - 1.26 | 2 tab / d x 5; 1½ tab / d x 2 | 650 mg/wk |
| 1.27 - 1.30 | 2 tab / d x 6; 1½ tab / d x 1 | 675 mg/wk |
| 1.31 - 1.35 | 2 tab / day | 700 mg/wk |
| 1.36 - 1.40 | 2 tab / d x 6; 2½ tab / d x 1 | 725 mg/wk |
| 1.41 - 1.45 | 2 tab / d x 5; 2½ tab / d x 2 | 750 mg/wk |
| 1.46 - 1.49 | 2 tab / d x 4; 2½ tab / d x 3 | 775 mg/wk |
| 1.50 - 1.54 | 2½ tab/ d x 4; 2 tab / d x 3 | 800 mg/wk |
| 1.55 - 1.59 | 2½ tab/ d x 5; 2 tab / d x 2 | 825 mg/wk |
| 1.60 - 1.64 | 2½ tab/ d x 6; 2 tab / d x 1 | 850 mg/wk |
| 1.65 - 1.69 | 2½ tab/ d | 875 mg/wk |
| 1.70 - 1.73 | 2½ tab/ d x 6; 3 tab / d x 1 | 900 mg/wk |
| 1.74 - 1.78 | 2½ tab/ d x 5; 3 tab / d x 2 | 925 mg/wk |
| 1.79 - 1.83 | 2½ tab/ d x 4; 3 tab / d x 3 | 950 mg/wk |
| 1.84 - 1.88 | 3 tab/ d x 4; 2½ tab / d x 3 | 975 mg/wk |
| 1.89 - 1.92 | 3 tab/ d x 5; 2½ tab / d x 2 | 1000 mg/wk |
| 1.93 - 1.97 | 3 tab/ d x 6; 2½ tab / d x 1 | 1025 mg/wk |
| 1.98 - 2.02 | 3 tab/ d x 7 | 1050 mg/wk |



| 2.03 - 2.07 | 3 tab/ d x 6; 3½ tab / d x 1 | 1075 mg/wk |
|-------------|------------------------------|------------|
| 2.08 - 2.11 | 3 tab/ d x 5; 3½ tab / d x 2 | 1100 mg/wk |
| 2.12 - 2.16 | 3 tab/ d x 4; 3½ tab / d x 3 | 1125 mg/wk |
| 2.17 - 2.21 | 3½ tab/ d x 4; 3 tab / d x 3 | 1150 mg/wk |
| 2.22 - 2.26 | 3½ tab/ d x 5; 3 tab / d x 2 | 1175 mg/wk |
| 2.27 - 2.30 | 3½ tab/ d x 6; 3 tab / d x 1 | 1200 mg/wk |
| 2.31 - 2.35 | 3½ tab/ d x 7 | 1225 mg/wk |
| 2.36 - 2.40 | 3½ tab/ d x 6; 4 tab / d x 1 | 1250 mg/wk |
| 2.41 - 2.45 | 3½ tab/ d x 5; 4 tab / d x 2 | 1275 mg/wk |
| 2.46 - 2.49 | 3½ tab/ d x 4; 4 tab / d x 3 | 1300 mg/wk |
| 2.50 - 2.54 | 4 tab/ d x 4; 3½ tab / d x 3 | 1325 mg/wk |
| 2.55 - 2.59 | 4 tab/ d x 5; 3½ tab / d x 2 | 1350 mg/wk |
| 2.60 - 2.64 | 4 tab/ d x 6; 3½ tab / d x 1 | 1375 mg/wk |
| 2.65 - 2.69 | 4 tab/ d x 7 | 1400 mg/wk |
| 2.70 - 2.73 | 4 tab/ d x 6; 4½ tab / d x 1 | 1425 mg/wk |
| 2.74 - 2.78 | 4 tab/ d x 5; 4½ tab / d x 2 | 1450 mg/wk |
| 2.79 - 2.83 | 4 tab/ d x 4; 4½ tab / d x 3 | 1475 mg/wk |
| 2.84 - 2.88 | 4½ tab/ d x 4; 4 tab / d x 3 | 1500 mg/wk |
| 2.89 - 2.92 | 4½ tab/ d x 5; 4 tab / d x 2 | 1525 mg/wk |
| 2.93 - 2.97 | 4½ tab/ d x 6; 4 tab / d x 1 | 1550 mg/wk |
| 2.98 - 3.00 | 4½ tab/ d x 7 | 1575 mg/wk |

<sup>\*</sup>Patients exceeding a BSA of 3.00 m² should have their MP doses calculated on actual BSA with no maximum dose.



# APPENDIX IV: THIOGUANINE DOSING GUIDELINES

# THIOGUANINE 40 mg/m<sup>2</sup>

\*Patients exceeding a BSA of 3 m² should have their TG doses calculated on actual BSA with no maximum dose.

| <b>Body Surface Area</b> | Daily Dose (d) for 7 days | Cumulative Weekly |
|---|---|---|
| (m <sup>2</sup> )* | (1 tablet = 40 mg) | Dose |
| 0.27 - 0.3 | Use oral compounded suspension | |
| 0.31 - 0.34 | Use oral compounded suspension | |
| 0.35 - 0.38 | Use oral compounded suspension | |
| 0.39 - 0.41 | Use oral compounded suspension | |
| 0.42 - 0.45 | Use oral compounded suspension | |
| 0.46 - 0.48 | Use oral compounded suspension | |
| 0.49 - 0.54 | ½ tab / d x 7 | 140 mg/wk |
| 0.55 - 0.61 | ½ tab / d x 6; 1 tab / d x 1 | 160 mg/wk |
| 0.62 - 0.68 | ½ tab / d x 5; 1 tab / d x 2 | 180 mg/wk |
| 0.69 - 0.75 | ½ tab / d x 4; 1 tab / d x 3 | 200 mg/wk |
| 0.76 - 0.82 | 1 tab / d x 4; ½ tab / d x 3 | 220 mg/wk |
| 0.83 - 0.89 | 1 tab / d x 5; ½ tab / d x 2 | 240 mg/wk |
| 0.9 - 0.96 | 1 tab / d x 6; ½ tab / d x 1 | 260 mg/wk |
| 0.97 - 1.04 | 1 tab / d x 7 | 280 mg/wk |
| 1.05 - 1.11 | 1 tab / d x 6; 1½ tab / d x 1 | 300 mg/wk |
| 1.12 - 1.18 | 1 tab / d x 5; 1½ tab / d x 2 | 320 mg/wk |
| 1.19 - 1.25 | 1 tab/ d x 4; 1½ tab / d x 3 | 340 mg/wk |
| 1.26 - 1.32 | 1½ tab / d x 4; 1 tab / d x 3 | 360 mg/wk |
| 1.33 - 1.39 | 1½ tab / d x 5; 1 tab /d x 2 | 380 mg/wk |
| 1.4 - 1.46 | 1½ tab / d x 6; 1 tab / d x 1 | 400 mg/wk |
| 1.47 - 1.54 | 1½ tab /day | 420 mg/wk |
| 1.55 - 1.61 | 1½ tab / d x 6; 2 tab / d x 1 | 440 mg/wk |
| 1.62 - 1.68 | 1½ tab / d x 5; 2 tab / d x 2 | 460 mg/wk |
| 1.69 - 1.75 | 1½ tab / d x 4; 2 tab / d x 3 | 480 mg/wk |
| 1.76 - 1.82 | 2 tab / d x 4; 1½ tab / d x 3 | 500 mg/wk |
| 1.83 - 1.89 | 2 tab / d x 5; 1½ tab / d x 2 | 520 mg/wk |
| 1.9 - 1.96 | 2 tab / d x 6; 1½ tab / d x 1 | 540 mg/wk |
| 1.97 - 2.04 | 2 tab / day | 560 mg/wk |
| 2.05 - 2.11 | 2 tab / d x 6; 2½ tab / d x 1 | 580 mg/wk |
| 2.12 - 2.18 | 2 tab / d x 5; 2½ tab / d x 2 | 600 mg/wk |
| 2.19 – 2.25 | 2 tab / d x 4; 2½ tab / d x 3 | 620 mg/wk |
| 2.26 - 2.32 | 2½ tab / d x 4; 2 tab / d x 3 | 640 mg/wk |
| 2.33 - 2.39 | 2½ tab / d x 5; 2 tab / d x 2 | 660 mg/wk |
| 2.4 - 2.46 | 2½ tab / d x 6; 2 tab / d x 1 | 680 mg/wk |
| 2.47 - 2.54 | 2½ tab / d | 700 mg/wk |
| 2.55 - 2.61 | 2½ tab / d x 6; 3 tab / d x 1 | 720 mg/wk |
| 2.62 - 2.68 | 2½ tab / d x 5; 3 tab / d x 2 | 740 mg/wk |
| 2.69 - 2.75 | 2½ tab / d x 4; 3 tab / d x 3 | 760 mg/wk |
| 2.76 - 2.82 | 3 tab / d x 4; 2½ tab / d x 3 | 780 mg/wk |
| 2.83 - 2.89 | 3 tab / d x 5; 2½ tab / d x 2 | 800 mg/wk |
| 2.9 – 2.96 | 3 tab / d x 6; 2½ tab / d x 1 | 820 mg/wk |
| 2.97 - 3 | 3 tab / d x 7 | 840 mg/wk |



#### APPENDIX V: YOUTH INFORMATION SHEETS

# INFORMATION SHEET REGARDING RESEARCH STUDY (for children from 7 through 12 years of age)

# A trial to compare 2 ways to treat children with B-Lymphoblastic Leukemia (B-ALL) that has come back (relapsed) after the first treatment

- 1. We have been talking with you about your illness, B-ALL. You have received treatment for this B-ALL before. After doing tests, we have found that the cancer has come back in your bone marrow, brain or spinal cord, or testes. B-ALL that has come back after the first treatment is called relapse.
- 2. We are asking you to take part in a research study because you have B-ALL that has relapsed. A research study is when doctors work together to try out new ways to help people who are sick. In this study we are trying to learn more about how to treat B-ALL when it has come back after the first time it was treated. During this study, we want to test whether the relapsed B-ALL responds better to combination chemotherapy or a new drug called blinatumomab. The treatment that you get will depend on a process called random assignment. Random assignment is a lot like flipping a coin and you will have an equal chance of getting both treatment options.
- 3. Children and teens who are part of this study will be treated with either combination chemotherapy or a new drug called blinatumomab. It is possible that some children will get radiation to their brain or testes, depending on where the leukemia is found. Some children will also get a stem cell transplant.
- 4. Sometimes good things can happen to people when they are in a research study. These good things are called "benefits." We hope that a benefit to you of being part of this study is having the leukemia go away for as long as possible. But we don't know for sure if there is any benefit of being part of this study.
- 5. Sometimes bad things can happen to people when they are in a research study. These bad things are called "risks." The risks to you from this study are that you might experience more side effects from the combination chemotherapy or blinatumomab. Another risk is that the therapy on this study might not be as effective as other options. Other things may happen to you that we don't yet know about.
- 6. Your family can choose to be part of this study or not. Your family can also decide to stop being in this study at any time once you start. There may be other treatments for your illness that your doctor can tell you about. Make sure to ask your doctors any questions that you have.
- 7. We are asking your permission to collect additional blood and bone marrow. We want to see if there are ways to tell how the cancer will respond to treatment. These samples would be taken when other standard tests are being performed, so there would be no extra procedures. You can still be treated on this study even if you don't allow us to collect the extra blood samples for research.



# INFORMATION SHEET REGARDING RESEARCH STUDY (for teens from 13 through 17 years of age)

# A trial to compare 2 ways to treat children with B-Lymphoblastic Leukemia (B-ALL) that has come back (relapsed) after the first treatment

- 1. We have been talking with you about your illness, B-ALL. You have received treatment for this B-ALL before. After doing tests, we have found that the cancer has come back in your bone marrow, brain or spinal cord, or testes. B-ALL that has come back after the first treatment is called relapse.
- 2. We are asking you to take part in a research study because you have B-ALL that has relapsed. A research study is when doctors work together to try out new ways to help people who are sick. In this study we are trying to learn more about how to treat B-ALL when it has come back after the first time it was treated. During this study, we want to test whether the relapsed B-ALL responds better to combination chemotherapy or a new drug called blinatumomab. The treatment that you get will depend on a process called random assignment. Random assignment is a lot like flipping a coin and you will have an equal chance of getting both treatment options.
- 3. Children and teens who are part of this study will be treated with either combination chemotherapy or a new drug called blinatumomab. It is possible that some children will get radiation to their brain or testes, depending on where the leukemia is found. Some children will also get a stem cell transplant.
- 4. Sometimes good things can happen to people when they are in a research study. These good things are called "benefits." We hope that a benefit to you of being part of this study is having the leukemia go away for as long as possible. But we don't know for sure if there is any benefit of being part of this study.
- 5. Sometimes bad things can happen to people when they are in a research study. These bad things are called "risks." The risks to you from this study are that you might experience more side effects from the combination chemotherapy or blinatumomab. Another risk is that the therapy on this study might not be as effective as other options. Other things may happen to you that we don't yet know about.
- 6. Your family can choose to be part of this study or not. Your family can also decide to stop being in this study at any time once you start. There may be other treatments for your illness that your doctor can tell you about. Make sure to ask your doctors any questions that you have.
- 7. We are asking your permission to collect additional blood and bone marrow. We want to see if there are ways to tell how the cancer will respond to treatment. These samples would be taken when other standard tests are being performed, so there would be no extra procedures. You can still be treated on this study even if you don't allow us to collect the extra samples for research.



# APPENDIX VI: ADDITIONAL INFORMATION FOR BANKING FOR FUTURE RESEARCH CORRELATIVE BIOLOGY STUDY

### a) Rationale

The ability to collect leukemic and normal tissue samples for future research, and to link these samples to patient characteristics and outcomes, has been critical to recent seminal discoveries regarding the molecular basis of de novo ALL and relapsed ALL, and the relationship of specific molecular lesions with outcomes and response to targeted therapies. In the context of this protocol, we will seek consent from participants to provide material for banking for the purpose of performing retrospective studies to refine risk stratification, identify new targets for therapy, identify biomarkers to predict response, and to link host polymorphisms with various disease characteristics and toxicities.

# b) Aims and methods

These studies will be performed as stand-alone biology studies subject to review and approval in accordance with the NCTN policies. The following are general descriptions of the types of studies planned.

# • Leukemia genomic studies

Modern genomic studies of high risk ALL have identified novel genetic alterations in ALL that are associated with treatment failure. In particular, high frequencies of mutations have been described in genes involved in B lymphocyte development (*EBF1*, *IKZF1*, *PAX5*) and signaling (*BTLA*, *CD200*, *RAS*) and in cell cycle regulation (*CDKN2A/B*, *RB*, *TP53*). Limited genomic analyses of paired diagnosis and relapse ALL samples have also shed light upon the early origin and clonal nature of such leukemia-associated mutations. Other yet-undiscovered mutations likely contribute the pathogenesis of this heterogeneous group of malignancies, and comprehensive prospective evaluation of the genetic landscape of relapsed ALL has not been performed. We hypothesize that integration of genomic profiling data will provide important insights regarding the molecular pathogenesis of relapsed ALL and may identify potential therapeutic targets or identify novel mechanisms of resistance within the context of the agents employed. Total context of the agents employed.

We hypothesize that high-throughput genome-wide profiling via multiple non-overlapping techniques provide a comprehensive genetic and epigenetic "fingerprint" and will identify key alterations that contribute to the pathogenesis and progression of relapsed ALL. We further hypothesize that integration of these approaches will allow discovery of alterations that may also be present in *de novo* ALL and could ultimately be used for initial risk stratification and new treatment approaches.

Consenting patients will submit bone marrow and/or peripheral blood samples at study entry and, if applicable, at second relapse to the central COG Tissue Bank at Nationwide Children's Hospital for storage of viably cryopreserved cells and for isolation nucleic acids, including DNA and RNA. Nucleic acids isolated from relapse specimens will be stored for potential use for genomic profiling, which will include single nucleotide polymorphism (SNP) arrays, array-based gene expression profiles and/or quantitative RT-PCR-based gene expression analyses, methylation arrays, and/or comprehensive sequencing approaches (e.g., RNA-seq, whole exome sequencing), depending on currently available technologies and funding sources. Banked specimens subsequently will be distributed from the reference laboratories to the laboratories performing the individual correlative biology studies. Results from these correlative biology studies may ultimately facilitate (a) enhanced refinement of risk stratification for patients with relapsed ALL, (b) detection of previously-unsuspected subset specificity of blinatumomab, and (c) generation of additional hypotheses with respect to the underlying biology of relapsed ALL.



#### • Host polymorphism studies

There is substantial evidence that both inherited germline constitutional and somatically-acquired ALL-specific genomic variation may contribute to variations in response. Plood samples obtained during remission are requested specifically for the purpose of providing constitutional (germline) DNA from each patient. Several efforts are anticipated for study of how genomic variation (SNPs, copy number variations, DNA methylation and insertions/deletions) in the constitutional DNA may be associated with phenotypes in ALL. The phenotypes could include those related to probability of cure, response, adverse events or classification. Techniques for interrogation of DNA variation are constantly evolving, and thus these techniques vary but may include candidate polymorphism testing (eg, via Taqman, GoldenGate, or PCR/RFLP assays), candidate gene sequencing (eg, via next-generation technologies coupled with exon capture) or whole-genome sequencing (eg, via next-generation technologies, with or without capture).

#### • MRD by next generation sequencing (NGS)

Next-generation sequencing (NGS) offers the potential for highly sensitive and standardized detection of minimal residual disease (MRD) in ALL. In comparison to current PCR methods, NGS assays do not require the laborious generation and validation of patient-specific primers, resulting in improved turn-around time and reduced cost, and may provide improved specificity by direct enumeration of leukemia-derived sequences. Current flow cytometric methods for MRD detection rely on relatively subjective assessments by trained interpreters and are about 1 log less sensitive than PCR-based methods. To determine the suitability of NGS methods for routine MRD assessment in a clinical trial setting, we will sequence the variable regions of IGH in pretreatment and post-treatment samples. Both the presence and the frequency of the MRD clone relative to the total IGH repertoire will be noted.



# APPENDIX VII-A: CLINICAL SITE MANAGEMENT OF OUT-PATIENT TREATMENT USING CTEP-SUPPLIED BLINATUMOMAB

- PREPARED IV INFUSION BAGS MAY NOT BE CHANGED BY THE STUDY SUBJECT
- PREPARED INFUSION BAGS OR INTACT VIALS MUST NOT BE TRANSPORTED TO ANOTHER LOCATION BY THE STUDY SUBJECT

#### AGENT PREPARATION AND ADMINISTRATION OPTIONS

- Prepare all out-patient infusion bags at the registering/treating NCTN Network institution. Study subjects should return to the registering/treating institution for all infusion bag changes.
- For study subjects that cannot return to the registering/treating institution for infusion bag exchanges, the next preference would be for another NCTN Network institution that is participating on the trial and is closer to the subject's home take over responsibility for the study subject's protocol participation. In such cases, transfer of the subject's protocol registration to another participating investigator and institution should be considered.
- If transferring the subject's protocol registration to another participating investigator and trial site within the NCTN Network is not feasible, use of a local outpatient infusion center could be considered.
  - a. First preference would be for all infusion bags to be prepared by the registering/treating institution and shipped via overnight courier delivery service in a 2° to 8°C pre-qualified shipping container to the local out-patient infusion center.
  - b. The prepared infusion bags are stored at the local outpatient infusion center. The infusion center would perform each infusion bag change.
  - c. If the local outpatient infusion center will not administer prepared infusion bags admixed by the registering/treating institution, the registering/treating institution may provide intact vials of blinatumomab to the local outpatient infusion center, with infusion bags prepared and administered by the local outpatient infusion center staff.
  - d. In either case, the local outpatient infusion center would be managed as a satellite pharmacy of the registering/treating institution (see evaluation criteria below).
  - e. If physical transport of intact vials of blinatumomab from the registering/treating institution to the local infusion center by registering/treating institution or local infusion center staff is not possible, CTEP will allow shipment of the vials from the registering/treating institution to the local infusion center via overnight courier delivery service in a 2° to 8°C pre-qualified shipping container.
- If an outpatient infusion center is not an option, use of a **home health care service** provider can be considered.

Note: If a home health care agency is being considered to prepare and change the blinatumomab infusion bag, the drug company that provides blinatumomab will cover the costs associated with a home health care agency providing these services.



- a. The first preference would be for all outpatient infusion bags to be prepared by the registering/treating institution and shipped via overnight courier delivery service in a 2° to 8°C pre-qualified shipping container to the servicing home health care agency.
- b. The prepared infusion bags are stored by the home health care agency and each individual infusion bag transported to the subject's home by the home health care service nursing staff under refrigerated storage conditions for each infusion bag change.
- c. If home health care agency will not administer prepared infusion bags admixed by the registering/treating institution, the registering/treating institution may provide intact vials of blinatumomab to the home health care agency, with infusion bags prepared and administered by the home health care agency staff.
- d. In either case, the home health care agency would be managed as a satellite pharmacy of the registering/treating institution (see evaluation criteria below).
- e. If physical transport of intact vials of blinatumomab from the registering/treating institution to the home health care agency by registering/treating institution or home health care agency staff is not possible, CTEP will allow shipment of the vials from the registering/treating institution to the home health care agency via overnight courier delivery service in a 2° to 8°C pre-qualified shipping container.
- 5. If all options above are not feasible, shipping the prepared infusion bags directly to patient's home via overnight courier delivery service for administration by home healthcare agency staff is acceptable.
  - a. The prepared infusion bags are to be shipped in a 2° to 8°C pre-qualified shipping container containing one infusion bag per box. Example 1, if you are making 2 x 48 hour infusion bags, each infusion bag will be shipped in a separate 2° to 8°C pre-qualified shipping container. Example 2, if you are making a 2 x 96 hour infusion bags, each infusion bag will be shipped in a separate 2° to 8°C pre-qualified shipping container. The infusion of the 2<sup>nd</sup> 96 hour bag must be completed within 8 days (192 hrs) of preparation to avoid exceeding the expiration date. The number of infusion bags that may be prepared and shipped is dependent on the duration the shipping container used is qualified to maintain 2° to 8°C temperature.
  - b. Patients should NOT open the shipping container upon arrival. Shipping containers are to be stored in a secured area away from reach of children or pets.
  - c. Shipping containers must only be opened by the home health care service staff at the time of the infusion bag change. Only one shipping container should be opened at a time. If cold-chain management of the prepared infusion bag has been interrupted by opening of the shipping container or storage of the prepared infusion bag in the shipping container exceeds the duration of the qualified time the container will maintain 2° to 8°C temperature, the infusion bag should not be used.



The home health care service staff should immediately contact the registering/treating institution site pharmacy as indicated on the shipment form. Within 1 business day, the registering/treating institution site should send an email to the COG Industry Sponsored Trials office at <a href="mailto:istprogram@childrensoncologygroup.org">istprogram@childrensoncologygroup.org</a> with a copy to PMB/CTEP at <a href="mailto:PMBafterhours@mail.nih.gov">PMBB/CTEP</a> at <a href="mailto:storygroup.org">istprogram@childrensoncologygroup.org</a> to report all such occurrences of prepared, unusable infusion bags shipped to a patient's home.

- d. Form documenting the time of packaging in the shipping container, duration of time the container will maintain 2° to 8°C temperature and verification that cold-chain management was maintained prior to administration must be included in each shipping container and returned to registering/treating institution for documentation purposes. (See Appendix VII-B)
- e. Home health care service staff is to use GCP guidelines.

#### **EVALUATION OF POTENTIAL SATELLITE PHARMACY SITES**

When the registering/treating institution is considering use of a local infusion center or home health care agency as a satellite pharmacy, the following must be assessed by the registering/treating institution in relation to the suitability of the local infusion center or home health care agency:

- Ability to appropriately store (temperature and security) the intact agent vials and/or prepared infusion bags.
- Ability to provide documentation of controlled and monitored temperature storage conditions while the IND agent is in the local infusion center or home health care agency possession.
- Availability of appropriately trained staff to prepare doses in compliance with USP <797> guidelines and the protocol, to label infusion bags according to the protocol instructions and to store agent doses under appropriate controlled temperature conditions.
- For home health care agency services, the ability to transport each prepared dose individually to the subject's home under appropriate controlled storage conditions or the ability to assess and confirm that cold-chain management of prepared infusion bags shipped to the subject's home is maintained prior to administration.
- Availability of appropriately trained staff to administer the prepared doses and perform the infusion bag changes according to the protocol.
- Methods for proper disposal of the waste, empty vials, IV bags, etc. are in place.
- Plan for return of unused intact vials to the registering/treating institution is in place.
- Source documentation to confirm agent administration must be maintained by the local infusion center or home health care agency and must be provided to the registering/treating institution for incorporation into the patient's medical/research records and for audit purposes.
- Plan for handling missed doses is in place.
- Agent accountability must be maintained via use of the NCI Drug Accountability Record Form (DARF). The originating site must keep a Control DARF and the local infusion center or home health care agency would be required to maintain a Satellite DARF if receiving and storing supplies of intact vials or receiving and storing infusion bags prepared by the registering/treating institution. Maintenance of a Satellite DARF is not required by home health care agency staff for prepared infusions bags shipped to the subject's home.
- The DARF must be provided to the registering/treating institution for record keeping purposes and audits.



• Documentation of IRB coverage for the protocol must be maintained. The IRB of record for the site must be informed that the study subject may receive therapy administered by a non-research site (i.e., the local infusion center or home health care agency).

# TRAINING FOR ALL PARTICIPATING SITES

The Lead Network Group for the trial must work with participating sites to:

- a. Implement a training process for participating NCTN Network sites regarding blinatumomab preparation and administration. Documentation of participating site training must be submitted via RSS as a protocol specific requirement at the time of site activation for participation on the trial.
- b. Develop a plan for participating NCTN Network sites to assess and train local outpatient infusion centers or home health care agency for patient treatment if required and document training of such sites.
- c. Have a training manual available for local outpatient infusion centers or home health care agencies on the clinical trial, appropriate agent preparation, handling and administration requirements and appropriate record keeping requirements.
- d. Create a definitive written communication plan for use between registering/treating institution and the local outpatient infusion centers or home health care agency on an ongoing basis during subject's treatment regimen, including emergency contact information for the registering/treating institution and investigator.



# APPENDIX VII-B: SHIPMENT OF BLINATUMOMAB IV BAG FROM SITE/PHARMACY TO PATIENT'S HOME

| Γο be completed by Site/Pharma | cy: | | | | |
|---|---|---|---|---|---|
| From: (Investigator Name, Address) | | To Patient: (Pa | To Patient: (Patient Initials, Study ID No) | | |
| | | Patient In | | Study ID Number | |
| repare shipment of IV bag at 2° astructions (see shipping contain tummer or winter package preparation). | ner instructions) | ). Please take car | | | |
| Date of packaging [DD/MMM/YYYY] | Time of p | packaging | | packed by (initials) | |
| Please tick the boxes and fill | | | | | |
| | | hours | | - | ture is |
| ☐ Cooling elements for | provided box u | sed according to | manu | facturer's instruction | |
| o be completed by Ambulant/F | Iome Care Serv | vice Provider: | | | |
| Shipment box unopened and c | content intact? | YES | | | |
| | | NO | | | |
| IF NO, please comment_ | | | | | |
| Date and time shipment box of | pened: | (date) | | | (time) |
| Confirmed by: | | (date) | | | (time) |
| , | (print name, | signature) Amb | . Care | Service | (date) |
| If time box ope | ened minus tin | ne of packaging | excee | nd inform site immed<br>ds the time duration<br>IV bag and <u>inform s</u> | n the shipping |

CONFIDENTIAL



# APPENDIX VIII: ADDITIONAL INFORMATION FOR MRD CORRELATIVE BIOLOGY STUDY

#### a) Rationale

Minimal residual disease is known to be a powerful prognostic factor in childhood ALL. 1-5,12,20-22 Although the majority of work has been done in newly diagnosed ALL patients, several studies using both polymerase chain reaction methods 13,14,16-18 and flow cytometry 19,23 have shown that MRD is highly predictive of second marrow relapse.

Flow cytometric MRD results will be used for the following purposes in this study:

- For late B-ALL marrow and late B-ALL IEM patients, we will use end-Block 1 flow cytometric MRD levels of < 0.1% vs. ≥ 0.1% to define low risk group vs. intermediate risk group, respectively. The low risk group will be eligible for LR randomization. The intermediate risk group will be eligible for HR/IR Randomization.
- For the LR patients participating in LR randomization, we will use end-Block 2 MRD levels of < 0.01% vs.  $\ge 0.01\%$  as a randomization stratification criteria to ensure balanced randomization.
- For the IR and HR patients participating in HR/IR Randomization, we will use end-Block 1 MRD levels of <0.1% vs.  $\ge 0.1\%$  as a randomization stratification criteria to ensure balanced randomization.
- For HR/IR Randomization patients proceeding to HSCT, we will use the end-Block 3/pre-HSCT MRD level, the peri-engraftment MRD level and the day +100 MRD level to determine eligibility for rapid tapering of immunosuppression.
- In HR/IR Randomization, we will use flow cytometric MRD+ rates at the end of Blocks 2 and 3 as a secondary efficacy objective.

Amendment #10 incorporates the High Risk/Intermediate Risk randomization closure. Effective September 18, 2019, accrual and randomization on the HR/IR arms closed. At completion of Block 1, if patient is found to be HR/IR the patient comes off protocol therapy.

# b) Technique

Aliquots of fresh bone marrow specimens <u>at study entry and during therapy at various designated time</u> <u>points</u> (see study schema and TDMs) will be adjusted to suitable cell concentrations and stained with the following combinations of monoclonal antibodies in 6-color immunofluorescence:

Tube 1: CD20-FITC/CD10-PE/CD38-PerCP-Cy5.5/CD58-APC/CD19-PE-Cy7/CD45-APC-Cy7
Tube 2: CD9-FITC/CD13-PE+CD33-PE/CD34-PerCP-Cy5.5/CD10-APC/CD19-PE-Cy7/CD45-APC-Cy7

After incubation, samples will be lysed with ammonium chloride, fixed with 0.25% ultra pure formaldehyde, and washed once before analysis. Samples will be run on a Becton Dickinson FACSCanto. A minimum of 750,000 events will be collected, and data will be analyzed by software developed by Dr. Brent Wood, University of Washington that facilitates the hierarchical gating strategy useful for identifying phenotypically aberrant cells. In cases in which the above panels are not informative for detecting abnormal cells, additional markers including but not limited to CD15 and TdT will be added to the panel to help identify MRD populations. In addition, if the administration of blinatumomab creates difficulties in identifying leukemic cells by virtue of CD19 expression, cytoplasmic CD79a and/or CD22 will be used to aid gating.



# APPENDIX IX: ADDITIONAL INFORMATION FOR CRLF2 CORRELATIVE BIOLOGY STUDY

#### a) Rationale

Recent genomic studies of ALL have identified genomic alterations of CRLF2, which encodes the thymic lymphopoietin receptor (TSLPR) and which results in upregulation of CRLF2 as an important contributor to leukemic pathogenesis. 3-5.7 Upregulation may occur by gene alterations, most often fusing CRLF2 to either P2RY8 or IGH@, as well as rarely, a CRLF2 point mutation (F232C), 3-5.7 though there may also be as yet unrecognized mechanisms. In addition, patients with whose blasts show upregulated CRLF2 typically also have simultaneous activating mutations in kinase genes including IKZF1, JAK1 and JAK2, and as a result have abnormalities in signal transduction networks. 3.4.7 Our results suggested high risk children with overexpressed CRLF2 as detected by PCR have very poor outcome irrespective of whether structural rearrangements can be identified, while other studies have suggested that this is only true of patients with P2RY8-CRLF2 translocations.<sup>2,9</sup> Moreover, in our studies CRLF2 did not appear to be prognostically significant in standard risk patients. However, virtually nothing is known about CRLF2 overexpression in the relapse setting, and whether its expression has continued prognostic significance in this already poorrisk group of patients. In addition, because of the underlying kinase abnormalities in this patient population, these patients are potentially ideal candidates for treatment with novel signal transduction inhibitors. Assessing CRLF2 expression may help to identify patients who might be candidates for specific therapy in trials that may be developed as these agents mature.

# b) Technique

In conjunction with the immunophenotyping performed at study entry as a baseline for flow cytometric MRD testing, we will also quantify surface TSLPR expression and correlate with outcome.

#### c) Specific Aims

#### Aims:

- 1) To determine if the frequency of high CRLF2 expression (which correlates with CRLF2 genomic lesions) is higher in the first marrow relapse B-ALL patient population than in the initial diagnosis B-ALL patient population.
- 2) To determine if first marrow relapse B-ALL patients with high CRLF2 expression have an inferior outcome to those without high CRLF2 expression.

#### d) Power calculations

**Aim 1:** Comparison of the frequency of CRLF2 expression among B-ALL patients in first marrow relapse to that in newly diagnosed B-ALL patients.

From past COG studies for newly diagnosed B-ALL, it is estimated that 10% of standard risk (SR) and 21% of high risk (HR) patients will relapse. Assuming there are 2/3 SR and 1/3 HR newly diagnosed patients, it is estimated that around 49% and 51% of patients in first relapse will be NCI SR and HR, respectively. Given that about 7% and 12% of the SR and HR patients have high level CRLF2 expression via flow cytometery, the overall rate of high CRLF2 expression (which correlates with genomic lesions) in newly diagnosed B-ALL patients is about 10%.

The following table provides the power to detect a difference in rates of high CRLF2 expression between newly diagnosed and 1<sup>st</sup> relapse B-ALL patients when the rate of high CRLF2 expression of the 1<sup>st</sup> relapse patients is 13%, 15%, 18% and 20% (i.e. RR=1.3, 1.5, 1.8 and 2.0), respectively. The power calculations are based on a one-sample exact test at 5% significance levels (one-sided). A total of 426 B-ALL marrow relapse ALL patients [180 early (CR1<36 months) and 246 late (CR1 ≥36 months)] were considered in this power calculation.



| Significance<br>Level | Rate of high CRLF2 expression in relapse B-ALL pts (baseline rate = 10% among newly diagnosed pts) | Power (%) |
|---|---|---|
| 5% | 13% | 60.0 |
| | 15% | 92.4 |
| | 18% | 99.9 |
| | 20% | 100.0 |

**Aim 2:** Comparison of EFS in first marrow relapse B-ALL patients with high level CRLF2 expression vs. those without high level CRLF2 expression.

It is anticipated that a total of 180 early (CR1<36 months) and 246 late (CR1  $\geq$ 36 months) marrow B-ALL patients will be enrolled to AALL1331. According to past studies, the 3-year EFS of early and late marrow relapse patients are approximately 26% and 65%, respectively, giving an overall 3-year EFS of about 48%. Assuming the above rates of high-level CRLF2 expression and minimum 2 years of follow-up, the table gives powers for comparing EFS between patient groups with and without high level CRLF2 expression. The power calculations are based on the one-sided log-rank test at the 5% significance level.

| Significance | CRLF2 high rate for | Samp | le Size | 3-year E | FS rates | · |
|---|---|---|---|---|---|---|
| Level | 1 <sup>st</sup> relapsed pre-B<br>pts | CRLF2 | CRLF2- | CRLF2+ | CRLF2- | Power |
| 0.05 | 0.13 | 55 | 371 | 0.18 | 0.52 | 100.0 |
| | 0.13 | 55 | 371 | 0.20 | 0.52 | 99.9 |
| | 0.13 | 55 | 371 | 0.23 | 0.52 | 99.8 |
| | 0.13 | 55 | 371 | 0.26 | 0.51 | 99.0 |
| | 0.13 | 55 | 371 | 0.30 | 0.51 | 96.3 |
| | 0.13 | 55 | 371 | 0.33 | 0.50 | 88.8 |
| | 0.13 | 55 | 371 | 0.36 | 0.50 | 77.7 |
| | 0.13 | 55 | 371 | 0.39 | 0.49 | 55.1 |
| | 0.15 | 64 | 362 | 0.18 | 0.53 | 100.0 |
| | 0.15 | 64 | 362 | 0.20 | 0.53 | 100.0 |
| | 0.15 | 64 | 362 | 0.23 | 0.52 | 99.9 |
| | 0.15 | 64 | 362 | 0.26 | 0.52 | 99.6 |
| | 0.15 | 64 | 362 | 0.30 | 0.51 | 97.5 |
| | 0.15 | 64 | 362 | 0.33 | 0.51 | 93.5 |
| | 0.15 | 64 | 362 | 0.36 | 0.50 | 81.2 |
| | 0.15 | 64 | 362 | 0.39 | 0.50 | 65.0 |
| | 0.18 | 77 | 349 | 0.18 | 0.55 | 100.0 |
| | 0.18 | 77 | 349 | 0.20 | 0.54 | 100.0 |
| | 0.18 | 77 | 349 | 0.23 | 0.53 | 100.0 |
| | 0.18 | 77 | 349 | 0.26 | 0.53 | 99.9 |
| | 0.18 | 77 | 349 | 0.30 | 0.52 | 99.1 |
| | 0.18 | 77 | 349 | 0.33 | 0.51 | 95.7 |
| | 0.18 | 77 | 349 | 0.36 | 0.51 | 88.8 |



| 0.18 | 77 | 349 | 0.39 | 0.50 | 69.6 |
|------|----|-----|------|------|-------|
| 0.20 | 85 | 341 | 0.18 | 0.56 | 100.0 |
| 0.20 | 85 | 341 | 0.20 | 0.55 | 100.0 |
| 0.20 | 85 | 341 | 0.23 | 0.54 | 100.0 |
| 0.20 | 85 | 341 | 0.26 | 0.54 | 100.0 |
| 0.20 | 85 | 341 | 0.30 | 0.53 | 99.6 |
| 0.20 | 85 | 341 | 0.33 | 0.52 | 97.8 |
| 0.20 | 85 | 341 | 0.36 | 0.51 | 90.6 |
| 0.20 | 85 | 341 | 0.39 | 0.50 | 72.1 |



# APPENDIX X: ADDITIONAL INFORMATION FOR BLINATUMOMAB PHARMACODYNAMICS CORRELATIVE BIOLOGY STUDY

#### a) Rationale

For patients with relapsed/refractory ALL, response patterns to blinatumomab are essentially binary. Some patients have a striking response, with a systemic cytokine release syndrome (CRS, most notably IL-6) accompanying clearance of leukemic blasts and culminating in an MRD-negative remission, and others do not respond. <sup>10,11,83</sup> For patients that have received blinatumomab in the setting of MRD positivity (i.e., with very low tumor burden), response rates are generally higher and significantly less likely to be associated with CRS. <sup>4,5</sup> Attempts to correlate responses with various peripheral blood parameters (such as ALC and T-cell subset quantitation) have been largely unsuccessful in either setting, although the patient numbers have been limited. <sup>3</sup>

The bone marrow microenvironment contains various immunologic components that have been shown to either enhance or suppress cytotoxic T-cell effector response to tumor antigens. The bone marrow serves as a reservoir of memory T-cells with heightened antigen specificity compared to peripheral blood memory T-cells, and the bone marrow microenvironment is capable of effectively priming naïve T-cell responses.

86 However, the bone marrow is also a reservoir for suppressive regulatory CD4/CD25/FOXP3+ T-cells (T regs).

87 Comparative studies of bone marrow vs. peripheral blood in patients with myeloma have shown that marrow-infiltrating lymphocytes (MILs) are more effectively activated and expanded and are more capable of tumor-specific cytotoxicity than peripheral blood lymphocytes (PBLs).

88 In addition, bone marrow contains myeloid-derived suppressor cells (MDSCs) that have been shown to preferentially capture and present tumor associated antigens to T regs, resulting in tumor tolerance, and preventing the capture and presentation of these antigens by dendritic cells to activate tumor-specific cytotoxic effector T-cells.

89 IL-6 is among the key mediators that skews the marrow T-cell repertoire from T regs to cytotoxic effector T-cells.

As has been suggested by previous studies, lymphocyte populations and cytokine profiles in the peripheral blood may also provide insight into responses<sup>3</sup> and adverse effects<sup>11</sup>. Since our study will include more patients than any blinatumomab trial to date, our study may be particularly well-suited to detect these associations.

#### b) Hypotheses and specific aims

The overall objective of this correlative study is to generate new knowledge regarding the mechanisms that determine the observed heterogeneity of clinical responses to blinatumomab in relapsed ALL, for which there are currently no biomarkers. While this study is preliminary and will not by itself establish biomarkers of blinatumomab response, it may identify putative biomarkers that can then be evaluated for validation in future studies.

We hypothesize that the balance of enhancing vs. suppressive components of the cytotoxic T-cell effector response in the bone marrow microenvironment (which we will directly measure using flow cytometry and single-cell RNA sequencing, and infer functionally using ex-vivo response assays) may be playing a particularly important role in determining the presence or absence of clinical response to blinatumomab. Specifically, we hypothesize that the bone marrow of patients that respond to blinatumomab (i.e., achieve complete continuous remission after treatment with blinatumomab) will be characterized by a relative predominance of cytotoxic memory/effector T-cells over T regs and MDSCs, , and ex-vivo induction of apoptosis and cytokine production, while the opposite pattern will be characteristic of the bone marrow of non-responders (i.e., those that relapse after treatment with blinatumomab).



• <u>Specific Aim 1</u>: To determine if the balance of enhancing vs. suppressive components of the cytotoxic T-cell effector response in the bone marrow microenvironment at baseline correlates with disease free survival (DFS) in relapsed ALL patients treated with blinatumomab.

We further hypothesize that lymphocyte populations and cytokine profiles in the peripheral blood at baseline and at post-treatment time points (hours 6 and 12 on day 1, and once on days 2, 7, 14 and 21) may also provide insight into adverse effects and clinical response, and so we will collect peripheral blood for flow cytometric characterization of lymphocyte subsets (including T-cell subsets as above, as well as circulating normal B-cells) and isolate plasma for multiplex cytokine profiling (including IL-6, IL-2R, IL-8, IL-10, MCP-1, MIP-1B, and INF-γ).

• <u>Specific aim 2</u>: To determine if peripheral blood patterns of lymphocyte subsets and cytokines, both at baseline and at post-treatment time points, correlates with incidence of blinatumomabrelated reportable adverse events (see <u>Section 5.2</u>), and DFS in relapsed ALL patients treated with blinatumomab.

# c) Methods

• Processing, cryopreservation and quality control

Refer to Section 13.5 for specimen collection and shipment. All blood and marrow samples will first be centrifuged to allow isolation of plasma. Plasma will be stored in 250 uL aliquots and stored at -80 C for subsequent batched assays. Cell pellets will be diluted in HBSS and centrifuged over Lymphocyte Separation Medium (LSM) to isolate mononuclear cells, then suspended in cryoprotectant solution and viably cryopreserved in liquid nitrogen in aliquots of 10e6 cells for subsequent batched assays. Assays will be performed as cohorts of five patients have provided a complete set of samples.

The Brown laboratory routinely processes blood and marrow specimens from cooperative group clinical trials and performs a wide variety of assays using plasma and viably cryopreserved cells. Samples are generally received in the laboratory within 48 hours of collection and processed immediately. Plasma and cells are sufficiently stable in transport under these conditions for the proposed assays. The flow cytometric assays are routinely performed in the Pardoll laboratory, which is collaborating on this project and has provided the processing protocol described above.

Multiparameter flow cytometric measurement of lymphocyte subsets and MDSCs

Vials of viably cryopreserved marrow and blood cells will be thawed and washed and viable cells counted by trypan blue exclusion. Cells will then be stained with isotype controls and the following antibody panels, and analyzed in triplicate by flow cytometry

- o For lymphocyte subsets: CD3, CD4, CD8, CD19, CD20, CD45RO, CD45RA, HLADR, CD27, CD62L, CD25, CD28 and CD127.
- o For MDSCs (marrow only): Lin, HLA-DR, CD33, CD11b, CD14, CD15

The **endpoint** for this assay will be the <u>relative percentage</u> and <u>absolute number</u> (in cells/uL) and of each of the following:

- o T regs
- Naïve T-cells
- Memory T-cells (central vs. effector)
- Activated T-cells
- o B-cells
- o Monocytic MDSC (marrow only)
- o Granulocytic MDSC (marrow only)



# • Cytokine profiling in marrow and blood plasma

Vials of frozen plasma will be thawed and a panel of cytokines will be quantitated in triplicate using a custom cytometric bead array kit (custom BD CBA) designed to measure the following: IL-6, IL-2R, IL-8, IL-10, MCP-1, MIP-1B, and INF-γ. Isotype controls will serve as negative controls, and standard curves will be generated using control cytokine solutions.

The endpoint for this assay will be levels of each cytokine in pg/mL.

### • Single cell RNA-seq

We will use the 10X Genomics scRNASeq platform, which allows mRNA expression profiling of up to ~12,000 individual cells per sample, as an unbiased approach to decompose the cellular composition of the BM microenvironment.

The **endpoint** for this assay will be the relative percentage of each of the following:

- o T regs
- Naïve T-cells
- o Memory T-cells (central vs. effector)
- Activated T-cells
- o B-cells
- o Monocytic MDSC (marrow only)
- o Granulocytic MDSC (marrow only)

# • Functional ex vivo cytotoxic response assays to mimic in vivo response

We will co-incubate:

- Thawed cryopreserved patient BM samples, initially enriched for mononuclear cells by centrifugation over lymphocyte separation medium (with healthy donor BM, available through institutional banking protocols, as control);
- Human B-ALL CD19+ cell lines (REH, NALM6) as leukemia stimulation (with CD19-AML cellline HL60 as control); and
- o Blinatumomab (AMG 103) (with control BiTE MEC14 as control)

Co-culture for up to 24 hrs to allow for optimal T-cell activation and blinatumomab-mediated B-ALL killing. Harvest cells and measure cytotoxic effect of blinatumomab on the leukemia cell line using Annexin V staining in conjunction with CD19 staining to isolate B-ALL cells. The **endpoint** for this assay will be proportion of apoptotic (Annexin V positive) B-ALL cells (relative to normal controls).

Also, harvest cell culture supernatant to measure soluble cytokine protein expression using bead-based custom assays as above. The **endpoint** for this assay will be <u>levels of each cytokine in pg/mL</u> (relative to negative controls).

#### • Dynamic T-cell clonal repertoire (ImmunoSEQ)

Genomic DNA will be isolated from a small amount of each PB sample. We will send DNA for sequencing using the ImmunoSeq platform developed by Adaptive Biotechnologies, which uses genomic DNA to generate an absolute count of every TcR sequence present.



# • Rationale for selection of methods and laboratories

The methods described above are performed routinely in the Brown laboratory, and are likely to optimize the chances that the proposed studies will be successful.

## d) Analysis and Statistical Considerations

#### • Specific Aim 1:

For the flow and scRNASeq assays, we will calculate ratio (R) of enhancing to suppressive components in bone marrow microenvironment for each patient as follows:

```
R = (# Memory T-cells + # Activated T-cells)/(# T regs + # MDSC)
```

For the ex-vivo assays, we will calculate an apoptosis index (AI) as follows:

AI = (% apoptosis with blina)/(% apoptosis with control BiTE)

We will use logistic regression to model outcome (no relapse vs. relapse) as a function of R. The Benjamin-Hochberg procedure will be used to control for multiple comparisons.

The anticipated result is that R and AI are negatively correlated with risk of relapse (i.e., a higher ratio of enhancing to suppressive components, and higher ex-vivo apoptosis induction, will reduce risk of relapse). If this anticipated result is seen, multivariate analysis that includes known associations with relapse (duration of first remission, MRD, etc.) will be performed to determine whether the marrow microenvironment ratio adds anything independent to known predictors of relapse in blinatumomabtreated patients.

This analysis will be performed on the entire cohort of patients treated with blinatumomab, and also separately on the HR/IR cohort and on the LR cohort.

We anticipate that a total of 156 evaluable patients will be treated with blinatumomab on this study (Section 9.2), of which 72 will be HR/IR and 84 will be LR. We assume that we will have 90% compliance with submission of the marrow sample. We assume that about 10% of submitted samples will fail analysis for technical reasons. Thus, we expect that our sample size for R will be 127 (59 HR/IR and 68 LR).

Since we are proposing to use standard assays (flow cytometric and scRNASeq quantification of marrow cell subsets, and ex-vivo apopotosis) in a novel way (calculation of enhancing vs. suppressive components), we do not have *a priori* knowledge of the expected range of observed ratios. As such, these studies are exploratory and definitive power calculations are not possible. However, if we assume the log(R) and log(AI) follows a Gaussian distribution with a mean of 0 and standard deviation of 1 (i.e., a standard normal distribution), and assuming an overall relapse rate of 50% for the trial, a sample size of 127 will have 80% power to detect an effect size of 0.5, using a 2-sided significance level of 0.05. For example, if we assume patients who eventually relapse have a mean R/AI of 1 (log(R/AI) = 0), then we would be able to detect that patients who do not eventually relapse have a mean R/AI of >3.16 (log(R/AI) = 0.5) or a mean R/AI of < 0.316 (log(R/AI) = -0.5). This effect size is not unreasonable to expect. These calculations are based on methods from Hsieh, et al. Statist. Med. 17, 1623-1634 (1998).



The relationships between the ratios and rates of relapse will be described, and subsequent studies will be designed to validate these findings prospectively in the context of future clinical trials.

### • Specific Aim 2:

There are 12 variables to be determined for each blood sample (7 samples per patient):

- 1) Total T-cell number
- 2) CD4 count
- 3) CD8 count
- 4) Memory T-cell count
- 5) Activated T-cell count
- 6-12) Level of each of 7 individual cytokines

For each of the 12 variables, we will determine the baseline value (BV; hour 0) and the maximal change value (MCV; value at the post-treatment timepoint for which the variable has increased or decreased to the greatest degree). For the MCV, a landmark approach will be used in which all cases are followed for 21 days, and the maximal change observed up to that point will be used to predict outcome *from that point forward* for all patients who are still observable up to that landmark time point.

There are 2 outcomes of interest:

- 1) Presence or absence of blinatumomab-related reportable adverse event
- 2) No relapse vs. relapse

As a first level analysis, we will use logistic regression to model each of the 2 outcomes as a function of each of the 12 variable's BV, and each of the 12 variable's MCV. The Benjamin-Hochberg procedure will be used to control for multiple comparisons.

The anticipated results are:

- 1) BV of some subsets of T-cell counts (memory T-cells, e.g.) are positively correlated with the risk of blinatumomab-related reportable adverse events, and negatively correlated with risk of relapse.
- 2) MCV of a subset of cytokines (IL-6 and INF-γ, e.g.) is positively correlated with the risk of blinatumomab-related reportable adverse events, and negatively correlated with risk of relapse.

Subsequent levels of analysis will attempt to characterize combinations of T-cell subset counts and cytokine levels that may perform better than individual variables in modeling the outcomes of interest.

If any of the anticipated results are seen with respect to the relapse outcomes, multivariate analysis that includes known associations with relapse (duration of first remission, MRD, etc.) will be performed to determine whether any of the T-cell subset/cytokine variables adds anything independent to known predictors of relapse in blinatumomab-treated patients.

This analysis will be performed on the entire cohort of patients treated with blinatumomab, and also separately on the HR/IR cohort and on the LR cohort.

We anticipate that a total of 156 evaluable patients will be treated with blinatumomab on this study (Section 9.2), of which 72 will be HR/IR and 84 will be LR. We assume that we will have at least 90% compliance with submission of the blood samples, and that about 10% of submitted samples will fail analysis for technical reasons. Thus, we expect that our sample size will be 127 (59 HR/IR and 68 LR).



Since we are proposing to use standard assays (flow cytometric quantification of blood T-cell subsets and cytokines) in a novel way (combining variables to model risks of adverse events and relapse after treatment with blinatumomab), we do not have *a priori* knowledge of the expected ranges of values for most variables. As such, these studies are exploratory and definitive power calculations are not possible.

However, some estimates based on specific assumptions are possible. If we assume that the baseline value for memory T-cell count for the entire study population follows a Gaussian distribution with a mean of 500/uL and a standard deviation of 100/uL, and we assume an overall relapse rate of 50% for the trial, a sample size of 127 will have 80% power to detect an effect size of 50/uL, using a 2-sided significance level of 0.05. For example, if we assume patients who eventually relapse have a mean BV memory T-cell count of 500, then we would be able to detect that patients who do not eventually relapse have a mean BV T-cell count of 500, then we would be able to detect that patients who do not eventually relapse have a mean BV T-cell count of 500, then we would be able to detect that patients who do not eventually relapse have a mean BV T-cell count of 500, then we would be able to detect that patients who do not eventually relapse have a mean BV T-cell count of 500, then we would be able to detect that patients who do not eventually relapse have a mean BV T-cell count of 500, then we would be able to detect that patients who do not eventually relapse have a mean BV T-cell count of 500, then we would be able to detect that patients who do not eventually relapse have a mean BV T-cell count of 500, then we would be able to detect that patients who do not eventually relapse have a mean BV T-cell count of 500, then we would be able to detect that patients who do not eventually relapse have a mean BV T-cell count of 500, then we would be able to detect that patients who do not eventually relapse have a mean BV T-cell count of 500, then we would be able to detect that patients who do not eventually relapse have a mean BV T-cell count of 500, then we would be able to detect that patients who do not eventually relapse have a mean BV T-cell count of 500, then we would be able to detect that patients who do not eventually relapse have a mean BV T-cell count of 500, then w

The relationships between the variable(s) and rates of adverse events/relapse will be described, and subsequent studies will be designed to validate these finding prospectively in the context of future clinical trials.

For the ImmunoSEQ experiments, we will assay n=72 samples (pre- vs. day 14, n=36 patients, n=18 relapse, n=18 no relapse). We hypothesize that "no relapse" samples will selectively demonstrate oligoclonal expansion of specific TcR clones. We will analyze patterns of T-cell clonal repertoire at baseline and changes after therapy, and look for associations of identified patterns and relapse/no relapse outcome. For significant associations, baseline/post-treatment patterns will be assessed for diagnostic value (e.g., correlation of baseline TcR repertoire with response) to be subsequently tested as a predictive biomarker of response. These assays will be descriptive and hypothesis-generating.



# APPENDIX XI: ADDITIONAL INFORMATION FOR PROTEIN CELL STRESS PATHWAYS CORRELATIVE BIOLOGY STUDY

#### a) Rationale

Many excellent studies have focused on gene expression profiles in ALL. 51,52 However, changes in protein cell stress pathways and deregulated signal transduction pathways, have been much less well studied in ALL. There is an unmet need to learn more about chemotherapy-induced proteins expression changes in order to determine if specific proteins or protein clusters can help predict response to therapy. Specific protein expression patterns are likely to correlate with disease-free survival (DFS) and will enable us to identify specific populations at risk for relapse. Since it is very difficult to salvage patients after second relapse, one of the **goals** of this study is to determine which patients classified as low risk based on timing and site of relapse (Section 9.2) would benefit from being risk stratified instead into the high risk group. This would improve DFS in all patients with relapsed ALL. Relevant protein expression profiles will be validated in future COG trial for patients with relapsed ALL and (if the increase in correct risk assignment increases to meets statistical specifications) will be used, in conjunction with molecular classification systems, as an adjunct for risk assignment.

# b) Hypotheses and specific aims

We **hypothesize** that activation of cell stress pathways and signal transduction pathways deregulated in ALL will correlate with DFS, and that the expression of specific proteins or proteins clusters will identify patients classified as low risk patients that would benefit from more intensive therapy. We have two **specific aims** to address these hypotheses:

- 1. To determine if specific protein expression profiles, as determined by reverse-phase protein lysate array (RPPA) and phosphoflow cytometry, correlate with clinical outcome (DFS)
- 2. To determine if alterations in specific groups of cell stress proteins can be used to generate a "high-risk" protein expression signature that identifies patients stratified to the low-risk group (based on time and site of relapse) that would benefit from stratification into the high-risk group.

### c) The contributions that the proposed study will make to the current knowledge base

Little is known about the changes in cell stress proteins during chemotherapy. This analysis will contribute greatly to our current knowledge base by 1) determining if specific proteins or protein clusters correlate with response therapy, 2) increasing our knowledge about lymphoblast response to standard relapse chemotherapy, 3) allowing a better understanding of the biology-defined ALL subgroups, aiding the development of targeted therapies, and 4) allowing for the development of protein expression risk-classifiers that could be validated and utilized, along with gene expression profiling, to aid in risk stratification in subsequent relapsed clinical trials.

# d) Relevant preclinical data

- 1. <u>RPPA</u> The Kornblau lab has analyzed two cohorts of adult AML using RPPA. The first, with 539 samples from 258 patients, was probed with 51 antibodies. the second, with 747 samples from 539 patients, was probed with 194 antibodies <sup>91,92</sup> These samples demonstrated that there were recurrent patterns of protein expression that correlated with outcome. Recent studies have shown that the analysis of RPPA and single cell network profiling by phosphoflow to can be analyzed using recently developed computational methods to provide a combined protein expression predictor. <sup>93</sup>
- 2. Phosphoflow cytometry: Studies have demonstrated that phosphoflow analyses can be predictive of outcome in pediatric acute leukemia. As an example, Redell et al. identified that responsiveness to IL-6 in pediatric AML was associated with superior survival. 94

### e) Relevant data from previous clinical studies

1. RPPA: Our preliminary data shows that we can reliably assess post-chemotherapy protein activation. Using a test set of 32 validated RPPA antibodies, we assessed changes in protein



- expression in 27 COG pediatric leukemia patients following induction chemotherapy. We have determined that 1) CellSave tubes preserve protein expression profiles post-treatment, as shown by the relative stability of actin expression, but a decrease in p-AKT; and 2) that we can detect the heterogeneous patterns of changes in protein expression over time, including changes in AKT, m-TOR, MAPkinase and the FOXO3 pathway following treatment (Horton, Kornblau, personal communication).
- 2. Phosphoflow: Based upon phosphoflow studies from phase 1 COG and adult trials using these assays, 81.95 we anticipate that we can reliably identify signaling upregulation at baseline and during therapy using shipped specimens. In an institutional study of adults with AML treated with sirolimus and chemotherapy, inhibition of phosphorylated S6 correlated with clinical responses (Perl 2012).
- f) The comparability of the methods proposed to those previously used, and the likelihood that the resulting data will be able to be compared with existing data. Analysis of RPPA is currently being performed using the same methods in AAML1031, and so these results should be directly comparable. Analysis of signal transduction networks will use identical methods to those piloted in ADVL1011 and ADVL1114, and so these should be comparable as well.

### g) The reason for selection of the assay methodology.

- 1. RPPA is a technique which can quantitate protein expression from over 1000 patient samples on a single slide using validated antibodies. The sample requirements are quite small; analysis of protein panels can be accomplished with as little as 200,000 cells per patient. This is the only assay able to provide detailed analysis of protein expression with this number of cells. This technique is also relatively resistant to protein degradation during shipping time. Blood is collected into CellSave preservation tubes, which we have shown can stabilize protein expression for up to 72 hours (Horton et al manuscript in review).
- 2. Similarly, phosphoflow cytometry is a very sensitive and reproducible technique, analyzing signal transduction abnormalities and the level of the single cell. Phosphoflow can also be used to analyze samples both at baseline and following chemotherapy treatment. 95

#### h) The stability of the samples used for analysis:

Although no formal studies have been performed to determine stability, samples collected locally over the past 15 years from the Horton laboratory were examined by RPPA. There were no statistically significant differences in expression patterns or protein intensity based on the age of the sample (Kornblau, personal communication).

### i) Technical performance characteristics

1. Antibody validation: RPPA antibodies have gone through extensive testing prior to inclusion on the array, <sup>88</sup> including both analytic validation, and assay validation with clinically relevant samples. <sup>94</sup> Antibodies validated for RPPA demonstrate specificity of signal and, in the case of phosphorylation or cleavage sensitive antibodies, context-specific validation performed in baseline and stimulated samples. <sup>87</sup> Validation steps have included: 1) antibody specificity as determined by immunoblot, 2) appropriate induction of phosphorylation/cleavage in response to known inducing agents, 3) correlation of RPPA signal with immunoblot expression (R>0.5), 4) acceptable sigmoidal curve fit of signal with sample dilution (analyzed using Super-Curve), 5) variable slope normalization <sup>97</sup> and, in cases of high background, 6) topographical normalization. Slides with unacceptable variances will be redone. RPPA has acceptable intra-assay and inter-assay variability, with intra-assay coefficients of variation (COV) of 6-15% and established inter-assay reproducibility. We have established standard operating procedures (SOPs) for sample processing, cell sorting and RPPA, and laboratory staff in both the Horton and Kornblau labs are experienced with the procedure.



b. <u>Minimizing sample variability</u>: based on prior testing samples received within 72h of collection from the patient have very similar protein expression patterns. (Horton, manuscript in preparation). Samples for RPPA will be collected in CellSave preservation tubes and mailed by FedEx courier to maintain protein integrity.

#### j) A description of the positive and negative controls

Controls will include normal adult and pediatric bone marrow, ALL cell lines, and ALL cells stimulated with chemotherapy as described .91,92,98

# k) The experience that the investigators have with the assay

- 1. The Horton Laboratory will be collaborating with Dr. Steve Kornblau who has extensive experience with RPPA analysis of leukemia samples. 91,92,98
- 2. The Tasian laboratory has extensive experience with phosphoflow cytometry analyses of primary patient leukemia specimens and of xenografted pediatric ALL and AML specimens. 99-102

# 1) The methods of scoring and plan for analysis

- a. Overview: Statistical analyses will be performed in a stepwise manner. First, we will analyze dynamic changes in protein activations following chemotherapy in all patients. The purpose is to discover natural groupings based on proteomic data only and to analyze the response of different biologically relevant signal transduction pathways during treatment. Second, we will examine protein clustering stratified by risk group and genetic subtype using supervised clustering analysis. Third, once clinical outcome data become available, we will analyze differences between treatment groups as they relate to DFS. This analysis will include unsupervised clustering methods. Finally, we will generate a classifier(s) that best correlates with clinical outcome for the group as whole. While the primary objective of the study is DFS, we will also examine classifiers stratified by CR and relapse after study completion.
- b. <u>Statistical analysis</u>: *Supercurve* algorithms were used to generate a single value from the 5 serial dilutions.<sup>1</sup> Loading controls<sup>2</sup> and topographical normalization<sup>3</sup> procedures will account for protein concentration and background staining variations. Analysis using unbiased clustering, perturbation bootstrap clustering and principle component analysis was then performed as previously described.<sup>4</sup> We (SM Kornblau, KR Coombes (MDACC) and A. Qutub (Rice University) have developed a novel modification of the Gap statistic, named "stability Gap" for selecting the optimal number of patient clusters from the range of possible clusters <sup>103</sup> This will be utilized to select the optimal number of clusters for comparison in outcomes analysis. Analysis typically places samples into 3-7 clusters for further analysis.

Comparison of the protein levels between paired samples will be done by performing paired t-tests. Association between protein expression levels and categorical clinical variables will be assessed in R using standard t tests, linear regression or mixed-effects linear models. Association between continuous variable and protein levels will be assessed by using Pearson and Spearman correlation and linear regression. Bonferroni corrections were performed to account for multiple statistical parameters for calculating statistical significance. The Kaplan-Meier method was used to generate the survival curves. Univariate and multivariate Cox proportional hazard modeling will be performed to investigate association with survival with protein levels as categorized variables using Statistica version 10 software (StatSoft, Tulsa, OK).

Other methods of analysis may include: Hierarchical Clustering, Principal Component Analysis (PCA), Self-Organizing Maps (SOM) and other class discovery methods. <sup>104</sup> Cluster stability will be accessed using reproducibility measures, including GAP, <sup>105</sup> and Stability Gap (manuscript in preparation), as well as robustness and discrepancy indices. <sup>106</sup> Differentially expressed proteins



will be found using paired t-test as well as repeated measures, mixed effect ANOVA and ANOVA with contrasts. To determine if dynamic changes in specific protein pathways predict chemoresistance, we will use different regression and classification methods: Self Organizing Maps(SOM) (when no outcome is used), class prediction methods such as logistic regression, Support Vector Machine, <sup>107</sup> Random Forest, <sup>108</sup> Binary Tree Prediction, Bayesian Compound Covariate Predictor, and Discriminant analysis (http://linus.nci.nih.gov/techreport/Manual32.pdf).

#### Correlation of protein data with clinical variables

For Specific Aim 1, we will determine if there is a protein classifier prognostic for clinical outcome. After assignment of each patient to a risk group (based on time and site of relapse, n=403 low-risk, n=195 high-risk), samples will be stratified based on risk group and supervised clustering analysis will be performed based on clinical outcome variables (DFS).

For Specific Aim 2, we will determine which patients classified as low-risk (based on time and site of relapse) that would benefit from the more intensive chemotherapy given to high-risk patients (*i.e.*, reassignment to the high risk group). Following the generation of a risk-based protein expression classifier from all low-risk patients, further testing of the putative classifier will be based on performance characteristics using predefined cutpoints using ROC curves. Comparisons will be made using the AUC of ROC curves between standard risk stratification (time and site of relapse), MRD response, and the putative protein expression classifiers. Model overfitting and biased assessment of model performance will be minimized using bootstrap clustering as previously described <sup>91</sup>ROC curves will be generated for each stratification group, as well as for combinations of groups. Since attainment of CR following subsequent relapse is suboptimal, <sup>109,110</sup> and DFS is guarded following subsequent relapse, protein expression classifiers that maximize specificity with adequate sensitivity will be prioritized for further characterization.

#### m) The sites performing the correlative studies.

RPPA analysis will be performed in the Kornblau laboratory (MD Anderson Cancer Center, Houston TX) in collaboration with Dr. Horton. Phosphoflow analysis will be performed in the Tasian laboratory (Children's Hospital of Philadelphia).

#### n) Maintenance of quality control/assurance

Quality control will be maintained as previously described (Section i). 91.92,98

#### o) Marker prevalence:

Since the methods will analyze multiple proteins (RPPA) and signal transduction pathways (phosphoflow), the prevalence of each marker will vary.

# p) Estimate what proportion of patients on a therapeutic trial will have available sample for correlative study analysis; discuss possible biases.

Based on prior samples obtained for RPPA analysis from patients enrolled on the Phase 3 COG AML trial AAML1031, we estimate 40% of enrollments will provide an evaluable sample. As the most common reasons for sample dropout include technical issues (20% sample dropout due to sample quality, 40% due to samples not being drawn at site, 10% due to delays in shipping), lack of consent (10-15%), and insufficient lymphoblasts in peripheral blood to qualify for the study (20%). The latter 20% will have a bias toward high-risk disease and early marrow relapse.

# q) Specify how any cutpoints will be determined

Specific aim 1: Performance characteristics and cutpoints will be made by comparison of AUC for ROC curves of available classifiers including standard risk stratification (time to and site of relapse) and MRD status. Since the objective of this study is to improve DFS, and DFS are can be estimated by



both the hazard ratio and probability of relapse. These numbers will become available from AALL0433, AALL01P2, AALL04P2 and AALL07P1 prior to trial completion. In order to identify patients likely to relapse, without increasing the risk of overtreating patients that require minimal therapy to achieve DFS, we will choose classifiers that maximize the true positive rate (sensitivity) while maintaining adequate specificity using statistically meaningful and clinically relevant cutpoints.

Specific aim 2: To determine if alterations in specific cell stress proteins can be used to generate a "high-risk" protein expression signature that identifies patients stratified to the low-risk (based on time and site of relapse) group that would have benefited from stratification into the high-risk group. For analysis of clinical utility, assumptions are usually made based on prior clinical trials for a similar pediatric relapsed ALL cohort. However, previous relapsed ALL COG studies have used different risk assessments, making *a priori* cutpoint determination challenging. Therefore, we will present basic principles for determining cutpoints for protein expression classifiers.

To aid in determining specific cutpoints, data from the recently completed AALL0433 clinical trial will be used to determine the prevalence of relapse and DFS in a similar LR population.

Since our aim is to improve the detection of true high risk patients misclassified into the low-risk group, we are interested in both the sensitivity and specificity of a putative protein classifier. The clinical usefulness of a protein expression classifier is dependent the proportion of low-risk patients that relapse (which can be estimated from the AALL0433 trial), as well as the proportion of low-risk patients with the "high-risk" putative classifier (determined by this study). Depending on the change in DFS for those correctly identified as having a "high-risk" protein classifier, the relative risks that can be used to identify the clinical usefulness can be estimated. Once these estimates are known, we can estimate both absolute risk reduction and decrease in relative risk of a low-risk patient with a "high-risk" classifier. Our goal would be to identify a classification signature that outperforms the current method of risk stratification (time and site of relapse) and/or allowed for an absolute risk reduction of at least 5% in the low-risk group.

#### r) Specify the statistical power of the correlative study

#### Sample size for basis of power calculations:

Based on power size calculations (Section 9.2.2), we anticipate that the study will enroll 598 patients, including 195 high-risk and 403 low-risk patients (based on time and site of relapse). Based on sample retrieval rate of 36% (see Section p), we will have 215 patients for protein expression analysis. For specific aim 1, all evaluable patients with usable sample would be considered for analysis (n=215). For the second aim, patients in the low-risk group (n=403) would be eligible if we receive usable sample. Based on sample recruitment in AAML1031 (36%), we expect to collect usable sample for 145 of the 403 evaluable patients. Although all sample set are required to have a 0h sample, about 82% of samples have the full data set (i.e. sufficient material for RPPA (CellSave preservation tubes) and phospho-flow (heparin tubes) at 0h, 6h, and 24h). For measures of changes over time, we anticipate that we will have 176 patient sets for SA1 and 118 patients for SA2. If the unfolded protein response is of interest, we expect that 90% of patients will have sufficient material for transcript analysis (n=193 for SA1, n=130 for SA2).

A summary of sample size data is provided in Table XI-1:

In addition to determining the effect sizes (defined as the difference in the corresponding mean outcomes over a common standard deviation) of assays between treatment groups, we will also compare protein classifiers with clinical outcome (MRD status and EFS). For the analysis of data across time (0h, 6h and 24h) we do not know *a priori* the most relevant time points to compare. Short-term



differences could have returned to baseline by 24h, and may be most accurately estimated by changes between 0h and 6h. Long-term differences would be best measured by 0h-24h comparison. Complex changes, such as increase at 6h and decreases by 24h (seen with NF- $\kappa$ B after chemotherapy) are best measured using all three time points as descriptors. However, for simplicity we have provided the affect sizes for changes from 0h to 24h in Table XI-1.

| Table XI-1: Effect-size differences based on sample size for protein cell stress pathways | | |
|---|---|---|
| 1. RPPA and phospho-flow | Samples size (max) | Effect size * |
| studies | | |
| Baseline and change at 24h by | 135 (67/tx group) | 0.488 |
| treatment arm (blinatumomab | | |
| therapy vs non-blinatumomab | 110 (55/tx group) | 0.539 |
| therapy; randomized patients only) | | |
| Baseline and change at 24h by | All patients: | |
| MRD response (rate of MRD >= | 215 (84 MRD) >= 0.1% / 131 MRD | 0.393 |
| 0.1%: 62% for high-risk, 28% for | < 0.1%) for baseline comparisons. | |
| low-risk; 39% overall) | • | |
| | 176 (69 MRD >=0.1%/107 MRD < | 0.435 |
| | 0.1%) for changes over time. | |
| | , C | |
| | Low-risk: | |
| | 145 (41 MRD >=0.1%/ 104 MRD | |
| | < 0.1%) for baseline comparisons. | 0.520 |
| | • | |
| | 118 (33 MRD >=0.1%/85 MRD < | |
| | 0.1%) for changes over time. | 0.579 |
| | , | |
| Baseline and change at 24h by 3- | 135 (86 no event/49 with event) for | 0.505 |
| year DFS for randomized patients | baseline changes. | |
| (estimated 3-year DFS 64%) | | |
| • | 110 (70 no event/ 40 with event) | 0.560 |
| | For changes over time. | |
| A | 2 Abbassistions, one masse try = tweet | |

Assumptions: alpha = 0.05, beta = 0.2. Abbreviations: grp= group, tx = treatment

#### s) Corrections for multiple comparisons

We will use the Benjamini-Hochberg correction to account for multiple comparisons. 111

# t) Discuss how the results will have an impact on future studies.

This contribution will significantly impact future studies because it will add protein cell stress markers to the armamentarium of genetic mutations currently used to assess relapse risk, increasing the power of risk stratification, and identifying patients most likely to relapse and those most likely to benefit from therapies that target deregulated cell signaling pathways in relapsed ALL.

<sup>\*</sup> With this effect size, the study will have at least 80% power at 2-sided significance level of 0.05 to detect such difference given the corresponding sample size.



# APPENDIX XII: COG STEM CELL COMMITTEE CONSENSUS GUIDELINES FOR ESTABLISHING ORGAN STAGE AND OVERALL GRADE OF ACUTE GRAFT VERSUS HOST DISEASE (GVHD)

### Reporting Requirements for Acute GVHD in COG Studies

In an attempt to standardize reporting of acute GVHD, the COG Stem Cell Transplantation Committee has adopted a modification of guidelines that were originally developed at the University of Michigan.

**Table 1** outlines standard criteria for GVHD organ staging. However, confounding clinical syndromes (such as non-GVHD causes of hyperbilirubinemia) may make staging GVHD in a given organ difficult. In addition, timing of organ specific symptoms affects whether that symptom is more or less likely to be true GVHD. Please refer to **Tables 2 and 3** to assist you in deciding whether to attribute these clinical findings to GVHD, especially in situations where a biopsy is not possible. For additional help, please see the text which follows the tables. **Table 4** reviews the approach to assessing GVHD as acute, chronic, or the overlap between the two.

Finally, engraftment syndrome will be reported separately from the GVHD scoring presented below.

#### **Engraftment Syndrome**

A clinical syndrome of fever, rash, respiratory distress, and diarrhea has been described, just prior to engraftment in patients undergoing unrelated cord blood and mismatched transplantation. If, in the judgment of the local investigator, a patient experiences this syndrome, details of the event should be reported when requested in the study CRFs.

Modified Glucksberg Staging Criteria for Acute Graft versus Host Disease

Table 1 Organ Staging (See tables and text below for details)

| Stage | Skin | Liver (bilirubin) | Gut (stool output/day) |
|---|---|---|---|
| 0 | No GVHD rash | < 2 mg/dL | Adult: < 500 mL/day<br>Child: < 10 mL/kg/day |
| 1 | Maculopapular rash < 25% BSA | 2 - 3 mg/dL | Adult: 500 – 999 mL/day Child: 10 - 19.9 mL/kg/day Or persistent nausea, vomiting, or anorexia, with a positive upper GI biopsy. |
| 2 | Maculopapular rash<br>25 – 50% BSA | 3.1 - 6 mg/dL | Adult: 1,000 – 1,500 mL/day Child: 20 – 30 mL/kg/day |
| 3 | Maculopapular rash > 50% BSA | 6.1 - 15 mg/dL | Adult: > 1,500 mL/day<br>Child: > 30 mL/kg/day |
| 4 | Generalized erythroderma<br>plus bullous formation and<br>desquamation > 5% BSA | > 15 mg/dL | Severe abdominal pain with or without ileus, or grossly bloody stool (regardless of stool volume). |



For GI staging: The "adult" stool output values should be used for patients > 50 kg in weight. Use 3 day averages for GI staging based on stool output. If stool and urine are mixed, stool output is presumed to be 50% of total stool/urine mix (see Section 3.2).

For stage 4 GI: the term "severe abdominal pain" will be defined as:

- (a) Pain control requiring institution of opioid use, or an increase in on-going opioid use, PLUS
- (b) Pain that significantly impacts performance status, as determined by the treating MD.

If colon or rectal biopsy is +, but stool output is < 500 mL/day (< 10 mL/kg/day), then consider as GI stage 0.

There is no modification of liver staging for other causes of hyperbilirubinemia

### Overall Clinical Grade (based on the highest stage obtained):

Grade 0: No Stage 1 - 4 of any organ

**Grade I:** Stage 1 - 2 skin and no liver or gut involvement

**Grade II:** Stage 3 skin, or Stage 1 liver involvement, or Stage 1 GI **Grade III:** Stage 0 - 3 skin, with Stage 2 - 3 liver, or Stage 2 - 3 GI

Grade IV: Stage 4 skin, liver or GI involvement

# Table 2 Evaluating Liver GVHD in the Absence of Biopsy Confirmation (See Table 3.0 below)

Establishing liver GVHD with no skin or GI GVHD

| Establishing liver G ville with no skin or Gr G ville | | |
|---|---|---|
| No Skin/GI GVHD | Assume no liver GVHD, unless proven by biopsy | |
| Day 0 - 35 | | |
| No Skin/GI GVHD | If NO other etiology identified, NO | If other etiology identified or |
| Day 36 - 100 | improvement with stopping | improves with stopping hepatotoxic |
| | hepatotoxic medications/TPN: | drugs/TPN: |
| | Stage as liver GVHD | Do not stage as liver GVHD |

Establishing liver GVHD with skin or GI GVHD and other cause of hyperbilirubinemia

| Skin and/or GI GVHD | Worsening bilirubin level (includes | Stable or improving bilirubin after |
|---|---|---|
| present | worsening just prior to onset of skin | diagnosis of skin or GI GVHD, |
| | or GI tract GVHD) OR stable | irrespective of treatment: |
| | elevated bilirubin despite resolution | Do not stage as liver GVHD |
| | of non-GVHD cause of increased | |
| | bilirubin: | |
| | Stage as liver GVHD | |

Changing liver GVHD stage with other cause of hyperbilirubinemia

| Skin and GI GVHD | Liver GVHD staging is carried forward without increase in stage until other |
|---|---|
| stable, improving, or | disease process resolves (e.g., if TTP is diagnosed in the presence of stage 2 |
| absent | liver GVHD, the liver GVHD stage 2 is carried forward despite rising |
| | bilirubin level until TTP is resolved. If there is no liver GVHD – stage 0 – |
| | and new onset TTP, the stage 0 is carried forward until TTP is resolved). |



| Skin and/or GI GVHD | Liver GVHD is staged according to the Glucksberg criteria. The |
|---|---|
| worsening | elevated bili is attributed to GVHD alone. |
| | Thus, when skin or GI GVHD is worsening, there is no downgrading of liver GVHD staging for other causes of hyperbilirubinemia. (e.g., if TTP is diagnosed in the presence of stage 2 liver GVHD and worsening skin or GI GVHD, the liver is staged according to the actual bilirubin level even if some of the rise in bilirubin is attributed to TTP). |
| | Similarly, even if there is no liver GVHD at onset of a new process, (such as TPN cholestasis), but skin or GI GVHD worsen during that process, then liver GVHD is diagnosed and staged according to the height of the bilirubin. |
| | There is one exception to this: the diagnosis of TTP, with high LDH and unconjugated bilirubin precludes the diagnosis and staging of new liver GVHD in the absence of a confirmatory liver biopsy. |

Table 3 Evaluating GI GVHD in the Absence of Biopsy Confirmation (See Table 4.0 below)

Establishing GI GVHD with new onset diarrhea and no skin or liver GVHD

| No Skin/liver GVHD | Assume no GI GVHD, unless proven by biopsy | |
|---|---|---|
| Day 0 through | | |
| engraftment | | |
| No Skin/liver GVHD | NO other etiology of diarrhea | Any other etiology of diarrhea |
| Engraftment through | identified: | identified: |
| day 100 | Stage as GI GVHD | Do not stage as GI GVHD |

Establishing GI GVHD with pre-existing diarrhea and skin or liver GVHD

| Skin and/or liver GVHD | Worsening diarrhea (includes | Improving diarrhea after the |
|---|---|---|
| present | worsening just prior to onset of skin | diagnosis of skin or liver GVHD |
| | or liver GVHD) OR persistent | (irrespective of treatment) OR |
| | diarrhea despite resolution of non- | persistent diarrhea without resolution |
| | GVHD cause: | of underlying non-GVHD cause: |
| | Stage as GI GVHD | Do not stage as GI GVHD |

# Differentiating Acute GVHD, Chronic GVHD, and Overlap Syndrome

There is often confusion differentiating acute from chronic GVHD, especially in the setting of reduced intensity transplants, DLI and new prophylactic treatments. The NIH Working Group recently published new classifications for GVHD:


Table 4 Acute GVHD, Chronic GVHD, and Overlap Syndrome

| Category | Time of Symptoms after HCT or DLI | Presence of Acute<br>GVHD features | Presence of Chronic GVHD features |
|---|---|---|---|
| Acute GVHD | | | |
| Classic acute GVHD | ≤100 d | Yes | No |
| Persistent, recurrent, or late-onset acute GVHD | >100 d | Yes | No |
| Chronic GVHD | | | |
| Classic chronic GVHD | No time limit | No | Yes |
| Overlap syndrome | No time limit | Yes | Yes |

- Scoring of acute GVHD may need to occur past day 100. In particular, patients should continue to be scored for acute GVHD when classic acute GVHD symptoms (maculopapular rash, nausea, vomiting, anorexia, profuse diarrhea particularly if bloody and ileus) persist past day 100 or if identical symptoms previously scored as acute GVHD resolve and then recur within 30 days during immunosuppression taper but past day 100.
- Those patients being scored as having acute GVHD should NOT have diagnostic or distinctive signs of chronic GVHD.
- Patients with both acute and chronic symptoms should be diagnosed as having Overlap Syndrome and scored according to their chronic GVHD score.

### Further Explanation of Criteria presented in Tables 2 and 3

### 1.0 Assessment of Skin GVHD

1.1 Presence or Absence of Skin GVHD: Skin GVHD will be considered present if a rash characteristic of acute GVHD develops after allogeneic marrow transplantation involving more than 25% of the body surface not clearly attributable to causes such as drug administration or infection. The extent of the body surface area involved can be estimated by the "Rule of Nines". In estimating the extent of skin GVHD, the area involved is calculated for individual anatomic areas, such as the arm or leg, and then the total is derived from a simple summation. Areas that are non-blanching should not be considered involved regardless of the overlying color of the rash (red, brown, etc.). Limited distribution erythema (with the exception of palms and soles) in the absence of associated rash elsewhere on the body will not be considered GVHD.

#### 2.0 Assessment of Liver GVHD

## 2.1 Assessing for the Presence or Absence of Liver GVHD

- A. Hyperbilirubinemia (total bilirubin  $\geq 2.0 \text{ mg/dL}$ ) in the **absence** of other signs of acute GVHD in the skin or GI tract:
  - Day 0-35: If hyperbilirubinemia alone is present with no other signs of acute GVHD in other organ systems, acute GVHD will not be diagnosed based solely on laboratory abnormalities. Acute GVHD will be diagnosed if findings on histopathology studies of liver from a biopsy or autopsy are confirmatory.
  - ii) Day 35-100: If hyperbilirubinemia (must be conjugated bilirubin) is not improving or is exacerbated (especially if serum alkaline phosphatase is increased), in the absence of acute GVHD in other organ systems, no other etiologies are identified, and does not improve with discontinuation of hepatotoxic drugs, acute GVHD will be diagnosed. However, it is distinctly unusual to develop ascites or a coagulopathy in the early stages of acute GVHD of



the liver alone. In the absence of histopathology studies of liver from a biopsy or autopsy specimen, ascites or a coagulopathy secondary to liver dysfunction will be considered to indicate the presence of another disease process (e.g. veno-occlusive disease). Recommended non-invasive studies to define an etiology for hyperbilirubinemia are:

- a. Imaging of liver (CT or ultrasound)
- b. Hepatitis screen (only if ALT is elevated)
- c. PT
- d. Blood cultures
- e. Review of medication list for potentially hepatotoxic drugs
- f. Review of risk factors for viral liver infection (HSV, CMV, VZV, adenovirus, EBV, HBV, and HCV)
- g. Hemolysis screen
- B. Pre-existing hyperbilirubinemia clearly attributed to an etiology other than acute GVHD in the presence of signs of acute GVHD in other organ systems.
  - i) If pre-existing non-GVHD liver disease (documented clinically, by lab assessment, or by imaging studies) is stable or improving at the onset of signs of acute GVHD in other organs, then acute GVHD of the liver will not be considered to be present unless proven by liver biopsy or autopsy.
  - ii) If hyperbilirubinemia worsens several days before or at the time of onset of signs of acute GVHD in other organ systems, GVHD will be considered to be present unless histopathology studies of liver are available and negative on a biopsy during that time interval or autopsy results exclude GVHD.
  - iii) If hyperbilirubinemia persists and is not improving after resolution of a pre-existing non-GVHD liver disease process (e.g. localized infection of liver, systemic sepsis, biliary tract obstruction) when signs of acute GVHD are present in other organ systems or no other intervening cause has been diagnosed, then acute GVHD will be considered to be present in the absence of a new, clearly identifiable cause of non-GVHD liver disease or unless a liver biopsy or autopsy specimen is negative.
- C. Prior acute GVHD in liver with new onset of a disease process that exacerbates pre-existing or recently resolved hyperbilirubinemia:
  - i) If an etiology other than acute GVHD is clearly identified as causing or exacerbating hyperbilirubinemia and acute liver GVHD has been diagnosed and has been stable, improving, or resolved, then the liver will not be restaged for acute GVHD until the resolution or stabilizing of the concurrent disease process (i.e., the liver stage prior to the onset of the new disease process will be carried forward until the new disease process resolves). Example: Acute GVHD of the liver and gut is diagnosed on Day 20. Treatment of acute GVHD results in falling bilirubin levels to liver Stage 1. Sepsis or TTP develops with transient worsening of the hyperbilirubinemia. The liver stage is not increased, despite a higher bilirubin level, because the cause of worsening hyperbilirubinemia is attributed to sepsis or TTP.
  - ii) If an etiology other than acute GVHD is clearly identified as causing or exacerbating hyperbilirubinemia in the presence of already worsening acute liver GVHD <u>or</u> GVHD of the skin or GI tract is simultaneously worsening, then the liver GVHD will be staged according to the actual bilirubin level, even though another cause of hyperbilirubinemia is present.

### 3.0 Assessment of GVHD of the Gastrointestinal Tract

## 3.1 Assessing for the Presence or Absence of GVHD of the Gastrointestinal Tract

- A. Diarrhea (≥ 500 mL/day in adults or > 10 mL/kg in pediatric patients) in the absence of other signs of acute GVHD in other organ systems
  - i) Day 0-engraftment: If diarrhea alone is present without other signs of acute GVHD in other



organ systems, acute GVHD will not be considered present. Diarrhea will be attributed to acute GVHD if histopathology studies of gastrointestinal tract from a biopsy or autopsy are diagnostic.

- ii) Engraftment-day 100: If diarrhea persists and is not improving, is exacerbated, or develops de novo in the absence of acute GVHD in other organ systems, histopathology studies of gut biopsies or from autopsy specimens are not available, and no other etiologies are clearly identified, acute GVHD will be considered to be the cause. A stool specimen should be examined to rule out infectious causes (e.g. rotavirus, adenovirus, and C. difficile toxin). It is recommended, if at all possible, that biopsies be obtained for diagnostic purposes.
- B. Pre-existing diarrhea clearly attributed to an etiology other than acute GVHD in the presence of signs of acute GVHD in other organ systems:
  - i) If pre-existing diarrhea caused by a process other than GVHD has been documented clinically or by lab assessment and is stable or improving at the onset of signs of acute GVHD in the skin or liver, then acute GVHD of the intestine will not be considered to be present in the absence of biopsy confirmation or autopsy report.
  - ii) If diarrhea or gastrointestinal symptoms are already present, but worsen significantly at the time of onset of signs of acute GVHD in the skin or liver, GVHD will be considered present, unless biopsy or autopsy are negative.
  - iii) If diarrhea persists after resolution of a pre-existing disease process with signs of acute GVHD present in other organ systems, GVHD will be considered present, unless biopsy or autopsy are negative.
- C. Prior or present acute GVHD in other organ systems with new onset of diarrhea: If diarrhea is **clearly** attributable to an etiology other than acute GVHD (e.g., infection) and a history of acute GVHD exists or acute GVHD is present in other organ systems and is stable, then the gastrointestinal tract will not be evaluable for acute GVHD until the resolution or stabilizing of the other disease process (e.g., infection) in the absence of biopsy or autopsy confirmation.
- D. Persistent anorexia, nausea or vomiting in the absence of signs of acute GVHD in other organ systems:

Persistent anorexia, nausea or vomiting in the absence of other known causes of these symptoms will be considered Stage 1 acute GVHD if confirmed by endoscopic biopsy.

If a biopsy is not possible (e.g. secondary to thrombocytopenia) but the clinical findings are compatible with acute GVHD, then the patient will be treated and recorded as having acute GVHD.

## 3.2 Staging of the Gastrointestinal Tract for the Severity of Acute GVHD

The severity of gastrointestinal tract GVHD will be staged according to modified Glucksberg criteria. To minimize errors caused by large day-to-day variation, diarrhea volume is measured as an average over 3 days and reported as the volume in milliliters per day. When urinary mixing is noted the stool volume will be considered half of the total volume unless nursing staff is able to give a better estimate from direct observation. Abdominal cramps are considered significant for staging if the severity results in a clinical intervention (e.g. analgesia, fasting, etc.). Blood in the stools is considered significant if the blood is visible or hematochezia/ melena is present and not clearly attributed to a cause other than GVHD (e.g. epistaxis/ hemorrhoids).



#### APPENDIX XIII: CTEP AND CTSU REGISTRATION PROCEDURES

### CTEP INVESTIGATOR REGISTRATION PROCEDURES

Food and Drug Administration (FDA) regulations and National Cancer Institute (NCI) policy require all individuals contributing to NCI-sponsored trials to register and to renew their registration annually. To register, all individuals must obtain a Cancer Therapy Evaluation Program (CTEP) Identity and Access Management (IAM) account (<a href="https://ctepcore.nci.nih.gov/iam">https://ctepcore.nci.nih.gov/iam</a>). In addition, persons with a registration type of Investigator (IVR), Non-Physician Investigator (NPIVR), or Associate Plus (AP) (i.e., clinical site staff requiring write access to OPEN, RAVE, or TRIAD or acting as a primary site contact) must complete their annual registration using CTEP's web-based Registration and Credential Repository (RCR) (<a href="https://ctepcore.nci.nih.gov/rcr">https://ctepcore.nci.nih.gov/rcr</a>). Documentation requirements per registration type are outlined in the table below.

| Documentation Required | IVR | NPIVR | AP | A |
|---|---|---|---|---|
| FDA Form 1572 | • | • | | |
| Financial Disclosure Form | • | • | • | |
| NCI Biosketch (education, training, employment, license, and certification) | <b>~</b> | <b>~</b> | V | |
| HSP/GCP training | ~ | • | • | |
| Agent Shipment Form (if applicable) | • | | | |
| CV (optional) | • | ~ | • | |

An active CTEP-IAM user account and appropriate RCR registration is required to access all CTEP and CTSU (Cancer Trials Support Unit) websites and applications. In addition, IVRs and NPIVRs must list all clinical practice sites and IRBs covering their practice sites on the FDA Form 1572 in RCR to allow the following:

- Added to a site roster
- Assigned the treating, credit, consenting, or drug shipment (IVR only) tasks in OPEN
- Act as the site-protocol PI on the IRB approval
- Assigned the Clinical Investigator (CI) role on the Delegation of Tasks Log (DTL).

Additional information can be found on the CTEP website at <a href="https://ctep.cancer.gov/investigatorResources/default.htm">https://ctep.cancer.gov/investigatorResources/default.htm</a>. For questions, please contact the RCR Help Desk by email at <a href="mailto:RCRHelpDesk@nih.gov">RCRHelpDesk@nih.gov</a>.



## **CTSU REGISTRATION PROCEDURES**

This study is supported by the NCI Cancer Trials Support Unit (CTSU).

## **Downloading Site Registration Documents:**

Site registration forms may be downloaded from the [insert study number] protocol page located on the CTSU members' website. Permission to view and download this protocol and its supporting documents is restricted and is based on person and site roster assignment housed in the CTSU RSS.

- Go to <a href="https://www.ctsu.org">https://www.ctsu.org</a> and log in to the members' area using your CTEP-IAM username and password
- Click on the Protocols tab in the upper left of your screen
- Either enter the protocol # in the search field at the top of the protocol tree, or
- Click on the By Lead Organization folder to expand
- Click on the COG link to expand, then select trial protocol #[insert study number]

Click on LPO Documents, select the Site Registration documents link, and download and complete the forms provided.

## **Requirements For AALL1331 Site Registration:**

- IRB approval (For sites not participating via the NCI CIRB; local IRB documentation, an IRB-signed CTSU IRB Certification Form, Protocol of Human Subjects Assurance Identification/IRB Certification/Declaration of Exemption Form, or combination is accepted )
- IROC Credentialing Status Inquiry (CSI) Form

NOTE: For studies with a radiation and/or imaging (RTI) component, the enrolling site must be aligned to a RTI provider. To manage provider associations access the Provider Association tab on the CTSU website at <a href="https://www.ctsu.org/RSS/RTFProviderAssociation">https://www.ctsu.org/RSS/RTFProviderAssociation</a>, to add or remove associated providers. Sites must be linked to at least one IROC credentialed provider to participate on trials with an RT component.

## **Submitting Regulatory Documents:**

Submit required forms and documents to the CTSU Regulatory Office, where they will be entered and tracked in the CTSU RSS.

Regulatory Submission Portal: <u>www.ctsu.org</u> (members' area) → Regulatory Tab → Regulatory Submission

When applicable, original documents should be mailed to: CTSU Regulatory Office 1818 Market Street, Suite 3000 Philadelphia, PA 19103

Institutions with patients waiting that are unable to use the Portal should alert the CTSU Regulatory Office immediately at 1-866-651-2878 in order to receive further instruction and support.

## **Checking Your Site's Registration Status:**

You can verify your site registration status on the members' section of the CTSU website. (Note: Sites will not receive formal notification of regulatory approval from the CTSU Regulatory Office.)



- Go to <a href="https://www.ctsu.org">https://www.ctsu.org</a> and log in to the members' area using your CTEP-IAM username and password
- Click on the Regulatory tab at the top of your screen
- Click on the Site Registration tab
- Enter your 5-character CTEP Institution Code and click on Go

Note: The status given only reflects compliance with IRB documentation and institutional compliance with protocol-specific requirements as outlined by the Lead Network. It does not reflect compliance with protocol requirements for individuals participating on the protocol or the enrolling investigator's status with the NCI or their affiliated networks.



#### APPENDIX XIV: POSSIBLE DRUG INTERACTIONS

The lists below <u>do not</u> include everything that may interact with chemotherapy. Study Subjects and/or their Parents should be encouraged to talk to their doctors before starting any new medications, using over-the-counter medicines, or herbal supplements and before making a significant change in diet.

### **Cyclophosphamide**

### Drugs that may interact with cyclophosphamide

- Allopurinol
- Amiodarone
- Carbamazepine
- Cyclosporine
- Digoxin
- Efavirenz
- Etanercept
- Hydrochlorothiazide
- Lumacaftor
- Mifepristone
- Pentostatin
- Rifampin
- Ritonavir
- Warfarin

#### Food and supplements that may interact with cyclophosphamide

- St. John's Wort
- Drinks, food, supplements, or vitamins containing "flavonoids" or other "antioxidants"

## **Cyclosporine**

### Drugs that may interact with cyclosporine

- Antibiotics
  - O Clarithromycin, erythromycin, nafcillin, rifapentin, rifampin, telithromycin
- Antidepressants and antipsychotics
  - Aripiprazole, citalopram, clozapine, escitalopram, fluoxetine, fluoxamine, lurasidone, nefazodone, paliperidone, quetiapine, thioridazine, ziprasidone
- Antifungals
  - O Amphotericin, caspofungin, fluconazole, itraconazole, isavuconazole, ketoconazole, posaconazole, voriconazole
- Anti-inflammatory, arthritis, or pain medications
  - Aspirin, celecoxib, hydroxychloroquine, ibuprofen, indomethacin, ketorolac, leflunomide, naproxen, meloxicam, oxaprozin, sulindac, tofacitinib, tolmetin
- Anti-rejection medications
  - Mycophenolate, sirolimus, tacrolimus



- Antiretrovirals and antivirals
  - Atazanavir, darunavir, delavirdine, efavirenz, etravirine, fosamprenavir, indinavir, letermovir, lopinavir, nelfinavir, nevirapine, ritonavir, saquinavir, Stribild, telaprevir, tipranavir
- Anti-seizure medications
  - O Carbamazepine, phenobarbital, phenytoin, primidone
- Cholesterol medications
  - O Atorvastatin, lovastatin, pravastatin, rosuvastatin, simvastatin, ezetimibe, fenofibrate, gemfibrozil, colesevelam, griseofulvin
- Heart medications
  - O Aliskiren, amiodarone, dronedarone, carvedilol, digoxin, diltiazem, eplerenone, verapamil, captopril, enalapril, lisinopril, ramipril
- Kidney medications
  - O Acetazolamide, amiloride, spironolactone, triamterene
- Some chemotherapy (be sure to talk to your doctor about this)
- Many other drugs, including the following:
  - Ambrisentan, bosentan, sitaxentan, aprepitant, allopurinol, colchicine, danazol, fluoxymesterone, modafinil, methyltestosterone, omeprazole, oxandrolone, mifepristone, natalizumab, pimozide, butabarbital, secobarbital, ivacaftor, octreotide

## Food and supplements that may interact with cyclosporine

- Alfalfa
- Black cohosh
- Echinacea
- Grapefruit, grapefruit juice, Seville oranges, star fruit
- Red Yeast Rice
- St. John's Wort

### Cytarabine (by vein)

### Drugs that may interact with cytarabine

• Clozapine, flucytosine, leflunomide, natalizumab

#### Food and supplements that may interact with cytarabine

Echinacea

#### **Dexamethasone**

## Drugs that may interact with dexamethasone

- Antibiotics
  - O Ciprofloxacin, levofloxacin, moxifloxacin, clarithromycin, erythromycin, nafcillin, rifabutin, rifampin, telithromycin
- Antidepressants and antipsychotics
  - Aripiprazole, buproprion, citalopram, clozapine, escitalopram, fluvoxamine, lurasidone, nefazodone, quetiapine
- Antifungals



- o Caspofungin, fluconazole, itraconazole, ketoconazole, posaconazole, voriconazole
- Arthritis medications
  - o Leflunomide, tofacitinib
- Anti-rejection medications
  - O Cyclosporine, sirolimus, tacrolimus
- Antiretrovirals and antivirals
  - O Atazanavir, darunavir, delaviridine, efavirenz, etravirine, fosamprenavir, indinavir, lopinavir, nelfinavir, nevirapine, rilpivirine, ritonavir, saquinavir, Stribild, telaprevir, tipranavir
- Anti-seizure medications
  - O Carbamazepine, oxcarbazepine, phenobarbital, phenytoin, primidone
- Heart medications
  - O Amiodarone, amlodipine, dronedenarone, verapamil
- Some chemotherapy (be sure to talk to your doctor about this)
- Some oral contraceptives or birth control medications
- Many other drugs, including the following:
  - O Aprepitant, artemether/lumefantine, aspirin, deferasirox, ibuprofen, ivacaftor, lomitapide, mifepristone, natalizumab, nimodipine, praziquantel, warfarin

## Food and supplements that may interact with dexamethasone

- Echinacea
- St. John's Wort
- Grapefruit, grapefruit juice, Seville oranges, star fruit

## **Etoposide**

### Drugs that may interact with etoposide

- Antibiotics
  - O Clarithromycin, erythromycin, nafcillin, rifapentin, rifampin, telithromycin
- Antidepressants and antipsychotics
  - o Clozapine, nefazodone
- Antifungals
  - o Fluconazole, itraconazole, ketoconazole, posaconazole, voriconazole
- Arthritis medications
  - Leflunomide, tofacitinib
- Anti-rejection medications
  - Cyclosporine
- Antiretrovirals and antivirals
  - O Atazanavir, darunavir, delaviridine, efavirenz, etravirine, fosamprenavir, indinavir, lopinavir, nelfinavir, nevirapine, ritonavir, saquinavir, Stribild®, telaprevir
- Anti-seizure medications
  - O Carbamazepine, fosphenytoin, phenobarbital, phenytoin, primidone
- Heart medications
  - o Amiodarone, dronedenarone, verapamil
- Some chemotherapy (be sure to talk to your doctor about this)
- Many other drugs, including the following:
  - O Aprepitant, atovaquone, bosentan, deferasirox, ivacaftor, lomitapide, mifepristone, modafinil, natalizumab, pimozide



### Food and supplements that may interact with etoposide

- Echinacea
- Glucosamine
- St. John's Wort
- Grapefruit, grapefruit juice, Seville oranges, star fruit

### **Fludarabine**

#### Drugs that may interact with fludarabine

• Clozapine, leflunomide, natalizumab, pentostatin, tofacitinib

## Food and supplements that may interact with fludarabine

Echinacea

### Leucovorin

### Drugs that may interact with leucovorin

- Glucarpidase
- Some antiepileptics (fosphenytoin, phenobarbital, phenytoin, primidone)
- Trimethoprim

### Food and supplements that may interact with leucovorin

Folic acid

#### **Methotrexate (by mouth or by vein)**

### Drugs that may interact with methotrexate

- Some antibiotics (amoxicillin, chloramphenicol, ciprofloxacin, penicillin, piperacillin, tetracycline, trimethoprim/sulfamethoxazole)
- Some anti-inflammatory drugs (aspirin, ibuprofen, naproxen, ketorolac, sulfasalazine, sulindac)
- Some heartburn medications (esomeprazole, lansoprazole, omeprazole, pantoprazole)
- Several other specific agents, including the following: amiodarone, clozapine, cyclosporine, eltrombopag, fosphenytoin, gemfibrozil, leflunomide, phenytoin, pimecrolimus, probenecid, pyrimethamine, ranolazine, retinoids, teriflunomide, theophylline, tolvaptan, warfarin



### Food and supplements that may interact with methotrexate

- Alcohol
- Echinacea
- Some vitamins, including those that contain folic acid or high doses of vitamin C

### **Mercaptopurine**

### Drugs that may interact with mercaptopurine

- Artiritis medications: leflunomide, tofacitinib
- Other medications, such as adalimumab, allopurinol, azathioprine, certolizumab pegol, clozapine, etanercept, febuxostat, golimumab, infliximab, natalizumab, olsalazine, sulfasalazine, warfarin

### Food and supplements that may interact with mercaptopurine

Echinacea

### **Mitoxantrone**

## Drugs that may interact with mitoxantrone

- Aripiprazole
- Clozapine
- Cyclosporine
- Eltrombopag
- Leflunomide
- Natalizumab
- Tofacitinib

#### Food and supplements that may interact with mitoxantrone

• Echinacea

#### Mycophenolate mofetil

### Drugs that may interact with mycophenolate mofetil

- Antacids such as aluminum hydroxide, magnesium hydroxide
- Arthritis medications such as leflunomide, tofacitinib
- Some antibiotics and antiviral medications (be sure to talk to your doctor about this)
- Some heartburn medications including esomeprazole, lansoprazole, omeprazole, pantoprazole
- Other medications such as cholestyramine, cyclosporine, natalizumab, oral contraceptives ("birth control"), probenecid, rifabutin, rifampin, rifapentine, sevelamer, tolvaptan, teriflunomide

#### Food and supplements that may interact with mycophenolate mofetil

- Echinacea
- Vitamins and supplements containing magnesium



#### <u>Pegaspargase</u>

### Drugs that may interact with pegaspargase

• Leflunomide, natalizumab, pegloticase, tofacitinib

### Food and supplements that may interact with pegaspargase

Echinacea

### **Tacrolimus**

### Drugs that may interact with tacrolimus

- Antibiotics
  - O Clarithromycin, erythromycin, nafcillin, rifapentin, rifampin, telithromycin
- Antidepressants and antipsychotics
  - Citalopram, clozapine, escitalopram, nefazodone, paliperidone, quetiapine, thioridizine, ziprasidone
- Antifungals
  - O Caspofungin, fluconazole, isavuconazole, itraconazole, ketoconazole, posaconazole, voriconazole
- Anti-inflammatory, arthritis, or pain medications
  - o Leflunomide, tofacitinib
- Anti-rejection medications
  - o Cyclosporine, sirolimus
- Antiretrovirals and antivirals
  - O Atazanavir, darunavir, delaviridine, efavirenz, etravirine, fosamprenavir, indinavir, lopinavir, nelfinavir, nevirapine, ritonavir, saquinavir, Stribild®, telaprevir, tipranavir
- Anti-seizure medications
  - o Carbamazepine, fosphenytoin, phenobarbital, phenytoin, primidone
- Heart medications
  - O Amiodarone, diltiazem, dronedenarone, disopyramide, procainamide, propafenone, quinidine, ranolazine, sotalol, verapamil
- Kidney medications
  - o Amiloride, spironolactone, triamterene
- Stomach and reflux medications
  - O Dexlansoprazole, esomeprazole, lansoprazole, omeprazole, rabeprazole
- Some chemotherapy (be sure to talk to your doctor about this)
- Many other drugs, including the following:
  - O Aprepitant, bosentan, cobicistat, colchicine, conivaptan, mifepristone, modafinil, natalizumab, pimozide

#### Food and supplements that may interact with tacrolimus

- Echinacea
- St. John's Wort
- Grapefruit, grapefruit juice, Seville oranges, star fruit



### **Thioguanine**

### Drugs that may interact with thioguanine

- Arthritis medications: leflunomide, tofacitinib
- Other medications, such as adalimumab, allopurinol, azathioprine, certolizumab pegol, clozapine, etanercept, golimumab, infliximab, natalizumab, olsalazine, sulfasalazine

### Food and supplements that may interact with thioguanine

• Echinacea

#### **Thiotepa**

#### Drugs that may interact with thiotepa

- Arthritis medications like leflunomide or tofacitinib
- Other medications like bupropion, clozapine, efavirenz, methadone, promethazine, or natalizumab

### Food and supplements that may interact with thiotepa

Echinacea

#### Vincristine

#### Drugs that may interact with vincristine

- Antibiotics
  - O Clarithromycin, erythromycin, nafcillin, rifapentin, rifampin, telithromycin
- Antifungals
  - o Fluconazole, itraconazole, isavuconazole, ketoconazole, posaconazole, voriconazole
- Arthritis medications
  - o Leflunomide, tocilizumab, tofacitinib
- Anti-rejection medications
  - o Cyclosporine
- Antiretrovirals and antivirals
  - Atazanavir, boceprevir, darunavir, delaviridine, efavirenz, etravirine, fosamprenavir, indinavir, lapatinib, lopinavir, nelfinavir, nevirapine, ritonavir, saquinavir, Stribild®, telaprevir, tenofovir, tipranavir
- Anti-seizure medications
  - O Carbamazepine, fosphenytoin, phenobarbital, phenytoin, primidone
- Heart medications
  - O Amiodarone, carvedilol, diltiazem, dronedenarone, propafenone, quinidine, ranolazine, verapamil
- Some chemotherapy (be sure to talk to your doctor about this)
- Many other drugs, including the following:



O Aprepitant, bosentan, cobicistat, conivapatan, deferasirox, fosnetupitant, ivacaftor, mifepristone, modafinil, natalizumab, nefazodone, netupitant

# Food and supplements that may interact with vincristine

- Echinacea
- St. John's Wort
- Grapefruit, grapefruit juice, Seville oranges, star fruit



#### **REFERENCES:**

- 1. Nguyen K, Devidas M, Cheng SC, et al: Factors influencing survival after relapse from acute lymphoblastic leukemia: a Children's Oncology Group study. Leukemia 22:2142-50, 2008
- 2. Handgretinger R, Zugmaier G, Henze G, et al: Complete remission after blinatumomabinduced donor T-cell activation in three pediatric patients with post-transplant relapsed acute lymphoblastic leukemia. Leukemia 25:181-4, 2012
- 3. Klinger M, Brandl C, Zugmaier G, et al: Immunopharmacologic response of patients with B-lineage acute lymphoblastic leukemia to continuous infusion of T cell-engaging CD19/CD3-bispecific BiTE antibody blinatumomab. Blood 119:6226-33, 2012
- 4. Topp MS, Gokbuget N, Zugmaier G, et al: Long-term follow-up of hematologic relapse-free survival in a phase 2 study of blinatumomab in patients with MRD in B-lineage ALL. Blood 120:5185-7, 2012
- 5. Topp MS, Kufer P, Gokbuget N, et al: Targeted therapy with the T-cell-engaging antibody blinatumomab of chemotherapy-refractory minimal residual disease in B-lineage acute lymphoblastic leukemia patients results in high response rate and prolonged leukemia-free survival. J Clin Oncol 29:2493-8, 2011
- 6. Lia Gore, Gerhard Zugmaier, Rupert Handgretinger, et al: Cytological and molecular remissions with blinatumomab treatment in second or later bone marrow relapse in pediatric acute lymphoblastic leukemia (ALL). J Clin Oncol 31, 2013 (suppl; abstr 10007). Published on Meeting Library (<a href="http://meetinglibrary.asco.org">http://meetinglibrary.asco.org</a>).
- 7. Raetz EA, Borowitz MJ, Devidas M, et al: Reinduction platform for children with first marrow relapse of acute lymphoblastic Leukemia: A Children's Oncology Group Study[corrected]. J Clin Oncol 26:3971-8, 2008
- 8. Tallen G, Ratei R, Mann G, et al: Long-term outcome in children with relapsed acute lymphoblastic leukemia after time-point and site-of-relapse stratification and intensified short-course multidrug chemotherapy: results of trial ALL-REZ BFM 90. J Clin Oncol 28:2339-47, 2010
- 9. Parker C, Waters R, Leighton C, et al: Effect of mitoxantrone on outcome of children with first relapse of acute lymphoblastic leukaemia (ALL R3): an open-label randomised trial. Lancet 376:2009-17, 2010
- 10. Weinshilboum R: Thiopurine pharmacogenetics: clinical and molecular studies of thiopurine methyltransferase. Drug Metab Dispos 29:601-605, 2001
- 11. Teachey DT, Rheingold SR, Maude SL, et al: Cytokine release syndrome after blinatumomab treatment related to abnormal macrophage activation and ameliorated with cytokine-directed therapy. Blood 121:5154-7, 2013
- 12. Paganin M, Zecca M, Fabbri G, et al: Minimal residual disease is an important predictive factor of outcome in children with relapsed 'high-risk' acute lymphoblastic leukemia. Leukemia 22:2193-200, 2008
- 13. Attarbaschi A, Mann G, Panzer-Grumayer R, et al: Minimal residual disease values discriminate between low and high relapse risk in children with B-cell precursor acute lymphoblastic leukemia and an intrachromosomal amplification of chromosome 21: the Austrian and German acute lymphoblastic leukemia Berlin-Frankfurt-Munster (ALL-BFM) trials. J Clin Oncol 26:3046-50, 2008
- 14. Eckert C, Biondi A, Seeger K, et al: Prognostic value of minimal residual disease in relapsed childhood acute lymphoblastic leukaemia. Lancet 358:1239-41, 2001
- 15. Lew G, Lu X, Yanofsky R, et al: The significance of minimal residual disease (MRD) in relapsed childhood B-lymphoblastic leukemia (B-ALL): A report from Children's Oncology Group (COG) protocol AALL0433.
- 16. Barredo JC, Devidas M, Lauer SJ, et al: Isolated CNS relapse of acute lymphoblastic leukemia treated with intensive systemic chemotherapy and delayed CNS radiation: a pediatric oncology group study. J Clin Oncol 24:3142-9, 2006



- 17. Ritchey AK, Pollock BH, Lauer SJ, et al: Improved survival of children with isolated CNS relapse of acute lymphoblastic leukemia: a pediatric oncology group study. J Clin Oncol 17:3745-52, 1999
- 18. Goulden N, Langlands K, Steward C, et al: PCR assessment of bone marrow status in 'isolated' extramedullary relapse of childhood B-precursor acute lymphoblastic leukaemia. Br J Haematol 87:282-5, 1994
- 19. Neale GA, Pui CH, Mahmoud HH, et al: Molecular evidence for minimal residual bone marrow disease in children with 'isolated' extra-medullary relapse of T-cell acute lymphoblastic leukemia. Leukemia 8:768-75, 1994
- 20. Schrappe M, Zimmermann M, Moricke A, et al: Dexamethasone in Induction Can Eliminate One Third of All Relapses in Childhood Acute Lymphoblastic Leukemia (ALL): Results of An International Randomized Trial in 3655 Patients (Trial AIEOP-BFM ALL 2000). ASH Annual Meeting Abstracts 112:7-, 2008
- 21. Silverman LB, Gelber RD, Dalton VK, et al: Improved outcome for children with acute lymphoblastic leukemia: results of Dana-Farber Consortium Protocol 91-01. Blood 97:1211-8, 2001
- 22. Gaynon PS, Trigg ME, Heerema NA, et al: Children's Cancer Group trials in childhood acute lymphoblastic leukemia: 1983-1995. Leukemia 14:2223-33, 2000
- 23. Hijiya N, Liu W, Sandlund JT, et al: Overt testicular disease at diagnosis of childhood acute lymphoblastic leukemia: lack of therapeutic role of local irradiation. Leukemia 19:1399-403, 2005
- 24. Sirvent N, Suciu S, Bertrand Y, et al: Overt testicular disease (OTD) at diagnosis is not associated with a poor prognosis in childhood acute lymphoblastic leukemia: results of the EORTC CLG Study 58881. Pediatr Blood Cancer 49:344-8, 2007
- 25. van den Berg H, de Groot-Kruseman HA, Damen-Korbijn CM, et al: Outcome after first relapse in children with acute lymphoblastic leukemia: a report based on the Dutch Childhood Oncology Group (DCOG) relapse all 98 protocol. Pediatr Blood Cancer 57:210-6, 2011
- 26. van den Berg H, Langeveld NE, Veenhof CH, et al: Treatment of isolated testicular recurrence of acute lymphoblastic leukemia without radiotherapy. Report from the Dutch Late Effects Study Group. Cancer 79:2257-62, 1997
- 27. Dordelmann M, Reiter A, Zimmermann M, et al: Intermediate dose methotrexate is as effective as high dose methotrexate in preventing isolated testicular relapse in childhood acute lymphoblastic leukemia. J Pediatr Hematol Oncol 20:444-50, 1998
- 28. Freeman AI, Weinberg V, Brecher ML, et al: Comparison of intermediate-dose methotrexate with cranial irradiation for the post-induction treatment of acute lymphocytic leukemia in children. N Engl J Med 308:477-84, 1983
- 29. Tsuchida M, Ohara A, Manabe A, et al: Long-term results of Tokyo Children's Cancer Study Group trials for childhood acute lymphoblastic leukemia, 1984-1999. Leukemia 24:383-96, 2010
- 30. Bader P, Kreyenberg H, Henze GH, et al: Prognostic value of minimal residual disease quantification before allogeneic stem-cell transplantation in relapsed childhood acute lymphoblastic leukemia: the ALL-REZ BFM Study Group. J Clin Oncol 27:377-84, 2009
- 31. Sramkova L, Muzikova K, Fronkova E, et al: Detectable minimal residual disease before allogeneic hematopoietic stem cell transplantation predicts extremely poor prognosis in children with acute lymphoblastic leukemia. Pediatr Blood Cancer 48:93-100, 2007
- 32. Knechtli CJ, Goulden NJ, Hancock JP, et al: Minimal residual disease status before allogeneic bone marrow transplantation is an important determinant of successful outcome for children and adolescents with acute lymphoblastic leukemia. Blood 92:4072-9, 1998
- 33. Pulsipher MA, Langholz B, Wall DA, et al: The Relationship of Acute Gvhd and Preand Post-Transplant Flow-MRD to the Incidence and Timing of Relapse in Children Undergoing Allogeneic Transplantation for High Risk ALL: Defining a Target Population and Window for Immunological Intervention to Prevent Relapse. ASH Annual Meeting Abstracts 120:470-, 2012



- 34. Bader P, Kreyenberg H, Hoelle W, et al: Increasing mixed chimerism is an important prognostic factor for unfavorable outcome in children with acute lymphoblastic leukemia after allogeneic stem-cell transplantation: possible role for pre-emptive immunotherapy? J Clin Oncol 22:1696-705, 2004
- 35. Rettinger E, Willasch AM, Kreyenberg H, et al: Preemptive immunotherapy in childhood acute myeloid leukemia for patients showing evidence of mixed chimerism after allogeneic stem cell transplantation. Blood 118:5681-8, 2011
- 36. Horn B, Soni S, Khan S, et al: Feasibility study of preemptive withdrawal of immunosuppression based on chimerism testing in children undergoing myeloablative allogeneic transplantation for hematologic malignancies. Bone Marrow Transplant 43:469-76, 2009
- 37. Schwartz GJ, Gauthier B: A simple estimate of glomerular filtration rate in adolescent boys. J Pediatr 106:522-6, 1985
- 38. Relling MV, Pui CH, Sandlund JT, et al: Adverse effect of anticonvulsants on efficacy of chemotherapy for acute lymphoblastic leukaemia. Lancet 356:285-90, 2000
- 39. Bermudez M, Fuster JL, Llinares E, et al: Itraconazole-related increased vincristine neurotoxicity: case report and review of literature. J Pediatr Hematol Oncol 27:389-92, 2005
- 40. Ariffin H, Omar KZ, Ang EL, et al: Severe vincristine neurotoxicity with concomitant use of itraconazole. J Paediatr Child Health 39:638-9, 2003
- 41. Przepiorka D, Blamble D, Hilsenbeck S, et al: Tacrolimus clearance is age-dependent within the pediatric population. Bone Marrow Transplant 26:601-5, 2000
- 42. Stock W, Douer D, DeAngelo DJ, et al: Prevention and management of asparaginase/pegasparaginase-associated toxicities in adults and older adolescents: recommendations of an expert panel. Leuk Lymphoma 52:2237-53, 2011
- 43. Lee DW, Gardner R, Porter DL, et al: Current concepts in the diagnosis and management of cytokine release syndrome. Blood 124:188-95, 2014
- 44. Thorsten L, Peter M, Holger O, et al: CNS late-effects after ALL therapy in childhood. Part III: Neuropsychological performance in long-term survivors of childhood ALL: Impairments of concentration, attention, and memory\*†‡. Medical and Pediatric Oncology 38:320-328, 2002
- 45. Mulhern RK, Palmer SL: Neurocognitive late effects in pediatric cancer. Curr Probl Cancer 27:177-97, 2003
- 46. Harila-Saari AH, Paakko EL, Vainionpaa LK, et al: A longitudinal magnetic resonance imaging study of the brain in survivors in childhood acute lymphoblastic leukemia. Cancer 83:2608-17, 1998
- 47. Winick NJ, Bowman WP, Kamen BA, et al: Unexpected acute neurologic toxicity in the treatment of children with acute lymphoblastic leukemia. J Natl Cancer Inst 84:252-6, 1992
- 48. Wiedemann BC, Balis FM, Murphy RF, et al: Carboxypeptidase-G2, thymidine, and leucovorin rescue in cancer patients with methotrexate-induced renal dysfunction. J Clin Oncol 15(5):2125-34, 1997
- 49. DeAngelis LM, Tong WP, Lin S, et al: Carboxypeptidase G2 rescue after high-dose methotrexate. J Clin Oncol 14(7):2145-9, 1996
- 50. Brackett J, Schafer ES, Leung DH, et al: Use of allopurinol in children with acute lymphoblastic leukemia to reduce skewed thiopurine metabolism. Pediatr Blood Cancer 61:1114-7, 2014
- 51. Weinshilboum R. M, Sladek S. L: Mercaptopurine pharmacogenetics: monogenic inheritance of erythrocyte thiopurine methyltransferase activity. Am.J.Hum.Genet 32:651-662, 1980
- 52. Bostrom B, Erdmann G: Cellular pharmacology of 6-mercaptopurine in acute lymphoblastic leukemia. Am.J.Pediatr.Hematol.Oncol. 15:80-86, 1993
- 53. Lennard L, Lewis I. J, Michelagnoli M, et al: Thiopurine methyltransferase deficiency in childhood lymphoblastic leukaemia: 6-mercaptopurine dosage strategies. Med.Pediatr.Oncol. 29:252-255, 1997
- 54. Relling M. V, Hancock M. L, Rivera G. K, et al: Mercaptopurine therapy intolerance and heterozygosity at the thiopurine S-methyltransferase gene locus. J.Natl.Cancer Inst 91:2001-2008, 1999



- 55. Yates C. R, Krynetski E. Y, Loennechen T, et al: Molecular diagnosis of thiopurine S-methyltransferase deficiency: genetic basis for azathioprine and mercaptopurine intolerance. Ann.Intern.Med 126:608-614, 1997
- 56. Otterness D, Szumlanski C, Lennard L, et al: Human thiopurine methyltransferase pharmacogenetics: gene sequence polymorphisms. Clin.Pharmacol.Ther 62:60-73, 1997
- 57. Hon Y. Y, Fessing M. Y, Pui C.-H, et al: Polymorphism of the thiopurine S-methyltransferase gene in African Americans. Hum.Mol.Genet 8:371-376, 1999
- 58. Krynetski E. Y, Evans W. E: Genetic polymorphism of thiopurine S-methyltransferase: molecular mechanisms and clinical importance. Pharmacology 61:136-146, 2000
- 59. Van den Berg HW, Desai ZR, Wilson R, et al: The pharmacokinetics of vincristine in man: reduced drug clearance associated with raised serum alkaline phosphatase and dose-limited elimination. Cancer Chemother Pharmacol 8(2):215-9, 1982
- 60. Munzert G, Kirchner D, Ottmann O, et al: Constitutive NF-kappab/Rel activation in philadelphia chromosome positive (Ph+) acute lymphoblastic leukemia (ALL). Leukemia & lymphoma 45:1181-4, 2004
- 61. Vrooman, et al: Preliminary Results Of a Pharmacokinetic Study Of Intravenous Asparaginase Erwinia Chrysanthemi Following Allergy To E Coli-Derived Asparaginase In Children, Adolescents, and Young Adults With Acute Lymphoblastic Leukemia Or Lymphoblastic Lymphoma. ASH abstracts 2013, #3904 and also communication from Jazz pharmaceuticals and updated FDA labeling information, 2013
- 62. Freidlin B, Korn EL: A comment on futility monitoring. Control Clin Trials 23:355-66, 2002
- 63. Anderson JR: Adjusting interim monitoring for efficacy when full information is misspecified. COG Internal Paper
- 64. Dmitrienko A: Statistical monitoring of clinical trials: A unified approach. Michael A. Proschan, K. K. Gordon Lan and Janet Turk Wittes, Springer, New York, 2006. No. of pages: xiv+258. Price: \$74.95, £50.00, €69.50. ISBN: 978-0-387-30059-7. Statistics in Medicine 26:3822-3824, 2007
- 65. Gordon Lan KK, Demets DL: Discrete sequential boundaries for clinical trials. Biometrika 70:659-663, 1983
- 66. O'Brien PC, Fleming TR: A multiple testing procedure for clinical trials. Biometrics 35:549-56, 1979
- 67. Zhang J, Mullighan CG, Harvey RC, et al: Key pathways are frequently mutated in high-risk childhood acute lymphoblastic leukemia: a report from the Children's Oncology Group. Blood 118:3080-7, 2011
- 68. Mullighan CG, Su X, Zhang J, et al: Deletion of IKZF1 and prognosis in acute lymphoblastic leukemia. N Engl J Med 360:470-80, 2009
- 69. van Delft FW, Horsley S, Colman S, et al: Clonal origins of relapse in ETV6-RUNX1 acute lymphoblastic leukemia. Blood 117:6247-54, 2011
- 70. Hunger SP, Raetz EA, Loh ML, et al: Improving outcomes for high-risk ALL: translating new discoveries into clinical care. Pediatr Blood Cancer 56:984-93, 2011
- 71. Mullighan CG: New strategies in acute lymphoblastic leukemia: translating advances in genomics into clinical practice. Clin Cancer Res 17:396-400, 2011
- 72. Roberts KG, Mullighan CG: How new advances in genetic analysis are influencing the understandign and treatment of childhood acute leukemia. Current opinion in pediatircs 23:34-40, 2011
- 73. Kishi S, Cheng C, French D, et al: Ancestry and pharmacogenetics of antileukemic drug toxicity. Blood 109:4151-7, 2007
- 74. Yang JJ, Cheng C, Yang W, et al: Genome-wide interrogation of germline genetic variation associated with treatment response in childhood acute lymphoblastic leukemia. JAMA 301:393-403, 2009



- 75. Davies SM, Borowitz MJ, Rosner GL, et al: Pharmacogenetics of minimal residual disease response in children with B-precursor acute lymphoblastic leukemia: a report from the Children's Oncology Group. Blood 111:2984-90, 2008
- 76. Krajinovic M, Labuda D, Sinnett D: Glutathione S-transferase P1 genetic polymorphisms and susceptibility to childhood acute lymphoblastic leukaemia. Pharmacogenetics 12(8):655-8, 2002
- 77. Ansari M, Sauty G, Labuda M, et al: Polymorphisms in multidrug resistance-associated protein gene 4 is associated with outcome in childhood acute lymphoblastic leukemia. Blood 114:1383-6, 2009
- 78. Davies SM, Bhatia S, Ross JA, et al: Glutathione S-transferase genotypes, genetic susceptibility, and outcome of therapy in childhood acute lymphoblastic leukemia. Blood 100:67-71, 2002
- 79. Stanulla M, Schaeffeler E, Flohr T, et al: Thiopurine methyltransferase (TPMT) genotype and early treatment response to mercaptopurine in childhood acute lymphoblastic leukemia. JAMA 293:1485-9, 2005
- 80. Rocha JC, Cheng C, Liu W, et al: Pharmacogenetics of outcome in children with acute lymphoblastic leukemia. Blood 105:4752-8, 2005
- 81. Aplenc R, Glatfelter W, Han P, et al: CYP3A genotypes and treatment response in paediatric acute lymphoblastic leukaemia. Br J Haematol 122:240-4, 2003
- 82. French D, Yang W, Cheng C, et al: Acquired variation outweighs inherited variation in whole genome analysis of methotrexate polyglutamate accumulation in leukemia. Blood 113:4512-20, 2009
- 83. Handgretinger R, Zugmaier G, Henze G, et al: Complete remission after blinatumomabinduced donor T-cell activation in three pediatric patients with post-transplant relapsed acute lymphoblastic leukemia. Leukemia 25:181-4, 2011
- 84. Feuerer M, Beckhove P, Bai L, et al: Therapy of human tumors in NOD/SCID mice with patient-derived reactivated memory T cells from bone marrow. Nat Med 7:452-8, 2001
- 85. Feuerer M, Beckhove P, Garbi N, et al: Bone marrow as a priming site for T-cell responses to blood-borne antigen. Nat Med 9:1151-7, 2003
- 86. Di Rosa F, Santoni A: Bone marrow CD8 T cells are in a different activation state than those in lymphoid periphery. Eur J Immunol 32:1873-80, 2002
- 87. Zou L, Barnett B, Safah H, et al: Bone marrow is a reservoir for CD4+CD25+ regulatory T cells that traffic through CXCL12/CXCR4 signals. Cancer Res 64:8451-5, 2004
- 88. Noonan K, Matsui W, Serafini P, et al: Activated marrow-infiltrating lymphocytes effectively target plasma cells and their clonogenic precursors. Cancer Res 65:2026-34, 2005
- 89. Serafini P, Mgebroff S, Noonan K, et al: Myeloid-derived suppressor cells promote cross-tolerance in B-cell lymphoma by expanding regulatory T cells. Cancer Res 68:5439-49, 2008
- 90. Bettelli E, Carrier Y, Gao W, et al: Reciprocal developmental pathways for the generation of pathogenic effector TH17 and regulatory T cells. Nature 441:235-8, 2006
- 91. Tibes R, Qiu Y, Lu Y, et al: Reverse phase protein array: validation of a novel proteomic technology and utility for analysis of primary leukemia specimens and hematopoietic stem cells. Mol Cancer Ther 5:2512-21, 2006
- 92. Kornblau SM, Tibes R, Qiu YH, et al: Functional proteomic profiling of AML predicts response and survival. Blood 113:154-64, 2009
- 93. York H, Kornblau SM, Qutub AA: Network analysis of reverse phase protein expression data: characterizing protein signatures in acute myeloid leukemia cytogenetic categories t(8;21) and inv(16). Proteomics 12:2084-93, 2012
- 94. Redell MS, Ruiz MJ, Gerbing RB, et al: FACS analysis of Stat3/5 signaling reveals sensitivity to G-CSF and IL-6 as a significant prognostic factor in pediatric AML: a Children's Oncology Group report. Blood 121:1083-93, 2013



- 95. Perl AE, Kasner MT, Shank D, et al: Single-cell pharmacodynamic monitoring of S6 ribosomal protein phosphorylation in AML blasts during a clinical trial combining the mTOR inhibitor sirolimus and intensive chemotherapy. Clin Cancer Res 18:1716-25, 2012
- 96. Espina V, Woodhouse EC, Wulfkuhle J, et al: Protein microarray detection strategies: focus on direct detection technologies. J Immunol Methods 290:121-33, 2004
- 97. Neeley ES, Kornblau SM, Coombes KR, et al: Variable slope normalization of reverse phase protein arrays. Bioinformatics 25:1384-9, 2009
- 98. Kornblau SM, Qutub A, Yao H, et al: Proteomic profiling identifies distinct protein patterns in acute myelogenous leukemia CD34+CD38- stem-like cells. PLoS One 8:e78453, 2013
- 99. Maude SL, Tasian SK, Vincent T, et al: Targeting JAK1/2 and mTOR in murine xenograft models of Ph-like acute lymphoblastic leukemia. Blood 120:3510-8, 2012
- 100. Tasian SK, Doral MY, Borowitz MJ, et al: Aberrant STAT5 and PI3K/mTOR pathway signaling occurs in human CRLF2-rearranged B-precursor acute lymphoblastic leukemia. Blood 120:833-42, 2012
- 101. Tasian SK, Li Y, Ryan T, et al: In Vivo Efficacy of PI3K Pathway Signaling Inhibition for Philadelphia Chromosome-Like Acute Lymphoblastic Leukemia. Blood 122(21): ASH Annual Meeting 2013 abstract #672, 2013
- 102. Gill S and Tasian SK, Ruella M, Shestova O, et al: Efficacy against Human Acute Myeloid Leukemia and Myeloablation of Normal Hematopoiesis in a Mouse Model Using Chimeric Antigen Receptor-Modified T-Cells. Blood 123: accepted for publication, 2014
- 103. SM Kornblau CH, YH Qiu, SY Yoo, N Xhang, TM Kadia, A Ferrajoli, KR Coombes, AA Qutub: Hippo Pathway (HP) activity in AML: different prognostic implications of TAZ vs. YAP inactivation by phosphorylation. Blood (2013), 2013
- 104. Dupuy A, Simon RM: Critical review of published microarray studies for cancer outcome and guidelines on statistical analysis and reporting. J Natl Cancer Inst 99:147-57, 2007
- 105. Tibshirani R, Walther G, T. H: Estimating the number of data clusters via the gap statistic. J.R.Statist.Doc.B. 63:10-20, 2001
- 106. McShane LM, Radmacher MD, Freidlin B, et al: Methods for assessing reproducibility of clustering patterns observed in analyses of microarray data. Bioinformatics 18:1462-9, 2002
- 107. Hsu CW, Lin CJ: A comparison of methods for multiclass support vector machines. IEEE Trans Neural Netw 13:415-25, 2002
- 108. Statnikov A, Wang L, Aliferis CF: A comprehensive comparison of random forests and support vector machines for microarray-based cancer classification. BMC Bioinformatics 9:319, 2008
- 109. Belgaumi AF, Al-Seraihy A, Siddiqui KS, et al: Outcome of risk adapted therapy for relapsed/refractory acute lymphoblastic leukemia in children. Leuk Lymphoma 54:547-54, 2013
- 110. Reismuller B, Peters C, Dworzak MN, et al: Outcome of children and adolescents with a second or third relapse of acute lymphoblastic leukemia (ALL): a population-based analysis of the Austrian ALL-BFM (Berlin-Frankfurt-Munster) study group. J Pediatr Hematol Oncol 35:e200-4, 2013
- 111. Benjamini Y, Y. H: Methods of assessing reporducibiolity of clustering patterns observed in analysis of microarray data. Journal of the Royal Statistical Society B. 57:289-300, 1995